

# CLI 00125 ReCePI PROTOCOL, v8.0

A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

**April 6, 2023** 

NCT03459287

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

## **PROTOCOL**

TITLE: A Randomized, Double-Blinded, Controlled, Parallel Group,

Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures

(the ReCePI study)

**SPONSOR:** Cerus Corporation

1220 Concord Avenue Concord, CA 94520, USA

(925) 288-6000

PROTOCOL NUMBER: CLI 00125

**DATE:** April 6, 2023 Amendment 8.0

**IDE NUMBER:** BB-IDE 13803

**MEDICAL MONITOR:** Christine Ernst, MD, PhD

Sr. Director, Clinical Research and Medical Affairs

Cerus Corporation (925) 288-6259

Richard J. Benjamin MD, PhD

Chief Medical Officer Cerus Corporation (925) 288-6020

MANAGER (or sponsor

Paulette Niemyski

contact):

Sr. Clinical Trial Manager

Cerus Corporation (925) 288-6000

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

## **SYNOPSIS**

| Name of Sponsor/Company: | | Individual S<br>Referring to | • | (For National Authority Use only) |
|---|---|---|---|---|
| | | of the Dossi | | Ose omy) |
| Name of Finishe | Name of Finished Product: | | | |
| Not applicable | | | | |
| Name of Active Ingredient: | | Page: | | |
| Red Blood Cells treated with the INTERCEPT Blood System | | | | |
| Title of Study: | A Randomized, Double-Blir<br>Study to Evaluate the Effica<br>Blood Cells in Patients unde<br>study) | Blood System for Red | | |
| Investigators / S | tudy Sites/Blood Centers: 15- | -20 clinical sit | es and up to 4 bloo | d centers |
| Publication (refe | erence): NA | | | |
| - " | years): To Be Determined (Trollment: November 21, 2018 | · · | of development: 3 | |
| Date of last con | npleted: TBD | | | |

## **Objective:**

The objective of this study is to evaluate the efficacy and safety of red blood cell (RBC) transfusion for support of acute anemia in cardiovascular surgery patients based on the clinical outcome of renal impairment following transfusion of RBCs treated with the INTERCEPT Blood System for Red Blood Cells compared to patients transfused with conventional RBCs.

## Methodology:

The study is a prospective, multicenter, randomized, double-blinded, active controlled, parallel-design, non-inferiority study.

## **Primary Endpoints:**

#### **Primary**

Efficacy:

The primary efficacy endpoint is the proportion of patients who have received at least one study transfusion with a diagnosis of renal impairment defined as:

 Any raised serum creatinine (sCr) level, occurring after transfusion of a study RBC, of ≥0.3 mg/dL (or 26.5 μmol/L) from the pre-surgery baseline within 48±4 hours of the end of surgery.

## Safety:

The primary safety endpoints are:

• Proportion of patients with any treatment-emergent adverse events (TEAEs) possibly, probably or

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| Name of Sponsor/Company: | Individual Study Table Referring to Part of the Dossier | (For National Authority |
|---|---|---|
| CERUS CORPORATION | | Use only) |
| Name of Finished Product: | Volume: | |
| Not applicable | | |
| Name of Active Ingredient: | Page: | |
| Red Blood Cells treated with the INTERCEPT Blood System | | |

definitely related to study RBC transfusion through 28 days after the last study transfusion; and

• Proportion of patients with treatment-emergent antibodies with confirmed specificity to INTERCEPT RBCs by the end of study (i.e., 75±15 days after the last study transfusion).

## **Study Procedures:**

## Screening/Recruitment

In order to minimize the number of patients who enroll in the study but do not require RBC transfusion, only patients with a relatively high likelihood to receive a RBC transfusion as determined by the Investigator (e.g., patients receiving aspirin, clopidogrel (or analogs) and/or GPIIb/IIIa inhibitors), or patients with a TRUST Score of  $\geq 3$  will be eligible for enrollment. Patients  $\geq 11$  years of age undergoing complex cardiac surgery may be identified through pre-operative scheduling procedures in advance of their surgery.

Patients undergoing urgent or emergent cardiac surgery are eligible for the study, subject to institutional review board (IRB) approval of an appropriate informed consent process.

All potentially eligible patients will be approached for study consent/assent within 30 days prior to their surgical procedure. Subjects who consent/assent to the study will be assigned a subject ID number and undergo screening.

Screening will include documentation of the patient's pre-surgical exposure to radiographic contrast media and number of prior pregnancies (females). Screening data may be derived from the medical record when performed within 30 days prior to their surgical procedure. Eligibility status and other study data including all TRUST components will be entered into the clinical database via an electronic data capture (EDC) system using electronic case report forms (eCRFs). Patients who fail eligibility for any or multiple inclusion/exclusion criteria may be rescreened for eligibility closer to the time of surgery.

## Randomization and Blinding

Eligible subjects will be randomized up to 7 days before or on the day of scheduled surgery (Day 0). An Interactive Web Response System (IWRS) will be used for electronic randomization of eligible patients. Randomization (in 1:1 ratio for Test:Control) stratified by site, pre-existing renal impairment (baseline sCr  $\geq$ 1.2 mg/dL vs. < 1.2 mg/dL), and cardiac surgery group (more at risk for renal complications vs. less at risk) will be employed. Screened subjects who receive a red cell transfusion prior to randomization will no longer be considered for randomization, and their participation in the study will end. Patients may be rescreened for eligibility closer to the time of surgery.

#### **Treatment**

Once a subject is randomized, only study RBCs (Test or Control, per the subject's randomization) should be dispensed and transfused during the acute transfusion support period (Day 0 to Day 7 post surgery, hospital discharge, or death, whichever is first), as clinically indicated and determined by the treating physician.

In rare exceptions where study RBCs are unavailable or patient's need for RBC transfusions exceeds the quantity of study RBCs in inventory at the hospital blood bank (e.g., during a Massive Transfusion Protocol), a

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| Name of Sponsor/Company: | Individual Study Table<br>Referring to Part<br>of the Dossier | (For National Authority<br>Use only) |
|---|---|---|
| CERUS CORPORATION | | |
| Name of Finished Product: | Volume: | |
| Not applicable | | |
| Name of Active Ingredient: | Page: | |
| Red Blood Cells treated with the INTERCEPT Blood System | | |

transfusion using non-study RBC (conventional) may be given to provide the patient with an appropriate and necessary treatment. In this case, a protocol deviation should be documented. If a study RBC transfusion is given after randomization before surgery commences, a protocol deviation should also be documented.

Treatment assessments will be divided into an acute transfusion support period starting the day of surgery (Day 0 up to Day 7) during which study RBC (Test or Control) are administered, a post-surgical follow-up period of a minimum of 28 days after the last study transfusion to collect additional safety data, a clinical assessment at day 30 after surgery specifically for mortality and RRT status, and a visit at day 75 ( $\pm$ 15) after the last study transfusion to assess mortality and RRT status, and collect samples for serological screening for antibodies specific to INTERCEPT RBCs.

In all patients, anesthesia and surgical procedures will be performed according to the local standards of care. Following the acute transfusion support period, subjects may receive conventional RBC components if additional transfusions are needed, as indicated by their treating physician.

## Study Assessments: Monitoring and Follow-up

Baseline through Acute Transfusion Support Period (Pre-Op Day -1 up to Post-Op Day 7)

A screen for antibodies specific for INTERCEPT RBCs should be performed every time that a routine IAT is performed during the acute 7-day study transfusion period.

A blood sample for sCr will be taken at  $48 \pm 4$  hours after completion of surgery for both transfused and non-transfused subjects., A sCr will be determined on a daily basis during the acute transfusion support period up to 7 days post-surgery. Other parameters including additional sCr will be collected on eCRFs only when available in the medical record.

Randomized subjects who do not receive an RBC transfusion following randomization within the first 48 hours after surgery will be discontinued from the study and replaced.

Daily sCr assessments will be recorded up to and including  $48 \pm 4$  hours for transfused and non-transfused subjects. Other post baseline laboratory parameters and adverse events (AEs) will not be collected for non-transfused subjects. Vital status will be reported for randomized and non-transfused subjects at the time of discontinuation.

Hemodynamic and laboratory measures will be assessed pre-operatively (Day -1, Baseline) and daily as available in the medical record from post-operative Day 1 through Day 7, hospital discharge or death, whichever occurs first. If a subject is discharged prior to Day 7 but returns to the study site for a standard of care visit on Day 7, blood samples should be obtained on that day for a complete blood count and sCr determination.

Hemodynamic parameters that will be collected if available, include heart rate, blood pressure, mean arterial pressure, central venous pressure (CVP), and peripheral oxygen saturation via pulse oximetry probe.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| Name of Sponsor/Company: | Individual Study Table<br>Referring to Part<br>of the Dossier | (For National Authority<br>Use only) |
|---|---|---|
| CERUS CORPORATION | | |
| Name of Finished Product: | Volume: | |
| Not applicable | | |
| Name of Active Ingredient: | Page: | |
| Red Blood Cells treated with the INTERCEPT Blood System | | |

Laboratory parameters that will be captured on eCRFs include BUN, creatinine, AST, ALT, fibrinogen, bilirubin, troponin, hemoglobin, and platelet counts.

Transfusion reactions (TRs), adverse events (AEs) and serious adverse events (SAEs) will be assessed on a daily basis and documented in the eCRF from the start of surgery or the start of the first study transfusion (whichever is first) through post-operative Day 7 and as available through day 28 after the last study transfusion. Vital status will be reported for randomized and non-transfused subjects at the time of discontinuation.

NOTE: The following applies to randomized transfused subjects only.

<u>Post-operative Day 8 (or Post-discharge, if earlier) through 28 Days After Last Study Transfusion.</u> Subjects will be monitored for TRs, AEs and SAEs following the 7-day acute transfusion support period, through 28 days after the last study transfusion or death, whichever occurs first, according to the local standard of care. In an outpatient setting, weekly telephone surveillance calls to the subject will be performed in order to collect safety events until the next follow-up visit.

## 28 (±3) Days After Last Study Transfusion or Premature Discontinuation from study.

Subjects who have been discharged should be scheduled for the follow up visit 28 (±3) days after the last study transfusion to obtain additional safety information, including patient-reported AEs/ SAEs; laboratory results including sCr, DAT/ IAT; a sample for HLA antibodies and antibodies specific to INTERCEPT RBCs will be obtained. All randomized subjects who receive any study RBC transfusion must have their vital status documented at this visit, or earlier, if the subject dies prior to the visit. If a subject has been discharged, other safety information (e.g., AEs and SAEs) may be obtained through medical records, the subject's physician, or a telephone interview with either the subject or a family member.

## 30 Days After Surgery

All randomized subjects who receive a study RBC transfusion must have their vital status and need for RRT (defined as hemodialysis or peritoneal dialysis) documented at Day 30 after surgery. RRT that is provided prophylactically during surgery while patient is on a bypass machine (the pump), does not meet this endpoint. The vital status and RRT assessment on Day 30 can be performed either from the medical records, from a phone call to the subject or family, or during the visit  $28\pm3$  days after the last study transfusion (only if the last study transfusion was given at day 2 or later in the acute transfusion support period).

## End of Study: 75 (±15 Days) After last Study Transfusion

75 ( $\pm 15$ ) days after the last study transfusion (End of Study), serum samples for antibodies specific for INTERCEPT RBCs will be obtained, either in hospital, at a clinic visitor or offsite. Mortality and the need for RRT will be assessed.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| Name of Sponsor/Company: | Individual Study Table<br>Referring to Part<br>of the Dossier | (For National Authority<br>Use only) |
|---|---|---|
| CERUS CORPORATION | | |
| Name of Finished Product: | Volume: | |
| Not applicable | | |
| Name of Active Ingredient: | Page: | |
| Red Blood Cells treated with the INTERCEPT Blood System | | |

## Data and Safety Monitoring Board (DSMB)

The study will be monitored by an independent Data and Safety Monitoring Board (DSMB). The primary mission of the DSMB is to ensure patient safety and review protocol compliance for data collection. The DSMB will be assembled by the Sponsor and composed of transfusion medicine and other experts as per the DSMB charter. DSMB members will be independent of the Sponsor.

## Interim Analysis and Early Stopping Rule

Aside from the blinded interim analysis for sample size re-estimation performed in October 2021, no other interim analysis is planned for this study to compare treatment differences with respect to efficacy or safety at any time prior to the completion of the study. Specific stopping rules, defined for safety considerations, are defined in Section 4.6 of the protocol.

#### **Number of patients:**

A total of at least 292 evaluable, randomized and transfused patients, 146 per arm, are planned to generate sufficient efficacy and safety data for the Test and Control components in patients undergoing cardiac surgery procedures.

For the primary efficacy endpoint, the proportion of patients with a  $\Delta sCr \ge 0.3$  mg/dL from pre-surgery baseline to within 48±4 hours after surgery, a non-inferiority test will be conducted to assess for treatment difference (Test – Control). By assuming an event rate of 30% in the Control group and no more than 50% increase from the Control rate as the non-inferiority margin, a sample size of 292 patients (146 per arm) will provide approximately 80% power to declare non-inferiority at the two-sided 0.05 alpha level, assuming the true treatment difference is zero.

#### Diagnosis and main criteria for inclusion:

## **Inclusion criteria:**

- 1. Age  $\geq$  11 years of age
- 2. Weight  $\geq 40 \text{ kg}$
- 3. Scheduled complex cardiac surgery or thoracic aorta surgery. The procedure may be performed either on or off cardiopulmonary bypass machine (CBP or "pump"). For the purposes of this protocol "Repeat procedure" means that the subject had a previous cardiac surgery. Procedures that qualify as complex cardiac surgery include but are not limited to, the following:
  - Single Vessel Coronary Artery Bypass Graft, first or repeat procedure
  - Multiple Coronary Artery Bypass Grafts, first or repeat procedure
  - Single Valve Repair or Replacement, first or repeat procedure
  - Multiple Valve Repair or Replacement, first or repeat procedure

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| Name of Sponsor/Company: | Individual Study Table Referring to Part of the Dossier | (For National Authority<br>Use only) |
|---|---|---|
| CERUS CORPORATION | | |
| Name of Finished Product: | Volume: | |
| Not applicable | | |
| Name of Active Ingredient: | Page: | |
| Red Blood Cells treated with the INTERCEPT Blood System | | |

- Surgery involving both Coronary Artery Bypass Graft(s) and Valve Repair(s), first or repeat procedure
- One or more of the following procedures, with or without Coronary Bypass Graft(s):
  - o left ventricular aneurysm repair
  - o ventricular and/or atrial septal defect repairs
  - o Batista procedure (surgical ventricular remodeling)
  - o surgical ventricular restoration
  - o congenital cardiac defect repair
  - o aortic procedures
  - o other cardiac surgery or thoracic aorta surgery types with a high probability of bleeding.
- 4. TRUST probability score (Alghamdi, Davis et al. 2006) ≥ 3, or currently on a regimen of aspirin (any dose), clopidogrel (or analogs) and/or GPIIb/IIIa inhibitors or at a high probability for need of a transfusion during or after surgery at the discretion of the Investigator
- 5. Female subjects of child-bearing potential must meet the 2 criteria below at screening:
  - Negative serum or urine pregnancy test
  - Use at least one method of birth control that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence or vasectomized partner
- 6. Signed and dated informed consent/assent form.

## Exclusion criteria:

- 1. Confirmed positive baseline serum/plasma antibody specific to INTERCEPT RBCs (S-303 specific antibody) screening panel prior to randomization.
- 2. Pregnant or breast feeding
- 3. Refusal of blood products or other inability to comply with the protocol in the opinion of the Investigator or the treating physician
- 4. Treatment with any medication that is known to adversely affect RBC viability, such as, but not limited to dapsone, levodopa, methyldopa, nitrofurantoin, and its derivatives, phenazopyridine and quinidine.
- 5. Planned cardiac transplantation
- 6. Active autoimmune hemolytic anemia

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| Name of Sponsor/Company: | Individual Study Table<br>Referring to Part<br>of the Dossier | (For National Authority<br>Use only) |
|---|---|---|
| CERUS CORPORATION | | |
| Name of Finished Product: | Volume: | |
| Not applicable | | |
| Name of Active Ingredient: | Page: | |
| Red Blood Cells treated with the INTERCEPT Blood System | | |

- 7. Left ventricular assist device (LVAD) or extracorporeal membrane oxygenation (ECMO) support pre-operatively or planned need post-operatively
- 8. Cardiogenic shock requiring pre-operative placement of an intra-aortic balloon pump (IABP) (NOTE: IABP done for unstable angina or prophylactically for low ejection fraction is not excluded).
- 9. Planned use of autologous or directed donations.
- 10. RBC transfusion during current hospitalization prior to enrollment and randomization (within 7 days).
- 11. Participation in an interventional clinical study concurrently or within the previous 28 days. This includes investigational blood products, pharmacologic agents, imaging materials (including dyes), surgical techniques, or devices. Observational studies of FDA cleared or approved products or nutrition, psychology, or socioeconomic issues are not grounds for exclusion.
- 12. Patients with a current diagnosis of either chronic kidney disease or acute kidney injury and with sCr ≥1.8 mg/dL at screening and patients requiring RRT. (NOTE: If sCr at screening is <1.8 mg/dL, a patient with a diagnosis of chronic or acute kidney injury alone is not excluded).
- 13. Patients with a current diagnosis of either chronic or acute hepatic insufficiency and with a total serum bilirubin ≥ 2.0 mg/dL (≥34.2 μmol/L). (NOTE: If total serum bilirubin at screening is <2.0 mg/dL, a patient with a diagnosis of chronic or acute hepatic failure alone is not excluded).
- 14. Pre-existing antibody(ies) to RBC antigens that may make the provision of compatible study RBC components difficult.
- 15. History of TRs requiring washed RBCs, volume reduced RBC, or RBCs with additive solution removed.
- 16. Patients with documented IgA deficiency or a history of severe allergic reactions to blood products.
- 17. Patients who require gamma-irradiated RBC blood components.
- 18. Positive DAT as defined below:

A polyspecific DAT reaction strength > 2+, or

A polyspecific DAT (any strength) in conjunction with pan-reactivity with a commercial IAT antibody screening panel that precludes the identification of underlying alloantibodies or indicates the presence of autoantibody.

## Test product, dose and mode of administration:

The test device is the INTERCEPT Blood System for RBC. The INTERCEPT treatment process uses amustaline and glutathione together with a processing solution in a single-use disposable set and results in pathogen and leukocyte inactivated RBCs suspended in SAG-M additive solution (INTERCEPT RBCs). The INTERCEPT treatment will be performed on leukoreduced RBC components prepared from whole blood

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| Name of Sponsor/Company: | Individual Study Table<br>Referring to Part<br>of the Dossier | (For National Authority<br>Use only) |
|---|---|---|
| CERUS CORPORATION | | |
| Name of Finished Product: | Volume: | |
| Not applicable | | |
| Name of Active Ingredient: | Page: | |
| Red Blood Cells treated with the INTERCEPT Blood System | | |

collections and suspended in AS-5 additive solution within 24 hours of collection. The test component is allogeneic INTERCEPT RBCs suspended in SAG-M and stored at 1°C to 6° for up to 35 days post-donation and administered intravenously. The treating physician will determine dose and schedule of RBC transfusions.

## Control product, dose and mode of administration:

The control transfusion component is a conventional leukoreduced RBC component in an FDA approved additive solution (AS-1, AS-3 or AS-5) stored at 1°C to 6°C for up to 35 days post-donation and administered intravenously. The Control RBC components will be handled and labeled in a manner to maintain blinding. The treating physician will determine dose and schedule of RBC transfusions.

#### **Criteria for evaluation:**

#### **Efficacy:**

The primary efficacy endpoint is the proportion of patients, who have received at least one study transfusion with a diagnosis of renal impairment defined as:

• Any raised sCr level, occurring after transfusion of a study RBC, of ≥0.3 mg/dL (or 26.5 μmol/L) from the pre-surgery baseline within 48±4 hours of the end of surgery.

If any subject meets this criterion before receiving a study transfusion, that particular event will not be included in this analysis.

Secondary efficacy outcome measures include:

- The proportion of patients with a diagnosis of stage I, II or III Acute Kidney Injury (KDIGO 2012) based on changes in sCr levels from pre-surgery baseline and the need for renal replacement therapy (RRT) post-surgery.
- Mortality or the need for RRT by 30 days post-surgery.

## **Safety:**

The primary safety outcome measures are the:

- Proportion of patients with any treatment-emergent adverse events (TEAEs) possibly, probably or definitely related to study RBC transfusion through 28 days after the last study transfusion; and
- Proportion of patients with treatment emergent antibodies with confirmed specificity to INTERCEPT RBCs by end of study (i.e., 75±15 days after the last study transfusion).

Additional safety assessments will include:

- Treatment-emergent AEs through 28 days after the last study transfusion.
- Treatment-emergent SAEs through 28 days after the last study transfusion.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| Name of Sponsor/Company: | Individual Study Table<br>Referring to Part<br>of the Dossier | (For National Authority<br>Use only) |
|---|---|---|
| CERUS CORPORATION | | |
| Name of Finished Product: | Volume: | |
| Not applicable | | |
| Name of Active Ingredient: | Page: | |
| Red Blood Cells treated with the INTERCEPT Blood System | | |

- Transfusion reactions (as defined by the CDC National Healthcare Safety Network [NHSN] Hemovigilance Module protocol) through 28 days after last study transfusion.
- Treatment-emergent immunization to RBC allo-antigens through 28±3 days after the last study transfusion.
- Treatment-emergent immunization to HLA allo-antigens through 28±3 days after the last study transfusion.

#### Statistical methods:

For the primary efficacy endpoint, the treatment difference (Test – Control) and its two-sided 95% confidence interval (CI) will be estimated from Cochran-Mantel-Haenszel (CMH) test stratified by baseline sCr (sCr  $\geq$ 1.2 mg/dL vs. < 1.2 mg/dL) and cardiac surgery group (more at risk for renal complications vs. less at risk) performed. The upper bound of the two-sided 95% CI will be compared with the 50% of the observed Control rate. Non-inferiority will be achieved if the upper bound is less than the 50% of the observed Control rate. For the non-inferiority test, the null and alternative hypotheses (H0 and H1, respectively) will be formulated as follows:  $H_0: P_{Test} - P_{Control} \geq 50\% \times \hat{P}_{Control}$  vs.  $H_1: P_{Test} - P_{Control} < 50\% \times \hat{P}_{Control}$ ,

where  $P_{Test}$  and  $P_{Control}$  are the event rates for Test (INTERCEPT) and Control groups, respectively, and  $\hat{P}_{Control}$  is the observed Control rate.

Same CMH test will be used for assessment of treatment differences for the secondary efficacy endpoints. As a sensitivity analysis, logistic regression will be utilized to estimate the treatment differences after controlling for baseline sCr, cardiac surgery group performed and other covariates to be detailed in the statistical analysis plan (SAP). Treatment-emergent AEs (defined as AEs with an onset date/time that is on or after the start date/time of the first study transfusion) will be summarized by treatment group, system organ class (SOC), and preferred term.

Subgroup analysis by the randomization stratification variables (clinical site, pre-surgery renal impairment, and cardiac surgery group) and by demographic variables such as age group ( $\leq$ 18, 19 to 65, and >65 years old), sex, and race will be presented for primary and secondary efficacy endpoints. Additional subgroup analysis may also be presented as suggested by the data.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

## **TABLE OF CONTENTS**

| SY | NOPS | IS | 2 |
|---|---|---|---|
| 1 | LIS | T OF ABBREVIATIONS AND DEFINITIONS OF TERMS | 15 |
| 2 | BA | CKGROUND INFORMATION | 19 |
| | 2.1 | | |
| | 2.2 | Name and Description of the Investigational Product | 22 |
| | | 2.2.1 Description of Investigational Product | |
| | 2.3 | Summary of Nonclinical and Clinical Studies | |
| | | 2.3.1 Safety | |
| | | 2.3.2 Immunogenicity | |
| | | 2.3.3 Clinical Studies | 23 |
| | 2.4 | Summary of Potential Risks | 26 |
| | 2.5 | Description of and Rationale for Treatment | 27 |
| 3 | STU | UDY OBJECTIVES | 33 |
| 4 | INV | VESTIGATIONAL PLAN | 34 |
| | | Endpoints | |
| | | 4.1.1 Primary Endpoints | |
| | | 4.1.2 Secondary Endpoints | |
| | 4.2 | Study Design | |
| | 4.3 | Randomization and Blinding | 38 |
| | 4.4 | Treatment | 39 |
| | | 4.4.1 Test Product | 40 |
| | | 4.4.2 Control (reference) Product | 40 |
| | 4.5 | Subject Discontinuation | 40 |
| | | 4.5.1 Definitions | 41 |
| | | 4.5.1.1 Enrollment Pause | 41 |
| | | 4.5.1.2 Clinical Stop | |
| | | 4.5.1.3 Rules | |
| | | Accountability of Study Product | |
| | 4.7 | | |
| 5 | SEI | LECTION AND WITHDRAWAL OF SUBJECTS | 46 |
| | 5.1 | Subject Inclusion Criteria | 46 |
| | 5.2 | Subject Exclusion Criteria | 47 |
| | 5.3 | Subject withdrawal Criteria | 48 |
| | | 5.3.1 Discontinuation from study RBC transfusions | |
| | | 5.3.2 Early termination from Study | |
| 6 | TR | EATMENT OF SUBJECTS | 50 |
| | 6.1 | Treatment Plan | 50 |
| | | 6.1.1 Screening/Randomization (Day -30 to Day 0 Pre-Surgery) | 50 |

| | | 6.1.2 | Acute Transfusion Support Period (Surgery [Day 0] to Post-<br>operative Day 7, Hospital Discharge or Death, Whichever is First) | 51 |
|---|---|---|---|---|
| | | 6.1.3 | Post-operative Period (Day 8 [or Post-discharge, if earlier] through | |
| | | 0.1.5 | Day 28 After Last Study Transfusion) | |
| | | 6.1.4 | Day 28±3 After Last Study Transfusion or Early Termination | |
| | | 6.1.5 | Day 30 – After Surgery Assessment | |
| | | 6.1.6 | End of Study (75 ±15 Days After Last Study Transfusion) | |
| | | 6.1.7 | Assessments in Follow-up to a Reactive Antibody Test Specific for INTERCEPT RBCs | or |
| | 6.2 | Conco | | |
| | 6.3 | | omitant and Excluded Therapynent Compliance | |
| _ | | | <del>-</del> | |
| 7 | | | SSESSMENTS | |
| | 7.1 | - | Schedule of Assessments | |
| | 7.2 | | sment of Efficacy | |
| | | | Efficacy Parameters | |
| | | 7.2.2 | Methods and Timing of Efficacy Parameters | |
| | 7.3 | | sment of Safety | |
| | | 7.3.1 | J | |
| | | | 7.3.1.1 Definition of Adverse Event | |
| | | | 7.3.1.2 Definition of Serious Adverse Event | |
| | | | 7.3.1.3 Unexpected Adverse Event | |
| | | | 7.3.1.4 Definition of Unanticipated Adverse Device Effects | |
| | | | 7.3.1.5 Definition of Renal Impairment | |
| | | | 7.3.1.6 Definition of Acute Kidney Injury (AKI) | 68 |
| | | | 7.3.1.7 Renal Replacement Therapy | |
| | | | 7.3.1.8 Treatment-emergent HLA antibodies | |
| | | | 7.3.1.9 Definition of Culture Proven Sepsis/Septic Shock | |
| | | | | 09 |
| | | | 7.3.1.11 Suspected Hemolytic and Serologic Transfusion Reactions after Enrollment and Transfusion with Study | |
| | | | RBC Components | 72 |
| | | | 7.3.1.12 Abnormal Test Findings | |
| | | 7.3.2 | Methods and Timing of Safety Parameters | |
| | 7.4 | | ting Period | |
| | | | ding and Reporting Adverse Events | |
| | 7.5 | 7.5.1 | Assessing Severity of an Adverse Event | |
| | | 7.5.1 | Assessing Seriousness of an Adverse Event | |
| | | 7.5.2 | | |
| | | 7.5.3<br>7.5.4 | Assessing Causality of an Adverse Event | |
| | | | Assessing Relationship to the INTERCEPT Blood System Device | |
| | | 7.5.5 | Reporting Requirements | |
| | 7.0 | 7.5.6 | Reporting Device Malfunctions | |
| | 7.0 | Data a | and Safety Monitoring Board (DSMB) and Interim AnalysIs | ð2 |

| 8 | STA | ATISTICS | 83 |
|---|---|---|---|
| | 8.1 | Statistical Methods | 83 |
| | | 8.1.1 Efficacy Analysis | 83 |
| | | 8.1.2 Safety Analyses | 83 |
| | | 8.1.3 Subgroup Analyses | 83 |
| | 8.2 | Determination of Sample Size | 84 |
| | 8.3 | Criteria for Termination of the Study | 84 |
| | 8.4 | Handling of Dropouts or Missing Data | 84 |
| | 8.5 | Deviations from the Statistical Plan | 84 |
| | 8.6 | Selection of Subjects to be Analyzed | 84 |
| 9 | DIF | RECT ACCESS TO SOURCE DATA/DOCUMENTS | 86 |
| 10 | QU | ALITY CONTROL AND QUALITY ASSURANCE | 87 |
| | | Monitoring | |
| | 10.2 | 2 Investigational Product | 87 |
| 11 | ET | HICS | 88 |
| | 11.1 | Conduct of the Trial | 88 |
| | | 2 Patient Information and Consent | |
| | 11.3 | 3 Institutional Review Board (IRB)/Ethics Committee (EC) | 88 |
| | | 4 Confidentiality | |
| 12 | DA | TA HANDLING AND RECORD KEEPING | 90 |
| | 12.1 | Case Report Forms | 90 |
| | 12.2 | 2 Record Retention | 90 |
| 13 | | TERATURE REFERENCES | |
| 14 | | PENDICES | |
| • | 111 | | •••• |
| APF | END | IX 1: Transfusion Risk Understanding Scoring Tool (TRUST) | 95 |
| | | IX 2: Evaluation of Reactivity with INTERCEPT RBCs | |
| | | IX 3 CDC National Healthcare Safety Network Biovigilance Component | |
| | | Hemovigilance Module Surveillance Protocol v2.5.2 | 109 |
| APF | PEND | IX 4: Common Terminology Criteria for Adverse Events (CTCAE) | |
| | | Version 5.0 Published: November 27, 2017 | 140 |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

## LIST OF TABLES

| Table 2.1 Summary of Clinical Studies with INTERCEPT Blood System for RBCs | |
|---|---|
| Current Process | 24 |
| Table 2.2 Reanalysis of Cerus Studies RBC 3A01 and CLI 00070 Using Renal | |
| Impairment Based on Change in Serum Creatinine Levels within 48 hours | |
| of Cardiac Surgery | 31 |
| Table 4.1 Stopping Rules for INTERCEPT RBC-specific antibodies | 43 |
| Table 7.1a – Screening/Randomization | 57 |
| Table 7.1b - Baseline (Pre-Surgery) | 58 |
| Table 7.1c – Acute Transfusion Support Period | |
| Table 7.1d – Post-Operative Period | 61 |
| Table 7.1e - Follow-up Visits (Day 28±3, 30, and 75±15) | 62 |
| Table 7.2: Hematology and Chemistry Testing- Required (R) results and Where | |
| Available (WA) <sup>a</sup> results | 63 |
| Table 7.3 Some Differential Diagnoses of Hemolytic Transfusion Reactions | 71 |
| Table 7.4 Severity Assessment of Adverse Events | 79 |
| Table 7.5 Relationship between Investigational Product and Adverse Events | 80 |
| Table 7.6 Cerus Product Safety Contact Information | 81 |
| LIST OF FIGURES | |
| Figure 4.1 Study Design Schematic | 36 |
| Figure 4.2 Study Flowchart | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

## 1 LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| AABB | American Association of Blood Banks |
|---|---|
| ADL | Activities of Daily Living |
| AE | Adverse Event |
| AHG | Anti-human Globulin |
| AHTR | Acute Hemolytic Transfusion Reaction |
| AKI | Acute Kidney Injury |
| AKIN | Acute Kidney Injury Network |
| ALP | Alkaline Phosphatase |
| ALT | Alanine Transaminase |
| ANOVA | Analysis of Variance |
| ANCOVA | Analysis of Covariance |
| AS | Additive Solution |
| AST | Aspartate Aminotransferase |
| ATP | Adenosine Triphosphate |
| ATR | Acute Transfusion Reaction |
| BP | Blood Pressure |
| bpm | Beats per minute |
| BUN | Blood Urea Nitrogen |
| BVDV | Bovine Viral Diarrhea Virus |
| С | Celsius |
| CABG | Coronary Artery Bypass Graft |
| CBC | Complete Blood Count |
| CDC | Centers for Disease Control and Prevention |
| CFR | Code of Federal Regulations |
| CFU | Colony Forming Units |
| CI | Confidence Interval |
| CLIA | Clinical Laboratory Improvement Amendments |
| СМН | Cochran-Mantel-Haenszel |
| CMV | Cytomegalovirus |
| СРВ | Cardiopulmonary Bypass |
| CP2D | Citrate Phosphate Double Dextrose |
| CPD | Citrate Phosphate Dextrose |
| CRF | Case Report Form |
| CRO | Contract Research Organization |
| CSF | Cerebrospinal Fluid |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CVP | Central Venous Pressure |
| DAT | Direct Antiglobulin Test. Also referred to as the direct Coombs test. |

| ъ . | |
|---|---|
| Device<br>Malfunction | The failure of a medical device to function according to its requirements. |
| DHBV | Duck Hepatitis B Virus |
| DHTR | Delayed Hemolytic Transfusion Reaction |
| dL | Deciliter Deciliter |
| DNA | Deoxyribonucleic Acid |
| ds DNA | Double stranded DNA |
| 2,3-DPG | 2,3-Diphosphoglycerate |
| DSMB | Data and Safety Monitoring Board |
| DSTR | Delayed Serological Transfusion Reaction |
| EC | Ethics Committee |
| ECMO | Extracorporeal Membrane Oxygenation |
| eCRF | Electronic Case Report Form |
| EDC | Electronic Data Capture |
| EIA | Emerging Infectious Agents |
| EKG | Electrocardiogram |
| EOS | End of Study |
| F | Fahrenheit |
| FDA | Food and Drug Administration |
| FNHTR | Febrile Non-Hemolytic Transfusion Reaction |
| g | Gram |
| GCP | Good Clinical Practice |
| GSH | Glutathione |
| HA | Hemolytic anemia |
| Hb | Hemoglobin |
| HBV | Hepatitis B Virus |
| Hct | Hematocrit |
| HCV | Hepatitis C Virus |
| HELLP | A syndrome occurring in pregnancy. A combination of the breakdown of red blood cells (hemolysis: the H in the acronym, elevated liver enzymes (EL), and low platelet count (LP). |
| HIV | Human Immunodeficiency Virus |
| HLA | Human Leukocyte Antigen |
| HR | Heart rate |
| HSV | Herpes Simplex Virus |
| HTR | Hemolytic Transfusion Reaction |
| IABP | Intra-aortic Balloon Pump |
| IAT | Indirect Antiglobulin Test. Also referred to as the Indirect Coombs Test. |
| IBS | INTERCEPT Blood System (abbreviation used in preceding protocol versions) |
| ICF | Informed Consent Form |

| ICH | International Council on Harmonization |
|---|---|
| ICU | Intensive Care Unit |
| IEC | |
| | Independent Ethics Committee |
| IgA | Immunoglobulin A |
| IgG | Immunoglobulin G |
| IgM | Immunoglobulin M |
| INTERCEPT<br>Blood System for | Name of the current Cerus' Investigational device |
| RBCs | |
| INTERCEPT | Red blood cell component (s) that have been processed/treated with the |
| RBC(s) | INTERCEPT Blood System for Red Blood Cells (also known as |
| . , | INTERCEPT RBCs or S-303 (treated) RBCs) |
| IP | Investigational product |
| IRB | Institutional Review Board |
| IWRS | Interactive Web Response System |
| KDIGO | Kidney Disease Improving Global Outcomes |
| kg | Kilogram |
| LDH | Lactate Dehydrogenase |
| L | Liter |
| LVAD | Left Ventricular Assist Device |
| mg | milligram |
| mITT | Modified Intent-to-Treat |
| mL | Milliliter |
| mM | Millimole |
| μΜ | Micromole |
| MI | Myocardial Infarction |
| mm <sup>3</sup> | Cubic millimeter |
| mm Hg | Millimeter of mercury |
| N | Number |
| NBG | Normalized Background |
| NCI | National Cancer Institute |
| PaCO <sub>2</sub> | Partial pressure of carbon dioxide |
| PFU | Plaque Forming Unit |
| PP | Per Protocol |
| RBC | Red Blood Cell |
| ReCePI | Red Cell Pathogen Inactivation (acronym) |
| RIFLE | Risk, Injury, Failure, Loss of kidney function, and End-stage kidney |
| | disease classification |
| RNA | Ribonucleic Acid |
| ROS | Reactive oxygen species |
| RR | Respiratory rate |

| RRT | Renal Replacement Therapy |
|---|---|
| ssRNA | Single Stranded Ribonucleic Acid |
| S-300 | (N-(9-Acridinyl)-β-alanine). The primary decomposition product of S-303. |
| S-303 | Amustaline. [N,N-bis (2-chloroethyl)]-2-aminoethyl 3-[(acridin-9-yl) amino] propionate free base. May also refer to S-303 in solution (dissolved S-303 2HCl). |
| S-303•2HCl | S-303 in the salt form used for treating RBC components. |
| SAG- M | SAG-Mannitol: an RBC additive solution |
| SAE | Serious Adverse Event |
| SD | Standard deviation |
| SCD | Sickle Cell Disease |
| sCr | Serum creatinine |
| SIRS | Systemic Inflammatory Response Syndrome |
| SOC | System Organ Class (MedDRA) |
| SOP | Standard Operating Procedure |
| TACO | Transfusion Associated Circulatory Overload |
| TA-GVHD | Transfusion Associated Graft versus Host Disease |
| TEAE | Treatment Emergent Adverse Event |
| TR | Transfusion Reaction |
| TRALI | Transfusion Related Acute Lung Injury |
| TRS | Transfusion Related Sepsis |
| TRUST | Transfusion Risk Understanding Screening Tool |
| TTI | Transfusion-Transmitted Infection |
| UADE | Unanticipated Adverse Device Effect |
| ULN | Upper Limit of Normal |
| UO | Urinary output |
| U.S. | United States |
| USP | US Pharmacopeia |
| VSV | Vesicular Stomatitis Virus |
| WBC | White Blood Cells |
| WNV | West Nile Virus |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

## 2 BACKGROUND INFORMATION

## 2.1 GENERAL

Red blood cell (RBC) transfusion is a critical supportive therapy for healthcare. Patients and physicians assume, when required, blood transfusion will be available and safe. However, serious transfusion-transmitted infections (TTI) caused by viruses, bacteria and protozoa (Stramer 2009, MacLennan 2006); and fatal transfusion complications such as transfusion-associated graft-versus-host disease (TA-GVHD) still pose a threat to transfusion recipients (Kopolovic 2015). Currently, prevention of TTI includes pre-donation evaluation and selection of low-risk donors, followed by serologic and/or nucleic acid testing for selected known infectious pathogens.

The advent of testing has greatly reduced TTI from blood products, particularly viral disease, and sepsis associated with the transfusion of bacterially contaminated red cell blood components is generally regarded as a very rare event. However, from 1976 through September 1998, 26 fatalities thought to be secondary to contaminated whole blood or red cells were reported to the U.S. FDA (Lee 1999). The majority of deaths reported to the FDA involved Yersinia enterocolitica. The highest reported incidence of Y. enterocolitica contamination was reported in New Zealand, with an incidence rate of 1 in 65,000 and a fatality rate of 1 in 104,000 red cell units transfused (Theakston et al. 1997). Unrecognized cases, underreporting, and regional variation may account for observed differences in this incidence. Interestingly, passive reporting studies of bacterially contaminated red cells from the United States, France, and the United Kingdom that caused symptoms of infection show a relative paucity of Y. enterocolitica cases (Perez et al. 2001, Kuehnert et al. 2001, Serious Hazards of Transfusion report for 2000-2001). Of the reported deaths, one was due to a coagulase-negative Staphylococcus strain and seven were due to a variety of gram-negative organisms (including Serratia liquefaciens in three cases). These organisms are all capable of growth at refrigerated temperatures (1° to 6°C). Sepsis associated with the transfusion of red cells contaminated with gram-negative bacteria is typically severe and rapid in onset (Brecher and Hay 2005). Patients frequently develop high fever (temperatures as high as 109°F have been observed) and chills during or immediately following transfusion. From 1987 to February 1996, 20 recipients of Y. enterocolitica red cells were reported to the Centers for Disease Control (Cookson et al, 1996). Twelve of the 20 recipients died, and the median time to death was only 25 hours. Of the seven who developed disseminated intravascular coagulopathy, six died.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

Prospective bacterial cultures of whole blood or red cells, however, have shown a much higher incidence of bacterial contamination (Damgaard et al 2015). The organisms commonly cultured are Staphylococcus sp. or Propionibacterium sp.; those strains that have been reported to be isolated in association with adverse events linked to the transfusion of contaminated red cell concentrates include Pseudomonas sp., S. marcescens, Enterobacter sp., Klebsiella sp., S. epidermidis and B. cereus (Siblini et al 2004).

Newly-emerging infectious agents also remain important risks to blood safety. Estimates of per-unit and per-patient aggregate infectious risks for conventional RBCs, including known and potential emerging infectious agents (EIA, modeled based on chikungunya and dengue viruses) were calculated by Kleinman and Stassinopoulos (2015). Minimum and maximum per-unit risks were calculated as 0.0003% (1/323,000) and 0.12% (1/831), respectively. The minimum estimate is for known lower-risk pathogens while the maximal estimate also includes an EIA and endemic area Babesia sp. risk. For patients with hemoglobinopathies who receive repeated RBC transfusions such as sickle cell disease (SCD), at the minimum risk level it is estimated that approximately 1/450 (0.22%) of patients will acquire an infection during their entire course of transfusion therapy (approximately 30-50 years); at the maximum risk levels, infections risk increases to 43-45% for patients with hemoglobinopathies, or almost 1 in every 2 patients (Kleinman and Stassinopoulos 2015).

Leukoreduced RBC concentrates contain <5 x10<sup>6</sup> white blood cells (WBC) that may induce TA-GVHD and/or alloimmunization to human leukocyte antigen (HLA) antigens. Gamma irradiation can effectively prevent TA-GVHD in transfusion recipients. However, almost half the cases of TA-GVHD occur in patients in which their treating physicians failed to identify risk using current guidelines for blood irradiation, leading to substantial morbidity and mortality (Kopolovic 2015). Moreover, irradiation adversely affects post-transfusion RBC recovery (Dumont 2008) and is associated with raised extracellular potassium levels in the transfused concentrates.

To proactively address the risk of TTIs and TA-GVHD, Cerus has developed pathogen and leukocyte inactivation technology systems (INTERCEPT Blood System<sup>TM</sup>) for platelet and plasma components and is currently developing a system for RBC concentrates. These systems use nucleic acid-targeted compounds that intercalate into, and upon activation, covalently bind to nucleic acids of viruses, bacteria, parasites and leukocytes that may contaminate blood components, and form irreversible adducts and crosslinks thus preventing replication and TTI. This

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

process does not depend on or generate reactive oxygen species (ROS) which can damage cells and proteins. RBCs do not require nucleic acid for therapeutic function and thus retain therapeutic efficacy after pathogen inactivation treatment. INTERCEPT treated RBC (INTERCEPT RBCs) components should not require gamma irradiation because the treatment process inactivates donor white blood cells with a high safety margin (Castro et al. 2016). It is also possible that INTERCEPT treatment may interfere with antigen presentation by donor leukocytes, thereby reducing the incidence of HLA alloimmunization.

Conventional leukoreduced RBC concentrates include approximately 20-40 mL of residual plasma that contains serum proteins and immunoglobulins; these are implicated in allergic TRs and Transfusion Related Acute Lung Injury (TRALI). The INTERCEPT RBC process includes a terminal washing step that reduces the concentration of plasma proteins and may reduce the incidence of these reactions.

The INTERCEPT Blood System for RBCs inactivates a variety of bacteria, viruses and protozoa. The organisms evaluated to date include examples representing a range of different characteristics, such as enveloped (HIV and DHBV) and non-enveloped (Bluetongue virus), RNA genome (HIV and BVDV) and DNA genome (DHBV), and single stranded (HIV) and double stranded (DHBV) genomes. The bacteria evaluated represent Gram negative bacilli (Yersinia sp., Serratia sp., *E. coli*, Salmonella sp. and Pseudomonas sp.) and Gram positive cocci (*S. epidermidis* and *S. aureus*) that are significant especially for RBC transfusion. The protozoan parasites evaluated to date are *Plasmodium falciparum* and *Babesia microti*. INTERCEPT RBCs have demonstrated adequate viability in terms of in vivo recovery and lifespan for transfusion (Cancelas 2015), and a recently completed Phase 3 clinical study (CLI 00076) in cardiovascular surgery patients conducted in Europe has demonstrated that INTERCEPT RBCs possess in vitro characteristics comparable to untreated RBCs with a comparable safety profile (Brixner 2015, Rico 2015).

The proposed phase 3 study in patients undergoing complex cardiac surgery is intended to demonstrate that INTERCEPT RBCs are non-inferior to conventional RBCs with regard to clinical safety and clinical efficacy for transfusion support of acute anemia during surgery with potential hemodynamic instability. The study is designed to support the licensure of the INTERCEPT Blood System for Red Blood Cells.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

## 2.2 NAME AND DESCRIPTION OF THE INVESTIGATIONAL PRODUCT

The INTERCEPT Blood System for RBCs is an investigational medical device used to prepare pathogen and leukocyte inactivated RBC components for transfusion.

## 2.2.1 Description of Investigational Product

The investigational device is the INTERCEPT Blood System for Red Blood Cells. The pathogen reduction process begins with a unit of RBCs derived from whole blood that is separated according to local regulations and standard operating procedures at the Blood Centers. RBCs are suspended in additive solution-5 (AS-5). Leukocyte-reduction of whole blood or RBCs will be performed per manufacturer's instructions. The INTERCEPT Blood System process is performed on a single unit of leukoreduced RBC in AS-5.

For a detailed description of the investigational product, please refer to the Investigator's Brochure.

## 2.3 SUMMARY OF NONCLINICAL AND CLINICAL STUDIES

The INTERCEPT treatment process uses amustaline and glutathione together with a processing solution in a single-use disposable set to produce pathogen inactivated RBCs in SAG-M additive solution. Cerus' pre-clinical and clinical development program has evaluated the efficacy of amustaline for pathogen inactivation and safety profiles of treated RBCs and breakdown products with regard to systemic toxicity, genotoxicity and carcinogenicity in accordance with International Council on Harmonization (ICH) standards for RBCs development of pharmaceuticals. These data are presented in detail in the Investigator's Brochure.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

## **2.3.1** Safety

No physiologically relevant toxicity using INTERCEPT RBCs at doses higher than planned for this trial was observed in pre-clinical studies. Additional information about the toxicological evaluations of the treatment system is provided in detail in the Investigator's Brochure.

## 2.3.2 Immunogenicity

The mechanism of action of S-303 can also lead to reactions with macromolecules other than nucleic acids in the blood components, such as constituents of the red cell membrane. In early studies of the pathogen inactivation process for RBCs (referred to as "Original process") there was evidence of antibody formation directed against INTERCEPT RBCs (also referred to as S-303-specific RBC antibodies) in two patients participating in a chronic RBC transfusion study. In order to minimize these non-specific and unwanted reactions with RBC surface molecules, an increased level of the quencher, glutathione (GSH), has been included in the current, pathogen inactivation process (referred to as "Current process").

Additional information regarding the potential for immunogenicity, and the studies that have been conducted is provided in the Investigator's Brochure.

## 2.3.3 Clinical Studies

Four clinical studies have been completed with the current process of the INTERCEPT Blood System for RBCs. The studies are summarized in **Table 2.1** below and additional detail is provided in the Investigator's Brochure.

Table 2.1 Summary of Clinical Studies with INTERCEPT Blood System for RBCs Current Process

| Study ID | Number<br>of Study<br>Centers | Design | Study & Ctrl<br>Drugs (Dose,<br>route &<br>regimen) | Study<br>Objective | # subjects<br>(entered,<br>completed) | Diagnosis | Primary<br>Endpoint(s) | Main Findings |
|---|---|---|---|---|---|---|---|---|
| CLI00062<br>(RBC08001) | 2 | Randomized,<br>single blinded,<br>controlled, 2<br>period, cross-<br>over | Single<br>transfusion of<br>5-15 mL of <sup>51</sup> Cr-<br>labeled Test<br>(S-303) or<br>Control RBCs<br>(35 day storage),<br>intravenous | Recovery of<br>IBS treated<br>autologous<br>RBCs; safety<br>and<br>tolerability | 26/26 | Healthy adult<br>subjects | 24 hour recovery<br>and life span of 35<br>day old autologous<br>RBCs | IBS-treated RBCs met FDA recommended criteria for 24 hour recovery with no significant difference between IBS-treated and control RBC Survival was significantly different between Test (32.8 days) and Control (39.5 days) but T50 of Test was within published reference range (28-35 days) No physiologically meaningful differences at end of storage between Test and Control RBC |
| CLI00073 | | Single-blinded,<br>randomized<br>crossover | Single<br>transfusion<br>µ10-30 mL of<br>51Cr-labeled<br>Test (S-303) or<br>Control RBCs<br>(35 day storage),<br>intravenous | Compare<br>survival and<br>recovery of<br>autologous<br>S 303 RBCs<br>to<br>conventional<br>RBCs | 42 enrolled/<br>26 completed | Healthy<br>subjects | 24 hour post-<br>infusion dual label<br>recovery of<br>autologous RBCs<br>stored for 35 days | The 24-hour post-transfusion recovery (both dual- and single-label) of autologous IBS RBCs following infusion after 35-days of storage met all the FDA criteria for the evaluation of RBC products. No immunologic reactivity developed to Test RBC. |
| CLI00070 | 3 | Randomized,<br>controlled,<br>double blinded,<br>parallel | IBS treated or<br>untreated RBC<br>transfusions for<br>up to 7 days<br>starting on day<br>of surgery; dose<br>and frequency<br>per treating<br>physician | In vitro characterizati on of IBS RBCs relative to EU criteria for RBC for transfusion Obtain clinical data to support design of add'l studies | 87<br>randomized;<br>51 treated<br>(25Test,<br>26Control) | Patients undergoing complex cardiac surgery with high likelihood of requiring RBC transfusion | Primary in vitro endpoint Hb content/unit Primary clinical endpoint = safety Exploratory endpoints indicative of tissue oxygenation include renal or | IBS RBC demonstrated equivalence to untreated RBC regarding hemoglobin content; the proportion of IBS RBCs satisfying the EDQM guidelines was higher than for conventional RBCs. The incidence of renal insufficiency was 15.7% (Test 5, Control 3, p=0.41). The incidence of hepatic insufficiency was 2% (Test 1, Control 0, p=0.37). There was no statistical difference between Test and Control groups for the |

| Study ID | Number<br>of Study<br>Centers | Design | Study & Ctrl<br>Drugs (Dose,<br>route &<br>regimen) | Study<br>Objective | # subjects<br>(entered,<br>completed) | Diagnosis | Primary<br>Endpoint(s) | Main Findings |
|---|---|---|---|---|---|---|---|---|
| | | | | to support<br>registration of<br>IBS for RBC | | | hepatic<br>insufficiency and<br>6MWT | assessments of the 6MWT at the time of first ambulation post-surgery and at day 13 or discharge. |
| | | | | | | | | No statistical differences in the overall incidence of AE rates, or in possibly related AEs between Test and Control, with similar distribution of SAEs between groups. The events observed were those expected in this population. |
| CLI 00076 | 3 | Randomized,<br>controlled,<br>double blinded,<br>two-period,<br>crossover, non-<br>inferiority | Six transfusion episodes of Test (INTERCEPT) or Control RBC; each treatment period to include 2 wash-in episodes and 4 study transfusion episodes; subjects will be transfused to maintain the same target hemoglobin level specified by treating physician in each study period | Evaluate the efficacy and safety of INTERCEPT RBCs in subjects who require chronic transfusion support due to thalassemia major | 86<br>randomized,<br>81 treated | Subjects with thalassemia major who require chronic transfusion of RBC components | Hgb consumption during each efficacy evaluation period (episodes 4 to 6) measured as the Hgb mass transfused per subject adjusted for episode-specific body weight and duration (Hgb g/kg body weight/day). Incidence of a treatment-emergent antibody with confirmed specificity to INTERCEPT treated RBCs associated with clinically significant hemolysis | The non-inferiority of INTERCEPT RBC components for the primary efficacy endpoint was robustly achieved consistently for both the ITT and PP analysis groups. No treatment emergent antibodies to INTERCEPT RBC were detected. Adverse events were equally distributed between Test and Control periods. |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

## 2.4 SUMMARY OF POTENTIAL RISKS

The potential risks of this study include those adverse reactions that are recognized to occur following any transfusion of RBC components and could be anticipated to occur with either control or INTERCEPT-treated components including, but not limited to, delayed serologic transfusion reactions (DSTRs), acute hemolytic transfusion reactions (AHTRs), delayed hemolytic transfusion reactions (DHTRs), febrile non-hemolytic transfusion reactions (FNHTRs), allergic (urticarial) reactions, anaphylaxis, transfusion-related acute lung injury (TRALI), transfusion-associated circulatory overload (TACO), transfusion-related sepsis (TRS), or transfer of an infectious agent via transfusion/transfusion transmitted infection (TTI), respectively, transfusion- associated graft-vs-host disease (TA-GVHD), and allo-immunization to RBC and HLA antigens.

The development of antibodies to INTERCEPT RBCs, or to neoantigens formed as a result of acridine binding to red cells, could occur as a result of transfusion with INTERCEPT RBCs. Acridine-specific antibodies were observed in an early and current ongoing blinded studies (as described in the Investigator's Brochure) and many could be neutralized with acridine in solution, thereby defining specificity for this moiety. The occurrence of these antibodies was not associated with any clinical events or observations. The Current process has been optimized to decrease the likelihood of this event.

A screening study was performed to evaluate the prevalence of natural antibodies with specificity for INTERCEPT RBCs (SUD 00742). Five plasma samples from 998 subjects requiring chronic transfusion support for anemia and 12 plasma samples from 10,721 hospital subjects demonstrated low titer cross-reactions with INTERCEPT RBCs. The cumulative prevalence of cross-reactive antibodies to INTERCEPT RBCs was 0.15%. Each of the antibodies identified was characterized and none were found to be IgG<sub>1</sub> or IgG<sub>3</sub> subclass, the antibody subclasses most associated with physiologic hemolytic activity. The majority demonstrated specificity for acridine.

Several instances of treatment emergent antibodies with specificity for INTERCEPT RBCs were reported during the ongoing Phase III clinical investigations. In each event, the antibodies were shown to be non-clinically significant without evidence of patient harm. These studies remain blinded and it is not known whether the patients received Test of Control RBCs.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

Natural antibodies to INTERCEPT RBCs are expected to occur in ongoing clinical trials. Risk mitigation is in place to protect patients and further evaluate clinical significance. All study subjects are screened before enrollment for INTERCEPT RBC-specific antibodies and subjects with natural cross-reactive antibodies are excluded. Subjects are regularly screened during the study including at approximately 75 days after the last study RBC transfusion in all ongoing clinical trials. Subjects with treatment emergent antibodies are withdrawn from receiving study RBC and are fully evaluated for evidence of hemolysis. Stopping rules are in place related to the occurrence of delayed serological and hemolytic TRs associated with treatment emergent antibodies to INTERCEPT RBCs.

Additional risks associated with Control components, that INTERCEPT treatment is designed to reduce, include risk of infectious contamination by viral or protozoan agents, such as HIV, HCV, HBV, malaria, and emerging viruses such as Zika, Dengue and Chikungunya.

The risk of bacterial contamination is considered to be negligible with INTERCEPT RBC components and, although it has not been measured directly, is expected to be less than the risk of bacterial contamination with conventional RBC components, thus providing a potential benefit of receiving INTERCEPT-treated components.

Finally, human error, clerical error and transfusion of RBC to the wrong patient remain risks of red cell transfusion.

## 2.5 DESCRIPTION OF AND RATIONALE FOR TREATMENT

Patients undergoing cardiac surgery are an appropriate study population because (i) these patients commonly require multiple RBC transfusions for support of acute anemia and might be expected to manifest complications ascribed to exposure to allogeneic blood, (ii) cardiac surgery patients comprise a large group of recipients with acute anemia requiring RBC transfusion and on a national basis account for a significant proportion of blood component utilization, and (iii) following cardiopulmonary bypass surgery, patients are in a pro-inflammatory state which might make them particularly vulnerable to adverse consequences of RBC transfusion, especially decreased tissue and organ oxygenation. While other types of surgical patients receive blood for acute anemia, they are either difficult to study in a clinical trial setting (e.g., trauma patients) or they may have high rates of autologous blood transfusion use (e.g., orthopedic patients). Cardiac surgery is also one setting where a liberal RBC transfusion policy has been documented to increase overall survival, suggesting an important role in ensuring tissue oxygenation (Murphy 2015).

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

The acute nature of the transfusion support in the setting of surgical blood loss with many confounding variables unrelated to the properties of RBC components limits the utility of measuring post-transfusion hemoglobin increments, and other direct measures of therapeutic benefit (Weiskopf 1998). In addition, evaluation of RBC component therapeutic efficacy is challenging because no single endpoint adequately reflects RBC transfusion efficacy in acute anemia. However, a reasonable approach is to assess a single key organ system such as renal as the primary endpoint. Accordingly, the primary efficacy measure in the proposed study is renal impairment defined by changes in serum creatinine.

Lassnigg et al. (Lassnigg 2004, Lassnigg 2008) found that measuring repeat sCr concentrations within 48 hours of cardiothoracic surgery and determining the ΔsCr from pre-surgery baseline concentrations was the most effective discrimination method to find patients at risk for adverse postoperative outcomes, including mortality by Day 30 post-surgery. In independent studies at two different European institutions that incorporated all cardiac surgery patients who survived at least 48 hours post-surgery, they found that  $\Delta sCr$  concentrations declined in the majority of patients and was associated with the lowest mortality (1.8%). Minimal increases [0-0.5 mg/dL were associated with a more than doubled mortality in both centers (5%/6%). Used as a sole criterion, ΔsCr within 48 hours of surgery was more sensitive than the RIFLE (Mehta 2007) and AKIN (Bellomo 2004) definitions of Acute Kidney Injury (AKI) as a correlate of poor outcomes. The most important findings of these studies were that 1) even a small absolute increase in sCr in the postcardiac surgery setting confers an adverse prognosis and increases the risk of death; 2) a window of 48 hours following cardiac surgery was able to classify the risk groups; and 3) ease of use and early prediction ability of absolute sCr changes alone challenge the RIFLE and AKIN classifications in these patients.

Historically acute kidney injury (AKI) is known to complicate recovery from cardiac surgery in up to 30% of patients, and places patients at a 5-fold increased risk of death during hospitalization (O'Neal et al. 2016).

AKI has been validated as a predictor of adverse outcomes after cardiac surgery based on sCr assessment alone. Many analyses do not incorporate urinary output (UO) as a component of the AKI measure, especially in cardiac surgery patients. For example:

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

- Hobson et al. (Hobson 2009) describe 2973 cardiac surgery patients between 1992 and 2002 and define AKI as a ≥50% increase in sCr from pre-surgery baseline. Survival was worse among patients with AKI and was proportional to its severity, with an adjusted hazard ratio of 1.23 (95% CI 1.06 to 1.42).
- Loef et al. (Loef 2005) describe an association of in-hospital and long term mortality with post-operative sCr levels only, in 843 cardiac surgery patients in 1991 (hazard ratio of death 1.83;95% confidence interval 1.38 to 3.20).
- More recently, Zhou et al. (Zhou 2016) confirmed the association of AKI based only on sCr criteria, with higher mortality and longer length of stay in 1036 critically ill ICU patients.

AKI that requires renal replacement therapy occurs in 2–5 % of patients following cardiac surgery and is associated with 50 % mortality (O'Neal 2016). For those who recover from renal replacement therapy or even mild AKI, progression to chronic kidney disease in the ensuing months and years is more likely than for those who do not develop AKI. Renal ischemia, reperfusion, inflammation, hemolysis, oxidative stress, cholesterol emboli, and toxins are known to contribute to the development and progression of AKI. Transfusion with RBC may prevent AKI by ensuring tissue oxygenation during and after surgery, but is also hypothesized to exacerbate AKI by the release of non-transferrin bound iron, promotion of a pro-inflammatory state, impairment of tissue oxygen delivery, and exacerbation of tissue oxidative stress (Karkouti 2012). A comparison of AKI incidence using conventional and INTERCEPT-treated RBC in cardiac surgery therefore offers a sensitive predictive measure of the equivalence of long-term outcomes following acute RBC transfusion for both benefits and potential harms.

Lassnigg et al. (Lassnigg 2004, Lassnigg 2008) found an association of small changes in serum creatinine ( $\Delta$ sCr) in the first 48 hours after surgery with mortality by day 30, and an independent association of transfusion with adverse outcomes. In the ReCePI study we will enroll cardiac patients that are likely to require RBC transfusions using the Transfusion Risk Understanding Screening Tool (TRUST) Score (Alghamdi 2006), and these patients are more likely to suffer post-surgery renal impairment than patients who are less likely to require transfusion.

Cerus has completed two studies in cardiac surgery in patient populations similar to that proposed in ReCePI, and these data have been submitted to the FDA: RBC3A01, "S-303 Treated Red Blood Cell Use in Patients Requiring Acute Transfusion Support," (Benjamin et al. 2005) (submitted to the FDA on March 30, 2005 under IDE 7750/91) and CLI 00070, "A Randomized Controlled Double-Blind Phase 3

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

Study to Assess Characteristics of S-303 Treated RBC Components and Evaluate Safety and Efficacy in Patients Requiring Transfusion Support of Acute Anemia," (submitted to the FDA on 30 September 2016 [Reference IDE 13803/65]).

The above studies inform the selection of the proportion of patients that are likely to meet the criterion of raised  $\Delta sCr$  within 48 hours post the completion of cardiac surgery. A summary table (**Table 2.2**) provides the data from our analysis of studies RBC 3A01 and CLI 00070 that shows that the proportions of Control patients had  $\Delta sCr$  values within 48 hours of surgery completion as follows:  $\geq 0.1 mg/dL = 55\%$ ;  $\geq 0.2 mg/dL = 45\%$ ; and  $\geq 0.3 mg/dL = 30\%$ .

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

Table 2.2 Reanalysis of Cerus Studies RBC 3A01 and CLI 00070 Using Renal Impairment Based on Change in Serum Creatinine Levels within 48 hours of Cardiac Surgery

| | Valve | only | CABG Only | | Valve ar | nd CABG | All Patients | | |
|---|---|---|---|---|---|---|---|---|---|
| CLI 00070 | Test | Control | Test | Control | Test | Control | Test | Control | Total |
| | (N=10) | (N=8) | (N=12) | (N=13) | (N=3) | (N=5) | (N=25) | (N=26) | (N=51) |
| Cr Increase ≥0.1 mg/dL | 7 (70.0%) | 5 (62.5%) | 5 (41.7%) | 3 (23.1%) | 3 (100%) | 4 (80.0%) | 15 (60.0%) | 12 (46.2%) | 27 (52.9%) |
| Cr Increase ≥0.2 mg/dL | 6 (60.0%) | 3 (37.5%) | 2 (16.7%) | 3 (23.1%) | 3 (100%) | 4 (80.0%) | 11 (44.0%) | 10 (38.5%) | 21 (41.2%) |
| Cr Increase ≥0.3 mg/dL | 5 (50.0%) | 2 (25.0%) | 0 | 1 (7.7%) | 1 (33.3%) | 2 (40.0%) | 6 (24.0%) | 5 (19.2%) | 11 (21.6%) |

| | Valve | Only | CABG Only | | Valve ar | nd CABG | All Patients * | | |
|---|---|---|---|---|---|---|---|---|---|
| RBC 3A | Test | Control | Test | Control | Test | Control | Test | Control | Total |
| | (N=31) | (N=28) | (N=4) | (N=10) | (N=36) | (N=34) | (N=74) | (N=74) | (N=148) |
| Cr Increase ≥0.1 mg/dL | 16 (51.6%) | 14 (50.0%) | 3 (75.0%) | 6 (60.0%) | 24 (66.7%) | 21 (61.8%) | 45 (60.8%) | 43 (58.1%) | 88 (59.5%) |
| Cr Increase ≥0.2 mg/dL | 10 (32.3%) | 12 (42.9%) | 3 (75.0%) | 4 (40.0%) | 15 (41.7%) | 17 (50.0%) | 29 (39.2%) | 35 (47.3%) | 64 (43.2%) |
| Cr Increase ≥0.3 mg/dL | 7 (22.6%) | 10 (35.7%) | 2 (50.0%) | 3 (30.0%) | 10 (27.8%) | 10 (29.4%) | 20 (27.0%) | 25 (33.8%) | 45 (30.4%) |

| | Valve Only RBC 3A Test Control | | CABG Only | | | Valve ar | nd CABG | All Patients | | |
|---|---|---|---|---|---|---|---|---|---|---|
| CLI 00070 and RBC 3A | | | | Test | Control | Test | Control | Test | Control | Total |
| | (N=41) | (N=36) | | (N=16) | (N=23) | (N=39) | (N=39) | (N=99) | (N=100) | (N=199) |
| Cr Increase ≥0.1 mg/dL | 23 (56.1%) | 19 (52.8%) | | 8 (50.0%) | 9 (39.1%) | 27 (69.2%) | 25 (64.1%) | 60 (60.6%) | 55 (55.0%) | 115 (57.8%) |
| Cr Increase ≥0.2 mg/dL | 16 (39.0%) | 15 (41.7%) | | 5 (31.3%) | 7 (30.4%) | 18 (46.2%) | 21 (53.8%) | 40 (40.4%) | 45 (45.0%) | 85 (42.7%) |
| Cr Increase ≥0.3 mg/dL | 12 (29.3%) | 12 (33.3%) | | 2 (12.5%) | 4 (17.4%) | 11 (28.2%) | 12 (30.8%) | 26 (26.3%) | 30 (30.0%) | 56 (28.1%) |

#### Notes:

<sup>\*</sup> Included patients with "Other" type of surgery.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

Based on these data, Cerus proposed a non-inferiority design in ReCePI to rule out an increase of  $\Delta sCr \ge 0.3 \,\text{mg/dL}$  more than 50% from the Control rate with approximately 80% power and one-sided alpha of 2.5%. This is based on a Control rate of  $\Delta sCr \ge 0.3 \,\text{mg/dL}$  of 30%. At least 292 subjects will be randomized and transfused. Randomization (in 1:1 ratio for Test:Control) stratified by site, pre-existing renal impairment (stratum with either  $sCr \ge 1.2 \,\text{mg/dL}$  or  $sCr < 1.2 \,\text{mg/dL}$  at baseline), and cardiac surgery risk level (high or low risk stratum group 1 or 2, respectively) will be employed.

As per Lassnigg et al (2004 and 2008) patients who die within 48 hours of the end of surgery and have received at least one study transfusion will be included in the modified intent-to-treat (mITT) analysis but excluded from the per protocol analysis. Patients who have not received a study transfusion within 48 hours of surgery will be excluded from the analysis and replaced.

Additional endpoints will include mortality or the need for RRT (defined as hemodialysis or peritoneal dialysis) by Day 30 post-surgery; and AKI as defined by modified Kidney Disease Improving Global Outcomes (KDIGO) criteria. Any RRT that is provided prophylactically during surgery while patient is on a bypass machine does not meet this endpoint. The vital status and RRT assessment on Day 30 after surgery can be performed either from the medical records, from a phone call to the subject or family, or during the visit 28 +/- 3 days after the last study transfusion if the window covers 30 days after surgery time point.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

## 3 STUDY OBJECTIVES

The objective of this study is to evaluate the efficacy and safety of RBC transfusion for support of acute anemia in cardiovascular surgery patients based on the clinical outcome of renal impairment following transfusion of RBCs treated with the INTERCEPT Blood System for Red Blood Cells compared to patients transfused with conventional RBCs.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

## 4 INVESTIGATIONAL PLAN

## 4.1 ENDPOINTS

## 4.1.1 Primary Endpoints

The primary efficacy endpoint is the proportion of patients, who have received at least one study transfusion with a diagnosis of renal impairment defined as:

• Any raised sCr level, occurring after transfusion of a study RBC, of ≥0.3 mg/dL (or 26.5 μmol/L) from the pre-surgery baseline within 48±4 hours of the end of surgery.

If any subject meets this criterion before receiving a study transfusion, that particular event will not be included in the primary endpoint analysis. The treatment comparison for the primary efficacy endpoint will be assessed by a non-inferiority test (Test–Control) with a non-inferiority margin of 50% increase from the Control rate and two-sided 0.05 alpha level. Patients who receive a study transfusion but die within 48 hours after surgery will be included in the mITT analysis but excluded from the per protocol analysis.

The primary safety endpoints are:

- Proportion of patients with any treatment-emergent adverse events (TEAEs) possibly, probably or definitely related to study RBC transfusion through 28 days after the last study transfusion; and
- Proportion of patients with treatment-emergent antibodies with confirmed specificity to INTERCEPT RBCs by end of study (i.e., 75±15 days after the last study transfusion).

TEAEs by definition will comprise all untoward medical events occurring after the start of the first study RBC transfusion and during the study (i.e., adverse events, serious adverse events, unanticipated adverse device effects, TRs and within 28 days post last study RBC transfusion). The primary safety endpoint is focused on possibly, probably or definitely related adverse events to the study RBC transfusion, because these patients have many adverse events which are unrelated to study RBC transfusion.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

## 4.1.2 Secondary Endpoints

- <u>Efficacy</u>: Secondary efficacy endpoints include:
  - The proportion of patients with a diagnosis of stage I, II or III Acute Kidney Injury (KDIGO 2012) based on changes in sCr levels from pre-surgery baseline and the need for renal replacement therapy (RRT) post-surgery.
  - o Mortality or the need for RRT by 30 days post completion of surgery.

<u>Safety</u>: Assessment of additional safety parameters in post-surgical subjects transfused with INTERCEPT RBCs compared with subjects transfused with conventional RBCs, include:

- Treatment-emergent AEs through 28 days after the last study transfusion.
- Treatment-emergent SAEs through 28 days after the last study transfusion.
- Transfusion reactions (as defined by the CDC National Healthcare Safety Network [NHSN] Hemovigilance Module protocol) through 28 days after last study transfusion.
- Treatment-emergent immunization to RBC allo-antigens through  $28 \pm 3$  days after the last study transfusion.
- Treatment-emergent immunization to HLA allo-antigens through 28±3 days after the last study transfusion.
**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

#### 4.2 STUDY DESIGN

The study is a prospective, multicenter, randomized, double-blinded, active controlled, parallel-design, non-inferiority study. **Figure 4.1** shows the study design and **Figure 4.2** shows the clinical study flowchart.



Figure 4.1 Study Design Schematic

- (1) Primary efficacy endpoint  $\Delta sCr \ge 0.3$  mg/dL from baseline assessed within 48±4 hours of the end of surgery.
- (2) Secondary efficacy endpoint of mortality or need for RRT assessed on Day 30 post-surgery

Figure 4.2 Study Flowchart



#### 4.3 RANDOMIZATION AND BLINDING

Potentially eligible subjects will be screened and will be considered for randomization. If a subject is screened and receives a RBC transfusion prior to randomization, that subject will no longer be considered for randomization, and their participation in the study will end. Patients may be rescreened for eligibility closer to the time of surgery. An Interactive Web Response System (IWRS) will be used for electronic randomization of eligible patients. Following screening and prior to surgery (up to 7 days before surgery or day of surgery but before start of surgical procedure), the subject's eligibility status will be re-checked and entered in the eCRF. If eligible, the subject will be randomized with a 1:1 ratio for Test:Control within his/her randomization stratum. Randomization will be stratified by site, pre-existing renal impairment (sCr ≥1.2 mg/dL vs. < 1.2 mg/dL), and surgery group based on less (# 1-3 below) vs. more (#4-7 below) risk for renal complications (based on Mehta 2006 and expert opinion).

#### Less Risk

- 1. Single Vessel Coronary Artery Bypass Graft, first or repeat procedure
- 2. Multiple Coronary Artery Bypass Grafts, first or repeat procedure
- 3. Single Valve Repair or Replacement, first or repeat procedure

### More Risk

- 4. Multiple Valve Repair or Replacement, first or repeat procedure
- 5. Surgery involving both Coronary Artery Bypass Graft(s) and Valve Repair(s), first or repeat procedure
- 6. One or more of the following procedures, with or without Coronary Bypass Graft(s):
  - Left ventricular aneurysm repair,
  - Ventricular and/or atrial septal defect repairs,
  - Batista procedure (surgical ventricular remodeling),
  - Surgical ventricular restoration,
  - Congenital cardiac defect repair,
  - Aortic procedures,
- 7. Other complex cardiac surgery or thoracic aorta surgery procedures not listed above

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

Patients undergoing urgent or emergent cardiac surgery are eligible for the study, subject to institutional review board (IRB) approval of an appropriate informed consent process.

Randomized subjects who do not receive any study RBC transfusions within the first 48 hours after completion of surgery will be discontinued from study and replaced. Serum Creatinine up to and including  $48 \pm 4$  hours post-surgery will be collected.

Other post baseline laboratory parameters and Adverse events (AEs) will not be collected for non-transfused subjects. Vital status will be reported for randomized and non-transfused subjects at the time of discontinuation.

Only appropriate blood bank staff and unblinded delegates who monitor the production of the RBC components will be able to access the treatment arm assignment. Selected Blood Center staff will not be blinded due to their role required for collection, preparation, and releasing of Test and Control RBC components for transfusion to study subjects. An unblinded study monitor will review and verify source data collected at the blood banks. Operating room staff, surgical staff, ICU staff and others caring for participating patients, as well as the sponsor (and delegates) will be blinded to treatment assignment. Study RBC components will be labeled in a manner to maintain the blind. In order to protect the blind, on the day of planned transfusion, the final product (test and control) will be transferred by the Blood Bank unblinded personnel into a commercially available RBC storage container (Fenwal<sup>TM</sup> Transfer Pack<sup>TM</sup> Container – 600mL, product code 4R2023) using a sterile docking technique. Blood transferred into an ancillary container should be stored at 1°C to 6°C and transfused within 7 days of transfer.

#### 4.4 TREATMENT

Eligible subjects will be consented/provide assent and randomized to receive either INTERCEPT RBCs (Test) or conventional RBCs (Control) which will be transfused as needed starting from surgery at Day 0 until study post-operative Day 7, hospital discharge or death, whichever is first.

Treatment assessments will be divided into an acute transfusion support period starting on the day of surgery (Day 0) until post-operative Day 7, hospital discharge, or death, whichever is first, and a post-surgical follow-up visit ( $28\pm3$  days) after the last study transfusion to collect additional safety data. A sample for sCr determination will be taken at  $48\pm4$  hours after the end of surgery to document the primary efficacy endpoint. For non-transfused subjects, a blood sample for sCr will be drawn at  $48\pm4$  hours post-surgery. Patient status with regard to mortality and RRT on Day 30 post surgery will be documented. Anesthesia and surgical procedures will be performed according to the local standards of the institution.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

Study RBC components will be ordered and administered to study subjects by treating physicians, according to the local standards of care. Following the post-surgery 7-day acute transfusion support period, subjects will receive conventional RBC components if additional transfusions are needed, as indicated by their treating physician.

#### 4.4.1 Test Product

The INTERCEPT treatment will be performed on leukoreduced RBC components prepared from citrate phosphate dextrose (CPD) anticoagulated whole blood and suspended in AS-5 additive solution (input) within 24 hours of collection. The test component is allogeneic INTERCEPT treated RBC components prepared following the Instructions for Use for the INTECEPT Blood System for RBCs (SPC-EN 00581-AW) and stored in SAG-M at 1°C to 6°C for up to 35 days post-donation and administered intravenously. Test RBC components will be released to clinical inventory after review of the batch production record associated with the INTERCEPT treatment process.

# 4.4.2 Control (reference) Product

The Control transfusion component is CPD or citrate phosphate double dextrose (CP2D) anticoagulated whole blood derived conventional leukoreduced RBC components suspended in an FDA approved additive solution (e.g., AS-1, AS-3 or AS-5) and stored at 1°C to 6°C for up to 35 days post-donation and administered intravenously. The Control RBC components will be handled and labeled in a manner to maintain blinding. Control RBC components will be released to clinical inventory after review of the batch production record associated with the trial.

#### 4.5 SUBJECT DISCONTINUATION

The following groups of subjects will not be eligible for study enrollment or will be discontinued from the study and may be replaced.

- Screened subjects who receive an RBC transfusion before undergoing randomization will not be eligible for study enrollment.
- Screened subjects who are not randomized before their surgery begins will not be eligible for enrollment.
- Randomized subjects who do not undergo surgery within 7 days of randomization, will be discontinued 7 days after randomization. Patients may be re-screened for eligibility and randomization closer to the time of surgery.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

Randomized subjects who do not receive a study RBC transfusion within the first 48  $\pm 4$  hours after surgery will be discontinued and replaced and will not be followed any longer. For non-transfused subjects, a blood sample for sCr will be drawn at  $48 \pm 4$  hours. Daily sCr assessments will be recorded up to and including  $48 \pm 4$  hours post surgery. Other post baseline laboratory parameters and Adverse events (AEs) will not be collected for non-transfused subjects. Vital status will be recorded at the time of discontinuation.

• Enrollment Pause and Stopping Rules

#### 4.5.1 Definitions

#### 4.5.1.1 Enrollment Pause

"Enrollment Pause" means that new patients will not be consented or provide assent for the study and subjects already screened will not be randomized. Subjects already randomized and receiving study RBC transfusions will continue to receive study transfusions with IAT crossmatch with each RBC component and a new screen for antibodies specific to INTERCEPT RBCs every third day to optimize protection of enrolled recipients. The FDA will be notified of all DSTRs specific to INTERCEPT RBCs.

#### 4.5.1.2 Clinical Stop

"Clinical Stop" means complete cessation of recruitment activities and all study transfusions, thus stopping the active study transfusion phase of the study. Study participants will continue receiving non-study conventional transfusions as needed. All safety monitoring tasks will continue as per protocol.

#### 4.5.1.3 Rules

The study may be temporarily paused or definitively stopped based on, but not limited to, the following rules/considerations:

- Poor/slow accrual: The goal is to recruit at least 292 patients in the study. The study may be stopped by the Sponsor if enrollment rates are not deemed acceptable or financially sustainable.
- Safety
- The DSMB will review safety data and make recommendations as per the current version of the DSMB Charter including interpretation of the stopping rules.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

• The major safety concern in this trial is the possible development of antibodies specific to INTERCEPT RBCs that causes accelerated RBC clearance, as evidence of an acute or delayed hemolytic transfusion reaction (AHTR or DHTR). The study will be stopped if one subject who has been exposed to INTERCEPT RBC demonstrates a confirmed antibody with specificity to INTERCEPT RBCs and experiences a clinically significant HTR with overt intravascular or extravascular hemolysis as assessed by the Investigator and reviewed by the DSMB.

Stopping rules due to the occurrence of INTERCEPT RBC-specific DSTRs, DHTRs, AHTRs or hyperhemolysis syndrome are followed after discussion with Sponsor in the event of a positive antibody specific for INTERCEPT RBCs.

**Table 4.1 Stopping Rules for INTERCEPT RBC-specific antibodies** 

| | Trigger | Sponsor<br>Action | Notify | | Enrollment | On<br>Study<br>Patients | Continuation | Additional actions | |
|---|---|---|---|---|---|---|---|---|---|
| | For INTERCEPT<br>RBC- Specific Abs | | IRB | FDA | DSMB | | I | | - |
| 1 | INTERCEPT RBC-<br>Specific DSTR with<br>no evidence of<br>hemolysis | Patient<br>Withdrawal | X | X | X | Continue | Continue <sup>1</sup> | - | Sponsor will notify DSMB and FDA of each INTERCEPT RBC-Specific Ab <sup>2</sup> . Investigation may include unblinding the treatment assignment |
| 2 | INTERCEPT RBC-<br>Specific DHTR (x1) | Clinical<br>Stop | X | X | X | Stop | Stop | After<br>Investigation<br>& discussion<br>with FDA &<br>DSMB | Investigate full hemolytic potential. Continuation contingent on outcome of investigation, including confirmation that the subject has been exposed to INTERCEPT (Test) RBCs, and on FDA agreement on resumption. |
| 3 | INTERCEPT RBC-<br>Specific AHTR (x1) | Clinical<br>Stop | X | X | X | Stop | Stop | After<br>Investigation<br>& discussion<br>with FDA &<br>DSMB | Stop study for an INTERCEPT RBC-specific single acute hemolytic reaction. Continuation contingent on outcome of investigation, including confirmation that the subject has been exposed to INTERCEPT (Test) RBC, and on FDA agreement on resumption. |

| | Trigger | Sponsor<br>Action | | Notify | y | Enrollment | On<br>Study<br>Patients | Continuation | Additional actions |
|---|---|---|---|---|---|---|---|---|---|
| | For INTERCEPT<br>RBC- Specific Abs | | IRB | FDA | DSMB | | | | - |
| 4 | INTERCEPT RBC-<br>Specific Hyper-<br>hemolysis Syndrome<br>(x1) | Clinical<br>Stop | X | X | X | Stop | Stop | With FDA release | Investigation may include unblinding the treatment assignment |

<sup>&</sup>lt;sup>1</sup> The DSMB would make a decision on whether or not to pause the study each time a DSTR occurs with INTERCEPT RBC specificity.

<sup>&</sup>lt;sup>2</sup> Applies to all INTERCEPT RBC-specific antibody examples shown in rows 1-4.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

#### 4.6 ACCOUNTABILITY OF STUDY PRODUCT

The Investigational Product includes both the INTERCEPT Blood System for RBCs, a medical device used to prepare pathogen inactivated RBC components for transfusion, and the investigational biological product, INTERCEPT RBCs in SAG-M.

The investigational device accountability will be verified by the unblinded study monitors throughout the duration of study. They will assure that the device components are under control at all times inclusive of shipment, storage, usage, and disposition.

The investigational biologic product will be produced by each Blood Center according to the Study RBC Processing Procedures and accountability will be tracked using the Blood Center's electronic data management system.

Both Test and Control RBC components are for the sole use of study participants. They may not be crossed back into general inventory at a blood center or clinical site. The disposition of all components prepared for the study (transfused, discarded or expired) will be recorded. The investigational biologic product accountability will be verified by the unblinded study monitors throughout the duration of study.

#### 4.7 SOURCE DATA

The subjects' medical records are the source data; the study data will be recorded in an EDC system using eCRFs. Data worksheets used during the preparation of study RBC components are considered the source data for processing study RBC components.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

# 5 SELECTION AND WITHDRAWAL OF SUBJECTS

#### 5.1 SUBJECT INCLUSION CRITERIA

The following conditions must be met before a subject may be randomized into the study.

- 1. Age  $\geq$  11 years old
- 2. Weight  $\geq$  40 kg
- 3. Scheduled complex cardiac surgery or thoracic aorta surgery. The procedure may be performed either on or off cardiopulmonary bypass machine (CPB or "pump"). For the purposes of this protocol "Repeat procedure" means that the subject had a previous cardiac surgery. Procedures that qualify as complex cardiac surgery include but are not limited to the following:
- Single Vessel Coronary Artery Bypass Graft, first or repeat procedure
- Multiple Coronary Artery Bypass Grafts, first or repeat procedure
- Single Valve Repair or Replacement, first or repeat procedure
- Multiple Valve Repair or Replacement, first or repeat procedure
- Surgery involving both Coronary Artery Bypass Graft(s) and Valve Repair(s), first or repeat procedure
- One or more of the following procedures, with or without Coronary Bypass Graft(s):
  - o left ventricular aneurysm repair,
  - o ventricular and/or atrial septal defect repairs,
  - o Batista procedure (surgical ventricular remodeling),
  - o surgical ventricular restoration,
  - o congenital cardiac defect repair
  - aortic procedures
  - o other cardiac surgery or thoracic aorta surgery types with a high probability of bleeding.
- 4. TRUST probability score (Alghamdi, Davis et al. 2006) ≥ 3, or currently on regimen of aspirin (any dose), clopidogrel (or analogs) and/or GPIIb/IIIa inhibitors, or at a high probability for need of a transfusion during or after surgery at the discretion of the Investigator.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

- 5. Female subjects of child-bearing potential who meet the 2 criteria below at screening:
  - A negative urine or serum pregnancy test
  - Use at least one method of birth control that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence or vasectomized partner.
- 6. Signed and dated informed consent/assent form.

#### 5.2 SUBJECT EXCLUSION CRITERIA

Patients will be excluded from this study if they meet any of the following criteria:

- 1. Confirmed positive baseline serum/plasma antibody specific to INTERCEPT RBCs (S-303 specific antibody) screening panel prior to randomization.
- 2. Pregnant or breast feeding.
- 3. Refusal of blood products or other inability to comply with the protocol in the opinion of the Investigator or the treating physician.
- 4. Treatment with any medication that is known to adversely affect RBC viability, such as, but not limited to dapsone, levodopa, methyldopa, nitrofurantoin, and its derivatives, phenazopyridine and quinidine.
- 5. Planned cardiac transplantation.
- 6. Active autoimmune hemolytic anemia.
- 7. Left ventricular assist device (LVAD) or extracorporeal membrane oxygenation (ECMO) support pre-operatively or planned need post-operatively.
- 8. Cardiogenic shock requiring pre-operative placement of an intra-aortic balloon pump (IABP) (NOTE: IABP done for unstable angina or prophylactically for low ejection fraction is not excluded).
- 9. Planned use of autologous or directed donations.
- 10. RBC transfusion during current hospitalization prior to enrollment and randomization (within 7 days).
- 11. Participation in an interventional clinical study concurrently or within the previous 28 days. This includes investigational blood products, pharmacologic agents, imaging materials (including dyes), surgical techniques, or devices. Observational studies of FDA cleared or approved products or nutrition, psychology, or socioeconomic issues are not grounds for exclusion.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

- 12. Patients with a current diagnosis of either chronic kidney disease or acute kidney injury and with sCr ≥1.8 mg/dL at screening and patients requiring RRT. (NOTE: If sCr at screening is <1.8 mg/dL, a patient with a diagnosis of chronic or acute kidney injury alone is not excluded).
- 13. Patients with a current diagnosis of either chronic or acute hepatic insufficiency and with a total serum bilirubin ≥ 2.0 mg/dL (≥34.2 µmol/L). (NOTE: If total serum bilirubin at screening is <2.0 mg/dL, a patient with a diagnosis of chronic or acute hepatic failure alone is not excluded).
- 14. Pre-existing RBC antibody that may make the provision of compatible study RBC components difficult.
- 15. History of TRs requiring washed RBCs, volume reduced RBCs, or RBCs with additive solution removed.
- 16. Patients with documented IgA deficiency or a history of severe allergic reactions to blood products.
- 17. Patients who require gamma-irradiated RBC blood components.
- 18. Positive DAT as defined below:

A polyspecific DAT reaction strength > 2+, or

A polyspecific DAT (any strength) in conjunction with pan-reactivity with a commercial IAT antibody screening panel that precludes the identification of underlying alloantibodies or indicates the presence of autoantibody.

#### 5.3 SUBJECT WITHDRAWAL CRITERIA

Study subjects are free to withdraw consent/assent or discontinue participation in the study at any time, without prejudice to further treatment. A patient's participation in the study may be terminated at any time at the discretion of the investigator if he/she feels it is in the patient's best interest. Randomized subjects who do not receive any study RBC transfusions from randomization to within the first 48 hours after surgery will be replaced.

# 5.3.1 Discontinuation from study RBC transfusions

Study RBC transfusions will be discontinued if the subject:

- Becomes pregnant.
- Is treated with a concurrent prescribed medication demonstrated to have caused hemolysis while on study.
- Develops an antibody with presumed or documented INTERCEPT RBC specificity and cannot be transfused further with INTERCEPT RBCs.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

• If INTERCEPT RBC-specific antibodies cannot formally be ruled out, or agglutination is visible for all the untreated RBC cells in the panel, (i.e., "panreactive").

If the subject is discontinued from study transfusions due to development of INTERCEPT RBC-specific antibody after receiving one or more study RBC transfusions, the subject should continue on study receiving only non-study RBC transfusions if needed and should complete all safety assessments, including the study  $75\pm15$  days post last transfusion follow-up visit. REF 01606 (S-303 Reactive Samples: Management of Patients and Samples) should be followed immediately after the INTERCEPT RBC-specific antibodies are identified. A specific data entry guidance is provided in CRF Completion Guidelines (CCGs) for the INTERCEPT RBC-specific antibody reactive test results.

#### **5.3.2** Early termination from Study

Upon early termination from study the tests required of the termination visit will be performed. If the subject is terminated from study (for any reason) before transfusion of any study RBC product, the subject will be replaced and no further follow up is required. For non-transfused subjects, a blood sample for sCr will be drawn at  $48 \pm 4$  hours. Daily sCr assessments will be recorded up to and including  $48 \pm 4$  hours post surgery. Other post baseline laboratory parameters and Adverse events (AEs) will not be collected for non-transfused subjects. Vital status will be recorded at the time of discontinuation. If the subject has received any study RBC product and it is possible, a physical examination, including general neurological examination, should be performed, concomitant medications and adverse events should be recorded, standard laboratory tests should be collected, and other blood samples should be obtained on day  $28 \pm 3$  and day  $75 \pm 15$  as described in the protocol.

If consent/assent for further follow-up is withdrawn, the subject should, at minimum, be asked to provide a blood sample at the time of withdrawal for sCr, DAT, IAT and INTERCEPT RBC-specific antibody screen.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

## 6 TREATMENT OF SUBJECTS

#### 6.1 TREATMENT PLAN

# 6.1.1 Screening/Randomization (Day -30 to Day 0 Pre-Surgery)

Patients will be identified through pre-operative scheduling procedures in advance of their complex cardiac surgery. Patients already hospitalized may be included.

Patients undergoing urgent or emergent cardiac surgery are eligible for the study, subject to institutional review board (IRB) approval of an appropriate informed consent process.

In order to minimize the number of patients who enroll in the study but do not require RBC transfusion, only patients with a relatively high likelihood to receive a transfusion as determined by the Investigator (e.g., patients currently on regimen of aspirin, clopidogrel (or analogs) and/or GPIIb/IIIa inhibitors), or patients with a TRUST score of ≥3 will be eligible for enrollment. A TRUST score of ≥3 corresponds to a high likelihood of requiring red cell transfusion within 96 hours of surgery. Study consent/assent will be sought in these eligible subjects within 30 days of their surgical procedure. Subjects who consent/assent to the study will be assigned a subject identification (ID) number and undergo screening.

The complete list of screening assessments are outlined in Table 7.1a. Data may be derived from the medical record where performed within 30 days prior to their surgical procedure. Blood samples for determination of HLA antibodies will also be collected at the screening visit and sent for testing at a specialty central laboratory. In certain situations, it is possible for a mobile medical professional, authorized by the sponsor and requested by site personnel, to conduct a home health service visit at a subject's home to collect screening assessments. Patients who fail eligibility for any or multiple inclusion/exclusion criteria may be rescreened for eligibility closer to the time of surgery.

All available components of the TRUST score (age, sex, Hb, weight, type of surgery, serum creatinine, surgical history and surgical task) will be collected on the case report form. The TRUST score (or the minimum and maximum possible TRUST scores, if there are any missing components) will be calculated according to the published algorithm (APPENDIX 1).

Eligible subjects will be randomized up to 7 days before or on the day of surgery, but prior to the start of surgery (i.e., induction of anesthesia). The adverse event collection period will begin at the beginning of surgery or the first study RBC transfusion, whichever is first.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

For non-transfused subjects, a blood sample for sCr will be drawn at  $48 \pm 4$  hours. Daily sCr assessments will be recorded up to and including  $48 \pm 4$  hours post surgery. Other post baseline laboratory parameters and Adverse events (AEs) will not be collected for non-transfused subjects. Vital status will be recorded at the time of discontinuation.

The complete list of baseline assessments to be performed pre-operatively on the day before or on the day of surgery before surgery commences are outlined in Table 7.1b.

# 6.1.2 Acute Transfusion Support Period (Surgery [Day 0] to Post-operative Day 7, Hospital Discharge or Death, Whichever is First)

The complete list of assessments to be performed during the acute transfusion support period are outlined in Table 7.1c.

During the acute transfusion support period (Day 0 to Day 7), hospital discharge or death, whichever is first, patients will be transfused with Test or Control RBCs. Induction and end of anesthesia are considered start and stop time of surgery. All transfusions administered through Day 7 will be of the assigned treatment arm as often as feasible without compromising patient care.

A screen for antibodies specific for INTERCEPT RBCs should be performed every time that a routine IAT is performed during the acute 7-day study transfusion period.

A blood sample for sCr will be taken at 48 ( $\pm$ 4 hours) after completion of surgery, and sCr will be determined on a daily basis during the acute transfusion support period up to 7 days post-surgery. Other parameters will be collected on eCRFs only when available in the medical record.

Randomized subjects who do not receive an RBC transfusion following randomization within the first 48 hours after surgery will be discontinued from the study and replaced.

For non-transfused subjects, a blood sample for sCr will be drawn at  $48 \pm 4$  hours. Daily sCr assessments will be recorded up to and including  $48 \pm 4$  hours post surgery. Other post baseline laboratory parameters and adverse events (AEs)Es) will not be collected for non-transfused subjects. Vital status will be recorded at the time of discontinuation.

Once a subject is randomized, in rare exceptions where study RBCs are unavailable or a subject's need for RBC transfusions exceeds the quantities of the prepared study RBCs (e.g., during a Massive Transfusion Protocol), non-study RBC (conventional) transfusion may be given to provide the subject with an appropriate and necessary treatment. Non-study RBC transfusion data is captured in the eCRF. In this case, a protocol deviation should be noted. Transfusions will be administered according to

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

local institutional policy and safety standards as ordered by the medical team for patient care needs. Anesthesia and surgical procedures will be performed according to the local standards of the institution.

Hemodynamic and laboratory results will be recorded daily from post-surgery through post-operative Day 7, hospital discharge or death, whichever occurs first. If an assessment is performed more than once in a day, the first set of results should be entered into the eCRF.

If a subject is discharged prior to the end of the acute transfusion support period (Day 7) but for any reason returns to the study site (e.g., re-hospitalization or standard care) within this acute transfusion support period, lab values routinely collected as standard of care should be recorded in the eCRF.

If multiple assessments (hemodynamic parameters, vital signs, laboratory parameters) are taken in a calendar day, the reported value for first collection of the day should be recorded in the eCRF with the exception of serum creatinine. Serum creatinine will be collected and recorded in the eCRF on a daily basis during the 7 day acute transfusion support period. If serum creatinine is measured multiple times in a day, the worst daily value should be recorded in the eCRF. In addition, a sample to measure sCr will be taken at 48±4 hours after the end of surgery and captured on a specific CRF page for that time-point.

For non-transfused subjects, a blood sample for sCr will be drawn at  $48 \pm 4$  hours hours post-surgery. Serum Creatinine up to and including  $48 \pm 4$  hours post-surgery will be collected.

Urine output (mL/kg/hour) will be recorded in the eCRF daily while a urinary catheter is in place.

Other assessments during this trial period include details related to the specific surgical procedure (type of procedure, start and end times, RBC components transfused, all other blood components transfused, estimated blood loss from the surgical procedure, concomitant medications, intraoperative cell recovery and reinfusion, hemodilution, and nadir temperature). Additionally, daily estimated blood loss from chest tube(s) and from other sources, and day of chest tube removal will be recorded. See Table 7.1c for a detailed list of study assessments.

AEs and SAEs, including TRs and protocol-specified AEs (see Section 7.3), will be assessed from the start of surgery or the start of the first study RBC transfusion (whichever is first) on a daily basis and documented in the eCRF through post-operative Day 7. Adverse events (AEs) will not be collected for non-transfused

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

subjects, but vital status will be recorded at the time of discontinuation. See Table 7.1c for a detailed list of study assessments.

NOTE: The following post-operative assessments apply to randomized transfused subjects only.

# 6.1.3 Post-operative Period (Day 8 [or Post-discharge, if earlier] through Day 28 After Last Study Transfusion)

The complete list of assessments to be performed during this post-operative period are outlined in Table 7.1d.

Laboratory results recorded in the eCRFs during this period will only be those assessed as clinically significant per the Investigator. Following the post-surgery 7-day acute transfusion support period, the post-operative period starts on Day 8 after surgery and goes through the Day 28±3 visit. Subjects will receive conventional non-study RBC components if additional transfusions are needed, as indicated by their treating physician.

Weekly telephone surveillance calls to the subject will be performed to collect AEs, SAEs and TRs. If a surveillance call falls on the same week as the Day 28±3 follow-up visit, the follow-up visit assessments will take precedent and a surveillance call is not required.

#### 6.1.4 Day 28±3 After Last Study Transfusion or Early Termination

The complete list of assessments to be performed during the Day 28±3 or Early Termination visit are outlined in Table 7.1e.

Subjects should be scheduled for a follow-up visit 28±3 days after the last study transfusion to obtain additional safety information, including subject-reported AEs, SAEs, and laboratory results. This visit may occur either in hospital, clinic visit, or offsite. In certain situations, it is possible for a mobile medical professional, authorized by the Sponsor and requested by site personnel, to conduct a home health service visit at a subject's home to collect these assessments. Blood samples for determination of HLA antibodies will also be collected at the visit and sent for testing at a specialty central laboratory. TRs, AEs and SAEs will be documented for 28 days after the last study transfusion, or earlier if the subject dies prior to Day 28 post last study RBC transfusion. If a subject has been discharged prior to Day 28 post last study RBC transfusion, the vital status, need for RRT and other safety information (e.g., AEs and SAEs) may be obtained through medical records, the subject's physician, or a telephone interview with either the subject or a family member.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

# 6.1.5 Day 30 – After Surgery Assessment

The complete list of assessments to be performed at Day 30 are outlined in Table 7.1e.

All randomized subjects who receive a study RBC transfusion must have their vital status and need for RRT (defined as hemodialysis or peritoneal dialysis) documented at Day 30 after surgery. RRT that is provided prophylactically during surgery while patient is on a bypass machine (the pump) does not meet this endpoint. The vital status and RRT assessment on Day 30 post surgery can be obtained either from the medical records, from a phone call to the subject or family, or during the visit  $28\pm3$  days after the last study transfusion (only if the last study transfusion was given at day 2 or later in the acute transfusion support period).

# 6.1.6 End of Study (75 ±15 Days After Last Study Transfusion)

The complete list of assessments to be performed at the 75  $\pm$ 15 day study visit are outlined in Table 7.1e.

Subjects should be scheduled for a second follow up visit on Day 75±15 days after the last study transfusion for vital status, need for RRT, and for assessment of INTERCEPT RBC-specific antibodies at end of study, either in hospital, clinic visit or off-site. In certain situations, it is possible for a mobile medical professional, authorized by the Sponsor and requested by site personnel, to conduct a home health service visit at a subject's home to collect these assessments. If the assessment of INTERCEPT RBC-specific antibodies is positive, the positive S-303 specific DSTR should be entered on the Adverse Event eCRF.

# 6.1.7 Assessments in Follow-up to a Reactive Antibody Test Specific for INTERCEPT RBCs

In the event of detection of treatment-emergent antibodies with specificity to INTERCEPT RBCs, the Investigator shall be instructed about specific laboratory and clinical assessments to be performed. See section 7.3.1.11 Suspected Hemolytic and Serologic TRs after Enrollment and Transfusion with Study RBC Components assessment of immune reactivity of INTERCEPT for more details.

#### 6.2 CONCOMITANT AND EXCLUDED THERAPY

Standard medical care according to local institutional standards will be provided to each subject. The following concomitant (or planned) therapies/procedures will exclude subjects from the current study:

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

- Left-ventricular assist device (LVAD) or Extracorporeal membrane oxygenation (ECMO) support pre-operatively or planned need post-operatively.
- Cardiogenic shock requiring pre-operative placement of an IABP (Note: IABP done for unstable angina or prophylactically for low ejection fraction is not excluded).
- Treatment with any medication that is known to adversely affect RBC viability, such as but not limited to, dapsone, levodopa, methyldopa, nitrofurantoin, and its derivatives, phenazopyridine and quinidine.
- Planned use of autologous or directed donations
- Patients who have received an RBC transfusion during current hospitalization prior to randomization (within 7 days)
- Subjects who have received investigational products, including investigational blood products, pharmacologic agents or imaging materials, within the prior 28 days will also be excluded.

# 6.3 TREATMENT COMPLIANCE

Treatment compliance will be overseen by the Investigator and study staff and relevant documentation will be recorded in the eCRF. Compliance will be monitored by the Sponsor and/or Sponsor's representatives by review of source documents. The study RBC components will be labeled and tracked through all stages of processing of Test and Control components, storage, issue, and transfusion.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

# 7 STUDY ASSESSMENTS

#### 7.1 STUDY SCHEDULE OF ASSESSMENTS

A screen for antibodies specific for INTERCEPT RBCs should be performed every time that a routine IAT is performed during the acute 7-day study transfusion period.

A blood sample for sCr will be taken at 48 (±4 hours) after completion of surgery, and sCr will be determined on a daily basis during the acute transfusion support period up to 7 days post-surgery. Other parameters will be collected on eCRFs only when available in the medical record.

For non-transfused subjects, a blood sample for sCr will be drawn at  $48 \pm 4$  hours and daily sCr assessments will be recorded up to and including  $48 \pm 4$  hours post surgery. All samples obtained for determination of human leukocyte antigen (HLA) will be stored for up to 1 year after the study has completed.

The study assessments used to evaluate both efficacy and safety are presented in Table 7.1a, Table 7.1b, Table 7.1c, Table 7.1d, Table 7.1e and 7.2.

| Table 7.1a – Screening/Randomization | | |
|---|---|---|
| Study Period – Screening Visit (Day -30 to Day 0 pre-surgery) | | |
| Assessment | | Superscripts Defined |
| Informed Consent/Assent | X | |
| Demographics | X | <sup>1.</sup> For Screening/Randomization purposes, data from medical records |
| Indication /Type of scheduled surgery | X | within 30 days prior to their surgical procedure may be used. |
| Medical, surgical, transfusion and medication history including radiographic contrast media within 7 days of surgery/ the need for irradiated RBC products | X | <sup>2.</sup> See <b>Table</b> 7.2: Hematology and Chemistry Testing for details on required labs. |
| Number of prior pregnancies (females) | X | |
| Physical examination including height and weight | X | |
| Vital signs (HR, BP, RR) <sup>1</sup> | X | |
| Concomitant medications | X | |
| EKG <sup>1</sup> | X | |
| Pregnancy test (if applicable) 1,2 | X | |
| Hematology panel <sup>1,2</sup> | X | |
| Blood chemistry <sup>1,2</sup> | X | |
| Blood type <sup>1</sup> | X | |
| DAT <sup>1</sup> , IAT <sup>1</sup> | X | |
| INTERCEPT RBC antibody screen (S-303-specific antibody screen) | X | |
| Sample for HLA antibodies | X | |
| TRUST score components | X | |
| Randomization <sup>#</sup> | X | *Eligible patients will be randomized up to 7 days before or on the day of surgery, but prior to the start of surgery (i.e., induction of anesthesia). |
| AEs/SAEs/TRs* | X | *The adverse event, serious adverse event and transfusion reaction collection period will begin at the start of surgery or the first study RBC transfusion, whichever is first. Adverse events (AEs) will not be collected for non-transfused subjects, but vital status will be recorded at the time of discontinuation. |

| Та | ble 7.1b | - Baseline (Pre-Surgery) |
|---|---|---|
| Study Period – Baseline (Day -1 or Day 0 Pre-Surgery) | | |
| Assessment | | |
| Vital signs (HR, BP, RR) <sup>3</sup> | X | <sup>2</sup> See <b>Table 7.2</b> : Hematology and Chemistry Testing for details on required labs. |
| Concomitant medications <sup>3</sup> | X | <sup>3</sup> .These assessments can be combined with screening assessments if |
| Pregnancy test (if applicable) <sup>2,3</sup> X | | screening visit is also on Day -1 or Day 0 Pre-Surgery. |
| Hematology panel <sup>2,3</sup> X | | <sup>4</sup> ·Data collected on eCRFs only as available from medical records if performed as Standard of Care. |
| Blood chemistry <sup>2, 3</sup> | X | performed as Standard of Care. |
| EKG <sup>3</sup> | X <sup>4</sup> | 5. Hemodynamic Parameters: Peripheral O <sub>2</sub> Saturation, Mean Arterial Pressure, Central Venous Pressure. |
| Hemodynamic Parameters <sup>5</sup> | X <sup>4</sup> | |
| Fibrinogen Troponin | X <sup>4</sup> | |
| AEs/ SAEs/TRs* | X | *The adverse event, serious adverse event and transfusion reaction collection period will begin at the start of surgery or the first study RBC transfusion, whichever is first. Adverse events (AEs) will not be collected for non-transfused subjects but vital status will be recorded at the time of discontinuation. |

# Table 7.1c – Acute Transfusion Support Period Study Period - Acute Transfusion Support Period (Surgery [Day 0] to Post-operative Day 7, hospital discharge or death, whichever is first)

| | is first) | | |
|---|---|---|---|
| Assessment | Day 0<br>Surgery | Day 1 - | Superscripts Defined |
| Vital signs (HR, BP, RR) | X | $X^6$ | <sup>2.</sup> See <b>Table 7.2</b> : Hematology and Chemistry Testing |
| Concomitant medications | X <sup>7</sup> | $X^6$ | for details on required labs. |
| EKG | X <sup>4</sup> | X <sup>4</sup> | 4. Data collected on eCRFs only as available from medical records if performed as Standard of Care. |
| Hematology panel <sup>2</sup> | X | X <sup>6</sup> | <sup>5.</sup> Hemodynamic Parameters, if available- Peripheral |
| Blood chemistry <sup>2</sup> | X | $X^6$ | O <sub>2</sub> Saturation, Mean Arterial Pressure <sup>4</sup> , Central Venous Pressure <sup>4</sup> |
| Serum Creatinine at 48±4 hours after end of surgery | | $X^{10}$ | 6. These assessments are required to be collected daily |
| Hemodynamic Parameters <sup>3</sup> | X <sup>5</sup> | X <sup>6</sup> | on Day 1 through Day 7 post surgery or until |
| Fibrinogen, Troponin | X <sup>4</sup> | X <sup>4</sup> | discharge. If subject returns after discharge for a postoperative standard of care visit, assessments |
| Urine output <sup>8</sup> | X | X <sup>6</sup> | will be collected in eCRFs on the appropriate study |
| Procedure details | X | | day. |
| Study RBC crossmatch and Study RBC transfusion(s)/data | X | X | <sup>7.</sup> Any drugs given to induce anesthesia or drugs given as a prophylactic in combination with anesthesia |
| DAT, IAT, INTERCEPT RBC antibody screen (S-303-specific antibody screen) <sup>9</sup> | X <sup>4</sup> | X <sup>4</sup> | prior to surgery do not need to be recorded. Medications given during anesthesia to |
| All other blood components (including non- study RBCs) transfused, if any | X | X | treat an AE/SAE need to be recorded. 8. Urine output data collected daily while a urinary |
| Estimated blood loss from surgery | X | | catheter is in place. The date entered should reflect the start of the collection and match the visit date. |
| Estimated blood loss from other source including chest tube(s) | | $X^6$ | 9. S-303 screen must be performed whenever a |
| AEs/ SAEs/TRs* | X | $X^6$ | routine RBC alloantibody screen (IAT) is |
| | | | performed during the transfusion period. 10. For non-transfused subjects, a blood sample for |
| | | | sCr will be drawn at 48 ± 4 hours. Daily sCr |

## Table 7.1c – Acute Transfusion Support Period Study Period - Acute Transfusion Support Period (Surgery [Day 0] to Post-operative Day 7, hospital discharge or death, whichever is first) Day 0 Day 1 -**Superscripts Defined Assessment** Surgery 7 assessments will be recorded up to and including $48 \pm 4$ hours post surgery. \* The adverse event, serious adverse event and transfusion reaction collection period will begin at the start of surgery or the first study RBC transfusion, whichever is first. AEs including protocol specified AEs, TRs and SAEs (see Section 7.3) are collected through 28 days after the last study transfusion; also collected daily during acute

transfusion support period. For non-transfused subjects, adverse events (AEs) will not be collected for non-transfused subjects, but vital status will be

recorded at the time of discontinuation.

| Table 7.1d – Post-Operative Period | | |
|---|---|---|
| Study Period- Post-operative Period Day 8 (or Post-discharge, if Earlier) to Day 28 after last study transfusion | | |
| Assessment | Day 8<br>through to<br>Day 28 post<br>last study Tx | Superscript Defined |
| Weekly telephone calls | X | <sup>2.</sup> See Table 7.2: Hematology and Chemistry Testing |
| Concomitant medications | $X^4$ | for details on required labs |
| Hematology panel <sup>2, 10</sup> | $X^4$ | 4. Data collected on eCRFs as available from medical |
| Blood chemistry <sup>2, 10</sup> | $X^4$ | records if performed as Standard of Care. |
| Hemodynamic Parameters <sup>5</sup> | $X^4$ | 5. Hemodynamic Parameters, if available- Peripheral |
| Fibrinogen, Troponin | $X^4$ | O <sub>2</sub> Saturation, Mean Arterial Pressure, Central Venous Pressure |
| Urine output <sup>8</sup> | X <sup>4</sup> | |
| All other blood components (including non- study RBCs) transfused, if any | $X^4$ | 8. Urine output data collected daily while a urinary catheter is in place. The date entered should reflect the start of the collection and match the visit date. |
| AEs/ SAEs/TRs* | X | <sup>10.</sup> Laboratory results recorded in the eCRFs during this period will only be those assessed as clinically significant by the Investigator. |
| | | * The adverse event, serious adverse event and transfusion reaction collection period will begin at the start of surgery or the first study RBC transfusion, whichever is first. AEs including protocol specified AEs, TRs and SAEs (see Section 7.3) are collected through 28 days after the last study transfusion; also collected daily during acute transfusion support period. Adverse events (AEs) will not be collected for non-transfused subjects, but vital status will be recorded at the time of discontinuation. |

| Table 7.1e - Follow-up Visits (Day 28±3, 30, and 75±15) | | | | |
|---|---|---|---|---|
| Study Period (Day 28±3, 30, and 75±15[End of Study]) | | | | |
| Assessment | 28±3 days<br>After last study<br>transfusion<br>or Early<br>Termination | 30 days<br>After<br>Surgery | End of Study<br>(75±15 Days<br>After Last<br>Study<br>Transfusion) | Superscripts Defined |
| Vital signs (HR, BP, RR) | X | - | | <sup>2.</sup> See <b>Table 7.2</b> : Hematology and |
| Concomitant medications | X | | | Chemistry Testing for details on |
| Hematology panel <sup>2</sup> | X | | | required labs |
| Blood chemistry <sup>2</sup> | X | | | * The adverse event, serious adverse |
| DAT, IAT | X | | | event and transfusion reaction |
| INTERCEPT RBC antibody screen (S-303-specific antibody screen) | X | | X | of surgery or the first study RBC transfusion, whichever is first. AEs |
| Sample for HLA antibodies | X | | | including protocol specified AEs, TRs |
| All other blood components (including non- study RBCs) transfused, if any | X | | | and SAEs (see Section 7.3) are collected through 28 days after the last |
| AEs/ SAEs/TRs * | X | | | study transfusion; also collected daily |
| | | | | during acute transfusion support period. Adverse events (AEs) will not be collected for non-transfused subjects, but vital status will be recorded at the time of discontinuation. |
| Documentation of vital status and need for RRT | X | X <sup>11</sup> | X | 11. Assess at Day 30 post surgery via clinic visit, medical record or phone call. Any RRT that is provided prophylactically during surgery while the subject is on a bypass machine does not meet this endpoint. |

Table 7.2: Hematology and Chemistry Testing- Required (R) results and Where Available (WA)<sup>a</sup> results

| | Screening / R | andomization | Acute Tran | sfusion Support Period | Post-operative Period | Follow-up Visit |
|---|---|---|---|---|---|---|
| Study Period | Baseline<br>(Pre-surgery) | | Day 7, hosp | Day 0] to Post-operative<br>bital discharge or death,<br>ichever is first) | | |
| Window | Day -30 to<br>Day -1 | Day -1 or<br>Day 0<br>pre- surgery <sup>g</sup> | Day 0<br>Surgery | Days 1 – 7, hospital<br>discharge or death | Days 8 to 28 after last study transfusion / death Laboratory results recorded in the eCRFs during this period will only be those assessed as clinically significant per the investigator. | 28±3 days after last<br>study transfusion or<br>Premature<br>Discontinuation<br>Visit |
| Pregnancy test (if applicable) | $R^{j}$ | $R^{j}$ | | | | |
| Hematology (CBC): | | | | | | |
| Hematocrit (Hct) | $R^{b}$ | WA | R | R <sup>d,e,i</sup> | WA | R |
| Hemoglobin (Hb) | $R^{b}$ | WA | R | R <sup>d,e,i</sup> | WA | R |
| Platelets (PLT) | $R^b$ | WA | R | R <sup>d,e,i</sup> | WA | R |
| RBC Count | $R^{b}$ | WA | R | R <sup>d,e,i</sup> | WA | R |
| WBC Count | $R^b$ | WA | R | R <sup>d,e,i</sup> | WA | R |
| Fibrinogen | | WA | WA | WA <sup>d</sup> | WA | |
| Troponin | | WA | WA | WA <sup>d</sup> | WA | |
| Blood chemistry: | | | | | | |
| Alkaline Phosphatase (ALP) | WA | WA | WA | WA <sup>d</sup> | WA | WA |
| Alanine Transaminase (ALT) | WA | WA | WA | WA <sup>d</sup> | WA | WA |
| Aspartate Aminotransferase (AST) | WA | WA | WA | WA <sup>d</sup> | WA | WA |
| Bicarbonate (CO <sub>2</sub> ) | WA | WA | WA | WA <sup>d</sup> | WA | WA |
| Blood Urea Nitrogen (BUN) | $R^b$ | R | $R^h$ | $R^{d,h,i}$ | WA | R |
| Calcium (Ca) | $R^{b}$ | WA | R | WA <sup>d</sup> | WA | R |
| Chloride (Cl) | R <sup>b</sup> | WA | R | WA <sup>d</sup> | WA | R |
| Creatinine (sCr) | $R^b$ | R | $\mathbb{R}^{h}$ | R <sup>c,e,f,h,i</sup> | WA | R |
| Glucose | $R^b$ | WA | R | R <sup>d,i</sup> | WA | R |
| Lactate Dehydrogenase (LDH) | WA | WA | WA | WA <sup>d</sup> | WA | WA |
| Potassium (K) | R <sup>b</sup> | WA | R | R <sup>d,i</sup> | WA | R |
| Sodium (Na) | R <sup>b</sup> | WA | R | R <sup>d,i</sup> | WA | R |

| | Screening / Ra | andomization | Acute Tran | sfusion Support Period | Post-operative Period | Follow-up Visit |
|---|---|---|---|---|---|---|
| Study Period | | Baseline<br>(Pre-surgery) | Day 7, hosp | Day 0] to Post-operative ital discharge or death, ichever is first) | | |
| Window | Day -30 to<br>Day -1 | Day -1 or<br>Day 0<br>pre- surgery <sup>g</sup> | Surgery Days 1 – 7, hospital discharge or death | | Days 8 to 28 after last study transfusion / death Laboratory results recorded in the eCRFs during this period will only be those assessed as clinically significant per the investigator. | 28±3 days after last<br>study transfusion or<br>Premature<br>Discontinuation<br>Visit |
| Total Bilirubin | R <sup>b</sup> | R | R | $R^{d,i}$ | WA | R |

#### Footnotes:

- <sup>a</sup> R= required testing and reporting.
  - WA=where available. Data collected on eCRFs as available from medical records if performed as Standard of Care.
- <sup>b</sup> For Screening/Randomization purposes, data from medical records within 30 days of surgery may be used as long as laboratory tests are performed again prior to surgery in order to establish baseline values and confirm the subject's continued trial eligibility.
- <sup>c</sup> A sample to measure sCr will be taken at 48±4 hours after the end of surgery and captured on a specific CRF page for that time-point. For non-transfused subjects, a blood sample for sCr will be drawn at 48 ± 4 hours.
- <sup>d</sup> If an assessment is performed more than once in a day, the first set of results should be entered into the eCRF.
- <sup>e</sup> If a subject is discharged prior to the end of the acute transfusion support period (Day 7) but for any reason returns to the study site (e.g., rehospitalization or standard care) within this acute transfusion support period, lab values routinely collected as standard of care should be recorded in the eCRF.
- f If serum creatinine is measured multiple times in a day, the worst daily value should be recorded in the eCRF.
- g These assessments can be combined with screening assessments if screening visit is also on Day -1 or Day 0 Pre-Surgery.
- h Assessments that contribute to the AKI should be measured at approximately the same time every day during the treatment period.
- <sup>i</sup> These assessments are required to be collected daily on Day 1 through Day 7 post surgery or until discharge. If subject returns after discharge for a postoperative standard of care visit, assessments will be collected in eCRFs on the appropriate study day.
- <sup>j</sup> Negative urine or serum pregnancy test.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

## 7.2 ASSESSMENT OF EFFICACY

# 7.2.1 Efficacy Parameters

The primary efficacy endpoint is the proportion of patients with a diagnosis of renal impairment defined as any increase in sCr  $\geq$ 0.3 mg/dL (or 26.5  $\mu$ mol/L) from the presurgery baseline within 48±4 hours after the completion of surgery. If any subject meets this criterion before receiving a study transfusion, that particular event will not be included in this analysis.

Treatment difference (Test–Control) will be compared between the subjects who were randomized to receive INTERCEPT RBCs vs. those randomized to receive conventional RBCs with a non-inferiority margin of 50% increase from the Control rate and two-sided 0.05 alpha level.

Secondary efficacy parameters that will be assessed include:

- The proportion of patients with a diagnosis of stage I, II or III Acute Kidney Injury (KDIGO 2012) based on changes in sCr levels from baseline and the need for renal replacement therapy (RRT) post-surgery.
- Mortality or the need for RRT by Day 30 post-surgery.

# 7.2.2 Methods and Timing of Efficacy Parameters

Hemodynamic and laboratory measures will be assessed pre-operatively (Day -1 or pre-operatively on the day of surgery) and daily from post-operative Day 1 through post-operative Day 7, hospital discharge or death, whichever occurs first. Serum creatinine will be determined on a daily basis during the acute transfusion support period and, in order to capture the primary efficacy endpoint, a sample for sCr will be taken also at 48±4 hours after the end of surgery.

The rest of the efficacy parameters will be collected only as available in the medical record (refer to Study Schedule of Assessments; Section 7.1).

An end of acute transfusion period a blood sample will be collected at Day 7, hospital discharge, or death, whichever occurs first. If a subject is discharged prior to Day 7 but returns to the study site for a standard of care visit on Day 7, blood samples should be obtained on that day for a complete blood count and sCr determination.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

#### 7.3 ASSESSMENT OF SAFETY

# 7.3.1 Safety Parameters

The primary safety outcome measures are the:

- Proportion of patients with any treatment-emergent adverse events (TEAEs) possibly, probably or definitely related to study RBC transfusion through 28 days after the last study transfusion.
- Proportion of patients with treatment emergent antibodies with confirmed specificity to INTERCEPT RBCs).

Additional safety assessments will include, but are not limited to:

- Treatment-emergent AEs through 28 days after the last study transfusion.
- Treatment-emergent SAEs through 28 days after the last study transfusion.
- Transfusion reactions (as defined by the CDC National Healthcare Safety Network [NHSN] Hemovigilance Module protocol) through 28 days after last study transfusion.
- Treatment-emergent immunization to RBC allo-antigens through 28±3 days after the last study transfusion.
- Treatment-emergent immunization to HLA allo-antigens through 28±3 days after the last study transfusion.

#### 7.3.1.1 Definition of Adverse Event

An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical (investigational) product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not related to the medicinal (investigational) product (ICH E2A II/A/1, 21 CFR 312.32).

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

#### 7.3.1.2 Definition of Serious Adverse Event

A Serious AE (SAE) is any untoward medical occurrence that at any dose results in any of the following outcomes:

- Death
- Life-threatening event (results in an immediate risk of death from the reaction as it occurred)
- Inpatient hospitalization or prolongation of existing hospitalization
- A persistent or significant disability/incapacity
- A congenital anomaly/birth defect
- Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient or subject and/or may require intervention to prevent one of the outcomes listed in this definition.

The terms "severe" and "serious" are not synonymous. Severity refers to the intensity of an adverse event (e.g., rated as mild, moderate, or severe, life-threatening or death according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) criteria). Severity and seriousness need to be assessed for each adverse event recorded on the eCRF.

SAE must be reported by the Investigator to the Sponsor immediately (i.e., no more than 24 hours) after learning of the event.

# 7.3.1.3 Unexpected Adverse Event

Any adverse event occurring in one or more subjects in a research protocol, the nature, severity, or frequency of which is not consistent with (a) the applicable product information (protocol, informed consent/assent, Investigator's Brochure or other product labeling), or (b) the expected natural progression of any underlying disease, disorder or condition of the subject experiencing the adverse event and the subject's predisposing risk factor profile for the adverse event.

# 7.3.1.4 Definition of Unanticipated Adverse Device Effects

Any serious adverse effect on health or safety or any life-threatening problem or death caused by, or possibly, probably or definitely related to a device, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan or application (including a supplementary plan or application), or

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

any other unanticipated serious problem associated with a device that relates to the rights, safety, or welfare of subjects (21 CFR 812.3(s)).

# 7.3.1.5 Definition of Renal Impairment

For the purposes of this study, renal impairment is defined as an increase in  $sCr \ge 0.3$  mg/dL from the pre-surgical baseline concentration.

# 7.3.1.6 Definition of Acute Kidney Injury (AKI)

For the purposes of this study, a definition of an acute kidney injury during the study is based on the Kidney Disease: Improving Global Outcomes (KDIGO) AKI workgroup definition (KDIGO 2012) criteria as:

- An increase sCr ≥50% of the pre-surgery baseline level within 7 days postsurgery, OR
- An increase in sCr ≥0.3 mg/dL (26.5 μmol/L) from pre-surgery baseline within 48 hours of surgery.

For the purposes of this study, acute kidney injury stages are defined as follows (KDIGO AKI workgroup):

| Stage 1 | Serum creatinine: 1.5–1.9 times baseline within 7 days after surgery |
|---|---|
| | OR |
| | $\geq$ 0.3 mg/dl ( $\geq$ 26.5 $\mu$ mol/L) increase within 48 hours of surgery |

- Stage 2 Serum creatinine: 2.0–2.9 times baseline within 7 days after surgery
- Stage 3 Serum creatinine: 3.0 times baseline within 7 days after surgery OR
  Increase in serum creatinine to ≥4.0 mg/dl (≥353.6 µmol/L)
  OR
  Initiation of renal replacement therapy

If a renal event during the study fulfills KDIGO laboratory criteria as specified above, this may constitute an AE/SAE of AKI as per Investigator's clinical judgement.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

# 7.3.1.7 Renal Replacement Therapy

For the purposes of this study RRT is defined as the institution of hemodialysis or peritoneal dialysis to treat acute or chronic renal failure associated with a decrease in glomerular filtration rate with or without fluid overload, severe acidosis, hyperkalemia or other electrolyte abnormalities. Dialysis performed solely to treat toxin/poisonings or performed preventatively during surgery while on a bypass machine, will not be considered RRT in the terms of meeting a secondary endpoint.

# 7.3.1.8 Treatment-emergent HLA antibodies

For the purposes of this study, HLA Class I and II antibody testing will be performed in a central laboratory according to the method described by Triulzi et al. (Triulzi 2009). Screening tests for anti-HLA Class I and II will be performed with multi-antigen bead kits (LabScreen LSM12, LabScreen Mixed, One Lambda, Canoga Park, CA) according to the manufacturer's instructions. Data will be using two different normalized background (NBG) ratio cut-offs. The data will be analyzed using the manufacturer's recommended cutoff of a NBG ratio of 2.2. The data will also be analyzed using NBG ratios of the mean plus three or five standard deviations of a log transformed distribution of values for plasma samples for non-transfused males, as described (Triulzi 2009).

# 7.3.1.9 Definition of Culture Proven Sepsis/Septic Shock

For the purposes of this study, transfusion related sepsis/septic shock is defined as a positive culture from blood and/or CSF and a study RBC product with matching bacterial strains, with at least 3 of the following signs of septic inflammatory response syndrome (SIRS) (Levy 2003):

- Temperature  $< 36^{\circ}$ C or  $> 38^{\circ}$ C
- Heart rate > 90 bpm
- Respiratory rate > 20 breaths/min or PaCO<sub>2</sub> < 32 mmHg
- White blood cell count  $> 12,000 \text{ or } < 4,000 \text{ cells/mm}^3 \text{ or } > 10\% \text{ bands}$

#### 7.3.1.10 Definition of Transfusion Reaction

A transfusion reaction is defined as an undesirable response or effect in a patient temporally associated with and possibly, probably or definitely related to the administration of blood or blood components. The current version of the CDC NHSN Hemovigilance Protocol definitions must be used when recording transfusion reaction

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

terms in this study (APPENDIX 3).

# 7.3.1.10.1 Clinically Significant Antibodies (Chapman et al. 2004)

Clinically significant antibodies are those that are capable of causing patient morbidity due to accelerated destruction of a significant proportion of transfused red cells.

# 7.3.1.10.2 Delayed Serological Transfusion Reaction (DSTR) (Ness et al. 1990; Garratty 2012)

The DSTRs are where a particular alloantibody can be shown to be present in the patient's plasma, on the transfused donor RBCs and/or in an eluate from these RBCs, but no clinical or laboratory signs of hemolytic anemia (HA) are present. Regardless of the mechanism, the persistence of a positive DAT does not correlate with the presence or absence of clinical hemolysis (Ness 1990).

The DSTR may be in the form of new antibodies or a rising titer of antibodies in patients with pre-existing antibodies (patients with pre-existing antibodies specific to INTERCEPT RBCs at baseline evaluation will be excluded in ReCePI). DSTR will be categorized as described in the NHSN Hemovigilance Protocol v 2.5.2 (APPENDIX 3).

# 7.3.1.10.3 Delayed Hemolytic Transfusion Reaction (DHTR) (Ness et al. 1990)

A DHTR is defined as a DSTR that showed clinical and/or laboratory evidence of hemolysis. Table 7.3 shows some differential diagnoses of hemolytic transfusion reactions. DHTR will be categorized as described in the CDC NHSN Hemovigilance Protocol v 2.5.2 (APPENDIX 3).

# 7.3.1.10.4 Acute Hemolytic Transfusion Reaction (AHTR) (Ness 1990)

An AHTR is defined as the rapid destruction of RBCs during, immediately after, or within 24 hours of cessation of transfusion. Clinical and laboratory signs of hemolysis are present AHTR will be categorized as described in the CDC NHSN Hemovigilance Protocol v 2.5.2 (APPENDIX 3).

#### 7.3.1.10.5 Hyper-hemolysis Syndrome

Hyperhemolysis is characterized by a hemolytic transfusion reaction that leads to a life-threatening anemia, with drops in Hb and Hct to levels markedly lower than those present before transfusion.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

# **Table 7.3 Some Differential Diagnoses of Hemolytic Transfusion Reactions**

# Immunologically caused hemolysis

Autoimmune hemolytic anemia

'Warm' antibody induced hemolytic anemia

Cold hemagglutinin disease

Paroxysmal cold hemoglobinuria

Drug induced immune hemolytic anemia

Passenger lymphocyte syndrome after stem cell or solid organ transplantation Hemolytic disease of a newborn

# Acute episodes of non-immunologically caused hemolysis

Hereditary erythrocyte defects

Defects of red blood cell (RBC) enzymes (e.g., glucose-6-phosphate dehydrogenase deficiency)

Hemoglobinopathies (e.g., sickle cell disease)

Thalassemia

Defects of RBC membrane

Congenital erythropoietic porphyria

# Paroxysmal nocturnal hemoglobinuria

Infections

Bacterial (bartonellosis; hemolytic-uremic syndrome caused by enterohemorrhagic Escherichia coli; severe infections by bacteria producing hemolyzing toxins (e.g., Clostridium perfringens)) Protozoal (malaria, babesiosis)

Mechanical hemolysis by artificial heart valves or by extracorporeal circulation

Thrombotic-thrombocytopenic purpura (Moschowitz disease)

HELLP syndrome during gravidity

Intoxications

Near drowning

Source: Strobel E. 2008.
**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

# 7.3.1.11 Suspected Hemolytic and Serologic Transfusion Reactions after Enrollment and Transfusion with Study RBC Components

# 7.3.1.11.1 Assessment of Immune Reactivity to INTERCEPT RBCs

At the time of RBC crossmatch and at specified times during the study [screening (Table 7.1a) during the acute transfusion support period (Table 7.1c) and at Day 28 ( $\pm 3$  days) and day 75 ( $\pm 15$  days) (**Table 7.1e**) post first study transfusion;], patient plasma/serum samples are tested for the presence of antibody specific to INTERCEPT RBCs. The RBC screening panel uses a gel card agglutination format and has been validated at the Blood Center of Wisconsin for this purpose. The primary RBC screening panel is composed of reagent RBCs from 3 blood group O donors and is analogous to routine screening panels used in regular blood banking practice. The secondary RBC screening panel is composed of reagent RBCs from 6 different blood group O donors and is analogous to secondary panels used in routine practice to identify antibody specificity for a range of common RBC allo-antigens and is used if reactivity is detected in the primary screening assay. The panel donors were specifically antigenphenotyped for major blood group systems similar to the commercially available reagent cells panels for antibody identification and differentiation. The primary and secondary RBC screening panel cells have been prepared as both INTERCEPT-treated and untreated RBCs. Each panel has three sets of RBCs made from the identical group O donors: untreated RBC; treated RBCs consisting of cells carrying a "high" level of S-303 (amustaline) adducts (comparable to the INTERCEPT RBCs prepared with the "Original process" and cells carrying a "low" level of S-303 (amustaline) adducts (representative of INTERCEPT RBCs prepared with the "Current process". The primary screening panel is designed as a sensitive screening test for both common RBC alloantibodies and for INTERCEPT RBC-specific antibodies. The secondary panel is designed to determine the specificity of any antibodies detected in the primary screen and to distinguish common RBC alloantibodies from INTERCEPT RBC-specific antibodies.

By including cells with both low and high acridine adducts there is an increased sensitivity for antibody against acridine adducts and, much in the same way that homozygous donors are used to produce commercially prepared red cells, there is a greater potential for detecting low affinity or low titer (weak) antibodies. Thus, the panels have the capability to detect an antibody specific to INTERCEPT RBCs even in the presence of alloreactivity from an intrinsic antigen.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

The patient samples are tested against the screening panel(s) of reagent RBCs to identify an antibody specific to INTERCEPT RBCs. The gel card agglutination test results are scored (0, weak positive, 1+, 2+, 3+, 4+) and the reactivity is classified as follows:

- If the antibody screening score is 0 for all the untreated and INTERCEPT RBCs on the primary RBC screening panel, the sample is considered "non-reactive" with no antibodies (neither an intrinsic alloantibody or INTERCEPT RBC-specific antibody) present in the patient's serum and thus no requirement for antibody identification with the secondary antibody identification panel. Neither the secondary RBC screening panel nor additional tests are required. The patient continues to receive study RBC components according to the protocol. In addition, each unit of study RBC is crossmatched to the patient's plasma using an antiglobulin (AHG) gel card test, providing a further level of protection to detect incompatibility, including that caused by INTERCEPT RBC-specific antibodies.
- If the results of the primary RBC screening panel show concordant 3/3, 2/3, or 1/3 reactive with BOTH the INTERCEPT treated reagent RBCs and the corresponding Control untreated RBCs, the sample will be considered "presumed allo-reactive" antibody to an intrinsic red cell antigen. The sample is tested against the secondary RBC screening panel to identify and confirm the specificity of the allo-antibody producing the reaction according to standard blood banking rules (reactivity with three RBC cells bearing the RBC antigen, and non-reactivity with three RBC that lack the antigen). If the antibody that is causing the agglutination is identified and confirmed, then the sample is considered "allo-reactive" for that RBC alloantigen. In this setting, lack of reactivity with all (at least three) INTERCEPT treated RBC cells that lack the RBC alloantigen, will rule out INTERCEPT RBC antibody specificity. The patient continues on study and will receive compatible (cross matched) study RBC components.
- If INTERCEPT RBC-specific antibodies cannot be ruled out, or agglutination is visible for all the untreated RBC cells in the panel, (i.e., "pan-reactive"), the patient will be discontinued from the study transfusions and followed up at planned visits for safety until study completion.
- If the primary RBC screening panel score is positive with 2/3 or 3/3 of the INTERCEPT RBCs carrying S-303 (amustaline) adducts at either 'high" and/or "low" level AND 0/3 with the corresponding Control untreated RBCs which lack S-303 adducts, the sample is classified as "reactive for -INTERCEPT RBC-specific antibodies" and the sample will be sent to the central testing lab for further characterization of specificity.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

Weak false positive reactions occur with serological tests due to variation in performance of the test and manual interpretation of the results (Aubuchon 2008). The provisos below are put in place to ensure that patients are not inappropriately withdrawn from the study and are in keeping with the current blood bank policies that repeat reactive results with a minimum of two tests are required for a positive test in serological viral marker assays.

Should only 1/3 INTERCEPT RBC cells in the primary panel test reactive for the S-303 labeled cells without reactivity for the untreated RBCs, that INTERCEPT RBC cell (at both high and low levels of surface bound acridine) and its untreated control will be considered "initially reactive" and the test will be repeated in duplicate on that cell only (of the three cells in the primary panel), and the secondary panel will also be tested. In this setting the secondary panel serves to increase the sensitivity for INTERCEPT RBC- specific antibodies by testing a larger number of INTERCEPT RBC cells. Negative reactivity to both repeat tests of the primary panel cell and negativity with the secondary panel will be considered a negative test. Reactivity in at least one of two repeat primary panel cells INTERCEPT RBC cells or any INTERCEPT RBC cell in the secondary panel without reactivity with the corresponding untreated RBC will be a considered positive test for INTERCEPT RBC reactivity. The sample will be sent for additional characterization at the Central immunohematology reference laboratory to include inhibition studies to determine specificity of observed reactivity. (see APPENDIX 2 for a Characterization plan for potential antibody to INTERCEPT RBCs- Addendum to the CLI 00125 Protocol).

The above-mentioned Central Laboratory protocol will ensure that the minimum criteria for discontinuation of a patient from study transfusions requires reactivity with at least two INTERCEPT RBC cells in the panel with no reactivity with the corresponding untreated control, or repeat reactivity with a single INTERCEPT RBC cell with an unreactive determination with its untreated control.

The patient will be followed up until completion of all study visits, and, if transfused with study RBCs, and evidence for clinical hemolysis will be investigated. A procedure, for patient and laboratory sample management for studies involving INTERCEPT Blood System for RBCs when a reactive S-303 result is obtained (S-303 Reactive Samples: Management of Patients and Samples; REF 01606), will be followed.

To discriminate whether an antibody with specificity for INTERCEPT RBCs is physiologically active or clinically significant, any one of the following criteria indicative of accelerated RBC clearance in the absence of active bleeding, organ-mediated RBC sequestration, severe erythroid hypoplasia or other concurrent medical

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

cause for acute anemia not associated with transfusion, should be present:

- a. During the first 7 days following transfusion, the patient's hemoglobin level has returned to the pre-transfusion level.
- b. During Days 8-14 following transfusion, patient's hemoglobin level has declined below the pre-transfusion hemoglobin level for this transfusion.

Beyond Day 14 post-transfusion, the assessment of a clinically significant change in the patient's post-transfusion hemoglobin level compared with prior responses for comparable hemoglobin doses transfused as judged by the Investigator.

Other clinical signs and symptoms that may be considered by the Investigator to judge whether accelerated RBC clearance is occurring, include:

# Extravascular hemolysis

- falling hematocrit
- increased unconjugated bilirubin ( $\geq 1.5$ -fold higher than the upper limit of normal)
- fever
- positive DAT
- micro-spherocytes on peripheral smear
- decreased or absent haptoglobin levels
- elevated reticulocyte count

# Intravascular hemolysis

- shock syndrome
- hypotension (BP lower than 90/60 mmHg)
- back pain
- plasma free hemoglobin increased
- increase in lactate dehydrogenase (LDH) ≥1.5-fold higher than the upper limit of normal (LDH ≥1.5×ULN)
- urine hemoglobin (hemoglobinuria)
- urine hemosiderin (hemosiderinuria)
- decreased or absent haptoglobin levels

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

- elevated reticulocyte count
- fragmented RBC on peripheral smear
- DAT may be positive

Plasma/serum samples for patients with confirmed antibodies specific to INTERCEPT RBCs (i.e., a DSTR, DHTR or any ATR) will be assessed for hemolytic potential according to a defined Central Laboratory protocol, provided to the sites and filed in the Investigator Site File (see APPENDIX 2) to define physiologic significance. For the purposes of this protocol, the development of a new antibody specific to INTERCEPT RBCs in the patient and with evidence of accelerated RBC clearance, in the absence of clinical alternative explanations (e.g., concomitant RBC alloantibodies, sickle cell disease, etc.) will be classified as a hemolytic transfusion reaction. All INTERCEPT RBC-specific antibodies and all hemolytic TRs will be reported to the FDA and DSMB.

# 7.3.1.11.2 Investigation of Hemolytic Potential

Investigation of the hemolytic potential of any INTERCEPT RBC-specific antibodies found in the ReCePI study will be conducted by a Central Laboratory according to the document titled "Evaluation of Reactivity with INTERCEPT RBC" provided to the sites and filed in the Investigator Site File and the protocol in APPENDIX 2. Patient samples will be managed using the supplemental instructions for patient and laboratory sample management for studies involving INTERCEPT Blood System for RBCs when a reactive S-303 result is obtained (S-303 Reactive Samples: Management of Patients and Samples; REF 01606) Possible studies may include:

- Antibody specificity via inhibition studies (inhibited by soluble acridine or not)
- Antibody characterization:
- Immunoglobulin isotype and IgG subclass (IgM, IgG<sub>1, 2, 3 or 4</sub>)
- Antibody titer
- Persistence and titer over time
- Thermal spectrum and phase of reaction
- Complement-mediated in vitro hemolysis
- Investigation of concurrent antibodies to intrinsic RBC allo-antigens
- Monocyte Monolayer Assay for clinical significance (Arndt and Garratty 2004)

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

# 7.3.1.12 Abnormal Test Findings

The criteria for determining whether an abnormal objective test finding should be reported as an adverse event are as follows:

- Test result is associated with accompanying symptoms, and/or
- Test result requires additional diagnostic testing or medical/surgical intervention, and/or
- Test result leads to a change in trial dosing or discontinuation from the study participation, significant additional concomitant drug treatment, or other therapy, and/or
- Test result is considered to be an adverse event by the Investigator or Sponsor.

Merely repeating an abnormal test, in the absence of any of the above conditions, does not constitute an adverse event. Any abnormal test result that is determined to be an error does not require reporting as an adverse event.

# 7.3.2 Methods and Timing of Safety Parameters

The use of intravenous radiographic contrast media will be documented starting 7 days prior to surgery, as will details related to the specific surgical procedure (type of procedure, start and end times), RBC components transfused, all other blood components transfused, estimated blood loss from the surgical procedure, concomitant medications, intraoperative cell recovery and reinfusion, hemodilution, and nadir temperature. Additionally, daily estimated blood loss from chest tube(s) and from other sources, and day of chest tube removal will be recorded. Safety events (TRs, AEs and SAEs) will be documented on a daily basis during the acute transfusion support period (through Day 7).

Subjects will continue to be monitored through a post-surgical follow-up period for up to 28 days after the last study transfusion, or death, whichever occurs first. During this period, subjects will be monitored for safety events. Blood samples for laboratory studies, DAT/IAT and for antibodies specific to INTERCEPT RBC- associated antigens will be obtained at 28±3 days after the last study transfusion and at end of study.

All samples obtained for determination of human leukocyte antigen (HLA) will be stored for up to 1 year after the study has completed.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

# 7.4 REPORTING PERIOD

All safety events will be collected from the start of surgery or the start of the first study transfusion (whichever is first) through 28 days after the last study transfusion or death, whichever is first.

Vital status and need for RRT of all subjects will be collected at 30 days after the end of surgery and at the end of study visit (Day  $75 \pm 15$  days).

Blood sample for assessment of sCr will be collected on post-operative day 2 (at  $48 \pm 4$  hours post end of surgery) for the primary endpoint. For non-transfused subjects, a blood sample for sCr will be drawn at  $48 \pm 4$  hours post-surgery.

Blood samples for assessment of INTERCEPT RBC-specific antibody, HLA antibodies and chemistry and hematology laboratory studies at 28±3 days after the last study transfusion.

Blood samples for assessment of INTERCEPT RBC-specific antibody will also be obtained 75  $\pm$ 15 days after the last study transfusion.

# 7.5 RECORDING AND REPORTING ADVERSE EVENTS

# 7.5.1 Assessing Severity of an Adverse Event

The Investigator will assess the severity of each adverse event based on the NCI Common Terminology Criteria for Adverse Events (CTCAE) (APPENDIX 4) and summarized in **Table 7.4**.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

# **Table 7.4 Severity Assessment of Adverse Events**

- **Grade 1**: Mild asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
- **Grade 2**: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL
- **Grade 3**: Severe or medically significant but not immediately life threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL
- Grade 4: Life-threatening consequences; urgent intervention indicated.

**Grade 5**: Death related to AE.

# Link to NCI CTCAE 5.0:

https://ctep.cancer.gov/protocoldevelopment/electronic\_applications/docs/CTCAE\_v5\_Quick\_Reference\_8.5x 11.pdf (APPENDIX 4)

Note the distinction between the severity and the seriousness of an adverse event. A severe event is not necessarily a serious event. For example, a headache may be severe (interferes significantly with patient's usual function) but would not be classified as serious unless it met one of the criteria for serious adverse events. Consistency between severity and seriousness assessments should be ensured by the Investigator.

# 7.5.2 Assessing Seriousness of an Adverse Event

The Investigator will assess if an AE resulted in any one or more of the following outcomes that result in classification of the event as an SAE: death, a life-threatening event (results in an immediate risk of death from the reaction as it occurred), inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity, a congenital anomaly/birth defect, or another important medical event (Section 7.3.1.2).

# 7.5.3 Assessing Causality of an Adverse Event

The Investigator's assessment of causality must be provided for all adverse events (serious and non-serious). An Investigator's causality assessment is the determination of whether there exists a reasonable possibility that the investigational product caused or contributed to an adverse event. If the Investigator does not know whether or not investigational product caused the event, then the event will be handled as "possibly related to investigational product" for reporting purposes.

Adverse events assessed by the Investigator to be related (possible, likely/probable) to the investigational product also must be evaluated as a Transfusion Reaction and classified per the CDC NHSN Hemovigilance Protocol (APPENDIX 3).

The standard nomenclature for defining the causal relationship between an AE and the

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

blinded study product transfused is listed in **Table 7.5**.

Table 7.5 Relationship between Investigational Product and Adverse Events

| Imputability Level | Explanation |
|---|---|
| Excluded | When there is conclusive evidence beyond reasonable doubt that the adverse event can be attributed to alternative causes |
| Unlikely | When the evidence is clearly in favor of attributing the adverse event to causes other than the study transfusion |
| Possible | When the evidence is indeterminate for attributing the adverse event to the study transfusion or an alternate cause |
| Likely/Probable | When the evidence is clearly in favor of attributing the adverse event to the study transfusion |
| Certain/Definite | When there is conclusive evidence beyond reasonable doubt that the adverse event can be attributed to the study transfusion |

# 7.5.4 Assessing Relationship to the INTERCEPT Blood System Device

The Clinical Investigator in collaboration with the blood transfusion service staff will assess whether there is a reasonable possibility that the INTERCEPT Blood System for Red Blood Cells medical device used for preparation and or processing of the blood component caused or contributed to an AE. Determination of whether there is a reasonable possibility that an INTERCEPT component caused or contributed to an AE includes assessing whether a device malfunction occurred during the preparation of the blinded study RBC component.

# 7.5.5 Reporting Requirements

The AE, SAE, and TR collection period will begin at the start of surgery or the first study RBC transfusion, whichever is first. AEs including protocol specified AEs, TRs, and SAEs (see Section 7.3) are collected daily during the acute transfusion support period and as reported through 28 days after the last study transfusion. Each AE is to be assessed to determine if it meets the criteria for an SAE. If an SAE occurs, expedited reporting will follow regional and international regulations, as appropriate. Adverse events (AEs) will not be collected for non-transfused subjects. Vital status will be reported for randomized and non-transfused subjects at the time of discontinuation.

If an SAE occurs, the Investigator must notify Cerus or its designated safety representative within 24 hours after becoming aware of the event by entering in the eCRF. When reporting SAEs to Cerus, the Investigator will ensure the report includes the severity, seriousness criteria or criterion, and causality assessments as detailed in section 7.5.

Recording the data directly into the eCRF is the preferred method to send this information to the

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

project contact for SAE receipt. In circumstances where the Investigator is unable to record the data on the eCRF, the Investigator must notify Cerus Product Safety via e-mail or the PPD Hotline within 24 hours of the site's awareness. Sponsor and Contract Research Organization (CRO) contact information is provided in **Table 7.6**.

**Table 7.6 Cerus Product Safety Contact Information** 

| Name, Title (Study Role) | Phone | Address |
|---|---|---|
| ePIP (protocol inquiries) | N/A | No longer used |
| PPD Safety Hotline<br>(SAE reporting if Medidata Rave is unavailable) | 800-201-8725 | N/A |
| Cerus Product Safety Team | N/A | ReCePISafety@cerus.com |
| Christine Ernst, MD, PhD Sr. Director, Clinical Research & Medical Affairs (Medical Monitor) | 925-288-6259 | cernst@cerus.com |
| Richard Benjamin, MD, PhD Chief Medical Officer (Back-up Medical Monitor) | 925 288-6020 | rbenjamin@cerus.com |

Investigators must also comply with local requirements for reporting SAEs to the Institutional Review Board/Ethics Committee (IRB/EC).

For all SAEs, the Investigator is obligated to pursue and provide information to Cerus or its representative in accordance with the timeframes for reporting specified above. In addition, an Investigator may be requested by Cerus or its designee to obtain specific additional follow-up information in an expedited fashion. This information may be more detailed than that captured on the adverse event case report form. In general, this will include a description of the adverse event in sufficient detail to allow for a complete medical assessment of the case and independent determination of possible causality. Information on other possible causes of the event, such as concomitant medications and illnesses must be provided. In the case of a patient death, a summary of available autopsy findings must be sent as soon as possible to Cerus or its designated representative.

# 7.5.6 Reporting Device Malfunctions

Blood centers are required to report any malfunctions of the INTERCEPT Blood System for RBCs medical device on the eCRFs. If a device malfunction impacts the

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

health of a person (patient, user or other) during the study, it may also be considered an AE/SAE. The Investigator must notify Cerus Product Safety. Sponsor contact information is provided in **Table 7.6**. If a device malfunction occurs at the participating hospitals sites, the site will complete a Device Malfunction Form.

# 7.6 DATA AND SAFETY MONITORING BOARD (DSMB) AND INTERIM ANALYSIS

The study data and safety will be monitored on a regular basis by an independent Data and Safety Monitoring Board (DSMB). The primary responsibility of the DSMB is to ensure patient safety and review protocol compliance for data collection. The DSMB will be assembled by the Sponsor and composed of transfusion medicine experts, surgeon(s) and a statistician. DSMB members will be independent of the Sponsor. The DSMB will review safety data and make recommendations according to the current DSMB charter.

Aside from the blinded interim analysis for sample size re-estimation performed in October 2021 that resulted in the reduction in study size from 600 to ≥292 patients, no other interim analysis is planned for this study to compare treatment differences with respect to efficacy or safety at any time prior to the completion of the study. Specific stopping rules, developed for safety considerations, are defined in Section 4.6.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

# 8 STATISTICS

# 8.1 STATISTICAL METHODS

# 8.1.1 Efficacy Analysis

For the primary efficacy endpoint, the treatment difference (Test – Control) and its two-sided 95% confidence interval (CI) will be estimated from Cochran-Mantel-Haenszel (CMH) test stratified by baseline sCr (sCr ≥1.2 mg/dL vs. < 1.2 mg/dL) and cardiac surgery group (more at risk for renal complications vs. less at risk) performed. The upper bound of the two-sided 95% CI will be compared with the 50% of the observed Control rate. Non-inferiority will be achieved if the upper bound is less than the 50% of the observed Control rate. For the non-inferiority test, the null and alternative hypotheses (H0 and H1, respectively) will be formulated as follows:

$$H_0: P_{Test} - P_{Control} \ge 50\% \times \hat{P}_{Control}$$
 vs.  $H_1: P_{Test} - P_{Control} < 50\% \times \hat{P}_{Control}$ 

where  $P_{Test}$  and  $P_{Control}$  are the event rates for Test (INTERCEPT) and Control groups, respectively, and  $\hat{P}_{Control}$  is the observed Control rate.

Same CMH test will be used for assessment of treatment differences for the secondary efficacy endpoints. As a sensitivity analysis, logistic regression will be utilized to estimate the treatment differences after controlling for baseline sCr, cardiac surgery group performed and other covariates to be detailed in the statistical analysis plan (SAP).

# 8.1.2 Safety Analyses

Treatment- emergent AEs (defined as AEs with an onset date/time that is on or after the start date/time of the first study transfusion) will be summarized by treatment group, system organ class (SOC), and preferred term. Descriptive summaries of safety measures will be based on observed data. No imputation of missing scores will be implemented.

# 8.1.3 Subgroup Analyses

Subgroup analysis by the randomization stratification variables (clinical site, presurgery renal impairment, and cardiac surgery group) and by demographic variables such as age group (≤18, 19 to 65, and >65 years old), sex, and race will be presented for primary and secondary efficacy endpoints.

Additional subgroup analysis may also be presented as suggested by the data.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

# 8.2 DETERMINATION OF SAMPLE SIZE

A total of at least 292 transfused subjects, approximately 146 per arm, are planned to generate sufficient efficacy and safety data for the Test and Control components in patients undergoing cardiac surgery procedures.

For the primary efficacy endpoint, a non-inferiority test will be conducted to assess for treatment difference (Test – Control). By assuming the proportion of patients with  $\Delta sCr \ge 0.3 \text{mg/dL}$  to be 30% in the Control arm and no more than 50% increase from the Control rate as the non-inferiority margin, a sample size of 292 patients (146 per arm) will provide approximately 80% power to declare non-inferiority at the two-sided 0.05 alpha level, assuming the true treatment difference is zero.

# 8.3 CRITERIA FOR TERMINATION OF THE STUDY

No statistical stopping rules for efficacy will be carried out for this trial. However, specific stopping rules for safety considerations based on development of specific immune reactivity to INTERCEPT RBCs and life-threatening or fatal adverse events will be implemented as described in **Section 4.6**.

The Sponsor may stop the trial for any reason; the reason for trial cessation will be documented.

# 8.4 HANDLING OF DROPOUTS OR MISSING DATA

For the primary analysis of the primary efficacy endpoint, missing data will be noted as such without imputation. Multiple imputation may be explored as an additional analysis.

# 8.5 DEVIATIONS FROM THE STATISTICAL PLAN

Any changes in the planned analyses specified in this protocol will be documented. The reasons for the modifications and when the changes were made will also be documented.

# 8.6 SELECTION OF SUBJECTS TO BE ANALYZED

The primary efficacy analysis group will be based on the modified intent-to-treat (mITT) population, including all randomized subjects who undergo cardiac surgery and receive one or more study RBC transfusions from randomization to within the first 48 hours post-surgery, hospital discharge, or death, whichever occurs first, and summarized under their assigned treatment group, regardless of the type of RBC components transfused.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

The safety analysis group will be based on the safety population and include all randomized subjects who have received any study transfusions during the study. Safety analyses will be performed using the Safety Population and summarizing by actual treatment group received.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

# 9 DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

Prior to participating in the study, the Investigator agrees to provide Cerus representatives or their designees direct access to source documents for trial-related monitoring and auditing. The quality representative(s) of the Sponsor may visit a clinical facility or blood center to ensure proper conduct of the protocol, recording of data, and maintenance of records.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

# 10 QUALITY CONTROL AND QUALITY ASSURANCE

# 10.1 MONITORING

During trial conduct, Cerus or its agent will conduct periodic monitoring visits to ensure that the protocol and Good Clinical Practices (GCPs) are being followed. The monitors may review source documents to confirm that the data recorded on eCRFs are accurate. The Investigator and institution will allow Cerus monitors or its agents and appropriate regulatory authorities direct access to source documents to perform this verification.

The trial site may be subject to review by the institutional review board (IRB)/independent ethics committee (IEC), and/or to quality assurance audits performed by Cerus and/or to inspection by appropriate regulatory authorities.

It is important that the Investigator(s) and their relevant personnel are available during the monitoring visits and possible audits or inspections and that sufficient time is devoted to the process.

# 10.2 INVESTIGATIONAL PRODUCT

Each red cell collection center and each processing center will be accountable for receipt and disposition of all investigational device inventory shipped to the site. All investigational devices used to manufacture the study RBC will be stored at the Blood Centers, in a secure area with access limited to authorized study personnel. Inventory records will be maintained and reviewed according to monitoring procedures.

An investigational device receiving, and dispensing record will be maintained by the Blood Centers to maintain control of investigational devices used during the study. Unused Investigational Product (IP), study RBC units, should not be returned to the Blood Center, but must be destroyed by the Hospital or Clinic Blood Bank according to the Hospital/Institution's Standard Operating Procedure (SOP). Destruction of any IP must be properly documented on the IP Accountability log.

Any device malfunction will be documented on the eCRFs. If an investigational device fails to perform in the expected manner, the Sponsor will be notified, and the event will be appropriately reported. If requested, defective devices will be returned to the Sponsor for inspection and analysis according to procedures.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

# 11 ETHICS

# 11.1 CONDUCT OF THE TRIAL

The trial will be conducted according to the protocol, the International Council on Harmonization E6 Good Clinical Practice (GCP), and applicable local/national regulatory requirements and laws.

# 11.2 PATIENT INFORMATION AND CONSENT

The informed consent/assent form must be agreed to by Cerus and the IRB/IEC and must be in compliance with ICH GCP, regional regulatory requirements, and legal requirements.

The Investigator must ensure that each trial patient, or his/her legally acceptable representative, is fully informed about the nature and objectives of the trial and possible risks associated with participation. The Investigator will obtain written informed consent/assent from each patient or the patient's legally acceptable representative before any trial-specific activity is performed. The informed consent/assent form used in this trial, and any changes made during the course of the trial, must be prospectively approved by both the IRB/IEC and Cerus before use. The investigator will retain the original of each patient's signed consent/assent form.

# 11.3 INSTITUTIONAL REVIEW BOARD (IRB)/ETHICS COMMITTEE (EC)

This protocol will be submitted to an appropriate central or local IRB/EC and its written unconditional approval obtained and submitted to Cerus or its designee before enrollment of the first subject.

Cerus will supply relevant data for Investigators to submit to the IRB/EC for the protocol's review and approval. Written verification of IRB/EC unconditional approval of the protocol and the subject Informed Consent Form (ICF)/assent form will be transmitted to Cerus or its designee prior to enrolling any subjects in the study. This approval must refer to the study by exact protocol title and number (including version), identify documents reviewed, and state the date of approval.

The Investigator must promptly report to the IRB/EC all changes in the research activity and all unanticipated problems involving risk to human subjects or others. This includes all SAEs that have resulted in an expedited safety report to the regulatory authorities (serious, unexpected AEs possibly related to investigational product). Concurrently, the Investigator must send the study Sponsor documentation of such IRB/EC notification. The Investigator must not make any changes in the research without IRB/EC approval

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

and Cerus approval, except where necessary to eliminate apparent immediate hazards to human subjects.

# 11.4 CONFIDENTIALITY

Individual subject medical information obtained as a result of this study is considered confidential, and disclosure to third parties other than those noted below is prohibited. Subject confidentiality will be further assured by utilizing subject identification code numbers to correspond to treatment data in the computer files.

However, such medical information may be given to the subject's personal physician, or to other appropriate medical personnel responsible for the subject's welfare.

In addition, data generated as a result of this study are to be available for inspection upon request by local health authority auditors, the Sponsor (including any person or companies that are working for or with or owned by the Sponsor [including monitors and auditors]), or by the IRB/EC. Therefore, absolute confidentiality cannot be guaranteed.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

# 12 DATA HANDLING AND RECORD KEEPING

# 12.1 CASE REPORT FORMS

An eCRF is required and should be completed for each included patient. The completed original eCRFs are the sole property of Cerus and should not be made available in any form to third parties, except for authorized representatives of Cerus or appropriate regulatory authorities, without written permission from Cerus.

It is the investigator's responsibility to ensure completion of, to review, and to approve all eCRFs. The eCRFs must be signed by the Investigator or by an authorized staff member. These signatures serve to attest that the information contained on the eCRFs is true. At all times, the investigator has final personal responsibility for the accuracy and authenticity of all clinical and laboratory data entered on the eCRFs. Patient source documents are the physician's patient records maintained at the trial site. In most cases, the source documents will be the hospital's or the physician's chart. In cases where the source documents are the hospital or the physician's chart, the information entered on the eCRFs must match those charts.

In some cases, the eCRF may also serve as the source document. In these cases, Cerus and the Investigator must prospectively document which items will be recorded in the source documents and for which items the eCRF will stand as the source document.

# 12.2 RECORD RETENTION

Investigators/institutions and the Sponsor shall maintain all study records required (by subpart 21CFR 812.140) during the investigation and for a period of 2 years after the latter of the following two dates: the date on which the investigation is terminated or completed, or the date that the records are no longer required for purposes of supporting a premarket approval application or a notice of completion of a product development protocol. Investigator/institution shall not destroy any such records prior to obtaining written permission from Cerus.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

# 13 LITERATURE REFERENCES

- 1. Arndt PA, Garratty G. A retrospective analysis of the value of monocyte monolayer assay results for predicting the clinical significance of blood group alloantibodies. Transfusion. 2004;44:1273-1281.
- 2. Alghamdi AA, Davis A, Brister S et al. Development and validation of Transfusion Risk Understanding Scoring Tool (TRUST) to stratify cardiac surgery patients according to their blood transfusion needs. Transfusion 2006; 46:1120-1129.
- 3. AuBuchon JP, de Wildt-Eggen J, Dumont LJ, Biomedical Excellence for Safer Transfusion C, Transfusion Medicine Resource Committee of the College of American P. Reducing the variation in performance of antibody titrations. Arch Pathol Lab Med 2008:132: 1194-201.
- 4. Bellomo R, Ronco C, Kellum JA, et al: Acute renal failure-Definition, outcome measures, animal models, fluid therapy and information technology needs: The Second International Consensus Conference of the Acute Dialysis Quality Initiative (ADQI) Group. Grit Care 2004; 8:R204-R212
- 5. Benjamin RJ, McCullough J, Mintz PD, Snyder E, Spotnitz WD, Rizzo RJ, Wages D, Lin JS, Wood L, Corash L, Conlan MG.2005. Therapeutic efficacy and safety of red blood cells treated with a chemical process (S-303) for pathogen inactivation: a Phase III clinical trial in cardiac surgery patients. Transfusion. 2005 Nov;45(11):1739-49.
- 6. Billings FT, Shaw AD. 2014. Clinical trial endpoints in acute kidney injury. Nephron Clin. Pract. 127(0):89-93.
- 7. Brecher ME and Hay SN. 2005. Bacterial Contamination of Blood Components. Clin Microbiol Rev 18(1), 195-204.
- 8. Brixner V, Kiessling AH, Madlener K et al. Clinical safety and efficacy of red blood cell components treated with the second generation S-303 pathogen and leukocyte inactivation system a randomized controlled double-blind phase 3 study in patients requiring transfusion support of acute anemia. Vox Sanguinis 2015; 109(S1):3C-S10-04. (oral presentation) [25th Regional Congress of the International Society of Blood Transfusion, 33rd Annual Conference of the British Blood Transfusion Society, London, United Kingdom Jun 27 Jul 1, 2015]
- 9. Cancelas J, Gottschall J, Rugg N et al. Red Blood Cells (RBC) Treated with the INTERCEPT Pathogen and Leukocyte Inactivation System and Stored for 35 Days Retain Viability. Transfusion 2015; Vol. 55 Supplement 3:158A-159A. (poster) [2015 American Association of Blood Banks Annual Meeting (AABB) Anaheim, Los Angeles, USA October 24 27, 2015]
- 10. Castro G, Green J, Stassinopoulos A. Effective inactivation of T-cells with S-303/GSH in human RBC as assessed by fluorescent limiting dilution assays (LDA). [Abstract P-216]. Vox Sanguinis 2016:111(Suppl. 1) 7-305.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

- 11. Chapman JF, Elliott C, et al. 2004. Guidelines for compatibility procedures in blood transfusion laboratories. Transfus Med 14(1): 59-73. doi:10.1111/j.0958-7578.2004.00482.x
- 12. Cookson ST, Arduino MJ, Aguero SM, Jarvis WR, and the *Yersinia* Study Group, Program Abstr. 36th Intersci. Conf. Antimicrob. Agents Chemother. abstr. 237, 1996.
- 13. Damgaard C, Magnussen K, Enevold C, et al.: Viable bacteria associated with red blood cells and plasma in freshly drawn blood donations. *PLoS One* 2015; 10: e0120826.
- 14. Dumont, LJ, and AuBuchon JP. Evaluation of proposed FDA criteria for the evaluation of radiolabeled red cell recovery trials. Transfusion 2008; 48(6): 1053-60.
- 15. FDA 2016. Recommendations for donor screening, deferral, and product management to reduce the risk of transfusion-transmission of Zika virus [Internet]. Silver Spring (MD):U.S. Department of Health and Human Services, Food and Drug Administration, Center for Biologics Evaluation and Research; 2016 [cited Jul 22, 2016]. Available from: http://www.fda.gov/downloads/BiologicsBloodVaccines/GuidanceComplianceRegulatoryInformation/Guidances/Blood/UCM486360.pdf
- 16. Garratty G. 2012. What is a Clinically Significant Antibody? ISBT Science Series 7: 54-57. doi:10.1111/j.1751-2824.2012.01594.x
- 17. Hillyer, C., C. Josephson, et al. (2003). Bacterial contamination of blood components: risk, strategies, and regulation: Joint ASH and AABB educational session in transfusion medicine. Hematology: 575-589.
- 18. Hobson, CE, Yavas S, et al. (2009). "Acute kidney injury is associated with increased long-term mortality after cardiothoracic surgery." Circulation 119(18): 2444-2453.
- 19. Karkouti, K. Transfusion and risk of acute kidney injury in cardiac surgery. Br J Anaesth 2012; 109 Suppl 1: i29-i38.
- 20. Kidney Disease: Improving Global Outcomes (KDIGO) Clinical Practice Guideline for Acute Kidney Injury. Kidney Int Suppl 2012; 2(Suppl 1):8; doi:10.1038/kisup.2012.1
- 21. Kleinman S and Stassinopoulos A. Risks associated with red blood cell transfusions: potential benefits from application of pathogen inactivation. Transfusion. 2015; 55(12): 2983-3000.
- 22. Kopolovic I, Ostro J, Tsubota H et al. A systematic review of transfusion-associated graft-versus- host disease. Blood 2015; 126(3): 406-414.
- 23. Kuehnert MJ, Roth VR, Haley NE et al. 2001. Transfusion-transmitted bacterial infection in the United States, 1998 through 2000. Transfusion 41:1493-1499.
- 24. Lassnigg A, Schmid ER, Hiesmayr M et al. Impact of minimal increases in serum creatinine on outcome in patients after cardiothoracic surgery: Do we have to revise current definitions of acute renal failure? Crit Care Med 2008; 36:1129-1137
- 25. Lassnigg A, Schmidlin D, Mouhieddine M et al. Minimal changes of serum creatinine predict prognosis in patients after cardiothoracic surgery: A prospective cohort study. J Am Soc Nephrol 2004; 1597-1605.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

- 26. Lee, J. 1999. U.S. Food and Drug Administration. Presented at the FDA/CBER Workshop on Bacterial Contamination of Platelets. www.FDA.gov
- 27. /CBER/minutes/bact092499.pdf.Levy MM, Fink MP, Marshall JC et al. SCCM/ESICM/ACCP/ATS/SIS International Sepsis Definitions conference. Critical Care Medicine 2003; 31:1250-1256.
- 28. Loef, B. G., A. H. Epema, et al. (2005). "Immediate postoperative renal function deterioration in cardiac surgical patients predicts in-hospital mortality and long-term survival." J Am Soc Nephrol 16(1): 195-200.
- 29. MacLennan S and Williamson LM. Risks of fresh frozen plasma and platelets. J Trauma 2006; 60 (6 Suppl):S46-50.
- 30. Mehta RH, MD, Grab JD, O'Brien SM, Bridges CR, Gammie JS, MD; Haan CK, Ferguson TB, Peterson ED, for the Society of Thoracic Surgeons National Cardiac Surgery Database Investigators. Bedside Tool for Predicting the Risk of Postoperative Dialysis in Patients Undergoing Cardiac Surgery Circulation. 2006;114:2208-2216.
- 31. Mehta RL, Kellum JA, Shah SV, et al: Acute Kidney Injury Network: Report of an initiative to improve outcomes in acute kidney injury. Crit Care 2007; 11:R31
- 32. Murphy GJ, Pike K, Rogers CA, Wordsworth S, Stokes EA, Angelini GD, Reeves BC, for the TITRe2 Investigators. Liberal or Restrictive Transfusion after Cardiac Surgery. N Engl J Med 2015; 372:997-1008.
- 33. Ness PM, Shirey RS, et al. 1990. The differentiation of delayed serologic and delayed hemolytic transfusion reactions: incidence, long-term serologic findings, and clinical significance. Transfusion 30(8): 688-693. doi:10.1046/j.1537-2995.1990.30891020325.x
- 34. O'Neal, J. B., A. D. Shaw, et al. Acute kidney injury following cardiac surgery: current understanding and future directions. Crit Care 2016; 20(1): 187
- 35. Perez P, Salmi LR, Follea G et al. 2001. Determinants of transfusion-associated bacterial contamination: results of the French BACTHEM case-control study. Transfusion 41:862-871.
- 36. Rico S, North AK, Lin J.S., Mufti N, Corash L. Cumulative Clinical Safety Experience In Acute Anemia Transfusion Support With the INTERCEPT System for Red Blood Cells (RBC). Vox Sanguinis 2015; 109 (Suppl. 2), 54 (poster P-093) [26th Regional Congress of the International Society of Blood Transfusion (ISBT) Bali, Indonesia – November 14 – 16, 2015]
- 37. SHOT, 2002. Serious Hazards of Transfusion. SHOT report for 2000-2001. Cumulative data 01/10/1995-30/09/2001) https://www.shotuk.org/shot-reports/
- 38. Siblini L, Lafeuillade B, Ros A, et al.: Influence of blood prestorage conditions and white blood cell filtration on the bacterial load of blood deliberately inoculated with Grampositive and Gram-negative pathogens. Vox Sang 2004; 87: 241-9.
- 39. Stramer SL, Hollinger FB, et al., Emerging infectious disease agents and their potential threat to 2525-2538.transfusion safety. Transfusion 2009; 49 Suppl 2: 1S-29S.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

- 40. Strobel E. Hemolytic Transfusion Reactions. Transfusion Medicine and Hemotherapy. 2008;35(5):346-353. doi:10.1159/000154811.
- 41. Theakston, E. P., A. J. Morris, S. J. Streat, B. W. Baker, and D. G. Wood- field. 1997. Transfusion transmitted Yersinia enterocolitica infection in New Zealand. Aust. N. Z. J. Med. 27:62–67T
- 42. Thygesen K, Alpert JS and White HD on behalf of the Joint ESC/ACC/AHA/WHF Task Force for the Redefinition of Myocardial Infarction. Universal definition of myocardial infarction. European Heart Journal 2007; 28:
- 43. Triulzi D, Kleinman S, Kakaiya R, Busch MP, et al. The effect of previous pregnancy and transfusion on HLA alloimmunization in blood donors: implications for a transfusion-related acute lung injury risk reduction strategy. Transfusion 2009; 49: 1825-35.
- 44. Weisbord SD, Gallagher M, Kaufman J. et al. Prevention of contrast-induced AKI: A review of published trials and design of the preservation of serious adverse events following angiography (PRESERVE) trial. Clin J Am Soc Nephrol 2013; 8:1618-1631.
- 45. Weiskopf RB, Viele MK, Feiner J et al. Human cardiovascular and metabolic response to acute, severe isovolemic anemia. JAMA 1998; 279(3):217-221.
- 46. Zhou, J., Y. Liu, et al. (2016). "A comparison of RIFLE, AKIN, KDIGO, and Cys-C criteria for the definition of acute kidney injury in critically ill patients." Int Urol Nephrol 48(1): 125-132.

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

# 14 APPENDICES

# APPENDIX 1: Transfusion Risk Understanding Scoring Tool (TRUST)

(Alghamdi AA, Davis A, Brister S, Corey P, Logan A. Development and validation of Transfusion Risk Understanding Scoring Tool (TRUST) to stratify cardiac surgery patients according to their blood transfusion needs. Transfusion 2006; 46:1120-1129.)

| Parameter | Finding | Points |
|---|---|---|
| Age of the patient in years | ≤ 65 years | 0 |
| | > 65 years | 1 |
| Sex | male | 0 |
| | female | 1 |
| hemoglobin | ≥ 13.5 g/dL | 0 |
| | < 13.5 g/dL | 1 |
| body weight in kilograms | ≥77 kilograms | 0 |
| | < 77 kilograms | 1 |
| elective surgery | yes | 0 |
| | no (non-elective) | 1 |
| serum creatinine | $\leq$ 1.36 mg/dL (120 $\mu$ mol/L) | 0 |
| | > 1.36 mg/dL (120 μmol/L) | 1 |
| history of previous cardiac surgery | no | 0 |
| | yes | 1 |
| surgical task | isolated | 0 |
| | Non-isolated (CABG + valve replacement, etc.) | 1 |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

# **Total TRUST Score** = SUM (points for all 8 parameters)

Interpretation:

minimum score: 0 maximum score: 8

The higher the score the greater the probability of requiring a blood transfusion.

| <b>Total Score</b> | Risk Group | Probability of Transfusion |
|--------------------|-------------------|----------------------------|
| 0 | baseline risk | < 20% |
| 1 | low risk | 20 - 39% |
| 2 | intermediate risk | 40 - 59% |
| 3 | high risk | 60 - 79% |
| 4 to 8 | very high risk | 80 - 100% |

X = (0.8377 \* (total score)) - 1.9503Probability of blood transfusion = 1 / (1 + EXP((-1) \* X))

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

# **APPENDIX 2: Evaluation of Reactivity with INTERCEPT RBCs**

# CHARACTERIZATION PLAN FOR POTENTIAL ANTIBODY TO INTERCEPT RBCs PROTOCOL Version 2 Addendum to CLI 00125 STUDY TITLE EVALUATION OF REACTIVITY WITH IBS RBC SPONSOR Cerus Corporation 2550 Stanwell Drive Concord, CA 94520, USA

# TEST SITE

Gregory A. Denomme, PhD, FCSMLS(D)
Director of Immunohematology &
Transfusion Services
BloodCenter of Wisconsin
638 N. 18th Street
Milwaukee, WI 53201-2178

Cerus Corporation 

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

PROTOCOL CLI 00125

# CHARACTERIZATION PLAN FOR POTENTIAL ANTIBODY TO INTERCEPT RBCs

#### 1.0 INTRODUCTION

The INTERCEPT Blood System for RBC uses the small molecule Amustaline to form covalent crosslinks within nucleic acids of contaminating pathogens and residual leukocytes, preventing their replication. Amustaline (also referred to as S-303) is a modular compound that decomposes by hydrolysis to the non-reactive compound S-300. Glutathione (GSH), a natural antioxidant, is included in the treatment process to quench unreacted S-303.

Clinical development of the INTERCEPT System for RBC initially involved a previous formulation and processing system (First Generation Process). During two Phase 3 studies (patients with acute anemia secondary to cardiovascular surgery (RBC 3A01) and patients with chronic anemia due to thalassemia or sickle cell disease (RBC 3B01) an unexpected cross-match reactivity specific to INTERCEPT RBCs was found in 2 patients in the chronic anemia study. The antibodies were low-titer (which declined to undetectable levels over 11 months) and were specific for the acridine moiety in S-303. Neither patient had demonstrable clinical evidence of accelerated red cell destruction in association with these antibodies (Benjamin et al. 2005). Follow-up evaluation demonstrated no adverse health effects and the potential for physiologic activity of the antiacridine antibody evaluated by a monocyte monolayer phagocytosis assay (Nance, et al. 1987; Arndt and Garratty 2004) indicated that these antibodies were unlikely to cause a hemolytic transfusion event. A Second Generation System was subsequently developed to reduce the density of INTERCEPT treatment-related membrane bound acridine adducts by increasing the concentration of the GSH quencher by 10-fold to 20 mM.

Using established routine methods, this document outlines the procedure for characterization of to any treatment-emergent antibody with confirmed specificity to IBS RBCs associated with clinically significant hemolysis.

At study entry and at specific times during the study, subject plasma/serum samples are tested for the presence of antibody against INTERCEPT RBC. The initial testing will be performed at the site with patient plasma or serum and Cerus Frozen Reagent RBCs using a commercial gel card IAT assay.

Cerus Corporation

CONFIDENTIAL


**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)


# CHARACTERIZATION PLAN FOR POTENTIAL ANTIBODY TO INTERCEPT RBCs

If a study site experiences positive reactivity/agglutination with patient plasma and INTERCEPT RBCs, an additional sample of plasma or serum will be sent to the central testing lab (BCW) for characterization.

#### 1.1 RESPONSIBILITIES

Clinical department management or a designated alternate at the hospital blood center and the Central Testing Laboratory at Blood Center of Wisconsin are responsible for implementing this procedure and revising it whenever necessary.

All trained personnel are responsible for performing this procedure to assure that quality standards are met.

#### 1.2 SCOPE AND OBJECTIVE

This document contains the procedure for characterization of positive reactivity with specificity (presumed or confirmed) against INTERCEPT treated RBC at any time during the study.

If a patient develops an antibody, the Investigator will collect patient samples (if possible, EDTA plasma and serum) and send them, along with the Patient Information form (FRM 00782) to the Blood Center of Wisconsin (BCW) who will act as the Central Testing Laboratory for antibody evaluation.

#### 2.0 MATERIALS AND METHOD

Lot numbers, serial numbers, and expiration dates will be recorded for all materials identified in this protocol.

- 10 x 75 mm borosilicate glass tubes (Kimble-Chase, Vineland, NJ)
- IgG gel cards, MDP081, Ortho Diagnostics, Raritan, NJ
- ID-Diluent 2, Ortho Diagnostics, Catalog number MTS9230
- Isotonic (0.85%) NaCl, EK Industries, Joliet, IL Product code 12441
- 9% w/v NaCl in H<sub>2</sub>O
- · 2.5% w/v NaCl in H20, lot numbers referenced in each appropriate section
- MLB2 Modified LISS, BioRad, Hercules, CA Reference number 8236100

Cerus Corporation 

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)


# CHARACTERIZATION PLAN FOR POTENTIAL ANTIBODY TO INTERCEPT RBCs

- Human Serum Albumin (HSA), Millipore, Kankakee, Illinois
- · Frozen Reagent RBC panels (Primary and Secondary panels)
- Monoclonal anti-acridine antibody positive control (2S-197-2M1, Antibody Solutions, Sunnyvale, CA. SPC-COA 00035)
- · 2-mercapto ethanol (Sigma Aldrich, M6250)

# For specificity determinations

- Cerus acridine compound S-300 (Lot number of compound will be recorded with the procedure)
- GSH (Identity/Code P/N 271) (Cerus SPC 00271)

#### Equipment

- · Ortho gel card incubator (Ortho Clinical; MTS9680) or equivalent
- Ortho Gel card centrifuge (Ortho Clinical; MTS5160) or equivalent

#### 3.0 REAGENT RBC PANELS

Reagent RBC panels have been prepared under contract from Cerus corp. from RBC components collected from different blood group O donors with defined red cell antigenic composition representative of the types of RBC antigens associated with clinically relevant immunologic reactions.

For the Primary "antibody detection" or "screening" panel, RBCs from 3 different donors were used and together, these 3 donor RBC components provided a reagent cell panel with a combination of intrinsic RBC antigens able to detect most clinically significant antibodies.

In addition to the "Primary 3 cell screening panel", a 6 donor RBC cell 
"Secondary identification panel" has been produced to aid identification of 
antibody should results from the Primary panel be equivocal or indeterminate. For 
the Secondary "antibody identification" panel, an additional 6 different donors 
were used, each again with specific antigen phenotypes to allow characterization 
of any positive response from the primary panel.

Cerus Corporation 

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

#### PROTOCOL CLI 00125

# CHARACTERIZATION PLAN FOR POTENTIAL ANTIBODY TO INTERCEPT RBCs

Thawing and use of Reagent frozen RBC is detailed in Cerus document INS 00593.

# 4.0 MOUSE MONOCLONAL ANTI-ACRIDINE ANTIBODY (POSITIVE CONTROL)

For each antibody analysis, a monoclonal anti-acridine antibody will be used as a positive control to demonstrate the detection of acridine on the surface of the frozen S-303 RBC panel cells. The monoclonal antibody was produced from a hybridoma obtained from a mouse immunized with KLH-conjugated S-197, a stable non-hydrolysable acridine analog of amustaline and specificity and sensitivity for acridine on the red cell surface has been extensively characterized (SUD 00734) The monoclonal antibody reacts with High and Low S303 treated RBC and fails to react with RBCs that had not been treated with INTERCEPT.

#### 5.0 PATIENT INFORMATION FORM

This information must be sent with the patient samples to the Central Testing Laboratory and include the following information:

- Patient identifier (patient ID number)
- Patient date of birth
- Patient Blood Group, including ABO and D (if available)
- Type of anticoagulant used and date of blood collection into anticoagulant
- IAT and DAT testing result
- Presence and identity of preexisting or newly acquired alloantibody against intrinsic red cell antigens
- Copies of laboratory worksheets of the tests performed identifying allo- or S-303 antibodies

Cerus Corporation 

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)


# CHARACTERIZATION PLAN FOR POTENTIAL ANTIBODY TO INTERCEPT RBCs

Any additional comments which may be useful to the Central Laboratory can be added to the last section of the form

#### 6.0 SAMPLES FOR ANALYSIS

Plasma or serum samples for antibody characterization will be prepared per Cerus INS 00733. The samples will be frozen and shipped to BCW (FRM 00781).

Gregory A. Denomme, PhD, FCSMLS(D)

Director of Immunohematology & Transfusion Services

Blood Center of Wisconsin

638 N. 18th Street, Milwaukee, WI 53201-2178

Notify the Central testing laboratory (BCW) that there is a World Courier delivery on the way by sending a copy of the Shipping Invoice by email or by FAX.

#### 7.0 SAMPLE ANAYSIS AT BCW

On arrival at BCW the plasma/serum sample will undergo extensive characterization to include confirmation of reactivity identified at the clinical site, characterization of antibody specificity, antibody titer, antibody type and subtype, and thermal amplitude. Allo-adsorption may be performed in cases with potential autoantibody and complement activations may be performed to characterize the hemolytic potential of IgM antibodies

All of the tests performed at BCW will be carried out according to their SOPs.

# 7.1 CONFIRMATION OF INTERCEPT RBC REACTIVITY WITH FROZEN RBC PANEL CELLS

The gel column agglutination technique developed and validated for use with human serum to detect antibodies to INTERCEPT RBC will be used in this characterization (VAL 00257).

As per manufacturer's recommendation,  $50~\mu L$  of Cerus Reagent RBC Primary panel cells at 0.8% hematocrit in ID-Diluent 2 (INS 00593) will be added to a

Cerus Corporation 

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)


# CHARACTERIZATION PLAN FOR POTENTIAL ANTIBODY TO INTERCEPT RBCs

column in the gel card followed by  $25~\mu L$  of patient plasma or serum and gel cards incubated at  $37^{\circ}C$  for 15 minutes in the gel card incubator (Ortho Clinical MTS 9680). After incubation, the gel cards are centrifuged with a speed of ~1000 rpm for 10 minutes (Ortho Clinical MTS 9650), the hemagglutination score will be noted as an indication of antibody bound to the RBCs (INS 00625). Using (i) High acridine, (ii) Low acridine, and (iii) untreated RBCs in a 3-cell screening procedure, reactivity to the INTERCEPT treated RBCs with no reactivity with corresponding untreated control cells is an indication that antibodies specific to S-303 RBC are present. Reactivity will also be confirmed by traditional LISS tube agglutination with and without AHG.

#### 7.2 ANTIBODY CHARACTERIZATION

#### 7.2.1 ANTIBODY TITER

Serial doubling dilutions of patient sample will be made using 6% albumin in saline as diluent to determine the positive reaction limit of the gel column agglutination assay using RBCs carrying both High and Low acridine adducts. The titer will be recorded as the inverse of the highest dilution that gave an observable, reproducible positive agglutination result with INTERCEPT treated RBCs. The accepted variation in strength of agglutination, particularly with weak reactivity, is +/- 1 doubling dilution (VAL 00257).

In conjunction, a series of doubling dilution will also be made of the murine monoclonal anti-S197 antibody as positive control using 6% albumin in saline as diluent.

#### 7.2.2 ANTIBODY SPECIFICITY BY HEMAGGLUTINATION INHIBITION

To establish specificity of patient sample reactivity, an acridine competition assay using agglutination inhibition (neutralization) with S-300 in solution (S-300 is the major acridine degradation product of INTERCEPT treated RBC) will be used (INS 00732).

Cerus Corporation 

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)


# CHARACTERIZATION PLAN FOR POTENTIAL ANTIBODY TO INTERCEPT RBCs

Patient plasma/serum (25  $\mu$ L) will be incubated with increasing concentrations of S-300 in 1.5 mL microcentrifuge tubes (5  $\mu$ L per tube) and incubated for 15 minutes at 37°C. During this time, 50  $\mu$ L of 0.8% INTERCEPT RBC (INS 00593) with high levels of acridine will be added to the upper well of the gel column. At the end of the incubation time (during which anybody in patient sample will bind to the free acridine), 25  $\mu$ L of the incubated plasma/S-300 mixture will be added to the INTERCEPT RBC in the gel card and incubated and centrifuged according to standard practice.

If the agglutination is reduced in an acridine dose-dependent manner this indicates that the antibody in the sample had specificity for acridine (S-300). As a positive control in each determination of specificity, incubation of compound with the monoclonal anti-S197 antibody will be included.

#### 7.2.3 IMMUNOGLOBULIN ISOTYPE

Gel column agglutination will be performed with monoclonal anti-IgG<sub>1</sub> & IgG<sub>3</sub> reagent in the gel cards. Reactivity in this card indicates the presence of an IgG<sub>1</sub>, IgG<sub>3</sub> or an IgM antibody. Absence of reactivity in samples that have previous reacted in anti IgG Gel cards, suggests the presence of an IgG<sub>2</sub> or IgG<sub>4</sub> subtype antibody. In order to exclude an IgM antibody, the procedure is performed with 'blank' or buffer only gel cards. Hemagglutination in a blank card (no anti-IgG, IgG1 or IgG3 reagent) is an indication that an IgM isotype antibody is present.

If an IgM antibody is suggested by the agglutination pattern in the buffer card, plasma will be treated with 2-Mercaptoenthanol (2-ME) to destroy the J-chain of IgM molecules. 2-ME treatment essentially destroys the ability of IgM to cause direct hemagglutination and will be used to further confirm the presence of IgM anti-S-303 in standard clinical tube test method. Both IgG<sub>1</sub> and IgG<sub>3</sub> isotype subclasses have the potential to activate complement and therefore the potential for causing hemolysis in vivo.

Cerus Corporation 

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)


# CHARACTERIZATION PLAN FOR POTENTIAL ANTIBODY TO INTERCEPT RBCs

#### 7.2.4 THERMAL AMPLITUDE TEST

An anti-S-303 antibody will be evaluated at different temperatures to determine the temperature range of reactivity. Standard tube tests will be performed at Room Temperature (RT) and at (or near) 37°C to determine the temperature range of reactivity. Antibodies that react at RT only are considered clinically insignificant. Antibodies that react at or near 37°C indicate the potential for binding at body temperature. Binding of antibodies at body temperature in vivo can result in their intra- or extravascular destruction, i.e. the potential for hemolysis.

#### 7.2.5 COMPLEMENT ACTIVATION

Some IgG antibodies may activate complement due to the initial binding to the RBCs, which can lead to hemolysis if this occurs in vivo. Tube tests can be performed to combine RBCs and serum at 37°C to determine if anti-S-303 antibodies can activate complement. These assays rely on an anti-globulin reagent that contains anti-C3b antibodies.

#### 7.2.6 COMPLEMENT-MEDIATED IN VITRO HEMOLYSIS

A bioassay can assess the direct potential for anti-S-303 to activate complement that proceeds to completion with an endpoint of hemolysis (Cunnion et al., 2016). In brief, serum or plasma are added in a calcium/magnesium buffer that facilitates complement activation through to C9 (complete hemolysis). The combined RBCs and serum are incubated at 37°C. Hemolysis is measured by optical density reading at 412nm. This in vitro hemolysis assay is a direct measure of the potential for hemolysis in vivo.

#### 7.2.7 MONOCYTE MONONUCLEAR ASSAY

The MMA is a sensitive and sophisticated in vitro measure of the clinical significance of antibodies to RBC. The MMA will be used to evaluate the hemolytic potential of antibodies with specificity for INTERCEPT RBCs identified in the clinical trial. MMA results, in some instances may prove inconclusive: Amdt and Garratty (2004) reported that "No patients with MMA

Cerus Corporation 

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)


# CHARACTERIZATION PLAN FOR POTENTIAL ANTIBODY TO INTERCEPT RBCs

results less than or equal to 5 percent had clinical signs of a reaction; one-third of patients with MMA results 5.1 to 20 percent versus two thirds with results greater than 20 percent had clinical signs of a Hemolytic Transfusion Reaction (HTR) after transfusion of incompatible blood." Based on these findings, Cerus will interpret the MMA results in the following way:

- INTERCEPT-RBC specific antibodies with an MMA of <5% will be declared "not clinically significant".
- INTERCEPT-RBC specific antibodies with an MMA of >20% will be declared "clinically significant".
- Should an emergent S-303 specific antibody prove to have an MMA result of 5.1-20 percent reactivity, indicative of a 30% of probability of clinical significance, Cerus will request a second patient sample taken at a later time point to seek further collaborative evidence of clinical significance, such as a rising titer, isotype class switch or increasing MMA reactivity.

#### 8.0 DEVIATIONS

Any deviations to the protocol or standard operating procedures during the performance of this study will be documented and included in the final report.

#### 9.0 DOCUMENTATION AND REPORT

Each run will be documented. Sampling and sample preparation will be recorded on data capture sheets. Upon completion of this protocol, a report for this study will be prepared.

# 10.0 DATA RETENTION

All raw data will be retained by BCW and copies will be provided to Cerus and retained in the Cerus Corporation archives, managed from 2550 Stanwell Drive, Concord, CA 94520.

Cerus Corporation 

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)


# CHARACTERIZATION PLAN FOR POTENTIAL ANTIBODY TO INTERCEPT RBCs

#### 11.0 COMPLIANCE

Unless otherwise stated, all procedures will be performed according to Cerus or BCW operating procedures.

#### REFERENCES

- Benjamin et al. 2005, "Therapeutic efficacy and safety of red blood cells treated with a chemical process (S-303) for pathogen inactivation: a Phase III clinical trial in cardiac surgery patients." Transfusion. 2005 Nov;45(11):1739-49.
- Nance, et al. 1987 "Predicting the clinical significance of red cell alloantibodies using a monocyte monolayer assay". TRANSFUSION 1987;27:449-452.
- Arndt and Garratty 2004, A retrospective analysis of the value of monocyte monolayerassay results for predicting the clinical significance of blood group alloantibodies. Transfusion Volume 44, September 2004Cunnion et al, Transfusion 2016;56:1845-8.

Cerus Corporation 

#### CHARACTERIZATION PLAN FOR POTENTIAL ANTIBODY TO INTERCEPT RBCs

#### APPENDIX 1 CERUS REFS

CLI 00033; RBC3A01

FRM 00782; "CLI 00126, PATIENT INORMATION TO ACCOMPANY SAMPLES FOR ANTIBODY INVESTIGATION AT CENTRAL TESTING LABORATORY

INS 00593; FREEZING AND THAWING OF RED BLOOD CELL SAMPLES

INS 00625; READING AND GRADING GEL CARD HEMAGGLTUINATION REACTION WITH CERUS FROZEN RED CELL PANELS

INS 00732 "AGGLUTINATION INHIBITION TO DETERMINE SPECIFICITY OF A POSITIVE REACTIVITY TO INTERCEPT TREATED RBCS IN CLI 00126"

INS 00733; PREPARATION OF SAMPLES FOR ANTIBODY CHARACTERIZATION AT A REFERENCE LABORATORY, CLI 00126"

FRM 00781 for "SHIPPING INVOICE FOR ANTIBODY TESTING SAMPLES FOR CLI 00126"

SPC-COA 00035; MOUSE MONOCLONAL ANTİBODY AGAİNST THE S-303 ANALOG, S-197 (2S197-2M1)

SUD 00734; INHÍBÍTÍON OF AGGLUTÍNATÍON WITH S-300 TO DETERMÍNE ACRÍDÍNE SPECÍFÍCÍTY OF A POSÍTÍVE REACTÍON TO INTERCEPT TREATED RBCS

VAL 00257; A VALIDATION STUDY FOR THE USE OF GEL COLUMN AGGLUTINATION TECHNOLOGY IN THE DETECTION OF IGG AND IGM SERUM AND PLASMA ANTIBODY TO S-303-TREATED RBCS

Cerus Corporation 

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

APPENDIX 3 CDC National Healthcare Safety Network Biovigilance Component Hemovigilance Module Surveillance Protocol v2.5.2

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)



# National Healthcare Safety Network Biovigilance Component Hemovigilance Module Surveillance Protocol

Division of Healthcare Quality Promotion

National Center for Emerging and Zoonotic Infectious Diseases

Centers for Disease Control and Prevention

Atlanta, GA, USA

 April 2018



**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)



NHSN Biovigilance Component Hemovigilance Module Surveillance Protocol v2.5.2 www.cdc.gov/nhsn

#### **Version History**

| Version Release Date | | Summary of Revisions |
|---|---|---|
| 1.0 | March 2009 | First version publicly released. |
| 1.1 | June 2010 | Revised background and text in main body of document. |
| | | Revised case definition criterion based on WG recommendations, pilot responses, |
| | | and CDC recommendations. |
| | | Updated FNHTR definition to allow reaction without documented fever. |
| | | Defined hypotension for infants and small children |
| | | Clarified TAGVHD probable and possible criteria. |
| 1.2 | July 2010 | Corrected definition of hypoxemia in glossary of terms. |
| 1.3 | June 2011 | Added version number and version history summary. |
| | | Summarized introduction and background sections for brevily |
| | | Reorganized surveillance methods section for ease of use. |
| | | Clarified reporting of "approved deviation" incidents. |
| | | Clarified use of "other" in adverse reaction reporting. |
| | | Clarified use of "doubtful" or "ruled out" in adverse reaction reporting. |
| | | Added denominator summary options to list of available analysis reports. |
| | | Replaced < and > signs with appropriate text for. |
| | | Added "cessation of" to time frame requirements in case definitions. |
| | | NEW probable case definition category for allergic reaction reporting. |
| | | Updated adult hypotensive reaction case definition to align with updated ISBT |
| | | definition. |
| | | NEW possible imputability category for DHTR. |
| | | DELETED possible case definition category for hypotensive reaction. |
| | | NEW probable imputability category for PTP reaction. |
| | | Updated and clarified imputability categories for TAGVHD reaction. |
| | | DELETED possible case definition category for TRALL. |
| | | Simplified imputability criteria for TTI. |
| | | Clarified case definition and impulability criteria for all adverse reactions. |
| 2.0 | January 2013 | Complete revision of organization and presentation of information |
| | | Major change in incident reporting requirements. With this release, only incidents that relate to an adverse patient reaction are required for participation. |
| | | Major change in adverse reaction reporting requirements. With this release, minor allergic reactions are no longer required for participation. |
| | | Combined the signs/symptoms with laboratory/radiology columns in case definition tables for clarity. Listed criteria in alphabetical order where possible for consistency and clarity. Moved general severity requirements from the appendix to the criteria tables where they were previously missing. |
| | | Re-ordered adverse reaction tables to put respiratory reactions first. |
| | | Added Imputability criteria of Doubtful, Ruled Out, and Not Determined to the case definition tables as OPTIONAL reporting categories. The reporting is not a change but including them in the table is new. They were added for clarity. |
| | | Added specific AHTR criteria to allow for reporting of non-immune mediated reactions. |
| | | Added a separate case definition table for Other and Unknown reactions. These categories are available for OPTONAL use. |
| | | Removed redundant and unnecessary appendices. |
| 2.1 | August 2013 | Minor revisions to verbiage throughout for clarity. |
| | 100000000000000000000000000000000000000 | Added definitions and illustration of surveillance key terms in Section 1. |
| | | Added clarification of surveillance vs. clinical definitions in Section 1. |
| | | Added less-specific case definition categories for OPTIONAL reporting of cases that do not fully meet CDC case criteria for the following reactions: hypotension, febrile non-hemolytic, acute hemolytic and delayed hemolytic. |

 April 2018



**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)



NHSN Biovigilance Component Hemovigilance Module Surveillance Protocol v2.5.2 www.cdc.gov/nhsn

| Version | Release Date Summary of Revisions | |
|---|---|---|
| | | Added a possible case definition category for TTI for OPTIONAL reporting of syndromic cases that are not laboratory confirmed. |
| 2.1.1 | September 2013 | Updated diagram in Section 1 and added version history for v2.0 and v2.1. |
| 2.1.2 | January 2014 | Updated the incident codes in Section 4 and included required reporting of discards and total crossmatch procedures on the Monthly Reporting Denominators form in Section 5. |
| 2.1.3 | August 2014 | Added a suggested citation for the surveillance protocol in Section 1. Updated the acute hemolytic case definition in Section 3 for clarity. Updated the reporting requirements in Section 5 for clarity. |
| 2.2 | January 2016 | Updated contact instructions for consistency in Section 1: User support |
| | | Updated version number in Section 1: Suggested Citation |
| | | Remove Root Cause Analysis Result from Section 4: Incident Glossary |
| | | Updated denominator report description to include Pathogen-reduced products in Section 5. Required Reporting |
| 2,3 | June 2016 | Updated denominator report description to include Table 3 description. |
| 24 | January 2017 | Section 1: Setting – Added additional Annual Facility form for Non-Acute Care Facilities to report. |
| | | Section 2: Annual Facility Survey – Added information about Non-Acute Care Facility Annual Facility Survey, Added links to the Annual Facility Survey – Non-Acute Care Facility form and table of instructions for clarity. |
| 2.5 | January 2018 | Section 1: Training, User Support, Data Reporting – Minor language changes for clarification |
| | | Section 3: Adverse Reaction Classification – Added information about module-<br>generated classification designations. |
| | | Adverse Reaction Glossary: Updated the definition of fever to be consistent with FNHTR criteria. |
| 2.5.2. | April 2018 | Section 4: Incident codes - UT 06 - "incompatible" replaced with "unapproved" |

 April 2018



**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)



NHSN Biovigilance Component Hemovigilance Module Surveillance Protocol v2.5.2 www.cdc.gov/nhsn

#### **Table of Contents**

| Section 1. Hemovigilance Module Surveillance Overview | 5 |
|---|---|
| Section 2. Hemovigilance Module Annual Facility Survey | 7 |
| Section 3: Hemovigilance Module Adverse Reactions | 8 |
| Adverse Reaction Case Classification Criteria Tables Transfusion-associated circulatory overload (TACO). Transfusion-related acute lung injury (TRALI) Transfusion-associated dyspnea (TAD). Allergic reaction | |
| Hypotensive transfusion reaction Febrile non-hemolytic transfusion reaction (FNHTR) Acute hemolytic transfusion reaction (AHTR) Delayed hemolytic transfusion reaction (DHTR) Delayed serologic transfusion reaction (DSTR) Transfusion-associated graft vs. host disease (TAGVHD) Post transfusion purpura (PTP) Transfusion-transmitted infection (TTI) Other or Unknown | 13<br>14<br>15<br>16<br>16<br>17<br>18<br>18<br>19 |
| Adverse Reaction Glossary | 23 |
| Section 4. Hemovigilance Module Incidents | 24 |
| Incident Codes | 25 |
| Occupation Codes | |
| Incident Glossary | |
| Section 5. Hemovigilance Module Denominators | 30 |

 April 2018



**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)



NHSN Biovigilance Component Hemovigilance Module Surveillance Protocol v2.5.2 www.cdc.gov/nhsn

#### Section 1. Hemovigilance Module Surveillance Overview

#### Purpose

The National Healthcare Safety Network (NHSN) Hemovigilance (HV) Module was created to implement national surveillance of transfusion-associated adverse events aimed at improving patient safety, minimizing morbidity and mortality of transfusion recipients, and identifying emerging complications and pathogens associated with blood transfusion.

#### Settings

The Hemovigilance Module may be used by any U.S. healthcare facility where blood components and manufactured blood products are transfused (e.g., adult or pediatric facilities, acute or non-acute care facilities). Surveillance must be performed facility-wide, including patient care areas for emergency, general medical, and surgical patients; obstetrics and gynecology; orthopedics, oncology, and other chronic diseases; and any other facility location where transfusions are administered.

#### Methods

The NHSN Hemovigilance Module requires comprehensive surveillance of patients and blood components throughout the transfusion process, from product receipt to administration to the patient. Participation in the NHSN Hemovigilance Module requires reporting of all adverse transfusion reactions and reaction-associated incidents that occur for patients transfused at or by your facility as well as a monthly summary of components transfused or discarded and patient samples collected for type and screen or crossmatch.

#### **Data Collection**

NHSN is a web-based application used by healthcare facilities to report surveillance data. Paper versions of all forms are used to collect data prior to data entry in the NHSN Hemovigilance Module. The paper forms are available on the <a href="NHSN Blood Safety Surveillance website">NHSN Blood Safety Surveillance website</a>. A link to the appropriate form(s) and their instructions is provided in the following sections for your convenience.

#### Training

Training presentations are available on the <a href="NHSN Blood Safety Surveillance website">NHSN Blood Safety Surveillance website</a> for self-paced training and must be reviewed prior to participating in the Hemovigilance Module. CDC also provides webinar and in-person training opportunities for current NHSN participants. These opportunities are communicated through the NHSN quarterly newsletter and emails from the Hemovigilance Team.

#### User Support

CDC is available to answer your questions about the Surveillance Protocol and to help navigate the NHSN web application. Please contact us at <a href="mailto:nhsn@cdc.gov">nhsn@cdc.gov</a>. Type **HEMOVIGILANCE** in the subject line for quickest routing to the Hemovigilance Team.

#### Suggested Citation for the Hemovigilance Module Surveillance Protocol

U.S. Centers for Disease Control and Prevention. The National Healthcare Safety Network (NHSN) Manual: Biovigilance Component v2.5. Atlanta, GA: Division of Healthcare Quality Promotion, National Center for Emerging and Zoonotic Infectious Diseases. Available at: <a href="http://www.cdc.gov/nhsn/PDFs/Biovigilance/BV-HV-protocol-current.pdf">http://www.cdc.gov/nhsn/PDFs/Biovigilance/BV-HV-protocol-current.pdf</a>. Accessed [enter date].

 April 2018



**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)



#### Key Terms (see Fig. 1)

- Adverse event: An unintended and undesirable occurrence before, during or after transfusion of blood or blood components. Adverse events include both incidents and adverse reactions.
- Adverse reaction: An undesirable response or effect in a patient temporally associated with the administration of blood or blood components. It may or may not be the result of an incident.
- Incident: Any error or accident that could affect the quality or efficacy of blood, blood components, or patient transfusions. It may or may not result in an adverse reaction in a transfusion recipient.
- Near miss: A subset of incidents that are discovered before the start of a transfusion that could
  have led to a wrongful transfusion or an adverse reaction in a transfusion recipient.

#### Data Reporting (See Fig. 1)

- . An annual facility demographic and practice survey for each calendar year of participation
- · ALL adverse reactions defined in this protocol that follow transfusion at or by your facility
- · ALL incidents (i.e., errors or accidents) associated with an adverse reaction
- The number of blood components transfused or discarded and patient samples collected for type and screen or crossmatch each month

Figure 1. Venn diagram of NHSN Hemovigilance Module surveillance terms.



**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)



NHSN Biovigilance Component Hemovigilance Module Surveillance Protocol v2.5.2 www.cdc.gov/nhsn

#### Section 2. Hemovigilance Module Annual Facility Survey

#### Required Reporting

Participating facilities must enter the Hemovigilance Module Annual Facility Survey at the time that they enroll or activate the Biovigilance Component and at the beginning of each calendar year thereafter. The survey is used by CDC to classify facilities for appropriate comparisons in aggregate data analyses and to learn more about common practices among transfusion services. The data collected in the survey covers the previous calendar year. For example, if the facility is enrolling in NHSN for the first time in October of 2013, report information for January 2012-December 2012 on the first Hemovigilance Module Annual Facility Survey. In January 2014, complete a new survey with data from January 2013-December 2013. CDC recommends collecting all survey information on a paper form before attempting to enter data into the web application.

As of January 2017, non-acute care facilities are able to report hemovigilance data to NHSN. Non-acute care facilities should complete Annual Facility Survey for Non-acute care facility 57.306. This form contains questions tailored to non-acute care facilities. Users may refer to the Non-Acute Care Facility Table of Instructions form 57.306 for detailed instruction about data collection.

#### Form

CDC 57.300 Hemovigilance Module Annual Facility Survey - Acute Care Facility

CDC 57.306 Hemovigilance Module Annual Facility Survey - Non-Acute Care Facility

#### Form Instructions

CDC 57.300 Hemovigilance Module Annual Facility Survey - Acute Care Facility Table of Instructions

CDC 57.306 Hemovigilance Module Annual Facility Survey - Non-Acute Care Facility Table of Instructions





**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)



NHSN Biovigilance Component Hemovigilance Module Surveillance Protocol v2.5.2 www.cdc.gov/nhsn

#### Section 3: Hemovigilance Module Adverse Reactions

#### Required Reporting

All CDC-defined transfusion-associated adverse reactions that are possibly, probably, or definitely related to a **transfusion performed by the participating facility** must be reported to NHSN. If a patient experiences more than one adverse reaction during or following the same transfusion episode, complete a separate form for each reaction. Adverse reaction reports should be entered into NHSN after an investigation of the reaction has been completed and imputability has been determined to the extent possible. Reports should be entered within 30 days of the month that the reaction occurred or when the investigation is completed.

#### **Optional Reporting**

Reporting suspected adverse reactions where imputability is determined to be doubtful or ruled out is not required. A facility may report reactions determined to be doubtful or ruled out in order to use NHSN to document transfusion reaction investigations each month. Adverse reactions that are not defined in the surveillance protocol may also be reported using the 'Other' and 'Unknown' adverse reaction categories; standard severity and imputability criteria are provided for that purpose.

#### Adverse Reaction Classification

Each CDC-defined transfusion-associated adverse reaction **must** be classified according to the reactionspecific case definition, severity, and imputability criteria printed in the protocol. It is imperative that every facility classify adverse reactions according to protocol definitions. Accurate classification will usually require a detailed review of the patient record.

To assist in classification, the Module will generate and assign designations for case definition, severity, and imputability based on signs, symptoms, and lab results entered in the investigation results section of the adverse reaction form.

Surveillance definitions are distinctly different from clinical definitions. Surveillance definitions are designed to capture data consistently and reliably in order to identify trends and inform quality improvement practices. The surveillance definitions are not intended as clinical diagnostic criteria or to provide treatment guidance.

#### **Defined Adverse Reactions**

- Transfusion-associated circulatory overload (TACO)
- Transfusion-related acute lung injury (TRALI)
- Transfusion-associated dyspnea (TAD)
- Allergic reaction (where severity is severe, life threatening, or death)
- Hypotensive transfusion reaction
- Febrile non-hemolytic transfusion reaction (FNHTR)
- Acute hemolytic transfusion reaction (AHTR)
- Delayed hemolytic transfusion reaction (DHTR)
- Delayed serologic transfusion reaction (DSTR)
- Transfusion-associated graft vs. host disease (TAGVHD)
- Post-transfusion purpura (PTP)
- Transfusion-transmitted infection (TTI)

#### Form

Adverse reaction forms are available at the NHSN Blood Safety Surveillance website.

#### Form Instructions

Adverse Reaction forms' Table of Instructions are available at the <u>NHSN Blood Safety Surveillance</u> <u>website</u>.

 April 2018



**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)



NHSN Biovigilance Component Hemovigilance Module Surveillance Protocol v2.5.2 www.cdc.gov/nhsn

#### Adverse Reaction Case Classification Criteria Tables

Transfusion-associated circulatory overload (TACO)

| Case Definition | Severity | Imputability |
|---|---|---|
| Definitive:<br>New onset or exacerbation | Non-severe:<br>Medical intervention (e.g. symptomatic | Definite:<br>No other explanations for circulatory |
| of 3 or more of the<br>following within 6 hours of<br>dessation of transfusion. | treatment) is required but lack of such would<br>not result in permanent damage or<br>impairment of a bodily function. | overload are possible. |
| <ul> <li>Acute respiratory distress (dyspnea,</li> </ul> | | Probable:<br>Transfusion is a likely contributor to |
| orthopnea, cough) Elevated brain | Severe:<br>Inpatient hospitalization or prolongation of | circulatory overload AND EITHER |
| natriuretic peptide<br>(BNP) | hospitalization is directly attributable to the<br>adverse reaction, persistent or significant | The patient received other fluids as<br>well |
| <ul> <li>Elevated central<br/>venous pressure<br/>(CVP)</li> </ul> | disability or incapacity of the patient occurs<br>as a result of the reaction, or a medical or<br>surgical intervention is necessary to | OR The patient has a history of cardiac insufficiency that could explain the |
| <ul> <li>Evidence of left heart failure</li> </ul> | preclude permanent damage or impairment of a body function. | circulatory overload, but<br>transfusion is just as likely to have<br>caused the circulatory overload. |
| <ul> <li>Evidence of positive<br/>fluid balance</li> </ul> | Life-threatening: | caused the circulatory overload. |
| <ul> <li>Radiographic<br/>evidence of<br/>pulmonary edema</li> </ul> | Major intervention required following the transfusion (e.g. vasopressors, inhubation, transfer to intensive care) to prevent death. | Possible:<br>The patient has a history of pre-<br>existing cardiac insufficiency that<br>most likely explains circulatory |
| Probable:<br>N/A | Death: | overload. |
| W.C. | The recipient died as a result of the | OPTIONAL |
| Possible:<br>N/A | adverse transfusion reaction. Death should be used if death is possibly, probably or definitely related to transfusion. If the patient died of a cause other than the transfusion, the severity of the reaction should be graded as appropriate | Doubtful:<br>Evidence is clearly in favor of a<br>cause other than the transfusion, but<br>transfusion cannot be excluded. |
| | given the clinical circumstances related to<br>the reaction. | Ruled Out:<br>There is conclusive evidence beyond<br>reasonable doubt of a cause other<br>than the transfusion. |
| | Not Determined:<br>The severity of the adverse reaction is | Man the Managard |
| | unknown or not stated. | Not Determined: |
| | | The relationship between the adverse reaction and the transfusion is unknown or not stated. |

 April 2018



**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)



NHSN Biovigilance Component Hemovigilance Module Surveillance Protocol v2.5.2 www.cdc.gov/nhsn

#### Transfusion-related acute lung injury (TRALI)

| Case Definition | Severity | Imputability |
|---|---|---|
| Definitive: | Non-severe: | Definite: |
| NO evidence of acute lung<br>injury (ALI) prior to<br>transfusion | Medical intervention (e.g. symptomatic treatment) is required but lack of such would not result in permanent damage or impairment of | There are no alternative risk factors for ALI present. |
| ALI onset during or within 6 hours of cessation of | a bodily function. | Probable:<br>N/A |
| transfusion | 202.00 | |
| AND | Severe: | 4000000 |
| Hypoxemia defined by any | Inpatient hospitalization or | Possible: |
| <ul> <li>PaO2/FiO2 less than or equal to 300 mm</li> </ul> | prolongation of hospitalization is<br>directly attributable to the adverse<br>reaction, persistent or significant | There is evidence of other causes for acute<br>lung injury such as: |
| Ha | disability or incapacity of the patient | Direct Lung Injury |
| <ul> <li>Oxygen saturation</li> </ul> | occurs as a result of the reaction, or a | Aspiration |
| less than 90% on | medical or surgical intervention is | Pneumonia |
| room air | necessary to preclude permanent | Toxic inhalation |
| Other clinical | damage or impairment of a body | Lung contusion |
| evidence | function. | Near drowning |
| AND | | Theat arouning |
| Radiographic evidence of | 7. 35 (1) St. 1 | Indirect Lung Injury |
| bilateral infiltrates | Life-threatening: | Severe sepsis |
| AND | Major intervention required following | Shock |
| No evidence of left atrial | the transfusion (e.g. vasopressors, | Multiple trauma |
| hypertension (i.e., | intubation, transfer to intensive care) | Burn injury |
| circulatory overload) | to prevent death. | Acute pancreatitis |
| | | <ul> <li>Cardiopulmonary bypass</li> </ul> |
| Probable: | Death: | Drug overdose |
| N/A | The recipient died as a result of the | |
| IN/A | adverse transfusion reaction. | OPTIONAL |
| | Death should be used if death is | Doubtful: |
| Possible:<br>N/A | possibly, probably or definitely<br>related to transfusion. If the patient<br>died of a cause other than the<br>transfusion, the severity of the | Evidence is clearly in favor of a cause other<br>than the transfusion, but transfusion cannot<br>be excluded. |
| | reaction should be graded as appropriate given the clinical | Ruled Out: |
| | circumstances related to the reaction. | There is conclusive evidence beyond |
| | circumstances related to the reaction. | reasonable doubt of a cause other than the transfusion. |
| | Not Determined: | 200-207 |
| | The severity of the adverse reaction | V-3-1 |
| | is unknown or not stated. | Not Determined:<br>The relationship between the adverse<br>reaction and the transfusion is unknown or<br>not stated. |

 April 2018



**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)



NHSN Biovigilance Component Hemovigilance Module Surveillance Protocol v2.5.2 www.cdc.gov/nhsn

#### Transfusion-associated dyspnea (TAD)

| Case Definition | Severity | Imputability |
|---|---|---|
| Definitive: Acute respiratory, distress occurring within 24 hours of cessation of transfusion | Non-severe: Medical intervention (e.g. symptomatic treatment) is required but lack of such would not result in permanent damage or impairment of a bodily function. | Definite:<br>Patient has no other conditions<br>that could explain symptoms. |
| AND | Taricino. | Probable: |
| Allergic reaction, TACO,<br>and TRALI definitions<br>are not applicable. | Severe:<br>Inpatient hospitalization or prolongation of<br>hospitalization is directly attributable to the | There are other potential causes<br>that could explain symptoms, but<br>transfusion is the most likely<br>cause. |
| Probable: | adverse reaction, persistent or significant disability<br>or incapacity of the patient occurs as a result of | |
| N/A | the reaction, or a medical or surgical intervention | Possible: |
| | is necessary to preclude permanent damage or<br>impairment of a body function. | Other present causes are most likely, but transfusion cannot be |
| Possible: | | ruled out. |
| N/A | And the second s | |
| | Life-threatening: | OPTIONAL |
| | Major intervention required following the<br>transfusion (e.g. vasopressors, intubation, transfer<br>to intensive care) to prevent death. | Doubtful: Evidence is clearly in favor of a cause other than the transfusion but transfusion cannot be excluded. |
| | Death: | Chalded |
| | The recipient died as a result of the adverse transfusion reaction. Death should be used if death is possibly, probably or definitely related to transfusion. If the patient died of a cause other than the transfusion, the severity of the reaction should be graded as appropriate given the clinical circumstances related to the reaction. | Ruled Out:<br>There is conclusive evidence<br>beyond reasonable doubt of a<br>cause other than the transfusion |
| | Not Determined:<br>The severity of the adverse reaction is unknown<br>or not stated. | Not Determined:<br>The relationship between the<br>adverse reaction and the<br>transfusion is unknown or not<br>stated. |

 April 2018



**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)



NHSN Biovigilance Component Hemovigilance Module Surveillance Protocol v2.5.2 www.cdc.gov/nhsn

#### Allergic reaction

Note: Minor allergic reactions (Non-severe) do not have to be reported to NHSN.

| Case Definition | Severity | Imputability |
|---|---|---|
| Case Definition Definitive: 2 or more of the following occurring during or within 4 hours of cessation of transfusion: • Conjunctival edema • Edema of lips, tongue and uvula • Erythema and edema of the periorbital area • Generalized flushing • Hypotension • Localized angioedema • Maculopapular rash • Pruritus (litching) • Respiratory distress; bronchospasm • Urticaria (hives) Probable: ANY 1 of the following occurring during or within 4 hours of cessation of transfusion: • Conjunctival edema • Edema of lips, tongue and uvula • Erythema and edema of the periorbital area • Localized angioedema • Maculopapular rash • Pruritus (litching) | Severity Severe, Life-threatening, Death: Involves respiratory and/or cardiovascular systems and presents like an anaphylactic reaction. There is anaphylaxis when, in addition to mucocutaneous symptoms, there are airway symptoms, hypotension, or associated symptoms like hypotenia and syncope. The respiratory signs and symptoms may be laryngeal (tightness in the throat, dysphagia, dysphonia, hoarseness, stridor) or pulmonary (dyspnea, cough, wheezing, bronchospasm, hypoxemia). Such a reaction usually occurs during or shortly after cessation of transfusion. Death should be used if death is possibly, probably or definitely related to transfusion. If the patient died of a cause other than the transfusion, the sevently of the reaction should be graded as appropriate given the clinical circumstances related to the reaction Not Determined: The severity of the adverse reaction is unknown or not stated. | Definite: Occurs during or within 2 hours of cessation of transfusion AND No other evidence of environmental, drug or dietary risks. Probable: Occurs during or within 2 hours of cessation of transfusion AND There are other potential causes present that could explain symptoms, but transfusion is the most likely cause. Possible: Occurs 2 - 4 hours after cessation of transfusion OR Other present causes are most likely, but transfusion cannot be ruled out. |
| OPTIONAL | OPTIONAL | OPTIONAL |
| Possible:<br>N/A | Non-severe: There is no immediate risk to the life of the patient, and the patient responds quickly to symptomatic treatment. | Doubtful: Evidence is clearly in favor of a cause other than the transfusion, but transfusion cannot be excluded. Ruled Out: There is conclusive evidence beyond reasonable doubt of a cause other than the transfusion. Not Determined: The relationship between the adverse reaction and the transfusion is unknown or not stated. |

 April 2018



**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)



NHSN Biovigilance Component Hemovigilance Module Surveillance Protocol v2.5.2 www.cdc.gov/nhsn

#### Hypotensive transfusion reaction

| Case Definition | Severity | Imputability |
|---|---|---|
| | Non-severe: | Definite: |
| Definitive: All other adverse reactions presenting with hypotension are excluded AND Hypotension occurs during or within 1 hour after cessation of transfusion. • Adults (18 years and older): Drop in systolic BP of greater than or equal to 30 mmHg and systolic BP less than or equal to 80 mmHg. • Infants, children and adolescents (1 year to less than 18 years old): Greater than 25% drop in systolic BP from baseline (e.g., drop in systolic BP of 120mmHg). • Neonates and small infants (less than 1 year old OR any age and less than 12 kg body weight): Greater than 25% drop in baseline value using whichever measurement is being recorded (e.g., mean BP). | | |
| N/A | graded as appropriate given the clinical circumstances | |
| OPTIONAL | related to the reaction. | OPTIONAL |
| Possible: | | Doubtful: |
| Hypotension occurs, does not meet the criteria above. Other, more specific reaction definitions do not apply. | Not Determined:<br>The severity of the adverse<br>reaction is unknown or not<br>stated. | Evidence is clearly in favor of a cause other than the transfusion, but transfusion cannot be excluded. Ruled Out: There is conclusive evidence beyond reasonable doubt of a cause other than the transfusion. Not Determined: |
| | | The relationship between the adverse reaction and the transfusion is unknown or not stated. |

 April 2018



**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)



NHSN Biovigilance Component Hemovigilance Module Surveillance Protocol v2.5.2 www.cdc.gov/nhsn

#### Febrile non-hemolytic transfusion reaction (FNHTR)

Note: Reactions may be classified as FNHTRs in the absence of fever if chills or rigors occur.

| Case Definition | Severity | Imputability |
|---|---|---|
| Definitive: Occurs during or within 4 hours of cessation of transfusion AND EITHER Fever (greater than or | Non-severe: Medical intervention (e.g. symptomatic treatment) is required but lack of such would not result in permanent damage or impairment of a bodily function. | Definite:<br>Patient has no other conditions<br>that could explain<br>signs/symptoms. |
| equal to 38°C/100.4°F<br>oral and a change of at<br>least 1°C/1.8°F) from pre-<br>transfusion value<br>OR<br>Chills/rigors are present. | Severe: Inpatient hospitalization or prolongation of hospitalization is directly attributable to the adverse reaction, persistent or significant disability or incapacity of the patient occurs as a result of the reaction, or a medical or surgical intervention is necessary to preclude | Probable: There are other potential causes present that could explain signs/symptoms, but transfusion is the most likely cause. Possible: |
| Probable:<br>N/A | permanent damage or impairment of a body function. | Other present causes are most likely, but transfusion cannot be ruled out. |
| OPTIONAL | Activities for the second | OPTIONAL |
| Possible:<br>FNHTR is suspected, but<br>reported symptoms and/or<br>available information are<br>not sufficient to meet the | Life-threatening: Major intervention required following the transfusion (e.g. vasopressors, intubation, transfer to intensive care) to prevent death. | Doubtful: Evidence is clearly in favor of a cause other than the transfusion, but transfusion cannot be excluded. |
| criteria defined above.<br>Other, more specific<br>adverse reaction definitions<br>do not apply. | Death: The recipient died as a result of the adverse transfusion reaction. Death should be used if death is possibly, probably or definitely related to transfusion. If the patient died of a cause other than the transfusion, the severity of the reaction should be graded as | Ruled Out:<br>There is conclusive evidence<br>beyond reasonable doubt of a<br>cause other than the transfusion. |
| | appropriate given the clinical circumstances related to the reaction. Not Determined: | Not Determined:<br>The relationship between the<br>adverse reaction and the<br>transfusion is unknown or not<br>stated. |
| | The severity of the adverse reaction is<br>unknown or not stated. | stateu. |

 April 2018



Title: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)



NHSN Biovigilance Component Hemovigilance Module Surveillance Protocol v2.5.2 www.cdc.gov/nhsn

Acute hemolytic transfusion reaction (AHTR)

Note: Report hemolytic reactions resulting from immune or non-immune causes, including when the recipient is intentionally transfused with incompatible blood components.

| Case Definition | Severity | Imputability |
|---|---|---|
| Definitive: | Non-severe: | Definite: |
| Occurs during, or within 24 hours of cessation of | Medical intervention (e.g. | ABO or other allotypic |
| transfusion with new onset of ANY of the following | symptomatic treatment) is | RBC antigen |
| signs/symploms: | required but lack of such would | incompatibility is known |
| Back/flank pain | not result in permanent | OR |
| Chills/rigors | damage or impairment of a | Only transfusion-related |
| <ul> <li>Disseminated intravascular coagulation (DIC)</li> </ul> | badily function. | (i.e., immune or non- |
| Epistaxis | | immune) cause of acute |
| Fever | | hemolysis is present. |
| <ul> <li>Hematuria (gross visual hemolysis)</li> </ul> | Severe: | |
| Hypotension | Inpatient hospitalization or | -3.00 |
| Oliguria/anuria | prolongation of hospitalization | Probable: |
| | is directly attributable to the | There are other |
| Pain and/or oozing at IV site | adverse reaction, persistent or | potential causes |
| Renal failure | significant disability or | present that could |
| AND | incapacity of the patient occurs | explain acute |
| 2 or more of the following: | as a result of the reaction, or a | hemolysis, but |
| <ul> <li>Decreased fibringen</li> </ul> | medical or surgical intervention | transfusion is the most |
| <ul> <li>Decreased haptoglobin</li> </ul> | is necessary to preclude | likely cause. |
| Elevated bilirubin | permanent damage or | |
| Elevated LDH | impairment of a body function. | |
| <ul> <li>Hemoglobinemia</li> </ul> | Contraction and account of the contraction of the c | Possible: |
| Hemoglobinuria | | Other causes of acute |
| <ul> <li>Plasma discoloration c/w hemolysis</li> </ul> | Life-threatening: | hemolysis are more |
| <ul> <li>Spherocytes on blood film</li> </ul> | Major intervention required | likely, but transfusion |
| AND EITHER | following the transfusion (e.g. | cannol be ruled out. |
| (IMMUNE-MEDIATED) | vasopressors, intubation, | 200000000000000000000000000000000000000 |
| Positive direct antiglobulin test (DAT) for anti-lgG or | transfer to intensive care) to | OPTIONAL |
| anti-C3 | prevent death. | Doubtful: |
| AND | 177 17 20 | Evidence is clearly in |
| Positive elution test with alloantibody present on the | | favor of a cause other |
| transfused red blood cells | Death: | than the transfusion, bu |
| OR | The recipient died as a result | transfusion cannot be |
| (NON-IMMUNE MEDIATED) | of the adverse transfusion | excluded. |
| Serologic testing is negative, and physical cause (e.g., | reaction. Death should be | excidied. |
| thermal, osmotic, mechanical, chemical) is confirmed. | used if death is possibly. | |
| (Standard Studies Control of Cont | probably or definitely related | Ruled Out: |
| Probable: | to transfusion. If the patient | There is conclusive |
| Meets signs and symptoms criteria for acute hemolysis. | died of a cause other than the | evidence beyond |
| AND EITHER | transfusion, the severity of the | reasonable doubt of a |
| (IMMUNE MEDIATED) | reaction should be graded as | cause other than the |
| Physical cause is excluded but serologic evidence is not | appropriate given the clinical | transfusion. |
| sufficient to meet definitive criteria | circumstances related to the | densiusium. |
| OR . | reaction. | |
| (NON-IMMUNE MEDIATED) | | Not Determined: |
| | CPC DCAP TO THE | |
| Physical cause is suspected and serologic testing is<br>negative. | Not Determined: | The relationship<br>between the adverse |
| OPTIONAL | The severity of the adverse | reaction and the |
| Possible: | reaction is unknown or not | transfusion is unknown |
| AHTR is suspected within 24 hours of cessation of | stated. | or not stated. |
| transfusion, but symptoms, test results, and/or information | - market | CO. A. A. A. S. C. C. C. |
| | 1 | |
| are not sufficient to meet the criteria defined above. Other, | | |

 April 2018



Title: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)



NHSN Biovigilance Component Hemovigilance Module Surveillance Protocol v2.5.2 www.cdc.gov/nhsn

Delayed hemolytic transfusion reaction (DHTR)

Note: Report all hemolytic reactions, including when the recipient is intentionally transfused with incompatible blood components.

| Case Definition | Severity | Imputability |
|---|---|---|
| Case Definition Definitive: Definitive: Desinitive direct antiglobulin test (DAT) for antibodies developed between 24 hours and 28 days after cessation of transfusion AND EITHER Positive elution test with alloantibody present on the transfused red blood cells OR Newly-identified red blood cell alloantibody in recipient serum AND EITHER Inadequate rise of post-transfusion hemoglobin level or rapid fall in hemoglobin back to pre-transfusion levels OR Otherwise unexplained appearance of spherocytes. Probable: Newly-identified red blood cell alloantibody demonstrated between 24 hours and 28 days after cessation of transfusion BUT Incomplete laboratory evidence to meet definitive case definition criteria. NOTE: Patient may be asymptomatic or have symptoms that are similar to but milder than AHTR; symptoms are not required to meet case definition | Non-severe: Medical intervention (e.g. symptomatic treatment) is required but lack of such would not result in permanent damage or impairment of a bodily function. Severe: Inpatient hospitalization or prolongation of hospitalization is directly attributable to the adverse reaction, persistent or significant disability or incapacity of the patient occurs as a result of the reaction, or a medical or surgical intervention is necessary to preclude permanent damage or impairment of a body function. Life-threatening: Major intervention required following the transfusion (e.g. vasopressors, intubation, transfer to intensive care) to prevent death. Death: The recipient died as a result of the adverse transfusion reaction. Death should be used if death is possibly, probably or definitely related to transfusion. | Imputability Definite: No other explanation for symptoms or newly-identified antibody is present. Probable: An alternate explanation for symptoms or newly-identified antibody is present, but transfusion is the most likely cause. Possible: Other explanations for symptoms or newly-identified antibody are more likely, but transfusion cannot be ruled out. |
| criteria. OPTIONAL | If the patient died of a cause other than the transfusion, the | OPTIONAL |
| Possible: DHTR is suspected, but reported symptoms, test results, and/or available information are not sufficient to meet the criteria defined above. Other, more specific adverse reaction definitions do not apply. | severity of the reaction should be graded as appropriate given the clinical circumstances related to the reaction. Not Determined: The severity of the adverse reaction is unknown or not stated. | Doubtful: Evidence is clearly in favor of a cause other than the transfusion, but transfusion cannot be excluded. Ruled Out: There is conclusive evidence beyond reasonable doubt of a cause other than the transfusion. Not Determined: The relationship between the adverse reaction and the transfusion is unknown or not stated. |

 April 2018



**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)



NHSN Biovigilance Component Hemovigilance Module Surveillance Protocol v2.5.2 www.cdc.gov/nhsn

# Delayed serologic transfusion reaction (DSTR)

Note: Delayed serologic reactions should only be reported for patients transfused by your facility.

| Case Definition | Severity | Imputability |
|---|---|---|
| Definitive: Absence of clinical signs of hemolysis AND Demonstration of new, clinically-significant antibodies against red blood cells BY EITHER Positive direct antiglobulin test (DAT) OR Positive antibody screen with newly identified RBC alloantibody. Probable: N/A Possible: N/A | Not Determined: Since this is by definition a reaction with no clinical symptoms, severity of the reaction cannot be graded. | Definite: New alloantibody is identified between 24 hours and 28 days after cessation of transfusion AND Transfusion performed by your facility is the only possible cause for seroconversion. Probable: New alloantibody is identified between 24 hours and 28 days after cessation of transfusion AND The patient has other exposures (e.g. transfusion by another facility or pregnancy) that could explain seroconversion, but transfusion by your facility is the most likely cause. Possible: New alloantibody is identified between 24 hours and 28 days after cessation of transfusion AND The patient was transfused by your facility, but other exposures are present that most likely explain |
| | | seroconversion. |
| | | OPTIONAL |
| | | Doubtful: Evidence is clearly in favor of a cause other than the transfusion, but transfusion cannot be excluded. |
| | | Ruled Out:<br>There is conclusive evidence beyond reasonable doubt<br>of a cause other than the transfusion. |
| | | Not Determined:<br>The relationship between the adverse reaction and the<br>transfusion is unknown or not stated. |

 April 2018



**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)



NHSN Biovigilance Component Hemovigilance Module Surveillance Protocol v2.5.2 www.cdc.gov/nhsn

#### Transfusion-associated graft vs. host disease (TAGVHD)

| Case Definition | Severity | Imputability |
|---|---|---|
| Definitive:<br>A clinical syndrome occurring from<br>2 days to 6 weeks after cessation of | Non-severe:<br>N/A | Definite:<br>WBC chimerism present in the absence of<br>alternative diagnoses. |
| transfusion characterized by: Characteristic rash: erythematous, maculopapular eruption centrally that spreads to extremities and may, in severe cases, progress to generalized erythroderma and hemorrhagic bullous formation. Diarrhea Fever Hepatomegaly Liver dysfunction (i.e., elevated ALT, AST, Alkaline | Severe: Patient had marked symptoms and responded to treatment. Life-threatening: Patient had severe symptoms and required life-saving treatment (e.g., immunosuppression). | Probable: WBC chimerism present BUT Other potential causes are present (e.g., stem cell transplantation). Possible: WBC chimerism not present or not done OR Alternative explanations are more likely (e.g., solid organ transplantation). |
| phosphatase, and bilirubin) Marrow aplasia | The recipient died as a result | OPTIONAL |
| Pancytopenia Pancytopenia AND Characteristic histological appearance of skin or liver biopsy. | of the adverse transfusion<br>reaction. Death should be<br>used if death is possibly,<br>probably or definitely<br>related to transfusion. If the<br>patient died of a cause other | Doubtful:<br>Evidence is clearly in favor of a cause<br>other than the transfusion, but transfusion<br>cannot be excluded. |
| Probable: Meets definitive criteria EXCEPT Biopsy negative or not done. | than the transfusion, the<br>severity of the reaction should<br>be graded as appropriate<br>given the clinical<br>circumstances related to the<br>reaction. | Ruled Out:<br>There is conclusive evidence beyond<br>reasonable doubt of a cause other than<br>the transfusion. |
| Possible:<br>N/A | Not Determined:<br>The severity of the adverse<br>reaction is unknown or not<br>stated. | Not Determined:<br>The relationship between the adverse<br>reaction and the transfusion is unknown or<br>not stated. |

 April 2018



**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)



NHSN Biovigilance Component Hemovigilance Module Surveillance Protocol v2.5.2 www.cdc.gov/nhsn

#### Post transfusion purpura (PTP)

| Case Definition | Severity | Imputability |
|---|---|---|
| Definitive: Alloantibodies in the patient directed against HPA or other platelet specific antigen detected at or after development of thrombocytopenia AND | Non-severe: Medical intervention (e.g. symptomatic treatment) is required but lack of such would not result in permanent damage or impairment of a bodily function. | Definite: Occurs 5-12 days post-transfusion AND Patient has no other conditions to explain thrombocytopenia. |
| Thrombocytopenia (i.e., decrease in platelets to less than 20% of pre-transfusion count). Probable: Alloantibodies in the patient directed against HPA or other platelet specific antigen detected at or after development of thrombocytopenia. AND Decrease in platelets to levels between 20% and 80% of pre-transfusion count. | Severe: Inpatient hospitalization or prolongation of hospitalization is directly attributable to the adverse reaction, persistent or significant disability or incapacity of the patient occurs as a result of the reaction, or a medical or surgical intervention is necessary to preclude permanent damage or impairment of a body function. Life-threatening: Major intervention required following the transfusion (e.g. vasopressors, | Probable: Occurs less than 5 or more than 12 days post-transfusion OR There are other potential causes present that could explain thrombocytopenia, but transfusion is the most likely cause. Possible: Alternate explanations for thrombocytopenia are more likely, but transfusion cannot be ruled out. |
| OPTIONAL | intubation, transfer to intensive care) to | OPTIONAL |
| Possible: PTP is suspected, but laboratory findings and/or information are not sufficient to meet defined criteria above. For example, the patient has a drop in platelet count to less than 80% of pre-transfusion count but HPA antibodies were not tested or were negative. Other, more specific adverse reaction definitions do not apply. | prevent death. Death: The recipient died as a result of the adverse transfusion reaction. Death should be used if death is possibly, probably or definitely related to transfusion. If the patient died of a cause other than the transfusion, the severity of the reaction should be graded as appropriate given the clinical circumstances related to the reaction. Not Determined: The severity of the adverse reaction is | Doubtful: Evidence is clearly in favor of a cause other than the transfusion, but transfusion cannot be excluded. Ruled Out: There is conclusive evidence beyond reasonable doubt of a cause other than the transfusion. Not Determined: The relationship between the adverse reaction and the transfusion is unknown or not stated. |

 April 2018



Title: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)



NHSN Biovigilance Component Hemovigilance Module Surveillance Protocol v2.5.2 www.cdc.gov/nhsn

| EL-Review Colonia, Total According | on-transmitted infe | |
|---|---|---|
| Case Definition | Severity | Imputability |
| Definitive: Laboratory evidence of a pathogen in the transfusion recipient. Probable: N/A | Non-severe: Medical intervention (e.g. symptomatic treatment) is required but lack of such would not result in permanent damage or impairment of a bodily function. Severe: Inpatient hospitalization or prolongation of hospitalization is directly attributable to the adverse reaction, persistent or significant disability or incapacity of the patient occurs as a result of the reaction, or a medical or surgical intervention is necessary to preclude permanent damage or impairment of a body function. | Definite: ONE or more of the pathogen in the transfused component Evidence of the pathogen in an additional component from the same donation Evidence of the pathogen in an additional component from the same donation Evidence of the pathogen in an additional recipient of a component from the same donation No other potential exposures to the pathogen could be identified in the recipient. AND EITHER Evidence that the recipient was not infected with the pathogen prior to transfusion OR Evidence that the identified pathogen strains are related by molecular or extended phenotypic comparison testing with statistical confidence (p<0.05). Probable: ONE or more of the following: Evidence of the pathogen in the transfused component Evidence of the pathogen in the donor at the time of donation Evidence of the pathogen in an additional component from the same donation. Evidence of the pathogen in an additional recipient of a component from the same donation. AND EITHER: Evidence that the recipient was not infected with this pathogen prior to transfusion OR No other potential exposures to the pathogen could be identified in the recipient. Possible: Case fails to meet definite, probable, doubtful, or ruled out imputability criteria. |
| | function. | |
| OPTIONAL | The Control of the Co | OPTIONAL |
| Possible: Temporally associated unexplained clinical illness consistent with infection, but no pathogen is detected in the recipient. Other, more specific adverse reactions are ruled out. Note: Possible cases cannot meet the definite or probable imputability criteria. | Life-threatening: Major intervention required following the transfusion (e.g., vasopressors, intubation, transfer to intensive care) to prevent death. Death: The recipient died as a result of the adverse transfusion reaction. Not Determined: The severity of the adverse reaction is unknown or not | Doubtful: Laboratory evidence that the recipient was infected with this pathogen prior to transfusion OR Evidence is clearly in favor of a cause other than transfusion, but transfusion cannot be excluded. Ruled Out: ALL of the following (where applicable): Evidence that the transfused component was negative for this pathogen at the time of transfusion Evidence that the donor was negative for this pathogen at the lime of donation Evidence that additional components from the same donation were negative for this pathogen OR There is conclusive evidence beyond reasonable doubt of a cause other than the transfusion. Not Determined: The relationship between the adverse reaction and the transfusion is unknown or not stated. |

 April 2018



**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)



NHSN Biovigilance Component Hemovigilance Module Surveillance Protocol v2.5.2 www.cdc.gov/nhsn

#### Transfusion-transmitted infection (TTI)

(continued

| | ratingens of well-documented importance in blood safety. |
|---|---|
| ١ | These pathogens have public health significance for hemovigilance, are well-documented blood stream |
| | pathogens, and/or are routinely screened for in blood donors. A full list of potentially infectious organisms is |
| | available in the drop down nathogen list in NHSN |

| Bacterial | Viral | Parasitic | Other |
|---|---|---|---|
| Enterobacter cloaçae Escherichia coli Klebsiella oxytoca Klebsiella preumoniae Pseudomonas aeruginosa Serratia marcescens Staphylococcus aureus Staphylococcus Eldermidis Staphylococcus (ugdunensis Syphilis (Treponema pallidum) Yersinia enterocolitica | Cytomegalovirus (CMV) Enterovirus spp. Epstein Barr (EBV) Hepatitis A Hepatitis B Hepatitis C Human Immunodeficiency Virus 1 (HIV-1) Human Immunodeficiency Virus 2 (HIV-2) Human Parvovirus B-19 Human T-Cell Lymphotropic Virus-1 (HTLV-1) Human T-Cell Lymphotropic Virus-2 (HTLV-2) West Nile Virus (WNV) Zika Virus (ZIKAVI) | Babesiosis (Babesia spp.)<br>Chagas disease<br>(Trypanosoma cruzi)<br>Malaria (Plasmodium spp.) | Creutzfeldt-<br>Jakob Disease<br>Variant (vCJD) |

#### Investigation triggers for potential transfusion-transmitted infections:

- Identification by testing (e.g., gram stain, other smear/staining, culture, or other method) of a bacterial, mycobacterial, or fungal pathogen in a recipient within the time period from exposure (i.e., transfusion) to onset of infection appropriate for the suspected pathogen.
- Identification of an unexpected virus in the transfusion recipient by testing (e.g., culture, direct fluorescent antibody, or polymerase chain reaction) within the time period from exposure (i.e., transfusion) to onset of infection appropriate for the suspected virus.
- Identification of an unexpected parasite in the recipient by testing (e.g., blood smear, histopathology, serologic testing, or polymerase chain reaction) within the time period from exposure (i.e., transfusion) to onset of infection appropriate for the suspected parasite.
- 4. Any of the above laboratory findings in the recipient unit upon residual testing.
- Unexplained clinical events occurring after transfusion that are consistent with transfusiontransmitted infection, such as:
  - a. Encephalitis, meningitis, or other unexplained central nervous system abnormalities.
  - b. Sepsis with or without multi-organ system dysfunction.
  - c. Hemolytic anemia and/or fever (e.g., in cases of transfusion-associated babesiosis or malaria).
  - d. Recipient death.
- For pathogens routinely screened in the blood donor, any infection in the recipient occurring within 6 months after transfusion if:
  - a. The index donation testing was negative but
  - b. The donor was subsequently found to be infected, and
  - c. The recipient had no pre-transfusion history of the same infection.

 April 2018



**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)



NHSN Biovigilance Component Hemovigilance Module Surveillance Protocol v2.5.2 www.cdc.gov/nhsn

#### Other or Unknown

Other: Use this option if the recipient experienced an adverse reaction that is not defined in the Hemovigilance Module surveillance protocol (e.g., transfusion-associated acute gut injury (TRAGI), transfusion-associated immunomodulation (TRIM), iron overload, microchimerism, hyperkalemia, thrombosis).

Unknown: Use this category if the patient experienced transfusion-related symptoms, but the medical event that caused those symptoms could not be classified.

Note: Reporting 'Other' and 'Unknown' reactions is not required by CDC.

| REPORTING OPTIONAL | | |
|---|---|---|
| Case Definition | Severity | Imputability |
| Not Applicable:<br>CDC does not<br>specifically define the<br>'Other' or 'Unknown'<br>adverse reaction | Non-severe: Medical intervention (e.g. symptomatic treatment) is required but lack of such would not result in permanent damage or impairment of a bodily function. | Definite: Conclusive evidence exists that the adverse reaction can be attributed to the transfusion. |
| categories, therefore<br>the case definition<br>criteria may only be<br>reported as N/A. | Severe: Inpatient hospitalization or prolongation of hospitalization is directly attributable to the adverse reaction, persistent or significant disability or incapacity of the patient occurs as a result of the reaction, or a medical or surgical intervention | Probable: Evidence is clearly in favor of attributing the adverse reaction to the transfusion. Possible: |
| | is necessary to preclude permanent damage or impairment of a body function. Life-threatening: | Evidence is indeterminate for<br>attributing the adverse reaction to<br>the transfusion or an alternate<br>cause. |
| | Major intervention required following the transfusion (e.g. vasopressors, intubation, transfer to intensive care) to prevent death. | Doubtful:<br>Evidence is clearly in favor of a<br>cause other than the transfusion, but<br>transfusion cannot be excluded. |
| | Death: The recipient died as a result of the adverse transfusion reaction. Death should be used if death is possibly, probably or definitely related to transfusion. If the patient died of a cause other than the transfusion, the severity of the reaction should be graded as appropriate given the clinical circumstances related to the reaction. | Ruled Out:<br>There is conclusive evidence<br>beyond reasonable doubt of a cause<br>other than the transfusion. |
| | Not Determined: The severity of the adverse reaction is unknown or not stated. | Not Determined:<br>The relationship between the<br>adverse reaction and the transfusion<br>is unknown or not stated. |

 April 2018



**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)



NHSN Biovigilance Component Hemovigilance Module Surveillance Protocol v2.5.2 www.cdc.gov/nhsn

#### **Adverse Reaction Glossary**

Antibodies often associated with AHTR, DHTR, DSTR:

| Anti-A | Anti-B | Anti-A,B | Anti-C | Anti-c | Anti-D | Anti-E | Anti-e | Anti-Fy <sup>a</sup> |
|---|---|---|---|---|---|---|---|---|
| | | Anti-Jkb | | | | | | |

**Bronchospasm (wheezing):** A contraction of smooth muscle in the walls of the bronchi and bronchioles, causing acute narrowing and obstruction of the respiratory airway. This constriction can result in a rasp or whistling sound while breathing.

Chills/rigors: A feeling of cold with shivering or shaking and pallor.

**Disseminated intravascular coagulation (DIC):** Bleeding disorder characterized by reduction in the factors involved in blood clotting due to their use in widespread clotting within the vessels. The intravascular clotting ultimately produces hemorrhage because of rapid consumption of clotting factors.

Edema: Swelling of soft tissues as a result of excessive fluid accumulation.

Epistaxis: Bleeding from the nose.

Fever: For the purposes of hemovigilance, greater than or equal to 38°C/100.4°F oral and a change of at least 1°C/1.8°F from pre-transfusion value.

Hematuria: Presence of blood or red blood cells in the urine.

Hemoglobinemia: The presence of free hemoglobin in the blood plasma.

Hemoglobinuria: Presence of free hemoglobin in the urine.

Hypoxemia: Abnormal deficiency in the concentration of oxygen in arterial blood, PaO2 / FiO2 less than or equal to 300 mm Hg OR oxygen saturation is less than 90% on room air.

Jaundice: New onset or worsening of yellow discoloration (icterus) of the skin or sclera (scleral icterus) secondary to an increased level of bilirubin.

Oliguria: New onset of decreased urinary output (less than 500cc output per 24 hours).

Other rash: Non-urticarial skin rash.

Pruritus: Itching.

**Shock:** A drop in blood pressure accompanied by a drop in cardiac output including rapid heart rate (increase to 100 beats per minute or more), rapid breathing, cutaneous vasoconstriction, pallor, sweating, decreased or scanty urine production, agitation and/or loss of consciousness that required fluid resuscitation, with or without inotropic support.

Shortness of breath (dyspnea): New onset or significant worsening of shortness of breath; or a significant increase in respiratory rate (with or without hypoxemia).

Urticaria (hives): Raised wheals on the skin.

 April 2018



**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)



NHSN Biovigilance Component Hemovigilance Module Surveillance Protocol v2.5.2 www.cdc.gov/nhsn

#### Section 4. Hemovigilance Module Incidents

#### Required Reporting

All incidents (i.e., accidents or errors) that are associated with a reported adverse reaction must be reported to NHSN using a detailed Incident form (CDC 57.305). If multiple incidents occur in association with an adverse reaction then report all. Incidents may occur before (e.g., wrong product released) or after (e.g., failure to report adverse reaction to blood bank) an adverse reaction. Each reaction must be reported using the detailed incident form; the incident result must be coded as 'Product transfused, reaction' to enter the associated patient identifier on the form. After the incident record is entered, the adverse reaction record must be linked to the incident record in the NHSN web application.

#### Incident Classification

Use the incident codes provided at the end of this section to classify incidents. If there is uncertainty then please contact NHSN User Support.

#### **Optional Reporting**

Any incident may be optionally reported to NHSN using the detailed Incident form (57.305) or the Monthly Incident Summary form (57.302). Approved deviations from standard operating procedure are not considered incidents because they did not occur by accident or in error. However, approved deviations may be optionally reported for a facility's use. Incidents that are optionally reported will not be aggregated or analyzed by CDC.

#### Form

CDC 57.305 Hemoviqilance Module Incident

#### Form Instructions

CDC 57.305 Hemovigilance Module Incident Table of Instructions

#### Summary Form (Optional)

CDC 57.302 Hemovigilance Module Monthly Incident Summary

#### Summary Form Instructions (Optional)

CDC 57.302 Hemovigilance Module Monthly Incident Summary Table of Instructions

 April 2018



Title: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)



NHSN Biovigilance Component Hemovigilance Module Surveillance Protocol v2.5.2 www.cdc.gov/nhsn

#### **Incident Codes**

Note: Incident codes are based on MERS TM (US) and TESS (Canada) incident classification schemes.

#### Product Check-In

(Transfusion Service)

Events that occur during the shipment and receipt of products into the transfusion service from the supplier, another hospital site, satellite storage, or clinical area

PC 00 Detail not specified

PC 01 Data entry incomplete/incorrect/not performed

PC 02 Shipment incomplete/incorrect

PC 03 Products and paperwork do not match

PC 04 Shipped/transported under inappropriate conditions

PC 05 Inappropriate return to inventory

PC 06 Product confirmation incorrect/not performed

PC 07 Administrative check not incorrect/not performed (record review/audit) PC 08 Product label incorrect/missing

#### **Product Storage**

(Transfusion Service)

Events that occur during product storage by the transfusion service.

US 00 Detail not specified

US 01 Incorrect storage conditions

US 03 Inappropriate monitoring of storage device US 04 Unit stored on incorrect shelf (e.g.,

ABO/autologous s/directed)

US 05 Incorrect storage location

#### **Inventory Management**

(Transfusion Service)

Events that involve quality management of the blood product inventory.

IM 00 Detail not specified

IM 01 Inventory audit incorrect/not performed

IM 02 Product status incorrectly/not updated online (e.g., available/discarded) IM 03 Supplier recall/traceback not appropriately

addressed/not performed IM 04 Product order incorrectly/not submitted to

supplier IM 05 Ouldated product in available inventory

IM 06 Recalled/quarantined product in available inventory

#### Product/Test Request

(Clinical Service)

Events that occur when the clinical service orders patient tests or blood products for transfusion.

PR 00 Detail not specified

PR 01 Order for wrong patient

PR 02 Order incompletely/incorrectly ordered (online order entry)

PR 03 Special processing needs not indicated (e.g., CMV negative, autologous)

PR 04 Order not done

PR 05 Inappropriate/unnecessary (intended) test ordered

PR 06 Inappropriate/unnecessary (intended) blood product ordered

PR 07 Incorrect (unintended) test ordered

PR 08 Incorrect (unintended) blood product ordered

#### Product/Test Order Entry

(Transfusion Service)

Events that occur when the transfusion service receives a patient order. This process may be excluded if clinical service uses online ordering.

OE 00 Detail not specified

OE 01 Order entered for wrong patient

OE 02 Order incompletely/incorrectly entered online

OE 03 Special processing needs not entered (e.g., CMV-, autologous)

OE 04 Order entry not done

OE 05 Inappropriate/unnecessary (intended) test order entered

OE 06 Inappropriate/unnecessary (intended) blood product order entered

OE 07 Incorrect (unintended) lest ordered

OE 08 Incorrect (unintended) blood product ordered

#### Sample Collection

(Service collecting the samples)

Events that occur during patient sample collection.

SC 00 Detail not specified

SC 01 Sample labeled with incorrect patient name

SC 02 Not labeled

SC 03 Wrong patient collected

SC 04 Collected in wrong tube type

SC 05 Sample QNS

SC 06 Sample hemolyzed

SC 07 Label incomplete/illegible/incorrect (other than patient name)

SC 08 Sample collected in error

SC 09 Requisition arrived without samples

SC 10 Wristband incorrect/not available

SC 11 Sample contaminated

 April 2018



**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)



NHSN Biovigilance Component Hemovigilance Module Surveillance Protocol v2.5.2 www.cdc.gov/nhsn

#### Incident Codes

ST 15 Sample test result misinterpreted

(continued)

Note: Incident codes are based on MERS TM (US) and TESS (Canada) incident classification schemes.

#### Sample Handling Sample Testing (continued) (Service collecting the samples) ST 16 Reagents used were Events that occur when a patient sample is sent for incorrect/inappropriate/expired/not properly OC'H testing. ST 17 ABO/Rh error caught on final check ST 18 Current/historical ABO/Rh mismatch SH 00 Detail not specified SH 01 Sample sent without requisition ST 19 Additional testing not performed SH 02 Requisition and sample label don't match ST 20 Confirmatory check incorrect/not performed (at SH 03 Patient ID incomplete/illegible on requisition time work performed) SH 04 No Patient ID on requisition SH 05 No phlebotomist/witness identification 21 Administrative check incorrect/not performed SH 06 Sample sent with incorrect requisition type (record review/audit) ST 22 Sample storage incorrect/inappropriate SH 07 Patient information (other than ID) missing/incorrect on requisition SH 08 Requisition sent without sample Product Manipulation/Processing/Testing SH 09 Data entry incorrect/incomplete/not performed (Transfusion Service) SH 10 Sample transport issue (e.g., sample Events that occur while testing, manipulating (e.g., broken/inappropriate conditions) pooling, washing, aliquoting, irradiating), processing, SH 11 Duplicate sample sent in error or labeling blood products. UM 00 Detail not specified Sample Receipt UM 01 Data entry incomplete/incorrect/not performed (Transfusion Service) UM 02 Record review incomplete/incorrect/not Events that occur when a sample is received by the performed UM 03 incorrect product (type) selected UM 04 incorrect product (patient) selected transfusion service. SR 00 Detail not specified SR 01 Sample accepted in error UM 05 Product labeled incorrectly (new/updated) SR 02 Historical review incorrect/not performed UM 06 Computer warning overridden in error or SR 03 Demographic review/ data entry incorrect/not outside SOP UM 07 Special processing needs not checked performed SR 04 Sample incorrectly accessioned UM 08 Special processing needs misunderstood or misinterpreted Sample Testing UM 09 Special processing needs performed (Transfusion Service) incorrectly UM 10 Special processing needs not performed Events that occur during patient sample testing by UM 11 Equipment problem/failure/not properly QC'd the transfusion service. UM 12 Reagents used were ST 00 Detail not specified ST 01 Data entry incomplete/incorrect/not performed incorrect/inappropriate/expired/not properly ST 02 Appropriate sample checks OC'd incomplete/incorrect/not performed UM 13 Confirmatory check incorrect/not performed (at time work performed) ST 03 Computer warning overridden in error or UM 14 Administrative check incorrect/not performed outside SOP ST 05 Sample test tube incorrectly accessioned (record review/audit) ST 07 Sample test tubes mixed up ST 09 Sample test tube mislabeled (wrong patient identifiers) ST 10 Equipment problem/failure/not properly QC'd ST 12 Sample testing not performed ST 13 Incorrect sample testing method chosen ST 14 Sample testing performed incorrectly

 April 2018



Title: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)



NHSN Biovigilance Component Hemovigilance Module Surveillance Protocol v2.5.2 www.cdc.gov/nhsn

#### **Incident Codes**

(continued)

Note: Incident codes are based on MERS TM (US) and TESS (Canada) incident classification schemes.

#### Request for Pick-up

(Clinical Service)

Events that occur when the clinical service requests pick-up of a blood product from the transfusion service.

- RP 00 Detail not specified
- RP 01 Request for pick-up on wrong patient
- RP 02 Incorrect product requested for pick-up
- RP 03 Product requested prior to obtaining consent
- RP 04 Product requested for pick-up, but patient not available
- RP 05 Product requested for pick-up, but IV not ready
- RP 06 Request for pick-up incomplete (e.g., patient ID/product type missing)
- RP 07 Pick-up slip did not match patient information on product

#### Product Issue

(Transfusion Service)

Events that occur when the transfusion service issues blood product to the clinical service

- Ul 00 Detail not specified
- UI 01 Data entry incomplete/incorrect/not performed
- UI 02 Record review incomplete/incorrect/not performed
- UI 03 Product issued for wrong patient
- UI 04 Product issued out of order
- Ul 05 Product issue delayed.
- UI 06 LIS warning overridden in error or outside SOP
- UI 07 Computer issue not completed
- UI 08 Issued visibly defective product (e.g. clots/aggregates/particulate matter)
- UI 09 Not/incorrect checking of unit and/or patient information
- Ul 10 Product transport issues (e.g., delayed) by transfusion service
- UI 11 Unit delivered to incorrect location by transfusion service
- Ul 12 Product transport issue (from transfusion
- service to clinical area)
  UI 18 Wrong product issued for intended patient (e.g. incompatible)
- Ul 19 Inappropriate product issued for patient (e.g., not irradiated, CMV+)
- UI 20 Confirmatory check incorrect/not performed (at time work performed)
- UI 21 Administrative check incorrect/not performed (record review/audit)
- UI 22 Issue approval not obtained/documented
- Ul 23 Receipt verification not performed (pneumatic tube issue)

#### Satellite Storage

(Clinical Service)

Events that occur while product is stored and handled by the clinical service.

- CS 00 Detail not specified
- CS 01 Incorrect storage conditions of product in clinical area
- CS 02 Incorrect storage location in the clinical area
- CS 03 Labeling issue (by clinical staff)
- CS 04 Floor/clinic did not check for existing products in their area
- CS 05 Product transport issues (to or between clinical areas)
- CS 06 Monitoring of satellite storage incorrect/incomplete/not performed
- CS 07 Storage tracking/documentation incorrect/incomplete/not performed

#### **Product Administration**

(Clinical Service)

Events that occur during the administration of blood products.

- UT 00 Detail not specified
- UT 01 Administered intended product to wrong patient
- UT 02 Administered wrong product to intended patient
- UT 03 Transfusion not performed in error
- UT 05 Bedside check (patient ID confirmation) incomplete/not performed
- UT 06 Transfused product with unapproved IV fluid
- UT 07 Transfusion delayed beyond pre-approved fimeframe
- UT 09 Transfused unsuitable product (e.g., outdated/inappropriately stored)
- UT 10 Administered components in wrong order UT 11 Appropriate monitoring of patient not
- performed UT 14 Transfusion volume too low (per order or SOP) UT 15 Transfusion volume too high (per order or
- SOP
- UT 16 Transfusion rate too slow (per order or SOP)
- UT 17 Transfusion rate too fast (per order or SOP)
- UT 18 Inappropriate preparation of product UT 19 Transfusion protocol not followed (not
- otherwise specified) UT 22 Order/consent check incorrect/not performed
- UT 23 Transfusion documentation incorrect/incomplete/not performed
- UT 24 Transfusion documentation not returned to
- transfusion service
- UT 26 Transfusion reaction protocol not followed

#### Other

MS 99 Other



 April 2018

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)



NHSN Biovigilance Component Hemovigilance Module Surveillance Protocol v2.5.2 www.cdc.gov/nhsn

#### **Occupation Codes**

| Laborato | ory | Addition | nal Occupation Types |
|---|---|---|---|
| IVT | IVT Team Staff | ATT | Attendant/Orderly |
| MLT | Medical Laboratory Technician | CSS | Central Supply |
| MTE | Medical Technologist | CSW | Counselor/Social Worker |
| PHL | Phlebotomist/IV Team | DIT | Dietician |
| Nursing | | DNA | Dental Assistant/Technician |
| LPN | Licensed Practical Nurse | DNH | Dental Hygienist |
| CNA | Nurse Anesthetist | DNO | Other Dental Worker |
| CNM | Certified Nurse Midwife | DNT | Dentist |
| NUA | Nursing Assistant | DST | Dental Student |
| NUP | Nurse Practitioner | FOS | Food Service |
| RNU | Registered Nurse | HSK | Housekeeper |
| Physicia | n | ICP | Infection Control Professional |
| FEL | Fellow | LAU | Laundry Staff |
| MST | Medical Student | MNT | Maintenance/Engineering |
| PHY | Attending/Staff Physician | MOR | Morgue Technician |
| RES | Intern/Resident | OAS | Other Ancillary Staff |
| Technicians | | OFR | Other First Responder |
| EMT | EMT/Paramedic | ОН | Occupational Health Professional |
| HEM | Hemodialysis Technician | OMS | Other Medical Staff |
| ORS | OR/Surgery Technician | OTH | Other |
| PCT | Patient Care Technician | OTT | Other Technician/Therapist |
| Other Pe | ersonnel | PAS | Physician Assistant |
| CLA | Clerical/Administrative | PHA | Pharmacist |
| TRA | Transport/Messenger/Porter | PHW | Public Health Worker |
| | | PLT | Physical Therapist |
| | | PSY | Psychiatric Technician |
| | | RCH | Researcher |
| | | RDT | Radiologic Technologist |
| | - | RTT | Respiratory Therapist/Technician |
| | | STU | Other Student |
| | | VOL | Volunteer |

 April 2018



**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)



NHSN Biovigilance Component Hemovigilance Module Surveillance Protocol v2.5.2 www.cdc.gov/nhsn

#### Incident Glossary

#### Incident Result

Product transfused; reaction (No recovery; harm):

A product related to this incident was transfused; the patient experienced an adverse reaction.

Product transfused; no reaction (No recovery; no harm):

A product related to this incident was transfused; the patient did not experience an adverse reaction.

No product transfused; unplanned recovery (Near miss; unplanned recovery):

No product related to this incident was transfused; the incident was discovered ad hoc, by accident, by human lucky catch, etc.

No product transfused; planned recovery (Near miss; planned recovery):

No product related to this incident was transfused; the incident was discovered through a standardized process or barrier designed to prevent errors.

 April 2018



**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)



NHSN Biovigilance Component Hemovigilance Module Surveillance Protocol v2.5.2 www.cdc.gov/nhsn

#### Section 5. Hemovigilance Module Denominators

#### Required Reporting

Facilities must report the total number of units and aliquots of specified blood components transfused and total number of discards each month. When reporting aliquots, the units from which they are made should **NOT** be counted as a transfused unit. The components transfused count should include autologous units. The total number of patient samples collected and total crossmatch procedures must also be reported. This form must be completed each month that surveillance is conducted and data can only be entered once the calendar month is over. For instance, February data must be entered after March 1st. Additionally, data cannot be entered for upcoming months.

#### Pathogen Reduced Blood Products

The total number of transfused units of blood components which are produced with pathogen-reduction technology (PRT) should be reported each month, if applicable. These PRT units are reported in Table 2 and are a subset of total number of units and aliquots transfused that are reported in Table 1. Table 3 relates to pathogen reduced apheresis platelets, if reported in table 2. For more guidance please refer to the Denominator QuickLearn on the <a href="https://www.number.org/numb

#### **Electronic Reporting**

In January 2017, the NHSN Hemovigilance Module can accept electronically reported denominator data via clinical documentation architecture (CDA). Compared to manual reporting, electronic reporting will decrease the time required for data collection and reporting, reduce data entry errors, and increase data granularity. In order to electronically report data, facilities' software system must have CDA functionality. For more information about electronic reporting and CDA, review CDA Frequently Asked Questions on the NHSN Blood Safety Surveillance website.

#### Form

CDC 57.303 Hemovigilance Module Monthly Reporting Denominators

#### Form Instructions

CDC 57.303 Hemovigilance Module Monthly Reporting Denominators Tables of Instructions

 April 2018



**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

APPENDIX 4: Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 Published: November 27, 2017

# Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0

Published: November 27, 2017

U.S. DEPARTMENT OF HEALTH AND HUMAN SERVICES

#### Common Terminology Criteria for Adverse Events (CTCAE) v5.0 Publish Date: November 27, 2017

#### Introduction

The NCI Common Terminology Criteria for Adverse Events is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term.

#### SOC

System Organ Class (SOC), the highest level of the MedDRA<sup>1</sup> hierarchy, is identified by anatomical or physiological system, etiology, or purpose (e.g., SOC Investigations for laboratory test results). CTCAE terms are grouped by MedDRA Primary SOCs. Within each SOC, AEs are listed and accompanied by descriptions of severity (Grade).

#### CTCAE Terms

An Adverse Event (AE) is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may <u>not</u> be considered related to the medical treatment or procedure. An AE is a term that is a unique representation of a specific event used for medical documentation and scientific analyses. Each CTCAE v4.0 term is a MedDRA LLT (Lowest Level Term).

#### Grades

Grade refers to the severity of the AE. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline:

Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.

Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting ageappropriate instrumental ADL\*.

Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL\*\*.

Grade 4 Life-threatening consequences; urgent intervention indicated.

Grade 5 Death related to AE.

A Semi-colon indicates 'or' within the description of the grade.

A single dash (-) indicates a Grade is not available. Not all Grades are appropriate for all AEs. Therefore, some AEs are listed with fewer than five options for Grade selection.

#### Grade 5

Grade 5 (Death) is not appropriate for some AEs and therefore is not an option.

#### Definitions

A brief Definition is provided to clarify the meaning of each AE term. A single dash (-) indicates a Definition is not available.

#### Navigational Notes

A Navigational Note is used to assist the reporter in choosing a correct AE. It may list other AEs that should be considered in addition to <u>or</u> in place of the AE in question. A single dash (-) indicates a Navigational Note has not been defined for the AE term

#### Activities of Daily Living (ADL)

- \*Instrumental ADL refer to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.
- \*\*Self care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.

<sup>1</sup> CTCAE v5.0 incorporates certain elements of the MedDRA terminology. For further details on MedDRA refer to the MedDRA MSSO Web site (https://www.meddra.org/);

#### **Table of Contents**

| Blood and lymphatic system disorders | 4 |
|---------------------------------------------------------------------|-----|
| Cardiac disorders | 6 |
| Congenital, familial and genetic disorders | 12 |
| Ear and labyrinth disorders | 13 |
| Endocrine disorders | 15 |
| Eye disorders | 18 |
| Gastrointestinal disorders | 24 |
| General disorders and administration site conditions | 44 |
| Hepatobiliary disorders | 48 |
| Immune system disorders | 51 |
| Infections and infestations | 53 |
| Injury, poisoning and procedural complications | 70 |
| Investigations | 84 |
| Metabolism and nutrition disorders | 91 |
| Musculoskeletal and connective tissue disorders | 95 |
| Neoplasms benign, malignant and unspecified (incl cysts and polyps) | 103 |
| Nervous system disorders | 104 |
| Pregnancy, puerperium and perinatal conditions | 114 |
| Psychiatric disorders | |
| Renal and urinary disorders | 119 |
| Reproductive system and breast disorders | 123 |
| Respiratory, thoracic and mediastinal disorders | 131 |
| Skin and subcutaneous tissue disorders | 142 |
| Social circumstances | 150 |
| Surgical and medical procedures | 151 |
| Vascular disorders | 152 |
| | | Blood and lymphatic system | disorders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Anemia | Hemoglobin (Hgb) <lln -="" 10.0<br="">g/dL; <lln -="" 6.2="" <lln<br="" l;="" mmol="">- 100 g/L</lln></lln> | Hgb <10.0 - 8.0 g/dL; <6.2 - 4.9<br>mmol/L; <100 - 80g/L | Hgb <8.0 g/dL; <4.9 mmol/L;<br><80 g/L; transfusion indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | erized by a reduction in the amount o<br>ath, palpitations of the heart, soft syst | | | nclude pallor of the skin and mucc | ous |
| Bone marrow hypocellular | Mildly hypocellular or <=25%<br>reduction from normal<br>cellularity for age | Moderately hypocellular or<br>>25 - <50% reduction from<br>normal cellularity for age | Severely hypocellular or >50 -<br><=75% reduction cellularity<br>from normal for age | Aplastic persistent for longer<br>than 2 weeks | Death |
| | terized by the inability of the bone ma | rrow to produce hematopoietic ele | ments. | | |
| Navigational Note: -<br>Disseminated intravascular<br>coagulation | - | Laboratory findings with no<br>bleeding | Laboratory findings and bleeding | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| risk of hemorrhage as the boo | terized by systemic pathological activa<br>dy is depleted of platelets and coagula | | which results in clot formation thro | ughout the body. There is an incre | ase in the |
| Navigational Note: - | >ULN and >Baseline | 1 | Steroids initiated | T | 1 |
| Eosinophilia | | l <sup>-</sup> | | l - | - |
| | terized by laboratory test results that i | ndicate an increased number of eo: | sinophils in the blood. | | |
| Navigational Note: - | | 1 | Languages and the | Liera | 1 p |
| Febrile neutropenia | | - | ANC <1000/mm3 with a single temperature of >38.3 degrees C (101 degrees F) or a sustained temperature of >=38 degrees C (100.4 degrees F) for more than one hour | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| F) for more than one hour. | terized by an ANC <1000/mm3 and a s | ingle temperature of >38.3 degrees | C (101 degrees F) or a sustained te | mperature of >=38 degrees C (100 | ).4 degrees |
| Navigational Note: - | 1 | | T = | Lieur | 1 |
| Hemolysis | Laboratory evidence of<br>hemolysis only (e.g., direct<br>antiglobulin test; DAT;<br>Coombs'; schistocytes;<br>decreased haptoglobin) | Evidence of hemolysis and<br>>=2 g decrease in hemoglobin | Transfusion or medical intervention indicated (e.g., steroids) | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder charact | terized by laboratory test results that i | ndicate widespread erythrocyte cel | l membrane destruction. | | |
| Navigational Note: - | | | | | |

| | | Blood and lymphatic system | disorders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Hemolytic uremic syndrome | - | - | Laboratory findings with clinical consequences (e.g., renal insufficiency, petechiae) | Life-threatening<br>consequences, (e.g., CNS<br>hemorrhage or<br>thrombosis/embolism or renal<br>failure) | Death |
| <b>Definition:</b> A disorder characteri<br><b>Navigational Note:</b> - | zed by a form of thrombotic microa | ngiopathy with renal failure, hemo | lytic anemia, and severe thrombocy | rtopenia. | |
| Leukocytosis | - | - | >100,000/mm3 | Clinical manifestations of<br>leucostasis; urgent<br>intervention indicated | Death |
| | zed by laboratory test results that i | ndicate an increased number of wh | ite blood cells in the blood. | | |
| Navigational Note: -<br>Lymph node pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteri | zed by a sensation of marked discor | mfort in a lymph node. | • | • | • |
| Navigational Note: - | | | | | |
| Methemoglobinemia | - | >ULN | Requiring urgent intervention | Life-threatening consequences | Death |
| Definition: A disorder characteri | zed by laboratory test results that i | ndicate increased methemoglobin i | n the blood. | | |
| Navigational Note: - | | | | | |
| Thrombotic thrombocytopenic purpura | - | - | Laboratory findings with dinical consequences (e.g., renal insufficiency, petechiae) | Life-threatening consequences, (e.g., CNS hemorrhage or thrombosis/embolism or renal failure) | Death |
| | zed by the presence of microangion<br>al disturbances. It is an acute or sub | | ytopenic purpura, fever, renal abno | rmalities and neurological abnorma | alities such |
| Navigational Note: - | | | | | |
| Blood and lymphatic system disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: -<br>Navigational Note: - | | | | | |

| | | Cardiac disorders | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Aortic valve disease | Asymptomatic valvular thickening with or without mild valvular regurgitation or stenosis by imaging | Asymptomatic; moderate regurgitation or stenosis by imaging | Symptomatic; severe<br>regurgitation or stenosis by<br>imaging; symptoms controlled<br>with medical intervention | Life-threatening<br>consequences; urgent<br>intervention indicated (e.g.,<br>valve replacement,<br>valvuloplasty) | Death |
| <b>Definition:</b> A disorder chara-<br><b>Navigational Note:</b> - | cterized by a defect in aortic valve func | tion or structure. | | | |
| Asystole | Periods of asystole; non-<br>urgent medical management<br>indicated<br>cterized by a dysrhythmia without card | - | - | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Navigational Note: - | cterized by a dysrnythrilla without card | пас егеситсаг асцуну. тургсану, ит | is is accompanied by cessation of the | pumping lunction of the neart. | |
| Atrial fibrillation | Asymptomatic, intervention not indicated | Non-urgent medical<br>intervention indicated | Symptomatic, urgent intervention indicated; device (e.g., pacemaker); ablation; new onset | Life-threatening<br>consequences; embolus<br>requiring urgent intervention | Death |
| originates above the ventric | cterized by a dysrhythmia without disco<br>les. | ernible P waves and an irregular ve | entricular response due to multiple re | eentry circuits. The rhythm disturb | ance |
| Navigational Note: -<br>Atrial flutter | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Symptomatic, urgent intervention indicated; device (e.g., pacemaker); ablation | Life-threatening<br>consequences; embolus<br>requiring urgent intervention | Death |
| atria. | cterized by a dysrhythmia with organiz | ed rhythmic atrial contractions wit | th a rate of 200-300 beats per minute | a. The rhythm disturbance originate | es in the |
| Navigational Note: - | | T | T: . | Lieut | I n d |
| Atrioventricular block complete | | Non-urgent intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker); new onset | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder chara- | cterized by a dysrhythmia with comple | te failure of atrial electrical impuls | e conduction through the AV node to | the ventrides. | |
| Navigational Note: - | | | | | |

| ### Actional Properties Figure Fig | | | Cardiac disorders | | | |
|---|---|---|---|---|---|---|
| degree not indicated indicated indicated indicated indicated paths that a delay in the time required for the conduction of an electrical impulse through the atrioventricular (AV) node beyond 0.2 seconds; prolongation of the PR interval greater than 200 milliseconds. Navigational Note: Cardiac arrest Life-threatening consequences; urgent intervention indicated intervention indicat | CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Definition: A disorder characterized by a dysrhythmia with a delay in the time required for the conduction of an electrical impulse through the atrioventricular (AV) node beyond 0.2 seconds; prolongation of the PR interval greater than 200 milliseconds. Navigational Note: Cardiac arrest Definition: A disorder characterized by cessation of the pumping function of the heart. Navigational Note: Chest pain - cardiac Mild pain Moderate pain; pain on exertion; limiting instrumental ADL; hemodynamically stable and exertion; limiting instrumental ADL; hemodynamically stable and exertion; unstable angina Definition: A disorder characterized by substernal discomfort due to insufficient myocardial exegenation e.g., angine pectoris. Navigational Note: Also consider Cardiac disorders: Myocardial infarction. Conduction disorder Mild symptoms; intervention Non-urgent medical intervention indicated consequences Definition: A disorder characterized by a pathological irregularities in the cardiac conduction system. Navigational Note: Present Present Asymptomatic with laboratory (e.g., BNP [B-Natriuretic Peptide]) or cardiac imaging abnormalities Asymptomatic with laboratory activity or exertion hospitalization; new onset of symptoms at rest or with minimal activity or exertion; hospitalization; new onset of symptoms or mechanical hemodynamic support) Definition: A disorder characterized by the inability of the heart to pump blood at an adequate volume to meet tissue metabolic requirements, or, the ability to do so only at an adequate volume to meet tissue metabolic requirements, or, the ability to do so only at an adequate volume to meet tissue metabolic requirements, or, the ability to do so only at an adequate volume to meet tissue metabolic requirements, or, the ability to do so only at an adequate volume to meet tissue metabolic requirements, or, the ability to do so only at an adequate volume | Atrioventricular block first | Asymptomatic, intervention | Non-urgent intervention | - | - | - |
| Seconds; prolongation of the PR interval greater than 200 milliseconds. Navigational Note: - Cardiac arrest | | | | | | |
| Navigational Note: - Cardiac arrest | | | | ion of an electrical impulse through | ı the atrioventricular (AV) node bey | ond 0.2 |
| Cardiac arrest | | interval greater than 200 millisecon | nds. | | | |
| Definition: A disorder characterized by cessation of the pumping function of the heart. Navigational Note: - Chest pain - cardiac | - | | | | | |
| Definition: A disorder characterized by cessation of the pumping function of the heart. Navigational Note: - Chest pain - cardiac Mild pain Moderate pain; pain on exertion; limiting instrumental ADL; hemodynamically stable angina Definition: A disorder characterized by substernal discomfort due to insufficient myocardial exygenation e.g., angina pectoris. Navigational Note: Also consider Cardiac disorders: Myocardial infarction. Conduction disorder Mild symptoms; intervention not indicated intervention indicated intervention indicated intervention indicated intervention indicated consequences Definition: A disorder characterized by pathological irregularities in the cardiac conduction system. Navigational Note: - Cyanosis Present Present Present Symptoms at rest or with minimal activity or exertion; hospitalization; new onset of symptoms Bymptoms at rest or with minimal activity or exertion; hospitalization; new onset of symptoms symptoms Death consequences; urgent intervention indicated (e.g., continuous IV therapy or mechanical hemodynamic support) Definition: A disorder characterized by the inability of the heart to pump blood at an adequate volume to meet tissue metabolic requirements, or, the ability to do so only at an | Cardiac arrest | - | - | - | | Death |
| Definition: A disorder characterized by cessation of the pumping function of the heart. Navigational Note: - Chest pain - cardiac | | | | | | |
| Navigational Note: - Chest pain - cardiac Mild pain Moderate pain; pain on exertion; limiting instrumental ADL; cardiac catheterization; new onset cardiac chest pain; unstable angina new onset cardiac chest pain; unstable angina new onset cardiac chest pain; unstable angina Definition: A disorder characterized by substernal discomfort due to insulficient myocardial oxygenation e.g., angina pectoris. Navigational Note: Also consider Cardiac disorders: Myocardial infarction. Conduction disorder Mild symptoms; intervention not indicated intervention indicated intervention indicated intervention indicated on sequences Definition: A disorder characterized by pathological irregularities in the cardiac conduction system. Navigational Note: - Pesent | | | | | intervention indicated | ļ |
| Mild pain Moderate pain; pain on exertion; limiting instrumental exertion; limiting instrumental palp; stable ADL; and a cardiac catheterization; new onset cardiac chest pain; unstable angina Pain at rest; limiting self care ADL; cardiac catheterization; new onset cardiac chest pain; unstable angina Pain at rest; limiting self care ADL; cardiac catheterization; new onset cardiac chest pain; unstable angina Pain at rest; limiting self care ADL; cardiac catheterization; new onset cardiac chest pain; unstable angina Pain at rest; limiting self care ADL; cardiac catheterization; new onset cardiac chest pain; unstable angina Pain at rest; limiting self care ADL; cardiac catheterization; new onset cardiac catheterization; new onset cardiac chest pain; unstable angina Pain at rest; limiting self care ADL; cardiac catheterization; new onset cardiac chest pain; unstable angina Pain at rest; limiting self care ADL; cardiac catheterization; new onset cardiac chest pain; unstable angina Pain at rest; limiting self care ADL; cardiac catheterization; new onset cardiac chest pain; unstable angina Pain at rest; limiting self cathetrization; new onset or Pain at rest; limiting self cathetrization; new onset or Pain at rest; lamiting self cathet | | zed b <b>y</b> cessation of the pumping fur | nction of the heart. | | | |
| exertion; limiting instrumental ADL; cardiac catheterization; new onset cardiac chest pain; unstable angina unstable angina pectoris. Definition: A disorder characterized by substernal discomfort due to insufficient myocardial exygenation e.g., angina pectoris. Navigational Note: Also consider Cardiac disorders: Myocardial infarction. Conduction disorder | • | | | | | |
| ADL; hemodynamically stable new onset cardiac chest pain; unstable angina Definition: A disorder characterized by substernal discomfort due to insufficient myocardial expgenation e.g., angina pectoris. Navigational Note: Also consider Cardiac disorders: Myocardial infarction. Conduction disorder Mild symptoms; intervention not indicated intervention indicated intervention indicated intervention indicated intervention indicated consequences Definition: A disorder characterized by pathological irregularities in the cardiac conduction system. Navigational Note: Cyanosis - Present Definition: A disorder characterized by a bluish discoloration of the skin and/or mucous membranes. Navigational Note: - Heart failure Asymptomatic with laboratory (e.g., BNP [B-Natriuretic Peptide]) or cardiac imaging abnormalities Symptoms with moderate activity or exertion hospitalization; new onset of symptoms intervention indicated (e.g., continuous IV therapy or mechanical hemodynamic support) Definition: A disorder characterized by the inability of the heart to pump blood at an adequate volume to meet tissue metabolic requirements, or, the ability to do so only at an | Chest pain - cardiac | Mild pain | | | - | - |
| Definition: A disorder characterized by substernal discomfort due to insufficient myocardial oxygenation e.g., angina pectoris. Navigational Note: Also consider Cardiac disorders: Myocardial infarction. Conduction disorder Mild symptoms; intervention Non-urgent medical intervention indicated intervention indicated intervention indicated consequences Definition: A disorder characterized by pathological irregularities in the cardiac conduction system. Navigational Note: Present | | | | | | |
| Definition: A disorder characterized by substernal discomfort due to insufficient myocardial expension e.g., angina pectoris. Navigational Note: Also consider Cardiac disorders: Myocardial infarction. Conduction disorder Mild symptoms; intervention not indicated intervention indicated intervention indicated intervention indicated intervention indicated consequences Definition: A disorder characterized by pathological irregularities in the cardiac conduction system. Navigational Note: - Cyanosis - Present Definition: A disorder characterized by a bluish discoloration of the skin and/or mucous membranes. Navigational Note: - Heart failure Asymptomatic with laboratory {e.g., BNP [B-Natriuretic Peptide]} or cardiac imaging abnormalities Pefinition: A disorder characterized by the inability of the heart to pump blood at an adequate volume to meet tissue metabolic requirements, or, the ability to do so only at an | | | ADL; hemodynamically stable | | | |
| Non-urgent medical intervention indicated (e.g., continuous IV therapy or mechanical hemodynamic support) Definition: A disorder characterized by the inability of the heart to pump blood at an adequate volume to meet tissue metabolic requirements, or, the ability to do so only at an | | | l | | | l |
| Conduction disorder Mild symptoms; intervention not indicated intervention indicated consequences Definition: A disorder characterized by pathological irregularities in the cardiac conduction system. Navigational Note: - Cyanosis - Present Definition: A disorder characterized by a bluish discoloration of the skin and/or mucous membranes. Navigational Note: - Heart failure Asymptomatic with laboratory (e.g., BNP [B-Natriuretic Peptide]) or cardiac imaging abnormalities Symptoms with moderate activity or exertion; hospitalization; new onset of symptoms intervention indicated (e.g., continuous IV therapy or mechanical hemodynamic support) Definition: A disorder characterized by the inability of the heart to pump blood at an adequate volume to meet tissue metabolic requirements, or, the ability to do so only at an | | • | | n e.g., angina pectoris. | | |
| not indicated intervention indicated intervention indicated consequences Definition: A disorder characterized by pathological irregularities in the cardiac conduction system. Navigational Note: - Present | | | | | | |
| Definition: A disorder characterized by pathological irregularities in the cardiac conduction system. Navigational Note: - Cyanosis - Present | Conduction disorder | | | | J | Death |
| Navigational Note: - Cyanosis - Present | | | • | intervention indicated | consequences | l |
| Cyanosis - Present | | zed b <b>y</b> pathological irregularities in | the cardiac conduction system. | | | |
| Definition: A disorder characterized by a bluish discoloration of the skin and/or mucous membranes. Navigational Note: - Heart failure | | | Γ= | | | |
| Navigational Note: - Heart failure Asymptomatic with laboratory (e.g., BNP [B-Natriuretic Peptide ]) or cardiac imaging abnormalities Asymptoms with moderate activity or exertion Asymptoms at rest or with minimal activity or exertion; hospitalization; new onset of symptoms Symptoms at rest or with minimal activity or exertion; hospitalization; new onset of symptoms Symptoms at rest or with Life-threatening consequences; urgent intervention indicated (e.g., continuous IV therapy or mechanical hemodynamic support) Definition: A disorder characterized by the inability of the heart to pump blood at an adequate volume to meet tissue metabolic requirements, or, the ability to do so only at an | • | - | | - | - | - |
| Heart failure Asymptomatic with laboratory (e.g., BNP [B-Natriuretic Peptide ]) or cardiac imaging abnormalities Pefinition: A disorder characterized by the inability of the heart to pump blood at an adequate volume to meet tissue metabolic requirements, or, the ability to do so only at an | Definition: A disorder characteri: | zed b <b>y</b> a bluish discoloration of the | skin and/or mucous membranes. | | | |
| (e.g., BNP [B-Natriuretic Peptide]) or cardiac imaging abnormalities Consequences; urgent intervention indicated (e.g., continuous IV therapy or mechanical hemodynamic support) Definition: A disorder characterized by the inability of the heart to pump blood at an adequate volume to meet tissue metabolic requirements, or, the ability to do so only at an | - | | | | | |
| Peptide ]) or cardiac imaging abnormalities hospitalization; new onset of symptoms intervention indicated (e.g., continuous IV therapy or mechanical hemodynamic support) Definition: A disorder characterized by the inability of the heart to pump blood at an adequate volume to meet tissue metabolic requirements, or, the ability to do so only at an | Heart failure | | | | | Death |
| abnormalities symptoms continuous IV therapy or mechanical hemodynamic support) Definition: A disorder characterized by the inability of the heart to pump blood at an adequate volume to meet tissue metabolic requirements, or, the ability to do so only at an | | | activity or exertion | | | |
| mechanical hemodynamic support) Definition: A disorder characterized by the inability of the heart to pump blood at an adequate volume to meet tissue metabolic requirements, or, the ability to do so only at an | | | | | , 3. | |
| Definition: A disorder characterized by the inability of the heart to pump blood at an adequate volume to meet tissue metabolic requirements, or, the ability to do so only at an | | abnormalities | | symptoms | | |
| Definition: A disorder characterized by the inability of the heart to pump blood at an adequate volume to meet tissue metabolic requirements, or, the ability to do so only at an | | | | | | |
| | | l li el e lette fel le e e | <b>!</b> | | | l |
| al avertion to the offling average up | | zed by the inability of the heart to p | oump blood at an adequate volume | to meet tissue metabolic requirem | ents, or, the ability to do so only at | an |
| elevation in the filling pressure. Navigational Note: If left sided use Cardiac disorders: Left ventricular systolic dysfunction; also consider Cardiac disorders: Restrictive cardiomyopathy, Investigations: Ejection fraction | | sa Cardiac disordare: Laft yeatricula | er evetalic duefunction; also conside | r Cardiac disarders: Restrictive core | liamyanathy Investigations: Fiastic | n fraction |
| Navigational Note: Their sided use Cardiac disorders: Ejectiventricular systolic dystunction; also consider Cardiac disorders: Restrictive Cardiac disorders: Ejection fraction decreased. | _ | se cararac ursor ders, Lert Veritricus | ar systeme dysiumedom, also conside | cal diac distributers, nestrictive card | nomyopauly, mivesugauons: Ejecuo | i i i delloi i |

| | | Cardiac disorders | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Left ventricular systolic<br>dysfunction | | - | Symptomatic due to drop in ejection fraction responsive to intervention | Refractory or poorly<br>controlled heart failure due to<br>drop in ejection fraction;<br>intervention such as<br>ventricular assist device,<br>intravenous vasopressor<br>support, or heart transplant<br>indicated | Death |
| | zed by failure of the left ventricle to | | | | |
| Mitral valve disease | r Investigations: Ejection fraction de<br>Asymptomatic valvular<br>thickening with or without<br>mild valvular regurgitation or<br>stenosis by imaging | Asymptomatic; moderate regurgitation or stenosis by imaging | Symptomatic; severe regurgitation or stenosis by imaging; symptoms controlled with medical intervention | Life-threatening<br>consequences; urgent<br>intervention indicated (e.g.,<br>valve replacement,<br>valvuloplasty) | Death |
| | zed b <b>y</b> a defect in mitral valve func | tion or structure. | • | • " | |
| Navigational Note: - | | | | | |
| Mobitz (type) II<br>atrioventricular block | Asymptomatic, intervention not indicated | Symptomatic; medical<br>intervention indicated | Symptomatic and incompletely controlled medically controlled with device (e.g., pacemaker); new onset | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| electrical impulse conduction the | zed by a dysrhythmia with relativel<br>rough the atrioventricular (AV) nod | | block of an atrial impulse. This is the | result of intermittent failure of atr | ial |
| Navigational Note: -<br>Mobitz type I | A | C | T C | 116- 4 | Death |
| vlobitz type i | Asymptomatic, intervention not indicated | Symptomatic; medical<br>intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker) | Life-threatening<br>consequences; urgent<br>intervention indicated | Deam |
| | zed by a dysrhythmia with a progre<br>on through the atrioventricular (AV | | or to the blocking of an atrial impuls | e. This is the result of intermittent f | allure of |

| | | Cardiac disorders | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Myocardial infarction | - | Asymptomatic and cardiac | Severe symptoms; cardiac | Life-threatening | Death |
| | | enzymes minimally abnormal | enzymes abnormal; | consequences; | |
| | | and no evidence of ischemic | hemodynamically stable; ECG | hemodynamically unstable | |
| | | ECG changes | changes consistent with | | |
| | | 1 | infarction | 1 | |
| | zed by gross necrosis of the myoca | rdium; this is due to an interruptior | of blood suppl <b>y</b> to the area. | | |
| Navigational Note: - | | | | | |
| Myocarditis | = | Symptoms with moderate | Severe with symptoms at rest | Life-threatening | Death |
| | | activity or exertion | or with minimal activity or | consequences; urgent | |
| | | | exertion; intervention | intervention indicated (e.g., | |
| | | | indicated; new onset of | continuous IV therapy or | |
| | | | symptoms | mechanical hemodynamic | |
| | | 1 | | support) | |
| | zed b <b>y</b> inflammation of the muscle | tissue of the heart. | | | |
| Navigational Note: - | | | 1 | | |
| Palpitations | Mild symptoms; intervention | Intervention indicated | - | - | - |
| | not indicated | 1 | | 1 | |
| | zed b <b>y</b> an unpleasant sensation of i | irregular and/or forceful beating of | the heart. | | |
| Navigational Note: - | | | | | |
| Paroxysmal atrial tachycardia | Asymptomatic, intervention | Non-urgent medical | Symptomatic, urgent | Life-threatening | Death |
| | not indicated | intervention indicated | intervention indicated; | consequences; incompletely | |
| | | | ablation | controlled medically; | |
| | | 1 | | cardioversion indicated | |
| | zed by a dysrhythmia with abrupt o | onset and sudden termination of at | ial contractions with a rate of 150- | 250 beats per minute. The rhythm | disturbance |
| originates in the atria. | | | | | |
| Navigational Note: - | | | | | |
| Pericardial effusion | = | Asymptomatic effusion size | Effusion with physiologic | Life-threatening | Death |
| | | small to moderate | consequences | consequences; urgent | |
| i i | | 1 | | intervention indicated | |
| <b>Definition:</b> A disorder characteriz | <br> <br> zed by fluid collection within the pa | <br>ericardial sac, usually due to inflami | <br>mation. | intervention indicated | l |
| Navigational Note: - | zed by fluid collection within the po | ericardial sac, usually due to inflam | mation. | | |
| | zed by fluid collection within the pa | <br>ericardial sac, usually due to inflam:<br> - | <br>mation.<br> - | intervention indicated Life-threatening | Death |
| Navigational Note: - | zed by fluid collection within the po | ericardial sac, usually due to inflami | <br>mation.<br> - | | Death |
| Navigational Note: - | zed by fluid collection within the po | ericardial sac, usually due to inflami | <br>mation.<br> - | Life-threatening | Death |
| Navigational Note: -<br>Pericardial tamponade | - | ericardial sac, usually due to inflame - ial pressure due to the collection of | - | Life-threatening consequences; urgent | Death |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Cardiac disorders | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Pericarditis | Asymptomatic, ECG or<br>physical findings (e.g., rub)<br>consistent with pericarditis | Symptomatic pericarditis (e.g., chest pain) | Pericarditis with physiologic<br>consequences (e.g.,<br>pericardial constriction) | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder character | rized by irritation to the layers of the | pericardium (the protective sac ar | ound the heart). | | |
| Navigational Note: - | | | | | |
| Pulmonary valve disease | Asymptomatic valvular<br>thickening with or without<br>mild valvular regurgitation or<br>stenosis by imaging | Asymptomatic; moderate regurgitation or stenosis by imaging | Symptomatic; severe<br>regurgitation or stenosis by<br>imaging; symptoms controlled<br>with medical intervention | Life-threatening<br>consequences; urgent<br>intervention indicated (e.g.,<br>valve replacement,<br>valvuloplasty) | Death |
| | rized b <b>y</b> a defect in pulmonar <b>y</b> valve | function or structure. | | | |
| Navigational Note: - | | | | | |
| Restrictive cardiomyopathy | Imaging findings only | Symptomatic without signs of<br>heart failure | Symptomatic heart failure or<br>other cardiac symptoms,<br>responsive to intervention;<br>new onset of symptoms | Refractory heart failure or<br>other poorly controlled<br>cardiac symptoms | Death |
| Definition: A disorder character | rized by an inability of the ventricles | to fill with blood because the myoc | ardium (heart muscle) stiffens and | loses its flexibility. | · |
| Navigational Note: - | · | · | | · | |
| Right ventricular dysfunction | Asymptomatic with laboratory<br>(e.g., BNP [B-Natriuretic<br>Peptide]) or cardiac imaging<br>abnormalities | Symptoms with moderate activity or exertion | Severe symptoms, associated<br>with hypoxia, right heart<br>failure; oxygen indicated | Life-threatening<br>consequences; urgent<br>intervention indicated (e.g.,<br>ventricular assist device);<br>heart transplant indicated | Death |
| Definition: A disorder character | rized by impairment of right ventricu | Ilar function associated with low eje | ection fraction and a decrease in m | otility of the right ventricular wall. | • |
| Navigational Note: - | | | | | |
| Sick sinus syndrome | Asymptomatic, intervention not indicated | Symptomatic, intervention<br>not indicated; change in<br>medication initiated | Symptomatic, intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder character | rized by a dysrhythmia with alternat | ing periods of bradycardia and atria | Il tachycardia accompanied by sync | ope, fatigue and dizziness. | ' |
| Navigational Note: - | | - | | - | |
| Sinus bradycardia | Asymptomatic, intervention not indicated | Symptomatic, intervention<br>not indicated; change in<br>medication initiated | Symptomatic, intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder character | rized by a dysrhythmia with a heart r | -<br>ate less than 60 beats per minute t | hat originates in the sinus node. | - | • |

| | Cardiac disorders | | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Sinus tachycardia | Asymptomatic, intervention | Symptomatic; non-urgent | Urgent medical intervention | - | - |
| | not indicated | medical intervention indicated | indicated | | |
| | erized by a dysrhythmia with a heart | rate greater than 100 beats per min | ute that originates in the sinus nod | e. | |
| Navigational Note: - | | | | | |
| Supraventricular tachycardia | Asymptomatic, intervention | Non-urgent medical | Symptomatic, urgent | Life-threatening consequences | Death |
| | not indicated | intervention indicated | intervention indicated | ļ., | ļ |
| | erized by a dysrhythmia with a heart | rate greater than 100 beats per mir | ute that originates above the ventr | icles. | |
| Navigational Note: | T | T | Т | Laza | |
| Tricuspid valve disease | Asymptomatic valvular | Asymptomatic; moderate | Symptomatic; severe | Life-threatening | Death |
| | thickening with or without | regurgitation or stenosis by | regurgitation or stenosis; | consequences, urgent | |
| | mild valvular regurgitation or | imaging | symptoms controlled with | intervention indicated (e.g., | |
| | stenosis | | medical intervention | valve replacement, | |
| | | 1 | l . | valvuloplasty) | l |
| | erized b <b>y</b> a defect in tricuspid valve fu | inction or structure. | | | |
| Navigational Note: - | T | | T | Take a second | |
| Ventricular arrhythmia | Asymptomatic, intervention | Non-urgent medical | Urgent intervention indicated | Life-threatening | Death |
| | not indicated | intervention indicated | | consequences; hemodynamic | |
| D-61-161 6 -11 | <br> | I as the assessment of a second | Į. | compromise | l |
| | erized by a dysrhythmia that originat | es in the ventrides. | | | |
| Navigational Note: - Ventricular fibrillation | 1 | | T | Liera e e | Death |
| ventricular fibrillation | - | - | - | Life-threatening | Death |
| | | | | consequences; hemodynamic | |
| Definition, A disauday above to | <br>erized by a dysrhythmia without disce | <br> | | compromise | l<br>Nama a fillea |
| ventricles. | anzed by a dysrnythma without disc | embre QR3 comprexes due to rapid | repeditive excitation of myocardial | libers without coordinated contrac | uon oi me |
| venuncies.<br>Navigational Note: - | | | | | |
| Ventricular tachycardia | 1 | Non-urgent medical | Symptomatic, urgent | Life-threatening | Death |
| ventricular tacriycarula | - | intervention indicated | intervention indicated | consequences; hemodynamic | Deaul |
| | | Intervention indicated | Intervendonnidicated | compromise | |
| Definition: A disorder characte | I<br>erized by a dysrhythmia with a heart | I<br>rate greater than 100 heats per min | I<br>uta that originates distal to the bur | | ı |
| Navigational Note: - | anzeu by a dysiniyu ii iila wilu ra neai c | rate greater triair 100 beats per iriir | ate diaconginates distal to die bul | idie of fils. | |
| Cardiac disorders - Other. | Asymptomatic or mild | Moderate: minimal, local or | Severe or medically significant | Life-threatening | Death |
| specify | symptoms; clinical or | noninvasive intervention | but not immediately life- | consequences; urgent | Deaul |
| opcon, | diagnostic observations only: | indicated; limiting age- | threatening; hospitalization or | intervention indicated | |
| | intervention not indicated | appropriate instrumental ADL | prolongation of existing | intervention indicated | |
| | inica veriabilitio ilidicated | appropriate instrumental ADE | hospitalization indicated: | | |
| | | | limiting self care ADL | | |
| Definition: - | 1 | 1 | I minding son care ADL | 1 | ı |
| Vavigational Note: - | | | | | |
| anaiPartollal Morel | | | | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | Congenital, familial and genetic disorders | | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Congenital, familial and<br>genetic disorders - Other,<br>specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: - | | | | | |
| Navigational Note: - | | | | | |

| | | Ear and labyrinth disord | lers | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Ear pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder charac | terized by a sensation of marked discor | mfort in the ear. | | | • |
| Navigational Note: - | | | | | |
| External ear pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder charac | terized by a sensation of marked discor | nfort in the external ear region. | | | |
| Navigational Note: - | | | | | |
| Hearing impaired | Adults enrolled on a Nonitoring Program (on a 1, 2, 4, 3, 6, and 8 lkHz audiogram): Threshold shift of 15 - 25 dB averaged at 2 contiguous test frequencies in at least one ear; Adults not enrolled on a Monitoring Program: Subjective change in hearing in the absence of documented hearing loss; | Adults enrolled on a Monitoring Program (on a 1, 2, 3, 4, 6, and 8 kHz audiogram): Threshold shift of >25 dB averaged at 2 contiguous test frequencies in at least one ear; Adults not enrolled on a Monitoring Program: Hearing loss with hearing aid or intervention not indicated; limiting instrumental ADL; | Adults enrolled on a Monitoring Program (on a 1, 2, 3, 4, 6, and 8 kHz audiogram): Threshold shift of >25 dB averaged at 3 contiguous test frequencies in at least one ear; therapeutic intervention indicated; Adults not enrolled on a Monitoring Program: Hearing loss with hearing aid or intervention indicated; Iimiting self care ADL; | Adults: Decrease in hearing to profound bilateral loss (absolute threshold x80 dB HL at 2 kHz and above); nonservicable hearing Pediatric: Audiologic indication for cochlear implant; > 40 dB HL (i.e., 45 dB HL or more); SNHL at 2 kHz and above | - |
| <b>Definition:</b> A disorder charac | Pediatric (on a 1, 2, 3, 4, 6, and 8 kHz audiogram): Threshold shift >20 dB hearing loss (HL) (i.e., 25 dB HL or greater); sensorineural hearing loss (SNHL) above 4 kHz (i.e., 6 or 8 kHz) in at least one ear | Pediatric (on a 1, 2, 3, 4, 6, and 8 kHz audiogram): Threshold shift > 20 dB at 4 kHz in at least one ear | Pediatric (on a 1, 2, 3, 4, 6, and 8 kHz audiogram): Hearing loss sufficient to indicate therapeutic intervention, including hearing aids; threshold shift >20 dB at 2 to < 4 kHz in at least one ear | structures. | |
| <b>Definition:</b> A disorder charac<br><b>Navigational Note:</b> - | one ear<br>terized by partial or complete loss of the | e ability to detect or understand so | least one ear | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Ear and labyrinth disord | ers | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Middle ear inflammation | Serous otitis | Serous otitis, medical<br>intervention indicated | Mastoiditis; necrosis of canal soft tissue or bone | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder characteri: | zed by inflammation (physiologic re | sponse to irritation), swelling and r | edness to the middle ear. | | |
| Navigational Note: - | | | | | |
| Tinnitus | Mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self<br>care ADL | - | - |
| | zed by noise in the ears, such as rin | ging, buzzing, roaring or clicking. | | | |
| Navigational Note: - | A AND I | L | | | |
| Vertigo | Mild symptoms | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL | - | - |
| Definition: A disorder characteri:<br>vertigo).<br>Navigational Note: - | zed by a sensation as if the external | world were revolving around the p | | himself were revolving in space (si | ubjective |
| Vestibular disorder | - | Symptomatic; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL | - | - |
| Definition: A disorder characteri: | zed b <b>y</b> dizziness, imbalance, nausea | , and vision problems. | | | . |
| Navigational Note: - | | | | | |
| Ear and labyrinth disorders -<br>Other, specify | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongalization of existing<br>hospitalization indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: - | • | • | - | • | ' |
| Navigational Note: - | | | | | |

| | | Endocrine disorders | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Adrenal insufficiency | Asymptomatic; clinical or | Moderate symptoms; medical | Severe symptoms; | Life-threatening | Death |
| | diagnostic observations only; | intervention indicated | hospitalization indicated | consequences; urgent | |
| | intervention not indicated | 1 | 1 | intervention indicated | 1 |
| | cterized by the adrenal cortex not prod | | sol and in some cases, the hormone | aldosterone. It may be due to | a disorder of |
| | ison's disease or primary adrenal insuff | iciency. | | | |
| Navigational Note: - | | | | | |
| Cushingoid | Mild symptoms; intervention | Moderate symptoms; medical | Severe symptoms, medical | - | - |
| | not indicated | intervention indicated | intervention or hospitalization | | |
| | 1 | 1 | indicated | I | 1 . |
| | cterized by signs and symptoms that re | semble Cushing's disease or syndro | me: buffalo hump obesity, striation | s, adiposity, hypertension, diab | etes, and |
| osteoporosis, usuall <b>y</b> due to | ex agenous corticosteroids. | | | | |
| Navigational Note: - | | | | | |
| Delayed puberty | = | No breast development by | No breast development by | = | - |
| | | age 13 yrs for females; testes | age 14 yrs for females; no | | |
| | | volume of <3 cc or no Tanner | increase in testes volume or | | |
| | | Stage 2 development by age | no Tanner Stage 2 by age 16 | | |
| | | 14.5 yrs for males | yrs for males; hormone | | |
| | ļ | I | replacement indicated | I | I |
| | cterized by unusually late sexual matur | ity. | | | |
| Navigational Note: - | | | | | |
| Growth accelerated | - | >= +2 SD (standard deviation) | - | - | - |
| | | above mid parental height or | | | |
| | | target height | 1 | l | 1 |
| <b>Definition:</b> A disorder charac | cterized by greater growth than expect | ed for age. | | | |
| Navigational Note: - | | | | | |
| Hyperparathyroidism | Mild symptoms; intervention | Moderate symptoms; medical | = | = | - |
| | not indicated | intervention indicated | | | |
| Definition: A disorder charac | cterized by an increase in production o | f parathyroid hormone by the parat | hyroid glands. This results in hyper | calcemia (abnormally high level | s of calcium in |
| the blood). | | | | | |
| Navigational Note: - | | | | | |
| -lyperthyroidism | Asymptomatic; clinical or | Symptomatic; thyroid | Severe symptoms; limiting self | Life-threatening | Death |
| | diagnostic observations only; | suppression therapy | care ADL; hospitalization | consequences; urgent | |
| | intervention not indicated | indicated; limiting | indicated | intervention indicated | |
| | | instrumental ADL | | 1 | |
| Definition: A disorder charac | cterized by excessive levels of thyroid h | ormone in the body. Common caus | es include an overactive thyroid gla | ind or thyroid hormone overdo: | se. |
| lavigational Note: - | • | • | . 3 | • | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Endocrine disorders | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Hypoparathyroidism | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; medical<br>intervention indicated | Severe symptoms; medical<br>intervention or hospitalization<br>indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder chara | cterized by a decrease in production of | -<br>parathyroid hormone by the parath | nyroid glands. | • | · |
| Navigational Note: - | | | | | |
| Hypophysitis | Asymptomatic or mild<br>symptoms; dinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder chara <b>Navigational Note:</b> - | cterized by inflammation and cellular in | filtration of the pituitary gland. | | | |
| Hypopituitarism | Asymptomatic or mild<br>symptoms; dinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder chara | cterized by a decrease in production of | hormones from the pituitary gland. | | | |
| Navigational Note: - | | | | | |
| Hypothyroidism | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; thyroid<br>replacement indicated;<br>limiting instrumental ADL | Severe symptoms; limiting self<br>care ADL; hospitalization<br>indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | cterized by a decrease in production of | thyroid hormone by the thyroid gla | nd. | | |
| Navigational Note: - | Physical signs of puberty with | Physical signs and biochemical | 1 | 1 | |
| Precocious puberty | no biochemical markers for<br>females <8 years and males <9<br>years | markers of puberty for<br>females <8 years and males <9 | - | - | - |
| <b>Definition:</b> A disorder chara for boys. | cterized by unusually early developmen | 1 1 | onset of sexual maturation begins ( | usually before age 8 for girls an | d before age 9 |
| Navigational Note: - | | | | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Endocrine disorders | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Testosterone deficiency | Asymptomatic; mild<br>symptoms with no<br>intervention indicated | Replacement therapy initiated | - | - | - |
| Definition: A disorder character | ized by low testosterone. | | | | |
| Navigational Note: - | | | | | |
| Virilization | Mild symptoms; intervention<br>not indicated | Moderate symptoms; medical<br>intervention indicated | - | - | - |
| Definition: A disorder character | ized by inappropriate masculinizati | on occurring in a female or prepube | rtal male. | | • |
| Navigational Note: - | | | | | |
| Endocrine disorders - Other,<br>specify | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: - | • | - | • | - | • |
| Navigational Note: - | | | | | |

| | | Eye disorders | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Blurred vision | Intervention not indicated | Symptomatic; moderate decrease in visual acuity (best corrected visual acuity 20/40 and better or 3 lines or less decreased vision from known baseline); limiting instrumental ADL | Symptomatic with marked decrease in visual acuity (best corrected visual acuity worse than 20/40 or more than 3 lines of decreased vision from known baseline, up to 20/200); limiting self care ADL | Best corrected visual acuity of<br>20/200 or worse in the<br>affected eye | - |
| Definition: A disorder chara | acterized by visual perception of unclear | or fuzzy images. | | • | • |
| Navigational Note: - | | | | | |
| Cataract | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; moderate decrease in visual acuity (best corrected visual acuity 20/40 and better or 3 lines or less decreased vision from known baseline); glare symptoms affecting instrumental ADL | Symptomatic with marked decrease in visual acuity (best corrected visual acuity worse than 20/40 or more than 3 lines of decreased vision from known baseline, up to 20/200); limiting self care ADL | Best corrected visual acuity of<br>20/200 or worse in the<br>affected eye | - |
| <b>Definition:</b> A disorder chara untreated. <b>Navigational Note:</b> - | acterized by partial or complete opacity | of the crystalline lens of one or both | n eyes. This results in a decrease in | visual acuity and eventual blindness | sif |
| Corneal ulcer | - | - | Corneal ulcer without perforation in the affected eye | Perforation in the affected eye | - |
| Definition: A disorder chara | acterized by an area of epithelial tissue lo | oss on the surface of the cornea. It i | • • | <ul> <li>s in the cornea and anterior chamb</li> </ul> | er. |
| Navigational Note: - | | | • | | |
| Dry eye | Asymptomatic; clinical or diagnostic observations only; symptoms relieved by lubricants | Symptomatic; moderate decrease in visual acuity (best corrected visual acuity 20/40 and better or 3 lines or less decreased vision from known baseline) | Symptomatic with marked decrease in visual acuity (best corrected visual acuity worse than 20/40 or more than 3 lines of decreased vision from known baseline, up to 20/200); limiting self care ADL | - | - |
| | acterized by dryness of the cornea and c | - · | | | |
| Navigational Note: If corne | al ulcer is present, grade under Eye diso | rders: Corneal ulcer. | | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Eye disorders | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Extraocular muscle paresis | Asymptomatic; clinical or diagnostic observations only | Unilateral paresis without double vision | Bilateral paresis or unilateral<br>paresis causing double vision<br>in peripheral gaze, but not in<br>central gaze | Bilateral paresis requiring<br>head turning to see beyond<br>central 60 degrees or double<br>vision in central gaze | - |
| <b>Definition:</b> A disorder characte <b>Navigational Note:</b> - | rized by incomplete paralysis of an e | xtraocular muscle. | | | |
| Eye pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Navigational Note: - | rized by a sensation of marked disco | mfort in the eye. | | | |
| Eyelid function disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; nonoperative intervention indicated; limiting instrumental ADL | Limiting self care ADL;<br>operative intervention<br>indicated | - | - |
| <b>Definition:</b> A disorder characte <b>Navigational Note:</b> - | rized by impaired eyelid function. | | • | • | |
| Flashing lights | Symptomatic but not limiting ADL | Limiting instrumental ADL | Limiting self care ADL | - | - |
| Definition: A disorder characte | rized by a sudden or brief burst of lig | ht | ! | • | |
| Navigational Note: Also consid | ler Eye disorders: Retinal tear or Reti | nal detachment | | | |
| Floaters | Symptomatic but not limiting<br>ADL | Limiting instrumental ADL | Limiting self care ADL | - | - |
| Definition: A disorder characte | rized by an individual seeing spots b | efore their eyes. The spots are shac | lows of opaque cell fragments in t | the vitreous humor or lens. | • |
| Navigational Note: Also consid | ler Eye disorders: Retinal tear or Reti | nal detachment | | | |
| Glaucoma | Less than 8 mmHg of elevated intraocular pressure (EIOP); no visual field deficit | EIOP which can be reduced to<br>21 mmHg or under with<br>topical medications and no<br>visual field deficit | EIOP causing visual field<br>deficits | Visual field deficit within the central 10 degrees of the visual field in the affected eye | - |
| Definition: A disorder characte | rized b <b>y</b> an increase in pressure in th | e eyeball due to obstruction of the | aqueous humor outflow. | | |
| Navigational Note: - | | | | | |

| | | Eye disorders | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Keratitis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; moderate decrease in visual acuity (best corrected visual acuity 20/40 and better or 3 lines or less decreased vision from known baseline) | Symptomatic with marked decrease in visual acuity (best corrected visual acuity worse than 20/40 or more than 3 lines of decreased vision from known baseline, up to 20/200); corneal ulcer; limiting self care ADL | Perforation; best corrected visual aculty of 20/200 or worse in the affected eye | - |
| <b>Definition:</b> A disorder characte | erized by inflammation to the cornea | of the eye. | | | |
| | der Eye disorders: Corneal ulcer | | | | |
| Night blindness | Symptomatic but not limiting<br>ADL | Symptomatic; moderate<br>decrease in visual acuity (best<br>corrected visual acuity 20/40<br>and better or 3 lines or less<br>decreased vision from known<br>baseline); limiting<br>instrumental ADL | Symptomatic with marked decrease in visual acuity (best corrected visual acuity worse than 20/40 or more than 3 lines of decreased vision from known baseline, up to 20/200); limiting self care ADL | Best corrected visual acuity of<br>20/200 or worse in the<br>affected eye | - |
| Definition: A disorder characte | erized by an inability to see clearly in | dim light. | | • | |
| Navigational Note: - | | | | | |
| Optic nerve disorder | Asymptomatic; clinical or diagnostic observations only | Moderate decrease in visual<br>acuity (best corrected visual<br>acuity 20/40 and better or 3<br>lines or less decreased vision<br>from known baseline) | Marked decrease in visual acuity (best corrected visual acuity worse than 20/40 or more than 3 lines of decreased vision from known baseline, up to 20/200) | Best corrected visual acuity of<br>20/200 or worse in the<br>affected eye | - |
| Definition: A disorder characte | erized by involvement of the optic ne | rve (second cranial nerve). | | | |
| Navigational Note: - | | | | | |
| Papilledema | Asymptomatic; no visual field deficit | Symptomatic; moderate<br>decrease in visual acuity (best<br>corrected visual acuity 20/40<br>and better or 3 lines or less<br>decreased vision from known<br>baseline) | Symptomatic with marked decrease in visual acuity (best corrected visual acuity worse than 20/40 or more than 3 lines of decreased vision from known baseline, up to 20/200) | Best corrected visual acuity of 20/200 or worse in the affected eye | - |
| | erized by swelling around the optic di | sc. | | | |
| Navigational Note: - | | | | | |

| | | Eye disorders | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Periorbital edema | Soft or non-pitting | Indurated or pitting edema;<br>topical intervention indicated | Edema associated with visual disturbance; increased intraocular pressure, glaucoma or retinal hemorrhage; optic neuritis; diuretics indicated; operative intervention indicated | | - |
| | rized by swelling due to an excessive | accumulation of fluid around the c | orbits of the face. | | |
| Navigational Note: - | | | | | |
| Photophobia | Symptomatic but not limiting<br>ADL | Limiting instrumental ADL | Limiting self care ADL | - | - |
| Definition: A disorder characte | rized by fear and avoidance of light. | | | | |
| Navigational Note: - | | | | | |
| Retinal detachment | - | - | Macular sparing<br>rhegmatogenous detachment | Macula-off rhegmatogenous<br>retinal detachment | - |
| Definition: A disorder characte | rized by the separation of the inner r | etina layers from the underlying pi | gment epithelium. | • | • |
| Navigational Note: - | | | | | |
| Retinal tear | No retinal detachment and<br>treatment not indicated | No retinal detachment and<br>treatment indicated | - | - | - |
| Definition: A disorder characte | rized by a small laceration of the reti | na, this occurs when the vitreous s | eparates from the retina. Symptom | s include flashes and floaters. | |
| Navigational Note: If retinal de | etachment is present, grade under E <b>y</b> | e disorders: Retinal detachment | | | |
| Retinal vascular disorder | - | Retinal vascular disorder<br>without neovascularization | Retinal vascular disorder with<br>neovascularization | - | = |
| Definition: A disorder characte | rized by pathological retinal blood ve | essels that adversely affects vision. | • | • | • |
| Navigational Note: If vitreous h | nemorrhage is present, report under | Eye disorders: Vitreous hemorrhag | e. | | |
| Retinopathy | Asymptomatic; clinical or diagnostic observations only | Symptomatic; moderate decrease in visual acuity (best corrected visual acuity 20/40 and better or 3 lines or less decreased vision from known baseline); limiting instrumental ADL | Symptomatic with marked decrease in visual acuity (best corrected visual acuity worse than 20/40 or more than 3 lines of decreased vision from known baseline, up to 20/200); limiting self care ADL | Best corrected visual acuity of<br>20/200 or worse in the<br>affected eye | - |
| <b>Definition:</b> A disorder involving | • | | | | |
| Navigational Note: If vitreous h | nemorrhage is present, report under | Eye disorders: Vitreous hemorrhag | e. | | |

| | | Eye disorders | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Scleral disorder | No change in vision from baseline | Symptomatic; moderate decrease in visual acuity (best corrected visual acuity 20/40 and better or 3 lines or less decreased vision from known baseline); limiting instrumental ADL | Symptomatic with marked decrease in visual acuity (best corrected visual acuity worse than 20/40 or more than 3 lines of decreased vision from known baseline, up to 20/200); limiting self care ADL | Best corrected visual acuity of<br>20/200 or worse in the<br>affected eye | - |
| Definition: A disorder charact | erized by involvement of the sclera o | f the eye. | | | |
| Navigational Note: - | | | | | |
| Uveitis | Anterior uveitis with trace cells | Anterior uveitis with 1+ or 2+ cells | Anterior uveitis with 3+ or<br>greater cells; intermediate<br>posterior or pan-uveitis | Best corrected visual acuity of 20/200 or worse in the affected eye | - |
| | erized by inflammation to the uvea o | f the eye. | | | |
| Navigational Note: - | | | | | |
| Vision decreased | - | Moderate decrease in visual acuity (best corrected visual acuity 20/40 and better or 3 lines or less decreased vision from known baseline) | Marked decrease in visual<br>acuity (best corrected visual<br>acuity worse than 20/40 or<br>more than 3 lines of<br>decreased vision from known<br>baseline, up to 20/200} | Best corrected visual acuity of 20/200 or worse in the affected eye | - |
| Definition: A disorder charact | terized by a decrease in visual acuity. | | • | • | |
| Navigational Note: If etiology | is known, use a more specific CTCAE | term. | | | |
| Vitreous hemorrhage | Intervention not indicated | Symptomatic; moderate decrease in visual acuity (best corrected visual acuity 20/40 and better or 3 lines or less decreased vision from known baseline); limiting instrumental ADL | Symptomatic with marked decrease in visual aculty (best corrected visual aculty worse than 20/40 or more than 3 lines of decreased vision from known baseline, up to 20/200); limiting self care ADL; vitrectomy indicated | Best corrected visual acuity of<br>20/200 or worse in the<br>affected eye | - |
| <b>Definition:</b> A disorder charact<br><b>Navigational Note:</b> - | erized by bleeding into the vitreous h | umor. | | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Eye disorders | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Watering eyes | Intervention not indicated | Symptomatic; moderate<br>decrease in visual acuity (best<br>corrected visual acuity 20/40<br>and better or 3 lines or less<br>decreased vision from known<br>baseline) | Marked decrease in visual acuity (best corrected visual acuity worse than 20/40 or more than 3 lines of decreased vision from known baseline, up to 20/200) | Best corrected visual acuity of 20/200 or worse in the affected eye | - |
| Definition: A disorder character<br>Navigational Note: - | ized by excessive tearing in the eyes | s; it can be caused by overproduction | on of tears or impaired drainage of t | he tear duct. | |
| Eye disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated; no<br>change in vision | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting<br>instrumental ADL; best<br>corrected visual acuity 20/40<br>and better or 3 lines or less<br>decreased vision from known<br>baseline | Severe or medically significant but not immediately sight-threatening; limiting self care ADL; decrease in visual acuity (best corrected visual acuity worse than 20/40 or more than 3 lines of decreased vision from known baseline, up to 20/200) | Sight-threatening consequences; urgent intervention indicated; best corrected visual acuity of 20/200 or worse in the affected eye | - |
| Definition: - | • | • | , , , , | • | |
| Navigational Note: - | | | | | |

| | | Gastrointestinal diso | rders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Abdominal distension | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; limiting instrumental ADL | Severe discomfort; limiting self care ADL | - | - |
| Definition: A disorder chara- | cterized by swelling of the abdomen. | | | | |
| Navigational Note: - | | | | | |
| Abdominal pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder chara- | cterized by a sensation of marked disco | omfort in the abdominal region. | • | - | · |
| Navigational Note: - | | | | | |
| Anal fissure | Asymptomatic | Symptomatic | Invasive intervention indicated | - | - |
| Definition: A disorder chara- | cterized by a tear in the lining of the an | nus. | • | • | • |
| Navigational Note: - | | | | | |
| Anal fistula | Asymptomatic | Symptomatic, invasive intervention not indicated | Invasive intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder character Navigational Note: - | cterized by an abnormal communicatio | n between the opening in the and | al canal to the perianal skin. | • | I |
| | cterized by an abnormal communicatio Mild symptoms; intervention not indicated | Moderate symptoms;<br>intervention indicated | Transfusion indicated; invasive intervention | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Navigational Note: -<br>Anal hemorrhage | Mild symptoms; intervention not indicated | Moderate symptoms;<br>intervention indicated | Transfusion indicated; | Life-threatening consequences; urgent | Death |
| Navigational Note: - Anal hemorrhage Definition: A disorder chara- | Mild symptoms; intervention | Moderate symptoms;<br>intervention indicated | Transfusion indicated; invasive intervention | Life-threatening consequences; urgent | Death |
| Navigational Note: -<br>Anal hemorrhage | Mild symptoms; intervention not indicated | Moderate symptoms;<br>intervention indicated | Transfusion indicated; invasive intervention | Life-threatening consequences; urgent | Death - |
| Navigational Note: - Anal hemorrhage Definition: A disorder chara Navigational Note: - Anal mucositis | Mild symptoms; intervention not indicated cterized by bleeding from the anal region Asymptomatic or mild symptoms; intervention not | Moderate symptoms; intervention indicated on. Symptomatic; medical intervention indicated; limiting instrumental ADL | Transfusion indicated; invasive intervention indicated; hospitalization Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent | Death |
| Navigational Note: - Anal hemorrhage Definition: A disorder chara- Navigational Note: - Anal mucositis Definition: A disorder chara- | Mild symptoms; intervention not indicated cterized by bleeding from the anal region Asymptomatic or mild symptoms; intervention not indicated | Moderate symptoms; intervention indicated on. Symptomatic; medical intervention indicated; limiting instrumental ADL of the mucous membrane of the | Transfusion indicated; invasive intervention indicated; hospitalization Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent | Death - |
| Navigational Note: - Anal hemorrhage Definition: A disorder chara- Navigational Note: - Anal mucositis Definition: A disorder chara- | Mild symptoms; intervention not indicated cterized by bleeding from the anal region Asymptomatic or mild symptoms; intervention not indicated cterized by ulceration or inflammation | Moderate symptoms; intervention indicated on. Symptomatic; medical intervention indicated; limiting instrumental ADL of the mucous membrane of the | Transfusion indicated; invasive intervention indicated; hospitalization Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent | Death - Death |
| Navigational Note: - Anal hemorrhage Definition: A disorder chara Navigational Note: - Anal mucositis Definition: A disorder chara Navigational Note: Report G Anal necrosis | Mild symptoms; intervention not indicated cterized by bleeding from the anal region Asymptomatic or mild symptoms; intervention not indicated cterized by ulceration or inflammation | Moderate symptoms; intervention indicated on. Symptomatic; medical intervention indicated; limiting instrumental ADL of the mucous membrane of the ders; Anal ulcer | Transfusion indicated; invasive intervention indicated; hospitalization Severe symptoms; limiting self care ADL anus. TPN or hospitalization indicated; invasive | Life-threatening consequences; urgent intervention indicated - Life-threatening consequences; urgent operative intervention | - |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Gastrointestinal disord | ders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Anal pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder chara | acterized by a sensation of marked disco | omfort in the anal region. | | | |
| Navigational Note: - | | | | | |
| Anal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function | Symptomatic and severely<br>altered GI function; non-<br>emergent operative<br>intervention indicated; TPN or<br>hospitalization indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Definition: A disorder chara | acterized by a narrowing of the lumen o | f the anal canal. | | | |
| Navigational Note: - | | | | | |
| Anal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function | Severely altered GI function;<br>TPN indicated; elective<br>invasive intervention<br>indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Definition: A disorder chara | acterized by a circumscribed, erosive les | ion on the mucosal surface of the a | anal canal. | | · |
| Navigational Note: - | | | | | |
| Ascites | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; invasive intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Definition: A disorder chara | acterized by accumulation of serous or h | nemorrhagic fluid in the peritoneal | cavity. | • | • |
| Navigational Note: - | • | | • | | |
| Belching | Increase from baseline | Intervention initiated<br>(including over the counter<br>medications) | - | - | - |
| Definition: To expel gas noi | sily from the mouth. | • | • | • | · |
| Navigational Note: Synony | m:Burping | | | | |
| Bloating | No change in bowel function<br>or oral intake | Symptomatic, decreased oral<br>intake; change in bowel<br>function | - | - | - |
| Definition: A disorder chara | acterized by subject-reported feeling of | uncomfortable fullness of the abdo | men. | - | • |
| Navigational Note: - | | | | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Gastrointestinal disord | ers | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Cecal hemorrhage | Mild symptoms; intervention<br>not indicated | Moderate symptoms;<br>intervention indicated | Transfusion indicated;<br>invasive intervention<br>indicated; hospitalization | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | acterized by bleeding from the cecum. | | | | |
| Navigational Note: -<br>Chellitis | Asymptomatic: clinical or | Note that the second second section is a second second section. | | _ | |
| Chellius | diagnostic observations only;<br>intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self<br>care ADL; intervention<br>indicated | - | - |
| Definition: A disorder chara | cterized by inflammation of the lip. | | • | | · |
| Navigational Note: - | | | | | |
| Chylous ascites | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical<br>intervention indicated (e.g.,<br>fat-restricted diet);<br>paracentesis or tube drainage<br>indicated | Severe symptoms; elective operative intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| <b>Definition:</b> A disorder chara <b>Navigational Note:</b> - | cterized by accumulation of milky fluid | in the peritoneal cavity. | | | |
| Colitis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Abdominal pain; mucus or blood in stool | Severe abdominal pain;<br>peritoneal signs | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | • | • | | | |
| <b>Definition:</b> A disorder chara | cterized by inflammation of the colon. | | | | • |
| <b>Definition:</b> A disorder chara <b>Navigational Note:</b> - | cterized by inflammation of the colon. | | | | · |
| | Asymptomatic | Symptomatic, invasive intervention not indicated | Invasive intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Navigational Note: -<br>Colonic fistula | <u> </u> | intervention not indicated | indicated | consequences; urgent | Death |
| Navigational Note: - Colonic fistula Definition: A disorder chara | Asymptomatic | intervention not indicated | indicated | consequences; urgent | Death |
| Navigational Note: - Colonic fistula Definition: A disorder chara Navigational Note: - Colonic hemorrhage | Asymptomatic Interized by an abnormal communication Mild symptoms; intervention | intervention not indicated n between the large intestine and a Moderate symptoms; | indicated nother organ or anatomic site. Transfusion indicated; invasive intervention | consequences; urgent intervention indicated Life-threatening consequences; urgent | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Gastrointestinal disord | lers | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Colonic obstruction Definition: A disorder chara | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated<br>icterized by blockage of the normal flow | Symptomatic; altered GI function of the intestinal contents in the co | Hospitalization indicated;<br>invasive intervention<br>indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Navigational Note: - | - | | | | |
| Colonic perforation | - | Invasive intervention not indicated | Invasive intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder chara<br><b>Navigational Note:</b> - | cterized by a rupture in the colonic wal | | | | |
| Colonic stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function | Severely altered GI function;<br>tube feeding or<br>hospitalization indicated;<br>elective operative<br>intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Definition: A disorder chara | cterized by a narrowing of the lumen of | the colon. | | | • |
| Navigational Note: - | | | | | |
| Colonic ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function | Severely altered GI function;<br>TPN indicated; elective<br>invasive intervention<br>indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Definition: A disorder chara | cterized by a circumscribed, erosive les | on on the mucosal surface of the c | olon. | • | • |
| Navigational Note: - | | | | | |
| Constipation | Occasional or intermittent<br>symptoms; occasional use of<br>stool softeners, laxatives,<br>dietary modification, or<br>enema | Persistent symptoms with<br>regular use of laxatives or<br>enemas; limiting instrumental<br>ADL | Obstipation with manual evacuation indicated; limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder chara | cterized by irregular and infrequent or | difficult evacuation of the bowels. | | | |
| Navigational Note: - | | | | | |
| Dental caries | One or more dental caries,<br>not involving the root | Dental caries involving the root | Dental caries resulting in<br>pulpitis or periapical abscess<br>or resulting in tooth loss | - | - |
| | cterized by the decay of a tooth, in whi | ch it becomes softened, discolored | and/or porous. | | • |
| Navigational Note: - | | | | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Gastrointestinal disord | ers | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Diarrhea | Increase of <4 stools per day<br>over baseline; mild increase in<br>ostomy output compared to<br>baseline | Increase of 4 - 6 stools per day<br>over baseline; moderate<br>increase in ostomy output<br>compared to baseline; limiting<br>instrumental ADL | Increase of >=7 stools per day<br>over baseline; hospitalization<br>indicated; severe increase in<br>ostomy output compared to<br>baseline; limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | cterized by an increase in frequency and | d/or loose or watery bowel movem | ents. | | |
| | Symptomatic (e.g., dry or thick sallva) without significant dietary alteration; unstimulated saliva flow >0.2 ml/min | Moderate symptoms; oral intake alterations (e.g., copious water, other lubricants, diet limited to purees and/or soft, moist foods); unstimulated saliva 0.1 to 0.2 ml/min oral cavity. | Inability to adequately aliment<br>orally; tube feeding or TPN<br>indicated; unstimulated saliva<br><0.1 ml/min | - | - |
| Navigational Note: - | | | | | |
| Duodenal fistula | Asymptomatic | Symptomatic, invasive intervention not indicated | Invasive intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | cterized by an abnormal communication | n between the duodenum and anot | her organ or anatomic site. | • | • |
| Navigational Note: -<br>Duodenal hemorrhage | Mild symptoms; intervention not indicated | Moderate symptoms;<br>intervention indicated | Transfusion indicated;<br>invasive intervention<br>indicated; hospitalization | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder chara- | cterized by bleeding from the duodenur | n. | | | |
| Navigational Note: - | | | | | |
| Duodenal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function | Hospitalization indicated;<br>invasive intervention<br>indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Definition: A disorder chara- | cterized by blockage of the normal flow | of stomach contents through the c | uodenum. | • | • |
| Navigational Note: - | | | | | |

| | | Gastrointestinal disord | ers | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Duodenal perforation | - | Invasive intervention not indicated | Invasive intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Navigational Note: - | cterized by a rupture in the duodenal w | rall. | | | |
| Duodenal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered Gl<br>function | Severely altered GI function;<br>tube feeding or<br>hospitalization indicated;<br>elective operative<br>intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Definition: A disorder charac | cterized by a narrowing of the lumen o | f the duodenum. | • | • | |
| Navigational Note: - | | | | | |
| Duodenal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical<br>intervention indicated;<br>limiting instrumental ADL | Severely altered GI function;<br>TPN indicated; elective<br>invasive intervention<br>indicated; limiting self care<br>ADL | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Definition: A disorder charac | ו<br>cterized by a circumscribed, erosive les | In on the mucosal surface of the d | | • | ı |
| Navigational Note: - | | | | | |
| Dyspepsia | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Severe symptoms; operative<br>intervention indicated | - | - |
| <b>Definition:</b> A disorder character heartburn, nausea and vomi <b>Navigational Note:</b> - | cterized by an uncomfortable, often pa<br>ting. | inful feeling in the stomach, resulti | ng from impaired digestion. Sympto | oms include burning stomach, bl | pating, |
| Dysphagia | Symptomatic, able to eat<br>regular diet | Symptomatic and altered eating/swallowing | Severely altered<br>eating/swallowing; tube<br>feeding, TPN, or<br>hospitalization indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder character Navigational Note: - | cterized by difficulty in swallowing. | • | • | | · |
| Enterocolitis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Abdominal pain; mucus or blood in stool | Severe or persistent<br>abdominal pain; fever; ileus;<br>peritoneal signs | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | cterized by inflammation of the small a<br>ing a known abnormality of the colon, i | | is. If reporting a documented infec | tion, use Infections and infestati | ons: |

| | | Gastrointestinal disord | ers | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade ! |
| Enterovesical fistula | Asymptomatic | Symptomatic, invasive<br>intervention not indicated | Invasive intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder charact | I<br>erized by an abnormal communication | n between the urinary bladder and | I<br>the intestine | intervendon macated | I |
| Navigational Note: - | carzed by an abriormal communicate | or between the armary bradder and | are mesarie. | | |
| Esophageal fistula | Asymptomatic | Symptomatic, invasive | Invasive intervention | Life-threatening | Death |
| | | intervention not indicated | indicated | consequences; urgent<br>intervention indicated | |
| <b>Definition:</b> A disorder charact | erized b <b>y</b> an abnormal communicatio | on between the esophagus and anot | her organ or anatomic site. | | |
| Navigational Note: - | | | | | |
| Esophageal hemorrhage | Mild symptoms; intervention | Moderate symptoms; | Transfusion indicated; | Life-threatening | Death |
| | not indicated | intervention indicated | invasive intervention | consequences; urgent | |
| D. finisian. 8 diameter de mars | <br>erized by bleeding from the esophage | | indicated; hospitalization | intervention indicated | ı |
| | erized by breeding from the esophago | ıs. | | | |
| Navigational Note: -<br>Esophageal necrosis | | Τ. | Inability to aliment adequately | Life-threatening | Death |
| sopriagearried usis | | · | by GI tract; invasive | consequences; urgent | Deaul |
| | | | intervention indicated | operative intervention | |
| | | | | indicated | |
| Definition: A disorder charact | erized by a necrotic process occurring | ; in the esophageal wall. | • | • | |
| Navigational Note: - | | | | | |
| Esophageal obstruction | Asymptomatic; clinical or | Symptomatic; altered GI | Hospitalization indicated; | Life-threatening | Death |
| | diagnostic observations only; | function; limiting instrumental | invasive intervention | consequences; urgent | |
| | intervention not indicated | ADL | indicated; limiting self care | intervention indicated | |
| | <u> </u> | I., | ADL | l | |
| | erized by blockage of the normal flow | v of the contents in the esophagus. | | | |
| Navigational Note: - | Lawre | The state of the state of | T | Г | |
| Esophageal pain | Mild pain | Moderate pain; limiting | Severe pain; limiting self care<br>ADL | - | - |
| Dafinisiana Aultanalan dan dan d | <br>erized by a sensation of marked disco | instrumental ADL | ADL | I | 1 |
| Definition: A disorder charact<br>Navigational Note: - | erized by a sensation of marked disco | ornior tin the esophageai region. | | | |
| Esophageal perforation | | Invasive intervention not | Invasive intervention | Life-threatening | Death |
| _sopriagear perioracorr | | indicated | indicated | consequences; urgent | Deadi |
| | | | | operative intervention | |
| | | 1 | | indicated | |
| Definition: A disorder charact | erized by a rupture in the wall of the | esophagus. | | • | • |
| Navigational Note: - | | · - | | | |

| | | Gastrointestinal disord | ers | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Esophageal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function | Severely altered GI function;<br>tube feeding or<br>hospitalization indicated;<br>elective operative<br>intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Definition: A disorder charac | cterized by a narrowing of the lumen o | f the esophagus. | | | |
| Navigational Note: - | | | | | |
| Esophageal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function; limiting instrumental<br>ADL | Severely altered GI function;<br>TPN indicated; elective<br>invasive intervention<br>indicated; limiting self care<br>ADL | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Definition: A disorder charac | cterized by a circumscribed, erosive les | ion on the mucosal surface of the e | sophageal wall. | • | · |
| Navigational Note: - | | | | | |
| Esophageal varices<br>hemorrhage | - | Self-limited; intervention not indicated | Transfusion indicated;<br>invasive intervention<br>indicated; hospitalization | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder charac | cterized by bleeding from esophageal v | arices. | | | • |
| Navigational Note: - | | | | | |
| Esophagitis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered<br>eating/swallowing; oral<br>supplements indicated | Severely altered<br>eating/swallowing; tube<br>feeding, TPN, or<br>hospitalization indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Definition: A disorder charac | cterized by inflammation of the esopha | geal wall. | | | |
| Navigational Note: - | | | | | |
| Fecal incontinence | Occasional use of pads required | Daily use of pads required | Severe symptoms; elective<br>operative intervention<br>indicated | - | - |
| Definition: A disorder charac | cterized by inability to control the esca | pe of stool from the rectum. | | | • |
| Navigational Note: - | | | | | |
| Flatulence | Mild symptoms; intervention<br>not indicated | Moderate; persistent;<br>psychosocial sequelae | - | - | - |
| Definition: A disorder charac | cterized by a discharge of excessive gas | from the lower GI tract. | | | |
| Navigational Note: - | | | | | |

| CTCAE Term | | | | | |
|---|---|---|---|---|---|
| CICAE IEIM | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Gastric fistula | Asymptomatic | Symptomatic, invasive intervention not indicated | Invasive intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | zed by an abnormal communication | n between the stomach and anothe | r organ or anatomic site. | | |
| Navigational Note: - | 1 | | | | |
| Gastric hemorrhage | Mild symptoms; intervention<br>not indicated | Moderate symptoms;<br>intervention indicated | Transfusion indicated;<br>invasive intervention<br>indicated; hospitalization | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder characteri | zed by bleeding from the gastric wa | all. | | | |
| Navigational Note: - | | | | | |
| Gastric necrosis | - | - | Inability to aliment adequately<br>by GI tract; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| <b>Definition:</b> A disorder characteri | zed by a necrotic process occurring | in the gastric wall. | | | |
| Navigational Note: - | | | | | |
| Gastric perforation | - | Invasive intervention not indicated | Invasive intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Definition: A disorder characteri | ized by a rupture in the stomach wa | ill. | | • | • |
| Navigational Note: - | | | | | |
| Gastric stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function | Severely altered GI function;<br>tube feeding or<br>hospitalization indicated;<br>elective operative<br>intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Definition: A disorder characteri | zed by a narrowing of the lumen of | the stomach. | | • | • |
| Navigational Note: - | | | | | |
| Gastric ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function; medical intervention<br>indicated; limiting<br>instrumental ADL | Severely altered GI function;<br>TPN indicated; elective<br>invasive intervention<br>indicated; limiting self care<br>ADL | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| <b>Definition:</b> A disorder characteri | zed b <b>y</b> a circumscribed, erosive lesi | on on the mucosal surface of the st | omach. | - | - |
| Navigational Note: - | | | | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Gastrointestinal disord | ers | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Gastritis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function; medical intervention<br>indicated | Severely altered eating or<br>gastric function; TPN or<br>hospitalization indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Definition: A disorder characte<br>Navigational Note: - | rized by inflammation of the stomad | h. | | | |
| Gastroesophageal reflux<br>disease<br><b>Definition:</b> A disorder characte | Mild symptoms; intervention<br>not indicated<br>rized by reflux of the gastric and/or o | Moderate symptoms; medical<br>intervention indicated<br>duodenal contents into the distal es | Severe symptoms; operative<br>intervention indicated<br>ophagus. It is chronic in nature and | -<br>l usually caused by incompetenc | e of the lower |
| esophageal sphincter, and may<br>Navigational Note: - | result in injury to the esophageal m | ucosal. Symptoms include heartbur | n and acid indigestion. | | |
| Gastrointestinal fistula | Asymptomatic | Symptomatic, invasive intervention not indicated | Invasive intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder characte<br><b>Navigational Note:</b> - | rized by an abnormal communication | n between any part of the gastroint | estinal system and another organ o | or anatomic site. | · |
| Gastrointestinal pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| | rized by a sensation of marked disco | mfort in the gastrointestinal region. | | | |
| Navigational Note: - | Land | Tarana and the | Larra I a a a a a a | Lucia | |
| Gastroparesis | Mild nausea, early satiety and<br>bloating, able to maintain<br>caloric intake on regular diet | Moderate symptoms; able to<br>maintain nutrition with<br>dietary and lifestyle<br>modifications; may need<br>pharmacologic intervention | Weight loss >=20% from<br>baseline; tube feeding or TPN<br>indicated; elective operative<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | - |
| | | | والمراجع وال | etric contents into the small into | |
| | rized by an incomplete paralysis of t | he muscles of the stomach wall resu | arring in derayed emptying or mega | ascric contents into the sinal inte | esune. |
| <b>Definition:</b> A disorder characte<br><b>Navigational Note:</b> -<br>Gingival pain | rized by an incomplete paralysis of ti<br>Mild pain | Moderate pain interfering | Severe pain; inability to | - | estine. |
| Navigational Note: -<br>Gingival pain | | Moderate pain interfering with oral intake | | | esune. |
| Navigational Note: -<br>Gingival pain | Mild pain | Moderate pain interfering with oral intake | Severe pain; inability to | - | estine. |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Gastrointestinal disord | ers | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Hemorrhoids | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; banding or<br>medical intervention indicated | Severe symptoms; invasive<br>intervention indicated | - | - |
| Definition: A disorder chara | acterized by the presence of dilated vein | s in the rectum and surrounding are | ea. | | |
| Navigational Note: - | | | | | |
| Ileal fistula | Asymptomatic | Symptomatic, invasive intervention not indicated | Invasive intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder chara | acterized by an abnormal communicatio | n between the ileum and another o | rgan or anatomic site. | | |
| Navigational Note: - | | | | | |
| Ileal hemorrhage | Mild symptoms; intervention<br>not indicated | Moderate symptoms;<br>intervention indicated | Transfusion indicated;<br>invasive intervention<br>indicated; hospitalization | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | acterized by bleeding from the ileal wall. | | | | |
| Navigational Note: - | | | | _ | |
| lleal obstruction | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI<br>function; limiting instrumental<br>ADL; naso-gastric tube<br>indicated | Hospitalization indicated;<br>invasive intervention<br>indicated; limiting self care<br>ADL; long intestinal tube<br>indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Definition: A disorder chara | acterized by blockage of the normal flow | of the intestinal contents in the ile | um. | • | |
| Navigational Note: - | | | | | |
| lleal perforation | - | Invasive intervention not indicated | Invasive intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Navigational Note: - | acterized by a rupture in the ileal wall. | | | | |
| Ileal stenosis | Asymptomatic; clinical or | Symptomatic; altered GI | Severely altered GI function; | Life-threatening | Death |
| | diagnostic observations only;<br>intervention not indicated | function | tube feeding or<br>hospitalization indicated;<br>elective operative<br>intervention indicated | consequences; urgent<br>operative intervention<br>indicated | |
| Definition: A disorder chara | acterized by a narrowing of the lumen o | f the ileum. | • | - | • |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Gastrointestinal disord | ers | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| lleal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered Gl<br>function | Severely altered GI function;<br>TPN indicated; elective<br>invasive intervention<br>indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Definition: A disorder character | rized b <b>y</b> a circumscribed, erosive lesi | on on the mucosal surface of the ile | eum. | • | |
| Navigational Note: - | | | | | |
| lleus | Asymptomatic and radiologic observations only | Symptomatic; altered Gl<br>function; bowel rest indicated | Severely altered GI function;<br>TPN indicated; tube<br>placement indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | rized by failure of the ileum to transp | port intestinal contents. | | | |
| Navigational Note: -<br>Intra-abdominal hemorrhage | - | Moderate symptoms;<br>intervention indicated | Transfusion indicated;<br>invasive intervention<br>indicated; hospitalization | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder character | ized by bleeding in the abdominal c | avit <b>y.</b> | | • | • |
| Navigational Note: - | | | | | |
| Jejunal fistula | Asymptomatic | Symptomatic, invasive intervention not indicated | Invasive intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder character | ized b <b>y</b> an abnormal communication | n between the jejunum and anothe | r organ or anatomic site. | • | • |
| Navigational Note: - | | | | | |
| Jejunal hemorrhage | Mild symptoms; intervention<br>not indicated | Moderate symptoms;<br>intervention indicated | Transfusion indicated;<br>invasive intervention<br>indicated; hospitalization | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder character | rized by bleeding from the jejunal wa | all. | | | • |
| Navigational Note: - | | | | | |
| Jejunal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function; limiting instrumental<br>ADL | Hospitalization indicated;<br>invasive intervention<br>indicated; limiting self care<br>ADL | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Definition: A disorder character | ized by blockage of the normal flow | of the intestinal contents in the jej | unum. | • | • |
| Navigational Note: - | | | | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Gastrointestinal disord | lers | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Jejunal perforation | - | Invasive intervention not indicated | Invasive intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Definition: A disorder character<br>Navigational Note: - | cterized by a rupture in the jejunal wall | | | | |
| Jeiunal stenosis | Asymptomatic; clinical or | Symptomatic: altered GI | S | Life-threatening | Death |
| Jejunai stenosis | Asymptomatic; cirilical or<br>diagnostic observations only;<br>intervention not indicated | function | Severely altered GI function;<br>tube feeding or<br>hospitalization indicated;<br>elective operative<br>intervention indicated | consequences; urgent operative intervention indicated | Deam |
| <b>Definition:</b> A disorder character Navigational Note: - | cterized by a narrowing of the lumen o | the jejunum. | • | • | · |
| Jejunal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN indicated; elective<br>invasive intervention | Life-threatening<br>consequences; urgent<br>operative intervention | Death |
| | | | indicated | indicated | |
| | <br>cterized by a circumscribed, erosive les | <br>ion on the mucosal surface of the je | | indicated | I |
| <b>Definition:</b> A disorder character Navigational Note: - Lip pain | cterized by a circumscribed, erosive les Mild pain | ion on the mucosal surface of the je Moderate pain; limiting instrumental ADL | | indicated | - |
| Navigational Note: -<br>Lip pain | Mild pain | Moderate pain; limiting instrumental ADL | ejunum. Severe pain; limiting self care | indicated | - |
| Navigational Note: -<br>Lip pain | • | Moderate pain; limiting instrumental ADL | ejunum. Severe pain; limiting self care | Indicated - | - |
| Navigational Note: -<br>Lip pain Definition: A disorder charac | Mild pain | Moderate pain; limiting instrumental ADL | ejunum. Severe pain; limiting self care | Life-threatening consequences; urgent intervention indicated | - Death |
| Navigational Note: -<br>Lip pain Definition: A disorder character Navigational Note: - Lower gastrointestinal hemorrhage | Mild pain cterized by a sensation of marked disco | Moderate pain; limiting instrumental ADL mfort of the lip. Moderate symptoms; intervention indicated | Severe pain; limiting self care ADL Transfusion indicated; invasive intervention indicated; hospitalization | Life-threatening consequences; urgent | -<br>Death |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Gastrointestinal disord | ers | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Mucositis oral | Asymptomatic or mild<br>symptoms; intervention not<br>indicated | Moderate pain or ulcer that<br>does not interfere with oral<br>intake; modified diet<br>indicated | Severe pain; interfering with<br>oral intake | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder charac<br>Navigational Note: - | cterized by ulceration or inflammation | of the oral mucosal. | | | |
| Nausea | Loss of appetite without alteration in eating habits | Oral intake decreased without significant weight loss, dehydration or malnutrition | Inadequate oral caloric or<br>fluid intake; tube feeding,<br>TPN, or hospitalization<br>indicated | - | - |
| | cterized by a queasy sensation and/or t | he urge to vomit. | | | |
| Navigational Note: - | | | | | |
| Obstruction gastric | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function; limiting instrumental<br>ADL | Hospitalization indicated;<br>invasive intervention<br>indicated; limiting self care<br>ADL | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| <b>Definition:</b> A disorder character Navigational Note: - | cterized by blockage of the normal flow | of the contents in the stomach. | | • | • |
| Oral cavity fistula | Asymptomatic | Symptomatic, invasive intervention not indicated | Invasive intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | cterized by an abnormal communicatio | n between the oral cavity and anoth | ner organ or anatomic site. | • | ' |
| Navigational Note: - | I amagina a sa | I and a second | I | T | |
| Oral dysesthesia | Mild discomfort; not<br>interfering with oral intake | Moderate pain; interfering<br>with oral intake | Disabling pain; tube feeding or<br>TPN indicated | - | - |
| Definition: A disorder charac | cterized by a burning or tingling sensati | on on the lips, tongue or entire mo | uth. | | |
| Navigational Note: - | | | | | |
| Oral hemorrhage | Mild symptoms; intervention<br>not indicated | Moderate symptoms;<br>intervention indicated | Transfusion indicated;<br>invasive intervention<br>indicated; hospitalization | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder charac | cterized by bleeding from the mouth. | · | : | = | • |
| Navigational Note: - | | | | | |
| Oral pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| <b>Definition:</b> A disorder character Navigational Note: - | cterized by a sensation of marked disco | mfort in the mouth, tongue or lips. | | • | ·<br> |

| | | Gastrointestinal disord | ders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Pancreatic duct stenosis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI<br>function | Severely altered GI function;<br>tube feeding or<br>hospitalization indicated;<br>elective operative<br>intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| <b>Definition:</b> A disorder character Navigational Note: - | terized by a narrowing of the lumen of | the pancreatic duct. | | | |
| Pancreatic fistula | Asymptomatic | Symptomatic, invasive intervention not indicated | Invasive intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder character Navigational Note: - | terized by an abnormal communicatio | n between the pancreas and anoth | er organ or anatomic site. | | |
| Pancreatic hemorrhage | Mild symptoms; intervention<br>not indicated | Moderate symptoms;<br>intervention indicated | Transfusion indicated;<br>invasive intervention<br>indicated; hospitalization | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder character Navigational Note: - | terized by bleeding from the pancreas | | • | • | · |
| Pancreatic necrosis | - | - | Tube feeding or TPN indicated; invasive intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Definition: A disorder charac | ।<br>terized by a necrotic process occurring | in the pancreas. | 1 | | ! |
| Navigational Note: - | | | | | |
| Pancreatitis | - | Enzyme elevation; radiologic findings only | Severe pain; vomiting;<br>medical intervention indicated<br>(e.g., analgesia, nutritional<br>support) | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder charac | terized b <b>y</b> inflammation of the pancre | as with no documented pancreas ir | nfection. | | • |
| Navigational Note: - | | | | | |
| Periodontal disease | Gingival recession or<br>gingivitis; limited bleeding on<br>probing; mild local bone loss | Moderate gingival recession<br>or gingivitis; multiple sites of<br>bleeding on probing;<br>moderate bone loss | Spontaneous bleeding; severe<br>bone loss with or without<br>tooth loss; osteonecrosis of<br>maxilla or mandible | - | - |
| | gingival tissue around the teeth. | | | | |
| Navigational Note: - | | | | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Gastrointestinal disord | lers | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Peritoneal necrosis | - | - | Tube feeding or TPN indicated; invasive intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Definition: A disorder cha<br>Navigational Note: - | racterized by a necrotic process occurring | ; in the peritoneum. | | | |
| Proctitis | Rectal discomfort. | Symptomatic (e.g., rectal | Severe symptoms; fecal | Life-threatening | Death |
| riocaus | intervention not indicated | discomfort, passing blood or<br>mucus); medical intervention<br>indicated; limiting<br>instrumental ADL | urgency or stool incontinence;<br>limiting self care ADL | consequences; urgent intervention indicated | Deau |
| Definition: A disorder cha<br>Navigational Note: - | racterized by inflammation of the rectum | | | | |
| Rectal fissure | Asymptomatic | Symptomatic | Invasive intervention indicated | - | = |
| | racterized by a tear in the lining of the re | ctum. | | - | |
| Navigational Note: - | | T | T | Luci | 1 5 4 |
| Rectal fistula | Asymptomatic | Symptomatic, invasive<br>intervention not indicated | Invasive intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | racterized by an abnormal communicatio | n between the rectum and another | organ or anatomic site. | | · |
| Navigational Note: -<br>Rectal hemorrhage | Mild symptoms: intervention | Moderate symptoms; | Transfusion indicated: | Life-threatening | Death |
| recearment nage | not indicated | intervention indicated | invasive intervention<br>indicated; hospitalization | consequences; urgent<br>intervention indicated | Deadi |
| <b>Definition:</b> A disorder cha | racterized by bleeding from the rectal wa | I and discharged from the anus. | , | The Control of the Control | ı |
| <b>Definition:</b> A disorder cha<br><b>Navigational Note:</b> - | acterized by bleeding from the rectal wa | I and discharged from the anus. | , | incorvenius i i i i i i i i i i i i i i i i i i | ı |
| | | Gastrointestinal disord | ers | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 9 |
| Rectal necrosis | - | - | Tube feeding or TPN indicated; invasive intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| <b>Definition:</b> A disorder char<br><b>Navigational Note:</b> - | acterized by a necrotic process occurring | in the rectal wall. | | | |
| Rectal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function; limiting instrumental<br>ADL | Hospitalization indicated;<br>invasive intervention<br>indicated; limiting self care<br>ADL | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| <b>Definition:</b> A disorder char<br><b>Navigational Note:</b> - | acterized by blockage of the normal flow | of the intestinal contents in the rec | ctum. | | |
| Rectal pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder char | acterized by a sensation of marked disco | mfort in the rectal region. | | • | · |
| Navigational Note: - | | | | | |
| Rectal perforation | - | Invasive intervention not indicated | Invasive intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| <b>Definition:</b> A disorder char<br><b>Navigational Note:</b> - | acterized by a rupture in the rectal wall. | | | | |
| Rectal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function | Severely altered GI function;<br>tube feeding or<br>hospitalization indicated;<br>elective operative<br>intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| | | 1 | intervention indicated | 1 | |
| | acterized by a narrowing of the lumen of | the rectum. | Intervention indicated | • | ı |
| <b>Definition:</b> A disorder char<br><b>Navigational Note:</b> -<br>Rectal ulcer | acterized by a narrowing of the lumen of Asymptomatic; clinical or | the rectum. Symptomatic; altered GI | Severely altered GI function; | Life-threatening | <u>'</u> |

| | | Gastrointestinal disord | ers | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Retroperitoneal hemorrhage | - | Self-limited; intervention indicated | Transfusion indicated;<br>invasive intervention<br>indicated; hospitalization | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder characteri | ized by bleeding from the retroperi | toneal area. | | • | • |
| Navigational Note: - | | | | | |
| Salivary duct inflammation | Slightly thickened saliva;<br>slightly altered taste (e.g.,<br>metallic) | Thick, ropy, sticky saliva;<br>markedly altered taste;<br>alteration in diet indicated;<br>secretion-induced symptoms;<br>limiting instrumental ADL | Acute salivary gland necrosis;<br>severe secretion-induced<br>symptoms (e.g., thick<br>saliva/oral secretions or<br>gagging); tube feeding or TPN<br>indicated; limiting self care<br>ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder characteri | ized by inflammation of the salivary | duct. | | | |
| Navigational Note: - | | | | | |
| Salivary gland fistula | Asymptomatic | Symptomatic, invasive<br>intervention not indicated | Invasive intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | ized b <b>y</b> an abnormal communicatio | n between a salivary gland and anot | ther organ or anatomic site. | | |
| Navigational Note: - | | | | Lie | |
| Small intestinal mucositis | Asymptomatic or mild<br>symptoms; intervention not<br>indicated | Symptomatic; medical<br>intervention indicated;<br>limiting instrumental ADL | Severe pain; interfering with<br>oral intake; tube feeding, TPN<br>or hospitalization indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder characteri | ized by ulceration or inflammation | of the mucous membrane of the sm | all intestine. | • | |
| Navigational Note: - | • | | | | |
| Small intestinal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function; limiting instrumental<br>ADL | Hospitalization indicated;<br>invasive intervention<br>indicated; limiting self care<br>ADL | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Definition: A disorder characteri | ized by blockage of the normal flow | of the intestinal contents of the sm | all intestine. | | |
| Navigational Note: - | | | | | |
| Small intestinal perforation | - | Invasive intervention not indicated | Invasive intervention indicated | Life-threatening consequences; urgent | Death |

# **Cerus Corporation**

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Gastrointestinal disord | ers | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Small intestinal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function | Symptomatic and severely<br>altered GI function; tube<br>feeding, TPN or<br>hospitalization indicated; non-<br>emergent operative<br>intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Definition: A disorder character | rized by a narrowing of the lumen of | the small intestine. | • | • | • |
| Navigational Note: - | | | | | |
| Small intestine ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function; limiting instrumental<br>ADL | Severely altered GI function;<br>TPN indicated; elective<br>invasive intervention<br>indicated; limiting self care<br>ADL | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Definition: A disorder character | rized by a circumscribed, erosive lesi | on on the mucosal surface of the sr | nall intestine. | • | • |
| Navigational Note: - | • | | | | |
| Stomach pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder character | rized by a sensation of marked disco | mfort in the stomach. | • | • | • |
| Navigational Note: - | | | | | |
| Tooth development disorder | Asymptomatic; hypoplasia of tooth or enamel | Impairment correctable with<br>oral surgery | Maldevelopment with<br>impairment not surgically<br>correctable; limiting self care<br>ADL | - | - |
| Definition: A disorder character | rized by a pathological process of the | e teeth occurring during tooth deve | lopment. | • | • |
| Navigational Note: - | | | | | |
| Tooth discoloration | Surface stains | - | - | - | - |
| Definition: A disorder character | rized by a change in tooth hue or tin | t. | • | • | • |
| Navigational Note: - | - | | | | |
| Toothache | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder character | rized by a sensation of marked disco | mfort in the tooth. | | | |
| Navigational Note: - | | | | | |

# **Cerus Corporation**

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Gastrointestinal disord | ers | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Typhlitis | - | - | Symptomatic (e.g., abdominal<br>pain, fever, change in bowel<br>habits with ileus); peritoneal<br>signs | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Definition: A disorder characte | rized by necrotizing enterocolitis in r | neutropenic patients. | | • | |
| Navigational Note: Also report | :Investigations:Neutrophil count dec | reased | | | |
| Upper gastrointestinal hemorrhage | Mild symptoms; intervention not indicated | Moderate symptoms;<br>intervention indicated | Transfusion indicated;<br>invasive intervention<br>indicated; hospitalization | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | rized by bleeding from the upper gas | trointestinal tract (oral cavit <b>y,</b> phar | ynx, esophagus, and stomach). | | |
| Navigational Note: - | | Latition 1 1 1 | T a 16 a41 3 | Lieur | 1 5 3 |
| Visceral arterial ischemia | - | Brief (<24 hrs) episode of<br>ischemia managed medically<br>and without permanent<br>deficit | Prolonged (>=24 hrs) or<br>recurring symptoms and/or<br>invasive intervention<br>indicated | Life-threatening<br>consequences; evidence of<br>end organ damage; urgent<br>operative intervention<br>indicated | Death |
| Definition: A disorder characte | rized by a decrease in blood supply o | due to narrowing or blockage of a vi | sceral (mesenteric) artery. | • | |
| Navigational Note: - | | | | | |
| Vomiting | Intervention not indicated | Outpatient IV hydration;<br>medical intervention indicated | Tube feeding, TPN, or<br>hospitalization indicated | Life-threatening consequences | Death |
| <b>Definition:</b> A disorder characte | rized by the reflexive act of ejecting | the contents of the stomach throug | h the mouth. | | |
| Navigational Note: - | | | | | |
| Gastrointestinal disorders -<br>Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: - | | | | | |
| Navigational Note: - | | | | | |

| | Ge | eneral disorders and administration | site conditions | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Chills | Mild sensation of cold; | Moderate tremor of the entire | Severe or prolonged, not | - | - |
| | shivering; chattering of teeth | body; narcotics indicated | responsive to narcotics | l | |
| | zed b <b>y</b> a sensation of cold that ofte | n marks a ph <b>y</b> siologic response to s | weating after a fever. | | |
| Navigational Note: - | | | | | |
| Death neonatal | - | - | - | Neonatal loss of life | - |
| <b>Definition:</b> Newborn death occur | rring during the first 28 days after b | irth. | | | |
| Navigational Note: - | | | | | |
| Death NOS | - | - | - | - | Death |
| Definition: Death that cannot be | attributed to a CTCAE term associa | ited with Grade 5. | | | |
| Navigational Note: If death is du | e to an AE (ex., Cardiac disorders: 0 | Cardiac arrest), report as a Grade 5 e | event under that AE. | | |
| Disease progression | = | = | - | - | Death |
| Definition: Death due to disease | progression that cannot be attribu- | ted to a CTCAE term associated wit | n Grade 5. | • | · · |
| Navigational Note: If death is du | e to an AE (ex., Cardiac disorders: 0 | Cardiac arrest), report as a Grade 5 | event under that AE. | | |
| Edema face | Localized facial edema | Moderate localized facial | Severe swelling; limiting self | - | - |
| | | edema; limiting instrumental | care ADL | | |
| | | ADL | | l | |
| | zed b <b>y</b> swelling due to excessive flu | id accumulation in facial tissues. | | | |
| Navigational Note: - | | | | | |
| Edema limbs | 5 - 10% inter-limb discrepancy | >10 - 30% inter-limb | >30% inter-limb discrepancy | - | - |
| | in volume or circumference at | discrepancy in volume or | in volume; gross deviation | | |
| | point of greatest visible | circumference at point of | from normal anatomic | | |
| | difference; swelling or | greatest visible difference; | contour; limiting self care ADL | | |
| | obscuration of anatomic | readily apparent obscuration | | | |
| | architecture on close | of anatomic architecture; | | | |
| | inspection | obliteration of skin folds; | | | |
| | | readily apparent deviation | | | |
| | | from normal anatomic | | | |
| | | contour; limiting instrumental | | | |
| 1 | I | ADL | | I | 1 |
| | zed by swelling due to excessive flu | id accumulation in the upper or low | er extremities. | | |
| Navigational Note: - | | | | | |

| | G | eneral disorders and administration | n site conditions | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Edema trunk | Swelling or obscuration of<br>anatomic architecture on<br>close inspection | Readily apparent obscuration<br>of anatomic architecture;<br>obliteration of skin folds;<br>readily apparent deviation<br>from normal anatomic<br>contour; limiting instrumental | Gross deviation from normal<br>anatomic contour; limiting self<br>care ADL | - | - |
| Definition, A disaudar dagestari | Tad by availing due to everyour fire | ADL | l | l | ļ |
| Navigational Note: - | zed by swelling due to excessive flu | iid accumulation in the trunk area. | | | |
| Facial pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteri<br>Navigational Note: - | zed by a sensation of marked disco | mfort in the face. | | | |
| Fatigue | Fatigue relieved by rest | Fatigue not relieved by rest;<br>limiting instrumental ADL | Fatigue not relieved by rest,<br>limiting self care ADL | = | - |
| Definition: A disorder characteri<br>Navigational Note: - | zed by a state of generalized weak | ness with a pronounced inability to | summon sufficient energy to accom | plish daily activities. | |
| Fever | 38.0 - 39.0 degrees C (100.4 -<br>102.2 degrees F) | >39.0 - 40.0 degrees C (102.3 -<br>104.0 degrees F) | >40.0 degrees C (>104.0<br>degrees F) for <=24 hrs | >40.0 degrees C (>104.0<br>degrees F) for >24 hrs | Death |
| Definition: A disorder characteri | zed by elevation of the body's tem | perature above the upper limit of no | ormal. | • | |
| Navigational Note: - | | | | | |
| Flu like symptoms | Mild flu-like symptoms present | Moderate symptoms; limiting<br>instrumental ADL<br>to those observed in patients with | Severe symptoms; limiting self care ADL | - | |
| cough. | zed by a group or symptoms simila | to those observed in patients with | rate na. remadaes lever, anns, bod | y acries, maraise, ross or appear | and dry |
| Navigational Note: Synonym: Flu | u, Influenza | | | | |
| Gait disturbance | Mild change in gait (e.g.,<br>wide-based, limping or<br>hobbling) | Moderate change in gait (e.g.,<br>wide-based, limping or<br>hobbling}; assistive device<br>indicated; limiting<br>instrumental ADL | Limiting self care ADL | - | - |
| <b>Definition:</b> A disorder characteri<br><b>Navigational Note:</b> - | zed by walking difficulties. | - | | - | |

| | G | eneral disorders and administratio | n site conditions | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Generalized edema | Noted on exam; 1+ pitting | Interfering with instrumental | Interferes with self care ADL; | Life-threatening consequences | - |
| | edema | ADLs; oral therapy initiated | intravenous therapy | | |
| | | 1 | indicated; skin breakdown | | |
| Definition: A disorder characte | rized by fluid accumulation in the tis | sues of the body including the skin. | | | |
| Navigational Note: - | | | | | |
| Hypothermia | - | 35 - >32 degrees C; 95 - >89.6 | 32 - >28 degrees C; 89.6 - | <=28 degrees C; 82.4 degrees | Death |
| | | degrees F | >82.4 degrees F | F; life-threatening | |
| | | | | consequences (e.g., coma, | |
| | | | | hypotension, pulmonary | |
| | | | | edema, acidemia, ventricular | |
| | | 1 | | fibrillation) | |
| <b>Definition:</b> A disorder characte | rized by an abnormally low body ten | nperature. Treatment is required w | hen the body temperature is 35C (9 | 5F) or below. | |
| Navigational Note: - | | | | | |
| Infusion site extravasation | Painless edema | Erythema with associated | Ulceration or necrosis; severe | Life-threatening | Death |
| | | symptoms (e.g., edema, pain, | tissue damage; operative | consequences; urgent | |
| | | induration, phlebitis) | intervention indicated | intervention indicated | |
| | rized by leakage of the infusion into | the surrounding tissue. Signs and s | ymptoms may indude induration, e | rythema, swelling, burning sensatio | n and |
| marked discomfort at the infus | ion site. | | | | |
| Navigational Note: - | T | | | T | |
| Injection site reaction | Tenderness with or without | Pain; lipodystrophy; edema; | Ulceration or necrosis; severe | Life-threatening | Death |
| | associated symptoms (e.g., | phlebitis | tissue damage; operative | consequences; urgent | |
| | warmth, erythema, itching) | I | intervention indicated | intervention indicated | l |
| | rized b <b>y</b> an intense adverse reaction | (usually immunologic) developing | at the site of an injection. | | |
| Navigational Note: - | | | | | |
| Localized edema | Localized to dependent areas, | Moderate localized edema | Severe localized edema and | - | - |
| | no disability or functional | and intervention indicated; | intervention indicated; | | |
| | impairment | limiting instrumental ADL | limiting self care ADL | l | |
| | rized by swelling due to excessive flu | | | | |
| | ng this term consider specific edema | | | | |
| | ma cerebral; Reproductive system ar | | ; Respiratory, thoracic and mediasti | nal disorders: Laryngeal edema or P | ulmonary |
| | tissue disorders: Periorbital edema; | | | | |
| Malaise | Uneasiness or lack of well | Uneasiness or lack of well | Uneasiness or lack of well | - | - |
| | being | being limiting instrumental | being limiting self-care ADL | | |
| | | ADL | | l | l |
| Definition: A disorder characte | rized by a feeling of general discomf | ort or uneasiness, an out-of-sorts fe | eeling. | | |
| Navigational Note: - | | | | | |

| | G | eneral disorders and administratio | n site conditions | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Multi-organ failure | - | - | Shock with azotemia and acid-<br>base disturbances; significant<br>coagulation abnormalities | Life-threatening consequences<br>(e.g., vasopressor dependent<br>and oliguric or anuric or<br>ischemic colitis or lactic<br>acidosis) | Death |
| | zed by progressive deterioration of | the lungs, liver, kidney and clotting | g mechanisms. | | |
| Navigational Note: - | | | | T | |
| Neck edema | Asymptomatic localized neck edema | Moderate neck edema; slight<br>obliteration of anatomic<br>landmarks; limiting<br>instrumental ADL | Generalized neck edema (e.g.,<br>difficulty in turning neck);<br>limiting self care ADL | Vascular or respiratory<br>impairment requiring urgent<br>intervention | - |
| <b>Definition:</b> A disorder characteri | zed by swelling due to an accumula | tion of excessive fluid in the neck. | | | |
| Navigational Note: - | | | | | |
| Non-cardiac chest pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteri | zed by a sensation of marked disco | mfort in the chest unrelated to a h | eart disorder. | | |
| Navigational Note: - | | | | | |
| Pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteri | zed by the sensation of marked dis | comfort, distress or agony. | | | |
| Navigational Note: Prior to using | g this term consider using a specific | body part pain term found through | hout the CTCAE (over 40 different p | ain terms). | |
| Sudden death NOS | - | - | - | - | Death |
| Definition: An unexpected death | n that cannot be attributed to a CTC | AE term associated with Grade 5. | • | | |
| Navigational Note: If death is du | ie to an AE (ex., Cardiac disorders: 0 | Cardiac arrest), report as a Grade 5 | event under that AE. | | |
| Vaccination site<br>lymphadenopathy | Local lymph node<br>enlargement | Localized ulceration;<br>generalized lymph node<br>enlargement | - | - | - |
| | zed by lymph node enlargement af | ter vaccination. | • | | • |
| Navigational Note: - | | | | | |
| General disorders and<br>administration site conditions<br>- Other, specify | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: - | | - | | • | • |
| Navigational Note: - | | | | | |

# **Cerus Corporation**

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Hepatobiliary disord | ers | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Bile duct stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered Gl<br>function; IV fluids indicated<br><24 hrs | Severely altered GI function;<br>invasive intervention<br>indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| <b>Definition:</b> A disorder character Navigational Note: - | terized by a narrowing of the lumen o | f the bile duct. | | | |
| Biliary fistula | - | Symptomatic, invasive intervention not indicated | Invasive intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder charac | terized by an abnormal communicatio | n between the bile ducts and anot | ther organ or anatomic site. | | |
| Navigational Note: - | | | | | • |
| Budd-Chiari syndrome | | Medical management indicated | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>asterixis; mild encephalopathy | Life-threatening<br>consequences; moderate to<br>severe encephalopathy; coma | Death |
| <b>Definition:</b> A disorder character Navigational Note: - | sterized by occlusion of the hepatic vei | ns and typically presents with abd | ominal pain, ascites and hepatomega | ly. | |
| Cholecystitis | - | Symptomatic; medical intervention indicated | Severe symptoms; invasive intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| <b>Definition:</b> A disorder character Navigational Note: - | terized by inflammation involving the | gallbladder. It may be associated v | with the presence of gallstones. | • | • |
| Gallbladder fistula | Asymptomatic | Symptomatic, invasive intervention not indicated | Invasive intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder character Navigational Note: - | terized by an abnormal communicatio | n between the gallbladder and an | other organ or anatomic site. | • | • |
| Gallbladder necrosis | - | - | - | Life-threatening<br>consequences; urgent invasive<br>intervention indicated | Death |
| Definition: A disorder charac | terized by a necrotic process occurring | in the gallbladder. | • | • | • |
| Navigational Note: - | | | | | |

| | | Hepatobiliary disord | ers | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Gallbladder obstruction | Asymptomatic; dinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function; IV fluids indicated<br><24 hrs | Symptomatic and severely<br>altered GI function; tube<br>feeding, TPN or<br>hospitalization indicated; non-<br>emergent operative<br>intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| | ized by blockage of the normal flow | of the contents of the gallbladder | | | |
| Navigational Note: - | | | | | |
| Gallbladder pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| | ized b <b>y</b> a sensation of marked disco | mfort in the gallbladder region. | | | |
| Navigational Note: - | | | | | |
| Gallbladder perforation | - | - | - | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder character | ized by a rupture in the gallbladder | wall. | 1 | | ' |
| Navigational Note: - | , , | | | | |
| Hepatic failure | - | - | Asterixis; mild<br>encephalopathy; drug-<br>induced liver injury (DILI);<br>limiting self care ADL | Life-threatening<br>consequences; moderate to<br>severe encephalopathy; coma | Death |
| Definition: A disorder character | ized by the inability of the liver to m | ■<br>netabolize chemicals in the body. I | aboratory test results reveal abnorm | ∎<br>nal plasma levels of ammonia, biliru | l<br>bin, lactic |
| | | | NR.) Drug-induced liever injury (DILI) | | , |
| Navigational Note: - | | | | | |
| Hepatic hemorrhage | Mild symptoms; intervention not indicated | Moderate symptoms;<br>intervention indicated | Transfusion indicated;<br>invasive intervention<br>indicated; hospitalization | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder character | ized by bleeding from the liver. | | | | |
| Navigational Note: - | _ | T | 1 | 1 126- 4 | DH- |
| Hepatic necrosis | - | - | | Life-threatening<br>consequences; urgent invasive<br>intervention indicated | Death |
| Definition: A disorder character | ized by a necrotic process occurring | in the hepatic parenchyma. | • | • | • |
| Navigational Note: - | | | | | |

| | | Hepatobiliary disorde | rs | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Hepatic pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder chara- | cterized by a sensation of marked disco | mfort in the liver region. | | - | |
| Navigational Note: - | | | | | |
| Perforation bile duct | - | - | Invasive intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Definition: A disorder chara- | cterized by a rupture in the wall of the | extrahepatic or intrahepatic bile du | ct. | | |
| Navigational Note: - | | | | | |
| Portal hypertension | - | Decreased portal vein flow | Reversal/retrograde portal<br>vein flow; associated with<br>varices and/or ascites | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder chara- | cterized b <b>y</b> an increase in blood pressui | re in the portal venous system. | | | |
| Navigational Note: - | | | | | |
| Portal vein thrombosis | - | Intervention not indicated | Medical intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder chara- | cterized by the formation of a thrombu | s (blood clot) in the portal vein. | • | • | • |
| Navigational Note: - | | | | | |
| Sinusoidal obstruction<br>syndrome | - | Blood bilirubin 2-5 mg/dL;<br>minor interventions required<br>(i.e., blood product, diuretic,<br>axygen) | Blood bilirubin >5 mg/dL;<br>coagulation modifier indicated<br>(e.g., defibrotide); reversal of<br>flow on ultrasound | Life-threatening<br>consequences (e.g.,<br>ventilatory support, dialysis,<br>plasmapheresis, peritoneal<br>drainage) | Death |
| Definition: A disorder chara- | cterized by severe hepatic injury as a re | sult of the blood vessels of the liver | r becoming inflamed and/or blocked | i. | |
| Navigational Note: - | | | | | |
| Hepatobiliar <b>y</b> disorders -<br>Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| _ | • | - | • | - | • |
| Definition: - | | | | | |

| | | Immune system disord | lers | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Allergic reaction | Systemic intervention not indicated | Oral intervention indicated | Bronchospasm;<br>hospitalization indicated for<br>clinical sequelae; intravenous<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder charact | erized by an adverse local or general | response from exposure to an aller | gen. | | |
| Navigational Note: If related t | to infusion, use Injury, poisoning and | procedural complications:Infusion | related reaction. Do not report both | 1. | |
| Anaphylaxis | · | | Symptomatic bronchospasm,<br>with or without urticaria;<br>parenteral intervention<br>indicated; allergy-related<br>edema/angioedema;<br>hypotension | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | erized by an acute inflammatory reac<br>t presents with breathing difficulty, di | | | | ersensitivity |
| Autoimmune disorder | Asymptomatic; serologic or | Evidence of autoimmune | Autoimmune reactions | Life-threatening | Death |
| Addrillianc disorder | other evidence of<br>autoimmune reaction, with<br>normal organ function;<br>intervention not indicated | reaction involving a non-<br>essential organ or function<br>(e.g., hypothyroidism) | involving major organ (e.g.,<br>colitis, anemia, myocarditis,<br>kidney) | consequences; urgent intervention indicated | Deadi |
| <b>Definition:</b> A disorder charact<br>own tissue constituents. | erized by loss of function or tissue de | struction of an organ or multiple or | gans, arising from humoral or cellul | ar immune responses of the individ | dual to his |
| Navigational Note: Prior to us | sing this term consider specific autoim | | | | |
| Cytokine release syndrome | Fever with or without constitutional symptoms | Hypotension responding to fluids; hypoxia responding to <40% O2 | Hypotension managed with<br>one pressor; hypoxia requiring<br>≥ 40% O2 | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder charact | erized by fever, tachypnea, headache | , tachycardia, hypotension, rash, ar | nd/or hypoxia caused by the release | of cytokines. | |
| Navigational Note: Also consi | der reporting other organ dysfunctior | ns including neurological toxicities s | such as: Psychiatric disorders: Halluc | inations or Confusion; Nervous sys | tem |
| disorders: Seizure, Dysphasia, | | | | | |
| 6 | Asymptomatic; clinical or | Moderate arthralgia; fever, | Severe arthralgia or arthritis;<br>extensive rash; steroids or IV | Life-threatening consequences; pressor or | Death |
| Serum sickness | diagnostic observations only;<br>intervention not indicated | rash, urticaria, antihistamines<br>indicated | fluids indicated | | |
| | diagnostic observations only;<br>intervention not indicated<br>erized by a delayed-type hypersensiti | indicated | fluids indicated | ventilatory support indicated | days |
| <b>Definition:</b> A disorder charact | intervention not indicated | indicated<br>vity reaction to foreign proteins de | fluids indicated<br>rived from an animal serum. It occur | ventilatory support indicated<br>s approximately six to twenty-one | |

# **Cerus Corporation**

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| Immune system disorders | | | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Immune system disorders -<br>Other, specify | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: - | | | | | |
| Navigational Note: - | | | | | |

| | | Infections and infestation | ons | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Abdominal infection | - | Oral intervention indicated (e.g., antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | cterized by an infectious process invol | ving the abdominal cavity. | | | |
| Navigational Note: - | | | | | |
| Anorectal infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder chara-<br><b>Navigational Note:</b> - | cterized by an infectious process invol | ving the anal area and the rectum. | | | |
| Appendicitis | - | - | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder characteristic Advisor of the Navigational Note: - | cterized by acute inflammation to the | vermiform appendix caused by a pat | hogenic agent. | | |
| Appendicitis perforated | - | - | Medical intervention<br>indicated; operative<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | r<br>cterized by acute inflammation to the<br>ndiceal wall rupture causes the release | | hogenic agent with gangrenous ch | nanges resulting in the rupture of | the |
| Navigational Note: - | • | • | | • | |
| Arteritis infective | - | - | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder chara- | cterized by an infectious process invol | ving an artery. | • | • | • |
| Navigational Note: - | | | | | |
| Bacteremia | - | Blood culture positive with no signs or symptoms | - | - | - |
| Definition: A disorder chara- | cterized by the presence of bacteria in | the blood stream. | • | - | • |
| Navigational Note: Consider | Infections and infestations: Sepsis (Gi | rades 3, 4 & 5) | | | |

| Infections and infectations | | | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Biliary tract infection | - | Oral intervention indicated (e.g., antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder characte<br><b>Navigational Note:</b> - | rized b <b>y a</b> n infectious process invol | ving the biliary tract. | | | |
| Bladder infection | - | Oral intervention indicated (e.g., antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | rized by an infectious process invol | ving the bladder. | | | |
| Navigational Note: -<br>Bone infection | - | Oral intervention indicated (e.g., antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder characte<br><b>Navigational Note:</b> - | erized by an infectious process invol | ving the bones. | • | • | • |
| Breast infection | - | Local infection with moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; severe infection;<br>axillary adenitis | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invol | • | 1 | • | 1 |
| Navigational Note: - | | | | | |
| Bronchial infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | rized by an infectious process invol | ving the bronchi. | | | · |
| Navigational Note: -<br>Catheter related infection | - | Localized; local intervention indicated; oral intervention indicated (e.g., antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder character <b>Navigational Note:</b> - | rized by an infectious process that | arises secondary to catheter use. | | - | • |

| | Infections and infestati | ons | | |
|---|---|---|---|---|
| Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| - | Localized; oral intervention indicated (e.g., antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| cterized b <b>y</b> an infectious process involv | ing the cecum. | | | |
| - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| cterized by an infectious process involv | ing the uterine cervix. | | | |
| Asymptomatic or mild symptoms; intervention not indicated | Symptomatic; moderate decrease in visual acuity (best corrected visual acuity 20/40 and better or 3 lines or less decreased vision from known baseline) | Symptomatic with marked decrease in visual aculty (best corrected visual aculty worse than 20/40 or more than 3 lines of decreased vision from known baseline, up to 20/200); limiting self care ADL | Best corrected visual acuity of<br>20/200 or worse in the<br>affected eye | - |
| cterized by inflammation, swelling and | redness to the conjunctiva of the ey | ye. | | |
| Infections and infestations: Conjunctiv | ritis infective if caused by infection | | | |
| | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | - |
| cterized by an infectious process involv | ing the conjunctiva. Clinical manifes | ,<br>stations include pink or red color in | the eyes. | |
| | - | • | - | |
| - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | cterized by an infectious process involved by an infectious process involved asymptoms; intervention not indicated cterized by inflammation, swelling and infections and infestations: Conjunctives | Grade 1 Grade 2 Localized; oral intervention indicated (e.g., antibiotic, antifungal, or antiviral) cterized by an infectious process involving the cecum. Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) cterized by an infectious process involving the uterine cervix. Asymptomatic or mild symptoms; intervention not indicated decrease in visual acuity (best corrected visual acuity 20/40 and better or 3 lines or less decreased vision from known baseline) cterized by inflammation, swelling and redness to the conjunctiva of the ellinfections and infestations: Conjunctivitis infective if caused by infection Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) cterized by an infectious process involving the conjunctiva. Clinical maniference in conjunctiva. | Grade 1 Grade 2 Grade 3 | Grade 1 Grade 2 Grade 3 Grade 4 |

| | Infections and infestati | ons | | |
|---|---|---|---|---|
| Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| - | - | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| terized b <b>y</b> an infectious process involv | ing a cranial nerve. | | | |
| Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; medical intervention indicated | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; IV<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated;<br>blindness | Death |
| terized by the reactivation of cytomes | alovirus (CMV). | • | • | • |
| :CMV | , | | | |
| - | Oral intervention indicated<br>(e.g., antibiotic, antifungal) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| terized by an infectious process involv | ing the use of a medical device. | • | • | • |
| - | Moderate symptoms; medical intervention indicated (e.g., oral antibiotics) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| terized by an infectious process involv | ing the duodenum. | • | • | • |
| - | - | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; severe changes in<br>mental status; self-limited | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | terized by an infectious process involv Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated terized by the reactivation of cytomeg: CMV - terized by an infectious process involv | terized by an infectious process involving a cranial nerve. Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated terized by the reactivation of cytomegalovirus (CMV). CONV Oral intervention indicated (e.g., antibiotic, antifungal) terized by an infectious process involving the use of a medical device. Moderate symptoms; medical intervention indicated (e.g., | - IV antiblotic, antifungal, or antiviral intervention indicated; invasive intervention or prolongation of existing hospitalization or prolongation of cytomegalovirus (CMV). - Oral intervention indicated (e.g., antifungal) - Moderate symptoms; medical intervention indicated but not immediately life-threatening; hospitalization or prolongation of existing hospitalization indicated intervention indicated - Oral intervention indicated (e.g., antifungal) - Moderate symptoms; medical intervention indicated (e.g., antifungal) - Woderate symptoms; medical intervention indicated intervention indicated; invasive intervention indicated; invasive intervention indicated; invasive intervention indicated intervention indicated intervention indicated. IV antibiotic, antifungal, or antiviral intervention indicated intervention indicated. - Woderate symptoms; medical intervention indicated intervention indicated. IV antibiotic, antifungal, or antiviral intervention indicated. | Grade 1 Grade 2 Grade 3 Grade 4 |

| Infections and infect ations | | | | |
|---|---|---|---|---|
| Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| - | | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| zed by an infectious process involvi | ng the brain and spinal cord tissues | | | |
| - | - | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| zed by an infectious process involvi | ng the endocardial layer of the hea | rt. | | |
| - | Local intervention indicated | Systemic intervention;<br>hospitalization indicated | Best corrected visual acuity of<br>20/200 or worse in the<br>affected eye | - |
| zed b <b>y</b> an infectious process involvi | ng the internal structures of the ey | e. | | • |
| - | per 24 hrs or duration of illness >48 hrs; moderate abdominal pain; oral intervention indicated (e.g., antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated;<br>profuse watery diarrhea with<br>signs of hypovolemia; bloody<br>diarrhea; fever; severe<br>abdominal pain;<br>hospitalization indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | ng the small and large intestines. | | | |
| | I | | Lie | T |
| Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; medical<br>intervention indicated | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; IV | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | zed by an infectious process involvi zed by an infectious process involvi zed by an infectious process involvi zed by an infectious process involvi difficile (c. diff, c. difficile). Asymptoms clinical or diagnostic observations only; | zed by an infectious process involving the brain and spinal cord tissues | Grade 1 Grade 2 Grade 3 | Grade 1 Grade 2 IV antiblotic, antifungal, or antiviral intervention indicated intervention; hospitalization indicated - Local intervention indicated - Local interve |

| | | Infections and infestati | ons | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Esophageal infection | - | Local intervention indicated<br>(e.g., oral antibiotic,<br>antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder chara<br><b>Navigational Note:</b> - | cterized by an infectious process involvi | ing the esophagus. | | | |
| Eye infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated;<br>enudeation | Death |
| | cterized by an infectious process involvi | ing the eye. | | | · |
| Navigational Note: -<br>Folliculitis | Covering <10% of the body<br>surface area; no intervention<br>indicated | Covering 10-30% of the body<br>surface area; topical<br>intervention initiated | >30% BSA; systemic intervention indicated | - | - |
| | cterized by inflammation or infection of | the hair follicles. | | | |
| Navigational Note: - | | I are a second second | T - " " " - | | |
| Fungemia | - | Moderate symptoms; medical intervention indicated | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated | - | - |
| Definition: A disorder chara | cterized by the presence of fungus in th | e blood stream. | , . | • | • |
| Navigational Note: - | | | | | |
| Gallbladder infection | - | Oral intervention indicated (e.g., antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | cterized by an infectious process involvi | ing the gallbladder. | | | |
| Navigational Note: - | | Laci | I 134 141 14 145 1 | Location | 1 5 2 |
| Gum infection | Local therapy indicated (swish and swallow) | Moderate symptoms; oral<br>intervention indicated (e.g.,<br>antibiotic, antifungal, or<br>antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder chara | cterized by an infectious process involvi | ing the gums. | | - | • |
| Navigational Note: - | | | | | |

| | | Infections and infestation | ons | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| | -<br>rized by an infectious process involvi | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, or antiviral) ing the liver. | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Navigational Note: - | T. A. 10 10 11 | Lagran and the second | I o | List of the second | T 6 11 |
| Hepatitis B reactivation | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; medical intervention indicated | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; IV<br>intervention indicated | Life-threatening consequences; urgent intervention indicated; severe decompensated liver function (e.g., coagulopathy, encephalopathy, coma) | Death |
| Definition: A disorder character | rized by the reactivation of hepatitis | B virus. | • | • | • |
| Navigational Note: - | | | | | |
| Hepatitis viral | Asymptomatic, intervention not indicated | Moderate symptoms; medical intervention indicated | Symptomatic liver<br>dysfunction; fibrosis by<br>biopsy; compensated<br>cirrhosis; hospitalization or<br>prolongation of existing<br>hospitalization indicated | Life-threatening consequences; severe decompensated liver function (e.g., coagulopathy, encephalopathy, coma) | Death |
| <b>Definition:</b> A disorder character <b>Navigational Note:</b> - | rized by a viral pathologic process in | volving the liver parenchyma. | | • | |
| Herpes simplex reactivation | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; medical intervention indicated | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; IV<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder character | rized by the reactivation of Herpes si | implex virus. | | • | , |
| Navigational Note: - | | • | | | |
| Infective myositis | - | Localized; local intervention<br>indicated (e.g., topical<br>antibiotic, antifungal, or<br>antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder character <b>Navigational Note:</b> - | rized by an infectious process involvi | ng the skeletal muscles. | | - | |

| Infections and infest ations | | | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Joint infection | - | Localized; local intervention<br>indicated; oral intervention<br>indicated (e.g., antibiotic,<br>antifungal, or antiviral);<br>needle aspiration indicated<br>(single or multiple) | Arthroscopic intervention indicated (e.g., drainage) or arthrotomy (e.g., open surgical drainage) | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder chara | acterized by an infectious process involv | ring a joint. | • | • | • |
| Navigational Note: - | | | | | |
| Kidney infection | - | Oral intervention indicated<br>(e.g., antibiotic, antifungal, or<br>antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder chara | acterized by an infectious process involv | ring the kidney. | • | • | • |
| Navigational Note: - | | | | | |
| Laryngitis | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | acterized by an inflammatory process in<br>optoms and no intervention, consider R | | disorders: Sore throat or Hoarsen | ess. | |
| Lip infection | Localized, local intervention indicated | Oral intervention indicated<br>(e.g., antibiotic, antifungal, or<br>antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | - | - |
| Definition: A disarder char- | acterized by an infectious process involv | ving the lips. | | • | • |
| Definition: A displace diale | | | | | |
| Navigational Note: - | | | | | |
| | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Navigational Note: -<br>Lung infection | -<br>acterized by an infectious process involv | intervention indicated (e.g.,<br>antibiotic, antifungal, or<br>antiviral) | antiviral intervention<br>indicated; invasive<br>intervention indicated | consequences; urgent | Death |

| Infections and infestations | | | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Lymph gland infection | - | Localized; oral intervention | IV antibiotic, antifungal, or | Life-threatening | Death |
| | | indicated (e.g., antibiotic, | antiviral intervention | consequences; urgent | |
| | | antifungal, or antiviral) | indicated; invasive | intervention indicated | |
| | | 1 | intervention indicated | 1 | |
| Definition: A disorder charac | terized by an infectious process involv | ring the lymph nodes. | | | |
| Navigational Note: - | | | | | |
| Mediastinal infection | = | - | IV antibiotic, antifungal, or | Life-threatening | Death |
| | | | antiviral intervention | consequences; urgent | |
| | | | indicated; invasive | intervention indicated | |
| | | | intervention indicated | | |
| Definition: A disorder charac | terized by an infectious process involved | ving the mediastinum. | • | • | • |
| Navigational Note: - | · | | | | |
| Meningitis | - | - | IV antibiotic, antifungal, or | Life-threatening | Death |
| - | | | antiviral intervention | consequences; urgent | |
| | | | indicated: invasive | intervention indicated | |
| | | | intervention indicated: focal | | |
| | | | neurologic deficit | | |
| Definition: A disorder charac | terized by acute inflammation of the | meninges of the brein and/or spinal | | • | |
| Navigational Note: - | cterized by acute irinarimation or the | neinges of the brain and or spinar | cora. | | |
| Mucosal infection | Localized, local intervention | Oral intervention indicated | IV antibiotic, antifungal, or | Life-threatening | Death |
| Mucosal infection | | | | | |
| | | leg antihiotic antifungal or | | | Deadi |
| | indicated | (e.g., antibiotic, antifungal, or | antiviral intervention | consequences; urgent | Deadi |
| | | (e.g., antibiotic, antifungal, or antiviral) | antiviral intervention indicated; invasive | | Deadi |
| Definition: A disorder charge | indicated | antiviral) | antiviral intervention | consequences; urgent | Death |
| | | antiviral) | antiviral intervention indicated; invasive | consequences; urgent | Deadi |
| Navigational Note: - | indicated trized by an infectious process involv | antiviral) ving a mucosal surface. | antiviral intervention<br>indicated; invasive<br>intervention indicated | consequences; urgent intervention indicated | |
| | indicated cterized by an infectious process involved. Asymptomatic; mild signs | antiviral) ving a mucosal surface. Moderate weakness or | antiviral intervention indicated; invasive intervention indicated | consequences; urgent intervention indicated Life-threatening | Death |
| Navigational Note: - | indicated terized by an infectious process involved. Asymptomatic; mild signs (e.g., Babinski's reflex or | antiviral) Ving a mucosal surface. Moderate weakness or sensory loss; limiting | antiviral intervention<br>indicated; invasive<br>intervention indicated | consequences; urgent intervention indicated Life-threatening consequences; urgent | |
| Navigational Note: -<br>Myelitis | indicated terized by an infectious process involved Asymptomatic; mild signs (e.g., Babinski's reflex or Lhermitte's sign) | antiviral) ving a mucosal surface. Moderate weakness or sensory loss; limiting instrumental ADL | antiviral intervention indicated; invasive intervention indicated Severe weakness or sensory loss; limiting self care ADL | consequences; urgent intervention indicated Life-threatening consequences; urgent intervention indicated | Death |
| Navigational Note: - Myelitis Definition: A disorder character | indicated terized by an infectious process involved. Asymptomatic; mild signs (e.g., Babinski's reflex or | antiviral) ving a mucosal surface. Moderate weakness or sensory loss; limiting instrumental ADL | antiviral intervention indicated; invasive intervention indicated Severe weakness or sensory loss; limiting self care ADL | consequences; urgent intervention indicated Life-threatening consequences; urgent intervention indicated | Death |
| Navigational Note: - Myelitis Definition: A disorder character Navigational Note: - | indicated cterized by an infectious process involved. Asymptomatic; mild signs (e.g., Babinski's reflex or Lhermitte's sign) cterized by inflammation involving the | antiviral) ving a mucosal surface. Moderate weakness or sensory loss; limiting instrumental ADL spinal cord. Symptoms include wea | antiviral intervention indicated; invasive intervention indicated Severe weakness or sensory loss; limiting self care ADL kness, paresthesia, sensory loss, m | consequences; urgent intervention indicated Life-threatening consequences; urgent intervention indicated | Death |
| Navigational Note: - Myelitis Definition: A disorder character | indicated cterized by an infectious process involved. Asymptomatic; mild signs (e.g., Babinski's reflex or Lhermitte's sign) cterized by inflammation involving the Localized, local intervention | antiviral) ving a mucosal surface. Moderate weakness or sensory loss; limiting instrumental ADL spinal cord. Symptoms include weather than the cord of the cord | antiviral intervention indicated; invasive intervention indicated Severe weakness or sensory loss; limiting self care ADL kness, paresthesia, sensory loss, m | consequences; urgent intervention indicated Life-threatening consequences; urgent intervention indicated | Death |
| Navigational Note: - Myelitis Definition: A disorder character Navigational Note: - | indicated cterized by an infectious process involved. Asymptomatic; mild signs (e.g., Babinski's reflex or Lhermitte's sign) cterized by inflammation involving the | antiviral) Ving a mucosal surface. Moderate weakness or sensory loss; limiting instrumental ADL spinal cord. Symptoms include weather than the cord of the cord. Symptoms include weather than the cord of the c | antiviral intervention indicated; invasive intervention indicated Severe weakness or sensory loss; limiting self care ADL kness, paresthesia, sensory loss, m IV antibiotic, antifungal, or antiviral intervention | consequences; urgent intervention indicated Life-threatening consequences; urgent intervention indicated | Death |
| Navigational Note: - Myelitis Definition: A disorder character Navigational Note: - | indicated cterized by an infectious process involved. Asymptomatic; mild signs (e.g., Babinski's reflex or Lhermitte's sign) cterized by inflammation involving the Localized, local intervention | antiviral) ving a mucosal surface. Moderate weakness or sensory loss; limiting instrumental ADL spinal cord. Symptoms include weather than the cord of the cord | antiviral intervention indicated; invasive intervention indicated Severe weakness or sensory loss; limiting self care ADL kness, paresthesia, sensory loss, m IV antibiotic, antifungal, or antiviral intervention indicated; invasive | consequences; urgent intervention indicated Life-threatening consequences; urgent intervention indicated | Death |
| Navigational Note: - Myelitis Definition: A disorder charact Navigational Note: - Nail infection | indicated cterized by an infectious process involved. Asymptomatic; mild signs (e.g., Babinski's reflex or Lhermitte's sign) cterized by inflammation involving the Localized, local intervention indicated | antiviral) ving a mucosal surface. Moderate weakness or sensory loss; limiting instrumental ADL spinal cord. Symptoms include weather of the cord of | antiviral intervention indicated; invasive intervention indicated Severe weakness or sensory loss; limiting self care ADL kness, paresthesia, sensory loss, m IV antibiotic, antifungal, or antiviral intervention | consequences; urgent intervention indicated Life-threatening consequences; urgent intervention indicated | Death |
| Navigational Note: - Myelitis Definition: A disorder charac Navigational Note: - Nail infection | indicated cterized by an infectious process involved. Asymptomatic; mild signs (e.g., Babinski's reflex or Lhermitte's sign) cterized by inflammation involving the Localized, local intervention | antiviral) ving a mucosal surface. Moderate weakness or sensory loss; limiting instrumental ADL spinal cord. Symptoms include weather of the cord of | antiviral intervention indicated; invasive intervention indicated Severe weakness or sensory loss; limiting self care ADL kness, paresthesia, sensory loss, m IV antibiotic, antifungal, or antiviral intervention indicated; invasive | consequences; urgent intervention indicated Life-threatening consequences; urgent intervention indicated | Death |

| | Infections and infest ations | | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Otitis externa | Localized, local intervention | Oral intervention indicated | IV antibiotic, antifungal, or | Life-threatening | Death |
| | indicated | (e.g., antibiotic, antifungal, or | antiviral intervention | consequences; urgent | |
| | | antiviral) | indicated; invasive | intervention indicated | |
| | | | intervention indicated | | |
| Definition: A disorder charact | erized by an infectious process involvi | ng the outer ear and ear canal. Cor | ntributory factors include excessive | water exposure (swimmer's ear | infection) and |
| cuts in the ear canal. Sympton | ns include fullness, itching, swelling ar | nd marked discomfort in the ear an | d ear drainage. | | |
| Navigational Note: Changes a | ssociated with radiation to external ea | ar (pinnae) are graded under Injury | , poisoning and procedural complic | cations: Dermatitis radiation | |
| Otitis media | - | Localized; oral intervention | IV antibiotic, antifungal, or | Life-threatening | Death |
| | | indicated (e.g., antibiotic, | antiviral intervention | consequences; urgent | |
| | | antifungal, or antiviral) | indicated; invasive | intervention indicated | |
| | | | intervention indicated | | |
| Definition: A disorder charact | erized by an infectious process involvi | ing the middle ear. | • | • | · |
| Navigational Note: - | | | | | |
| Ovarian infection | - | Localized; oral intervention | IV antibiotic, antifungal, or | Life-threatening | Death |
| | | indicated (e.g., antibiotic, | antiviral intervention | consequences; urgent | |
| | | antifungal, or antiviral) | indicated; invasive | intervention indicated | |
| | | | intervention indicated | | |
| Definition: A disorder charact | erized by an infectious process involvi | ing the ovary. | | - | · |
| Navigational Note: - | | | | | |
| Pancreas infection | - | - | IV antibiotic, antifungal, or | Life-threatening | Death |
| | | | antiviral intervention | consequences; urgent | |
| | | | indicated; invasive | intervention indicated | |
| | | 1 | intervention indicated | 1 | |
| Definition: A disorder charact | erized by an infectious process involvi | ing the pancreas. | | | - |
| Navigational Note: - | • | - | | | |

| | | Infections and infestati | ons | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Papulopustular rash | Papules and/or pustules covering <10% BSA, which may or may not be associated with symptoms of pruritus or tenderness | Papules and/or pustules covering 10-30% BSA, which may or may not be associated with symptoms of pruritus or tenderness; associated with psychosocial impact; limiting instrumental ADL; papules and/or pustules covering > 30% BSA with or without mild symptoms | Papules and/or pustules<br>covering >30% BSA with<br>moderate or severe<br>symptoms; limiting self-care<br>ADL; IV antibiotics indicated | Life-threatening<br>consequences | Death |
| Definition: A disorder charac | cterized by an eruption consisting of pa | pules (a small, raised pimple) and p | ustules (a small pus filled blister), t | typically appearing in face, scalp, | and upper |
| chest and back. Unlike acne, | this rash does not present with whiteh | eads or blackheads, and can be syn | nptomatic, with itchy or tender les | ions. | |
| Navigational Note: - | | | | | |
| Paron <b>y</b> chía | Nail fold edema or erythema;<br>disruption of the cutide | Local intervention indicated;<br>oral intervention indicated<br>(e.g., antibiotic, antifungal,<br>antiviral); nail fold edema or<br>erythema with pain;<br>associated with discharge or<br>nail plate separation; limiting<br>instrumental ADL | Operative intervention<br>indicated; IV antibiotics<br>indicated; limiting self care<br>ADL | | - |
| Definition: A disorder charac | cterized b <b>y</b> an infectious process involvi | ng the soft tissues around the nail. | | | |
| Navigational Note: - | | | | | |
| Pelvic infection | - | Moderate symptoms; oral<br>intervention indicated (e.g.,<br>antibiotic, antifungal, or<br>antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder character | cterized b <b>y</b> an infectious process involvi | ing the pelvic cavity. | | | |
| Navigational Note: - | | | | | |
| Penile infection | Localized, local intervention indicated | Oral intervention indicated<br>(e.g., antibiotic, antifungal, or<br>antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder charac | cterized b <b>y</b> an infectious process involvi | ing the penis. | • | - | • |
| Navigational Note: - | | | | | |

| | | Infections and infestati | ons | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Periorbital infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder charact | erized b <b>y</b> an infectious process involvi | ing the orbit of the eye. | | | |
| Navigational Note: - | | | | | |
| Peripheral nerve infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder charact | erized by an infectious process involvi | ing the peripheral nerves. | | | |
| Navigational Note: - | | | | | |
| Peritoneal infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder charact | erized by an infectious process involvi | ing the peritoneum. | | - | • |
| Navigational Note: - | | | | | |
| Pharyngitis | - | Oral intervention indicated (e.g., antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder charact | erized by inflammation of the throat. | | | | |
| Navigational Note: For Grade | 1 Consider Respiratory, thoracic and | mediastinal disorders: Sore throat | | | |
| Phlebitis infective | Localized, local intervention indicated | Oral intervention indicated<br>(e.g., antibiotic, antifungal, or<br>antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder charact | erized by an infectious process involvi | ing the vein. Clinical manifestations | include erythema, marked discor | nfort, swelling, and induration alo | ng the course |
| of the infected vein. | , , | 3 | • | . 3. | J |

# **Cerus Corporation**

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Infections and infestati | ons | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Pleural infection | - | Oral intervention indicated (e.g., antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder charac | terized b <b>y</b> an infectious process involv | ing the pleura. | | | |
| Navigational Note: - | | | | | |
| Prostate infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder charac | terized by an infectious process involv | ing the prostate gland. | • | • | • |
| Navigational Note: - | | 3 . 3 | | | |
| Rash pustular | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | - | - |
| Definition: A disorder charac | terized by a circumscribed and elevate | ed skin lesion filled with pus. | | • | • |
| Navigational Note: Synonym | : Boil | • | | | |
| Rhinitis infective | - | Localized; local intervention indicated | - | - | - |
| Definition: A disorder charac | terized by an infectious process involv | ing the nasal mucosal. | | • | · |
| Navigational Note: - | | | | | |
| Salivary gland infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder charac | terized by an infectious process involv | ing the salivary gland. | • | • | • |
| Navigational Note: - | | | | | |
| Scrotal infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder charac | terized by an infectious process involv | ing the scrotum. | | - | • |
| Navigational Note: - | | | | | |

| CTCAE Term Sepsis | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Sepsis | - | _ | -1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | | |
| | | | Blood culture positive with<br>signs or symptoms; treatment<br>indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder characterize<br><b>Navigational Note:</b> Includes SIRS. | | - | n that cause a rapidly progressing sy | stemic reaction that may lead t | o shock. |
| Shingles Definition: A disorder characterize | Localized, local intervention indicated | Local infection with moderate<br>symptoms; oral intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; IV<br>intervention indicated;<br>limiting self-care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Navigational Note: Synonym: Her | | Jaco Wilas. | | | |
| Sinusitis | - | Localized; oral intervention indicated (e.g., antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder characterize<br>Navigational Note: - | ed b <b>y</b> an infectious process involvi | ing the mucous membranes of the p | paranasal sinuses. | | |
| Skin infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder characterize | ed by an infectious process involvi | ing the skin such as cellulitis. | | • | • |
| Navigational Note: - | · | | | | |
| Small intestine infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |

| | | Infections and infestat | ions | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Soft tissue infection | - | Localized; oral intervention indicated (e.g., antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder chara | cterized by an infectious process invo | lving soft tissues. | | | |
| Navigational Note: - | | | | | |
| Splenic infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder chara | cterized by an infectious process invo | living the spleen. | • | • | • |
| Navigational Note: - | | | | | |
| Stoma site infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder chara<br><b>Navigational Note:</b> - | cterized by an infectious process invo | lving a stoma (surgically created ope | ning on the surface of the body). | • | · |
| Thrush | Asymptomatic; local<br>symptomatic management | Oral intervention indicated (e.g., antifungal) | IV antifungal intervention indicated | - | - |
| Definition: A disorder chara | cterized by a suspected candidal infe | ction involving an oral mucosal surfac | e. | | |
| Navigational Note: - | | | | | |
| Too th infection | - | Localized; local intervention<br>indicated (e.g., topical<br>antibiotic, antifungal, or<br>antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder chara | cterized by an infectious process invo | lving a tooth. | • | • | · |
| Navigational Note: - | | | | | |
| Tracheitis | - | Moderate symptoms; oral<br>intervention indicated (e.g.,<br>antibiotic, antifungal, or<br>antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder chara | cterized by an infectious process invo | lving the trachea. | | | |
| Delinition / Globi del Glaid | | | | | |

| | | Infections and infestati | ons | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Upper respiratory infection | - | Moderate symptoms; oral | IV antibiotic, antifungal, or | Life-threatening | Death |
| | | intervention indicated (e.g., | antiviral intervention | consequences; urgent | |
| | | antibiotic, antifungal, or | indicated; invasive | intervention indicated | |
| | | antiviral) | intervention indicated | | |
| Definition: A disorder character | rized by an infectious process involv | ing the upper respiratory tract (nos | e, paranasal sinuses, pharynx, laryn | x, or trachea). | |
| Navigational Note: - | | | | | |
| Urethral infection | = | Localized; oral intervention | IV antibiotic, antifungal, or | Life-threatening | Death |
| | | indicated (e.g., antibiotic, | antiviral intervention | consequences; urgent | |
| | | antifungal, or antiviral) | indicated; invasive | intervention indicated | |
| | | 1 " | intervention indicated | | |
| Definition: A disorder character | rized by an infectious process involv | ving the urethra. | • | • | • |
| Navigational Note: - | | | | | |
| Urinary tract infection | - | Localized; oral intervention | IV antibiotic, antifungal, or | Life-threatening | Death |
| • | | indicated (e.g., antibiotic, | antiviral intervention | consequences; urgent | |
| | | antifungal, or antiviral) | indicated: invasive | intervention indicated | |
| | | | intervention indicated | | |
| Definition: A disorder character | rized by an infectious process involv | ving the urinary tract most common | bly the bladder and the urethra | • | • |
| Navigational Note: - | inzed by an inneed day process in voice | ing are annually dues, most common | ny die bradder and die dreding. | | |
| Uterine infection | - | Moderate symptoms: oral | IV antibiotic, antifungal, or | Life-threatening | Death |
| | | intervention indicated (e.g., | antiviral intervention | consequences; urgent | |
| | | antibiotic, antifungal, or | indicated: invasive | intervention indicated | |
| | | antiviral) | intervention indicated | mico rondon maradesa | |
| Definition: A disorder character | rized by an infectious process involv | | | ial tissues | ' |
| Navigational Note: - | inzed by diffineed bd a process involv | ing the chaomed and remay exem | a to the myometriam and parametr | iai ussacs. | |
| Vaginal infection | Localized, local intervention | Oral intervention indicated | IV antibiotic, antifungal, or | Life-threatening | Death |
| 9 | indicated | (e.g., antibiotic, antifungal, or | antiviral intervention | consequences; urgent | |
| | The decou | antiviral) | indicated: invasive | intervention indicated | |
| | | andway | intervention indicated | intervention indicated | |
| Definition: A disorder character | rized by an infectious process involv | ving the vagina. | The state of the s | 1 | i |
| Navigational Note: - | | | | | |
| Viremia | - | Moderate symptoms; medical | Severe or medically significant | - | - |
| | | intervention indicated | but not immediately life- | | |
| | | | threatening; hospitalization or | I | |
| | | 1 | prolongation of existing | I | |
| | | 1 | hospitalization indicated | I | |
| Definition Adiamatan | 1 | <br> - | 1 nospitalization illustrated | ı | I |
| | rized by the presence of a virus in th | ne plood stream. | | | |
| Navigational Note: - | | | | | |

# **Cerus Corporation**

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Infections and infestati | ons | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Vulval infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process involv | ing the vulva. | | | |
| Navigational Note: - | | | | | |
| Wound infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention<br>indicated; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process involv | ing the wound. | | | |
| Navigational Note: - | | _ | | | |
| Infections and infestations -<br>Other, specify | Asymptomatic or mild<br>symptoms; dinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: - | • | - | • | - | • |
| Navigational Note: - | | | | | |

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade ! |
|---|---|---|---|---|---|
| Ankle fracture | Mild; non-operative | Limiting instrumental ADL; | Limiting self care ADL; elective | - | - |
| | intervention indicated | outpatient operative | operative intervention | | |
| | | intervention indicated | indicated requiring | | |
| | | | hospitalization | | |
| <b>Definition:</b> A finding of damag | e to the ankle ioint characterized by | a break in the continuity of the ar | kle bone. Symptoms include marked | discomfort, swelling and difficulty | moving the |
| affected leg and foot. | , | | | | |
| Navigational Note: - | | | | | |
| Aortic injury | - | Operative intervention not | Severe symptoms; limiting self | Life-threatening | Death |
| | | indicated | care ADL; repair or revision | consequences; evidence of | |
| | | | indicated | end organ damage; urgent | |
| | | | | operative intervention | |
| | | 1 | | indicated | |
| Definition: A finding of damag | e to the aorta. | • | 1 | | ' |
| Navigational Note: - | | | | | |
| Arterial injury | Asymptomatic diagnostic | Symptomatic; repair or | Severe symptoms; limiting self | Life-threatening | Death |
| | finding; intervention not | revision not indicated | care ADL; repair or revision | consequences; evidence of | |
| | indicated | | indicated | end organ damage; urgent | |
| | | | | operative intervention | |
| | | 1 | | indicated | |
| Definition: A finding of damag | e to an arterv. | • | ' | • | , |
| Navigational Note: - | | | | | |
| Biliary anastomotic leak | Asymptomatic diagnostic | Symptomatic; medical | Severe symptoms; invasive | Life-threatening | Death |
| | finding; intervention not | intervention indicated | intervention indicated | consequences; urgent | |
| | indicated | | | operative intervention | |
| | | 1 | | indicated | |
| <b>Definition:</b> A finding of leakage | e of bile due to breakdown of a bilia | ry anastomosis (surgical connectio | n of two separate anatomic structure | s). | |
| Navigational Note: - | | · - | | | |
| Bladder anastomotic leak | Asymptomatic diagnostic | Symptomatic; medical | Severe symptoms; invasive | Life-threatening | Death |
| | finding; intervention not | intervention indicated | intervention indicated | consequences; urgent | |
| | indicated | | | operative intervention | |
| | | 1 | | indicated | |
| <b>Definition:</b> A finding of leakage | e of urine due to breakdown of a bla | dder anastomosis (surgical connec | ction of two separate anatomic struct | ·<br>ures). | • |
| Navigational Note: - | | | • | , | |
| Bruising | Localized or in a dependent | Generalized | - | - | - |
| | area | 1 | | l | |

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Burn | Minimal symptoms; | Medical intervention: minimal | Moderate to major | Life-threatening | Death |
| Barri | intervention not indicated | debridement indicated | debridement or | consequences | Doggi |
| | The verteer he male acc | debriderierie iridicated | reconstruction indicated | consequences | |
| Definition: A finding of impaired | I<br>d integrity to the anatomic site of an | l<br>adverse thermal reaction. Burns o | | <br> cals direct heat electricity flames: | I<br>and |
| | e depends on the length and intensit | | | cais, all cee ricae, creedicity, harries | ana |
| Navigational Note: - | s depends on the rengal and intensit | y or exposure and arms arms provis | ion or a cauncile | | |
| Dermatitis radiation | Total and the same and the | Non-demonstration of the contract of the contr | NATIONAL ASSESSMENT OF THE PROPERTY OF THE PRO | 116- 4 | Death |
| Jermatius radiation | Faint erythema or dry | Moderate to brisk erythema; | Moist desquamation in areas<br>other than skin folds and | Life-threatening | Death |
| | desquamation | patchy moist desquamation, | | consequences; skin necrosis<br>or ulceration of full thickness | |
| | | mostly confined to skin folds | creases; bleeding induced by | | |
| | | and creases; moderate edema | minor trauma or abrasion | dermis; spontaneous bleeding | |
| | | | | from involved site; skin graft | |
| | | I | | indicated | |
| • | us inflammatory reaction occurring | | lly effective levels of ionizing radiat | ion. | |
| Navigational Note: Synonym: R | adiation induced skin toxicities (CTC | AE v3.0) | | | |
| Esophageal anastomotic leak | Asymptomatic diagnostic | Symptomatic; medical | Severe symptoms; invasive | Life-threatening | Death |
| | finding; intervention not | intervention indicated | intervention indicated | consequences; urgent | |
| | indicated | | | operative intervention | |
| | | | | indicated | |
| Definition: A finding of leakage | due to breakdown of an esophageal | anastomosis (surgical connection | of two separate anatomic structure | es). | |
| Navigational Note: - | | · - | | | |
| Fall | Minor with no resultant | Symptomatic; noninvasive | Hospitalization indicated; | - | - |
| | injuries; intervention not | intervention indicated | invasive intervention | | |
| | indicated | | indicated | | |
| <b>Definition:</b> A finding of sudden | movement downward, usually resul | ting in injury | | • | 1 |
| Navigational Note: - | ,, | | | | |
| Fallopian tube anastomotic | Asymptomatic; clinical or | Symptomatic: medical | Severe symptoms; invasive | Life-threatening | Death |
| leak | diagnostic observations only; | intervention indicated | intervention indicated | consequences; urgent | 20001 |
| icun. | intervention not indicated | incorvendor indicated | microcidon marcacca | operative intervention | |
| | indervendon not indicated | l | | indicated | 1 |

| | | Injury, poisoning and procedura | l complications | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Fallopian tube perforation | - | Invasive intervention not indicated | Invasive intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated (e.g., organ<br>resection) | Death |
| <b>Definition:</b> A disorder character<br><b>Navigational Note:</b> - | ized by a rupture of the fallopian tu | be wall. | | | |
| Fracture | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic but non-<br>displaced; immobilization<br>indicated | Severe symptoms; displaced<br>or open wound with bone<br>exposure; limiting self care<br>ADL; operative intervention<br>indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | ic injury to the bone in which the co<br>g this term consider specific fractur | | cedural complications: Ankle fractur | e, Hip fracture, Spinal fracture, o | or <b>W</b> rist |
| Gastric anastomotic leak | Asymptomatic diagnostic finding; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; invasive intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| <b>Definition:</b> A finding of leakage <b>Navigational Note:</b> - | due to breakdown of a gastric anast | comosis (surgical connection of tw | vo separate anatomic structures). | • | , |
| Gastrointestinal anastomotic<br>leak | Asymptomatic diagnostic finding; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; invasive intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| <b>Definition:</b> A finding of leakage <b>Navigational Note:</b> - | due to breakdown of a gastrointesti | nal anastomosis (surgical connec | tion of two separate anatomic struc | ures). | · |
| Gastrointestinal stoma<br>necrosis | - | Superficial necrosis;<br>intervention not indicated | Severe symptoms;<br>hospitalization indicated;<br>elective operative<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder character <b>Navigational Note:</b> - | ized by a necrotic process occurring | in the gastrointestinal tract stom | na. | | ·<br> |

| | | Injury, poisoning and procedural | complications | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Hip fracture | - | Hairline fracture; mild pain;<br>limiting instrumental ADL;<br>non-operative intervention<br>indicated | Severe pain; hospitalization or<br>intervention indicated for pain<br>control (e.g., traction);<br>operative intervention<br>indicated | Life-threatening<br>consequences; symptoms<br>associated with neurovascular<br>compromise | - |
| <b>Definition:</b> A finding of traumat<br><b>Navigational Note:</b> - | ic injury to the hip in which the cor | ntinuity of either the femoral head, f | emoral neck, intertrochanteric or su | ubtrochanteric regions is broken. | |
| Infusion related reaction | Mild transient reaction;<br>infusion interruption not<br>indicated; intervention not<br>indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics, IV fluids); prophylactic medications indicated for <=24 hrs | Prolonged (e.g., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement; hospitalization indicated for clinical sequelae | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder character<br>Navigational Note: - | rized by adverse reaction to the infl | usion of pharmacological or biologic | al substances. | | |
| Injury to carotid artery | - | Repair or revision not indicated | Severe symptoms; limiting self<br>care ADL (e.g., transient<br>cerebral ischemia); repair or<br>revision indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A finding of damage | to the carotid artery. | • | • | • | • |
| Navigational Note: - | | | | | |
| Injury to inferior vena cava | Asymptomatic diagnostic finding; intervention not indicated | Symptomatic; repair or revision not indicated | Severe symptoms; limiting self<br>care ADL; repair or revision<br>indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A finding of damage cava. | to the inferior vena | | | • | |
| Navigational Note: - | T | T | T | Lieu | |
| Injury to jugular vein | - | Repair or revision not indicated | Symptomatic limiting self care<br>ADL; repair or revision<br>indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A finding of damage | to the jugular vein. | - | • | • | • |
| Navigational Note: - | | | | | |

# **Cerus Corporation**

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Injury, poisoning and procedural | complications | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Injury to superior vena cava | Asymptomatic diagnostic finding; intervention not indicated | Symptomatic; repair or revision not indicated | Severe symptoms; limiting self<br>care ADL; repair or revision<br>indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A finding of damage | to the superior vena cava. | | | | |
| Navigational Note: - | | | | | |
| Intestinal stoma leak | Asymptomatic diagnostic finding; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; invasive intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| | of contents from an intestinal stom | a (surgically created opening on the | e surface of the body). | | |
| Navigational Note: - | | | | | |
| Intestinal stoma obstruction | - | Self-limited; intervention not indicated | Severe symptoms; IV fluids,<br>tube feeding, or TPN indicated<br>>=24 hrs; elective operative<br>intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Definition: A disorder characteri | zed by blockage of the normal flow | of the contents of the intestinal st | oma. | • | • |
| Navigational Note: - | | | | | |
| Intestinal stoma site bleeding | Minimal bleeding identified<br>on clinical exam; intervention<br>not indicated | Moderate bleeding; medical<br>intervention indicated | Transfusion indicated;<br>invasive intervention<br>indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder characteri | red by bleeding from the intestinal | stoma. | • | • | • |
| Navigational Note: - | | | | | |
| Intraoperative arterial injury | Primary repair of injured<br>organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A finding of damage | to an artery during a surgical proce | dure. | • | | · |
| Navigational Note: - | | | | | |
| Intraoperative breast injury | Primary repair of injured<br>organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A finding of damage <b>Navigational Note:</b> - | to the breast parenchyma during a | surgical procedure. | • | - | • |

| | | Injury, poisoning and procedura | i complications | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Intraoperative cardiac injury | - | - | Primary repair of injured | Life-threatening | Death |
| | | | organ/structure indicated | consequences; urgent | |
| | | 1 | | intervention indicated | |
| Definition: A finding of damage | e to the heart during a surgical pro- | cedure. | | | |
| Navigational Note: - | | | | | |
| Intraoperative ear injury | Primary repair of injured | Partial resection of injured | Complete resection or | Life-threatening | Death |
| | organ/structure indicated | organ/structure indicated | reconstruction of injured | consequences; urgent | |
| | | | organ/structure indicated; | intervention indicated | |
| | | | limiting self care ADL (e.g., | | |
| | | | impaired hearing; impaired | | |
| | | | balance) | I | |
| | e to the ear during a surgical proce | dure. | | | |
| Navigational Note: - | | | | | |
| Intraoperative endocrine | Primary repair of injured | Partial resection of injured | Complete resection or | Life-threatening | Death |
| injur <b>y</b> | organ/structure indicated | organ/structure indicated | reconstruction of injured | consequences; urgent | |
| | | | organ/structure indicated; | intervention indicated | |
| | | | 122-2 16 ADI | | |
| | 1 | | limiting self care ADL | 1 | |
| <b>Definition:</b> A finding of damage | ।<br>e to the endocrine gland during a s | <b>I</b><br>urgical procedure. | limiting self care AUL | 1 | I |
| <b>Definition:</b> A finding of damage <b>Navigational Note:</b> - | I<br>e to the endocrine gland during a s | urgical procedure. | IIMITING SEIT CARE AUL | I | |
| | e to the endocrine gland during a s Primary repair of injured | urgical procedure. Partial resection of injured | Complete resection or | Life-threatening | Death |
| Navigational Note: - | | • • | , , | Life-threatening consequences; urgent | Death |
| Navigational Note: -<br>Intraoperative gastrointestinal | Primary repair of injured | Partial resection of injured | Complete resection or reconstruction of injured organ/structure indicated; | | Death |
| Navigational Note: -<br>Intraoperative gastrointestinal | Primary repair of injured | Partial resection of injured | Complete resection or reconstruction of injured | consequences; urgent | Death |
| Navigational Note: -<br>Intraoperative gastrointestinal<br>injury | Primary repair of injured | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; | consequences; urgent | Death |
| Navigational Note: - Intraoperative gastrointestinal injury Definition: A finding of damage | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; | consequences; urgent | Death |
| Navigational Note: -<br>Intraoperative gastrointestinal<br>injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; | consequences; urgent | Death Death |
| Navigational Note: - Intraoperative gastrointestinal injury Definition: A finding of damage Navigational Note: - | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; limiting self care ADL | consequences; urgent intervention indicated | |
| Navigational Note: - Intraoperative gastrointestinal injury Definition: A finding of damage Navigational Note: - Intraoperative head and neck | Primary repair of injured organ/structure indicated to the gastrointestinal system du | Partial resection of injured organ/structure indicated ring a surgical procedure. Partial resection of injured | Complete resection or reconstruction of injured organ/structure indicated; limiting self care ADL Complete resection or | consequences urgent intervention indicated | |
| Navigational Note: - Intraoperative gastrointestinal injury Definition: A finding of damage Navigational Note: - Intraoperative head and neck | Primary repair of injured organ/structure indicated to the gastrointestinal system du | Partial resection of injured organ/structure indicated ring a surgical procedure. Partial resection of injured | Complete resection or reconstruction of injured organ/structure indicated; limiting self care ADL Complete resection or reconstruction of injured | consequences; urgent intervention indicated Life-threatening consequences; urgent | |
| Navigational Note: - Intraoperative gastrointestinal injury Definition: A finding of damage Navigational Note: - Intraoperative head and neck injury | Primary repair of injured organ/structure indicated to the gastrointestinal system du | Partial resection of injured organ/structure indicated ring a surgical procedure. Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; limiting self care ADL Complete resection or reconstruction of injured organ/structure indicated; | consequences; urgent intervention indicated Life-threatening consequences; urgent | |
| Navigational Note: - Intraoperative gastrointestinal injury Definition: A finding of damage Navigational Note: - Intraoperative head and neck injury Definition: A finding of damage | Primary repair of injured organ/structure indicated to the gastrointestinal system dustriance organ/structure indicated | Partial resection of injured organ/structure indicated ring a surgical procedure. Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; limiting self care ADL Complete resection or reconstruction of injured organ/structure indicated; | consequences; urgent intervention indicated Life-threatening consequences; urgent | |
| Navigational Note: - Intraoperative gastrointestinal injury Definition: A finding of damage Navigational Note: - Intraoperative head and neck injury | Primary repair of injured organ/structure indicated to the gastrointestinal system dustriance organ/structure indicated | Partial resection of injured organ/structure indicated ring a surgical procedure. Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; limiting self care ADL Complete resection or reconstruction of injured organ/structure indicated; | consequences; urgent intervention indicated Life-threatening consequences; urgent | |
| Navigational Note: - Intraoperative gastrointestinal injury Definition: A finding of damage Navigational Note: - Intraoperative head and neck injury Definition: A finding of damage Navigational Note: - | Primary repair of injured organ/structure indicated to the gastrointestinal system dustriance organ/structure indicated | Partial resection of injured organ/structure indicated ring a surgical procedure. Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; limiting self care ADL Complete resection or reconstruction of injured organ/structure indicated; limiting self care ADL | consequences; urgent intervention indicated Life-threatening consequences; urgent intervention indicated | Death |
| Navigational Note: - Intraoperative gastrointestinal injury Definition: A finding of damage Navigational Note: - Intraoperative head and neck injury Definition: A finding of damage Navigational Note: - | Primary repair of injured organ/structure indicated to the gastrointestinal system dustriance organ/structure indicated | Partial resection of injured organ/structure indicated ring a surgical procedure. Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; limiting self care ADL Complete resection or reconstruction of injured organ/structure indicated; limiting self care ADL Postoperative invasive | consequences; urgent intervention indicated Life-threatening consequences; urgent intervention indicated | Death |
| Navigational Note: - Intraoperative gastrointestinal injury Definition: A finding of damage Navigational Note: - Intraoperative head and neck injury Definition: A finding of damage Navigational Note: - Intraoperative hemorrhage | Primary repair of injured organ/structure indicated e to the gastrointestinal system du Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated ring a surgical procedure. Partial resection of injured organ/structure indicated regical procedure. | Complete resection or reconstruction of injured organ/structure indicated; limiting self care ADL Complete resection or reconstruction of injured organ/structure indicated; limiting self care ADL Postoperative invasive intervention indicated; | consequences; urgent intervention indicated Life-threatening consequences; urgent intervention indicated Life-threatening consequences; urgent intervention indicated | Death |
**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Injury, poisoning and procedura | l complications | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Intraoperative hepatobiliary<br>injury | Primary repair of injured<br>organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A finding of damage<br><b>Navigational Note:</b> - | to the hepatic parenchyma and/or | r biliary tract during a surgical proc | edure. | | |
| Intraoperative<br>musculoskeletal injury | Primary repair of injured organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | to the musculoskeletal system dur | ing a surgical procedure. | | | |
| Navigational Note: - | | | T | Tage 1 | |
| Intraoperative neurological<br>injury | Primary repair of injured<br>organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A finding of damage | to the nervous system during a su | rgical procedure. | | • | |
| Navigational Note: - | | | | | |
| Intraoperative ocular injury | Primary repair of injured<br>organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | to the eye during a surgical proced | dure. | | | · |
| Navigational Note: -<br>Intraoperative renal injury | Primary repair of injured organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | to the kidney during a surgical pro | cedure. | • | • | • |
| Navigational Note: -<br>Intraoperative reproductive<br>tract injury | Primary repair of injured organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A finding of damage<br>Navigational Note: - | to the reproductive organs during | a surgical procedure. | • | | • |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| Injury, poisoning and procedural complications | | | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Intraoperative respiratory<br>injury | Primary repair of injured<br>organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | to the respiratory system during a | surgical procedure. | | | · |
| Navigational Note: | 1 | | 1 | Link | |
| Intraoperative splenic injury | - | Primary repair of injured<br>organ/structure indicated | Resection or reconstruction of<br>injured organ/structure<br>indicated; limiting self care<br>ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | to the spleen during a surgical pro | cedure. | | | |
| Navigational Note: - | T = | T = | T | Liza | |
| Intraoperative urinary injury | Primary repair of injured<br>organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A finding of damage | to the urinary system during a sur | gical procedure. | | • | • |
| Navigational Note: - | | | | | |
| Intraoperative venous injur <b>y</b> | Primary repair of injured<br>organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | to a vein during a surgical procedu | ire. | | | |
| Navigational Note: - | | | | | |
| Kidney anastomotic leak | Asymptomatic diagnostic finding; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; invasive intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| <b>Definition:</b> A finding of leakage | of urine due to breakdown of a kic | lney anastomosis (surgical connect | ion of two separate anatomic structu | res). | |
| Navigational Note: - | | | | | |
| Large intestinal anastomotic<br>leak | Asymptomatic diagnostic finding; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; invasive intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| | due to breakdown of an anastomo | sis (surgical connection of two sep | arate anatomic structures) in the larg | ge intestine. | • |
| Navigational Note: - | | | | | |

| CTCAE Term | | Injury, poisoning and procedural of | • | | T |
|---|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Pancreatic anastomotic leak | Asymptomatic diagnostic | Symptomatic; medical | Severe symptoms; invasive | Life-threatening | Death |
| | finding; intervention not | intervention indicated | intervention indicated | consequences; urgent | |
| | indicated | | | operative intervention | |
| | 1 | I | | indicated | |
| | due to breakdown of a pancreatic a | nastomosis (surgical connection of t | two separate anatomic structures). | | |
| Navigational Note: - | | | | | |
| Pharyngeal anastomotic leak | Asymptomatic diagnostic | Symptomatic; medical | Severe symptoms; invasive | Life-threatening | Death |
| | finding; intervention not | intervention indicated | intervention indicated | consequences; urgent | |
| | indicated | | | operative intervention | |
| | 1 | 1 | | indicated | |
| Definition: A finding of leakage | due to breakdown of a pharyngeal a | anastomosis (surgical connection of | two separate anatomic structures) | | |
| Navigational Note: - | | | | | |
| Postoperative hemorrhage | Mild symptoms; intervention | Moderate bleeding requiring | Transfusion indicated of >=2 | Life-threatening | Death |
| | not indicated | transfusion < 2 units (10 cc/kg | units (10 cc/kg for pediatrics) | consequences; urgent | |
| | | for pediatrics) of pRBCs | pRBCs; invasive intervention | intervention indicated | |
| | | | indicated; hospitalization | | |
| Definition: A disorder character | ized by bleeding occurring after a su | urgical procedure. | | • | |
| Navigational Note: - | , | | | | |
| Postoperative thoracic | - | Extubated within 24 - 72 hrs | Extubated > 72 hrs | Life-threatening airway | Death |
| procedure complication | | postoperatively | postoperatively, but before | compromise; urgent | |
| ' | | l''' | tracheostomy indicated | intervention indicated (e.g., | |
| | | | • | tracheotomy or intubation) | |
| Definition: A finding of a previous | usly undocumented problem that o | cours after a thoracic procedure. | | | , |
| | , a | | | | |
| Navigational Note: - | | | | | |
| | Asymptomatic: reducible | Recurrent after manual | Severe symptoms: elective | Life-threatening | Death |
| | Asymptomatic; reducible | | Severe symptoms; elective operative intervention | Life-threatening | Death |
| | Asymptomatic; reducible | reduction; local irritation or | operative intervention | consequences; urgent | Death |
| | Asymptomatic; reducible | reduction; local irritation or<br>stool leakage; difficulty to fit | operative intervention<br>indicated; limiting self care | consequences; urgent operative intervention | Death |
| | Asymptomatic; reducible | reduction; local irritation or<br>stool leakage; difficulty to fit<br>appliance; limiting | operative intervention | consequences; urgent | Death |
| Prolapse of intestinal stoma | | reduction; local irritation or<br>stool leakage; difficulty to fit<br>appliance; limiting<br>instrumental ADL | operative intervention<br>indicated; limiting self care<br>ADL | consequences; urgent operative intervention indicated | Death |
| Prolapse of intestinal stoma Definition: A finding of protrusic | | reduction; local irritation or<br>stool leakage; difficulty to fit<br>appliance; limiting | operative intervention<br>indicated; limiting self care<br>ADL | consequences; urgent operative intervention indicated | Death |
| Prolapse of intestinal stoma Definition: A finding of protrusion Navigational Note: - | on of the intestinal stoma (surgically | reduction; local irritation or<br>stool leakage; difficulty to fit<br>appliance; limiting<br>instrumental ADL<br>y created opening on the surface of | operative intervention<br>indicated; limiting self care<br>ADL<br>the body) above the abdominal su | consequences; urgent<br>operative intervention<br>indicated<br>face. | Death |
| Prolapse of intestinal stoma Definition: A finding of protrusion Navigational Note: - | on of the intestinal stoma (surgically | reduction; local irritation or<br>stool leakage; difficulty to fit<br>appliance; limiting<br>instrumental ADL<br>created opening on the surface of<br>Local care or maintenance; | operative intervention indicated; limiting self care ADL the body) above the abdominal sure Dysfunctional stoma; elective | consequences; urgent operative intervention indicated face. | |
| Navigational Note: - Prolapse of intestinal stoma Definition: A finding of protrusic Navigational Note: - Prolapse of urostomy | on of the intestinal stoma (surgically<br>Asymptomatic; clinical or<br>diagnostic observations only; | reduction; local irritation or<br>stool leakage; difficulty to fit<br>appliance; limiting<br>instrumental ADL<br>y created opening on the surface of | operative intervention indicated; limiting self care ADL the body) above the abdominal sur Dysfunctional stoma; elective operative intervention or | consequences; urgent operative intervention indicated face. Life-threatening consequences; urgent | |
| Prolapse of intestinal stoma Definition: A finding of protrusion Navigational Note: - | on of the intestinal stoma (surgically | reduction; local irritation or<br>stool leakage; difficulty to fit<br>appliance; limiting<br>instrumental ADL<br>created opening on the surface of<br>Local care or maintenance; | operative intervention indicated; limiting self care ADL the body) above the abdominal sur Dysfunctional stoma; elective operative intervention or major stomal revision | consequences; urgent operative intervention indicated face. | |
| Prolapse of intestinal stoma Definition: A finding of protrusion Navigational Note: - | on of the intestinal stoma (surgically<br>Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | reduction; local irritation or<br>stool leakage; difficulty to fit<br>appliance; limiting<br>instrumental ADL<br>created opening on the surface of<br>Local care or maintenance; | operative intervention indicated; limiting self care ADL the body) above the abdominal sur Dysfunctional stoma; elective operative intervention or | consequences; urgent operative intervention indicated face. Life-threatening consequences; urgent | |

| | | Injury, poisoning and procedural | complications | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Radiation recall reaction<br>(dermatologic) | Faint erythema or dry<br>desquamation | Moderate to brisk erythema;<br>patchy moist desquamation,<br>mostly confined to skin folds<br>and creases; moderate edema | Moist desquamation in areas<br>other than skin folds and<br>creases; bleeding induced by<br>minor trauma or abrasion | Life-threatening<br>consequences; skin necrosis<br>or ulceration of full thickness<br>dermis; spontaneous bleeding<br>from involved site; skin graft<br>indicated | Death |
| | kin inflammatory reaction caused by<br>adiated skin and the symptoms disa | | | owing radiotherapy. The inflammato | ry reaction |
| Navigational Note: - | | | | | |
| Rectal anastomotic leak | Asymptomatic diagnostic finding; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; invasive intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Definition: A finding of leakage | due to breakdown of a rectal anasto | omosis (surgical connection of two | separate anatomic structures). | | |
| Navigational Note: - | | | | | |
| Seroma | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; simple<br>aspiration indicated | Symptomatic, elective invasive intervention indicated | - | - |
| <b>Definition:</b> A finding of tumor- | ike collection of serum in the tissues | | • | • | • |
| Navigational Note: - | | | | | |
| Small intestinal anastomotic<br>leak | Asymptomatic diagnostic finding; intervention not indicated | Symptomatic; medical<br>intervention indicated | Severe symptoms; invasive intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| <b>Definition:</b> A finding of leakage | due to breakdown of an anastomos | is (surgical connection of two separ | ate anatomic structures) in the sm | all bowel. | |
| Navigational Note: - | | · | | | |
| Spermatic cord anastomotic<br>leak | Asymptomatic diagnostic finding; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; invasive intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Definition: A finding of leakage | due to breakdown of a spermatic co | ord anastomosis (surgical connectio | n of two separate anatomic struct | ures). | |
| Navigational Note: - | | | | | |

| | | Injury, poisoning and procedural | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Spinal fracture | Mild back pain; | Moderate back pain; | Severe back pain; | Life-threatening | Death |
| | nonprescription analgesics | prescription analgesics | hospitalization or intervention | consequences; symptoms | |
| | indicated | indicated; limiting | indicated for pain control | associated with neurovascular | |
| | | instrumental ADL | (e.g., vertebroplasty); limiting | compromise | |
| | | 1 | self care ADL; disability | 1 | |
| <b>Definition:</b> A finding of trauma | tic injury to the spine in which the co | ontinuity of a vertebral bone is bro | ken. | | |
| Navigational Note: - | | | | | |
| Stenosis of gastrointestinal | - | Symptomatic; IV fluids | Severely altered GI function; | Life-threatening | Death |
| stoma | | indicated <24 hrs; manual | tube feeding, TPN or | consequences; urgent | |
| | | dilation at bedside | hospitalization indicated; | operative intervention | |
| | | | elective operative | indicated | |
| | | 1 | intervention indicated | | |
| Definition: A finding of narrow | ring of the gastrointestinal stoma (su | gically created opening on the sur | face of the body). | | |
| Navigational Note: - | | | | | |
| Stomal ulcer | Asymptomatic; clinical or | Symptomatic; medical | Severe symptoms; elective | - | - |
| | diagnostic observations only; | intervention indicated | operative intervention | | |
| | intervention not indicated | | indicated | | |
| Definition: A disorder characte | rized by a circumscribed, erosive les | ion on the jejunal mucosal surface | close to the anastomosis site followi | ing a gastroenterostom y procedure | |
| Navigational Note: - | - | | | | |
| Tracheal hemorrhage | Mild symptoms; intervention | Moderate symptoms; | Transfusion indicated; | Life-threatening | Death |
| | not indicated | intervention indicated | invasive intervention | consequences; urgent | |
| | | | indicated; hospitalization | intervention indicated | |
| Definition: A disorder characte | rized by bleeding from the trachea. | | | | |
| Navigational Note: - | | | | | |
| Tracheal obstruction | Partial asymptomatic | Symptomatic (e.g., noisy | Stridor or respiratory distress | Life-threatening airway | Death |
| | obstruction on examination | airway breathing), no | limiting self care ADL; invasive | compromise; urgent | |
| | (e.g., visual, radiologic or | respiratory distress; medical | intervention indicated (e.g., | intervention indicated (e.g., | |
| | endoscopic) | intervention indicated (e.g., | stent, laser) | tracheotomy or intubation) | |
| | | steroids); limiting | | | |
| | | instrumental ADL | | | |
| Definition: A disorder characte | erized by blockage of the lumen of th | e trachea. | | - | • |
| Navigational Note: - | | | | | |
| Tracheostomy site bleeding | Minimal bleeding identified | Moderate bleeding; medical | Transfusion indicated; | Life-threatening | Death |
| | on clinical exam; intervention | intervention indicated | invasive intervention | consequences; urgent | |
| | not indicated | | indicated | intervention indicated | |
| <b>Definition:</b> A disorder characte | rized by bleeding from the tracheos | tomy site. | • | • | • |
| Navigational Note: - | , | | | | |
| HanParioliai More: - | | | | | |

| | | Injury, poisoning and procedural | complications | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Ureterica nastomotic leak | Asymptomatic diagnostic finding; intervention not indicated | Symptomatic; medical<br>intervention indicated | Severe symptoms; invasive intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| <b>Definition:</b> A finding of leakage of <b>Navigational Note:</b> - | due to breakdown of a ureteral ana | stomosis (surgical connection of tw | o separate anatomic structures). | | |
| Urethral anastomotic leak | Asymptomatic diagnostic finding; intervention not indicated | Symptomatic; medical<br>intervention indicated | Severe symptoms; invasive intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| <b>Definition:</b> A finding of leakage of <b>Navigational Note:</b> - | due to breakdown of a urethral ana | stomosis (surgical connection of tv | vo separate anatomic structures). | | |
| Urostomy leak | Asymptomatic diagnostic finding; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; invasive intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| <b>Definition:</b> A finding of leakage of <b>Navigational Note:</b> - | of contents from a urostomy. | • | • | | • |
| Urostomy obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; dilation or<br>endoscopic repair or stent<br>placement indicated | Altered organ function (e.g., sepsis or hydronephrosis, or renal dysfunction); elective operative intervention indicated | Life-threatening<br>consequences; organ failure;<br>urgent operative intervention<br>indicated | Death |
| | ized by blockage of the urostomy. | • | • | • | • |
| Navigational Note: -<br>Urostomy site bleeding | Minimal bleeding identified<br>on clinical exam; intervention<br>not indicated | Moderate bleeding; medical intervention indicated | Transfusion indicated;<br>invasive intervention<br>indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder characteri<br>Navigational Note: - | zed by bleeding from the urostomy | site. | | | |
| Urostomy stenosis | | Symptomatic but no<br>hydronephrosis, sepsis, or<br>renal dysfunction; dilation or<br>endoscopic repair or stent<br>placement indicated | Symptomatic (e.g.,<br>hydronephrosis, or renal<br>dysfunction); elective<br>operative intervention<br>indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| <b>Definition:</b> A finding of narrowin<br><b>Navigational Note:</b> - | ng of the opening of a urostom <b>y.</b> | | | | |

CTCAE v5.0 – November 27, 2017 Back to TOC


**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Injury, poisoning and procedural o | complications | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Uterine anastomotic leak | Asymptomatic diagnostic finding; intervention not indicated | Symptomatic; medical<br>intervention indicated | Severe symptoms; invasive intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| <b>Definition:</b> A finding of leakage of <b>Navigational Note:</b> - | due to breakdown of a uterine anas | tomosis (surgical connection of two | separate anatomic structures). | | |
| Uterine perforation | - | Invasive intervention not indicated | Invasive intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder characteri<br><b>Navigational Note:</b> - | zed by a rupture in the uterine wall | | | | |
| Vaccination complication | Mild pain; erythema 2.5-5cm;<br>induration/swelling 2.5-5cm;<br>does not interfere with<br>activity | Moderate pain; Erythema 5.1-<br>10 cm; Induration/swelling<br>5.1-10 cm; lipodystrophy;<br>limiting instrumental ADL | Severe pain; Erythema > 10<br>cm; Induration/swelling > 10<br>cm; necrosis; limiting self care<br>ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | - |
| Definition: A disorder that occur | s after the injection of a substance | with antigenic properties, administ | ered to activate the immune syster | n. | • |
| Navigational Note: For systemic | vaccination complications, conside | r Immune system disorders: Allergi | creaction or Anaphylaxis. | | |
| Vaginal anastomotic leak | Asymptomatic diagnostic finding; intervention not indicated | Symptomatic; medical<br>intervention indicated | Severe symptoms; invasive intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Definition: A finding of leakage of | ue to breakdown of a vaginal anas | tomosis (surgical connection of two | separate anatomic structures). | • | • |
| Navigational Note: - | | | | | |
| Vas deferens anastomotic leak | Asymptomatic diagnostic finding; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| <b>Definition:</b> A finding of leakage of <b>Navigational Note:</b> - | due to breakdown of a vas deferens | anastomosis (surgical connection c | of two separate anatomic structure | s). | • |
| Vascular access complication | TPA administration into line<br>with no intent for systemic<br>therapy indicated | Device dislodgement,<br>blockage, leak, or malposition;<br>device replacement indicated | Pulmonary embolism, deep<br>vein or cardiac thrombosis;<br>intervention indicated (e.g.,<br>anticoagulation, lysis, filter,<br>invasive procedure) | Life-threatening<br>consequences with<br>hemodynamic or neurologic<br>instability | Death |
| • • | Isl <b>y</b> undocumented problem related | d to the vascular access site. | | | |
| Navigational Note: - | | | | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Injury, poisoning and procedural | complications | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Venous injury | Asymptomatic diagnostic finding; intervention not indicated | Symptomatic (e.g.,<br>claudication); repair or<br>revision not indicated | Severe symptoms; limiting self<br>care ADL; repair or revision<br>indicated | Life-threatening<br>consequences; evidence of<br>end organ damage; urgent<br>operative intervention<br>indicated | Death |
| <b>Definition:</b> A finding of damage: <b>Navigational Note:</b> - | to a vein. | | | | |
| Wound complication | Observation only; topical intervention indicated | Bedside local care indicated | Operative intervention indicated | Life-threatening consequences | Death |
| <b>Definition:</b> A finding of development | nent of a new problem at the site o | f an existing wound. | | | • |
| Navigational Note: Prior to using | g this term consider Injur <mark>y,</mark> poisonin | ng and procedural complications: W | found dehiscence or Infections and | infestations: Wound infection | |
| Wound dehiscence | Incisional separation,<br>intervention not indicated | Incisional separation, local care (e.g., suturing) or medical intervention indicated (e.g., analgesic) | Fascial disruption or<br>dehiscence without<br>evisceration; revision by<br>operative intervention<br>indicated | Life-threatening consequences; symptomatic hernia with evidence of strangulation; fascial disruption with evisceration; major reconstruction flap, grafting, resection, or amputation indicated | Death |
| <b>Definition:</b> A finding of separation | on of the approximated margins of a | a surgical wound. | | | |
| Navigational Note: Also conside | r Infections and infestations: Woun | | | | |
| Wrist fracture | Mild; non-operative intervention indicated | Limiting instrumental ADL;<br>outpatient operative<br>intervention indicated | Limiting self care ADL; elective<br>operative intervention<br>indicated requiring<br>hospitalization | - | - |
| <b>Definition:</b> A finding of traumation | c injury to the wrist joint in which th | ne continuity of a wrist bone is brok | cen. | | |
| Navigational Note: - | | | | | |
| Injury, poisoning and procedural complications - Other, specify | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: - | | | | | |
| Navigational Note: - | | | | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Investigations | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Activated partial<br>thromboplastin time<br>prolonged | >ULN - 1.5 x ULN | >1.5 - 2.5 x ULN | >2.5 x ULN; bleeding | - | - |
| | I<br>shoratory test results in which the n | I<br>ertiel thrombonlestin time is four | Indito be greater than the control value | Le As a possible indicator of coagu | Ionathy a |
| | in time (PTT) may occur in a variety | | | ac. As a possible maleator of coaga | ropadiy, a |
| Navigational Note: - | and the first state of the state of | | mary and order to a sautional | | |
| Alanine aminotransferase | >ULN - 3.0 x ULN if baseline | >3.0 - 5.0 x ULN if baseline | >5.0 - 20.0 x ULN if baseline | >20.0 x ULN if baseline was | - |
| increased | was normal; 1.5 - 3.0 x | was normal; >3.0 - 5.0 x | was normal; >5.0 - 20.0 x | normal; >20.0 x baseline if | |
| | baseline if baseline was | baseline if baseline was | baseline if baseline was | baseline was abnormal | |
| | abnormal | abnormal | abnormal | 1 | |
| Definition: A finding based on la | aboratory test results that indicate a | n increase in the level of alanine | aminotransferase (ALT or SGPT) in th | ne blood specimen. | • |
| Navigational Note: Also conside | er Hepatobiliar <b>y</b> disorders: Hepatic f | ailure | | | |
| Alkaline phosphatase | >ULN - 2.5 x ULN if baseline | >2.5 - 5.0 x ULN if baseline | >5.0 - 20.0 x ULN if baseline | >20.0 x ULN if baseline was | - |
| ncreased | was normal; 2.0 - 2.5 x | was normal; >2.5 - 5.0 x | was normal; >5.0 - 20.0 x | normal; >20.0 x baseline if | |
| | baseline if baseline was | baseline if baseline was | baseline if baseline was | baseline was abnormal | |
| | abnormal | abnormal | abnormal | 1 | |
| Definition: A finding based on la | aboratory test results that indicate a | an increase in the level of alkaline | phosphatase in a blood specimen. | • | • |
| Navigational Note: - | | | | | |
| Aspartate aminotransferase | >ULN - 3.0 x ULN if baseline | >3.0 - 5.0 x ULN if baseline | >5.0 - 20.0 x ULN if baseline | >20.0 x ULN if baseline was | - |
| increased | was normal; 1.5 - 3.0 x | was normal; >3.0 - 5.0 x | was normal; >5.0 - 20.0 x | normal; >20.0 x baseline if | |
| | baseline if baseline was | baseline if baseline was | baseline if baseline was | baseline was abnormal | |
| | abnormal | abnormal | abnormal | 1 | |
| Definition: A finding based on la | aboratory test results that indicate a | an increase in the level of asparta | e aminotransferase (AST or SGOT) in | n a blood specimen. | |
| Navigational Note: Also conside | er Hepatobiliary disorders: Hepatic f | ailure | | | |
| Blood antidiuretic hormone | Asymptomatic; clinical or | Symptomatic; medical | Hospitalization indicated | - | - |
| abnormal | diagnostic observations only; | intervention indicated | | 1 | |
| | intervention not indicated | | | 1 | |
| <b>Definition:</b> A finding based on la | aboratory test results that indicate a | bnormal levels of antidiuretic ho | mone in the blood specimen. | • | |
| Navigational Note: - | | | | | |
| Blood bicarbonate decreased | <lln and="" initiated<="" intervention="" no="" p=""></lln> | - | - | - | - |
| Definition: A finding based on la | aboratory test results that indicate a | decrease in levels of bicarbonate | in a venous blood specimen. | - | • |
| Navigational Note: Also conside | er Metabolism and nutrition disorde | re: Acidaeie ar Alkalaeie | ' | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Investigations | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Blood bilirubin increased | >ULN - 1.5 x ULN if baseline<br>was normal; > 1.0 - 1.5 x<br>baseline if baseline was<br>abnormal | >1.5 - 3.0 x ULN if baseline<br>was normal; >1.5 - 3.0 x<br>baseline if baseline was<br>abnormal | >3.0 - 10.0 x ULN if baseline<br>was normal; >3.0 - 10.0 x<br>baseline if baseline was<br>abnormal | >10.0 x ULN if baseline was<br>normal; >10.0 x baseline if<br>baseline was abnormal | - |
| Definition: A finding based on la | boratory test results that indicate a | n abnormall <b>y</b> high level of bilirubin | in the blood. Excess bilirubin is ass | ociated with jaundice. | |
| Navigational Note: Also conside | r Hepatobiliary disorders: Hepatic f | ailure | | | |
| Blood corticotrophin<br>decreased | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; medical<br>intervention indicated | Hospitalization indicated | - | = |
| Definition: A finding based on la | boratory test results that indicate a | n decrease in levels of corticotroph | in in a blood specimen. | | • |
| Navigational Note: - | | | | | |
| Blood gonadotrophin<br>abnormal | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; medical<br>intervention indicated;<br>limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A finding based on la | boratory test results that indicate a | bnormal levels of gonadotrophin h | ormone in a blood specimen. | • | · |
| Navigational Note: - | | | | | |
| Blood lactate dehydrogenase<br>increased | >ULN | - | - | - | - |
| Definition: A finding based on la | boratory test results that indicate in | ncreased levels of lactate dehydrog | enase in the blood specimen. | | |
| Navigational Note: - | | | | | |
| Blood prolactin abnormal | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting<br>instrumental ADL | - | - | - |
| Definition: A finding based on la | boratory test results that indicate a | -<br>bnormal levels of prolactin hormor | e in a blood specimen. | • | · |
| Navigational Note: - | | | | | |
| Carbon monoxide diffusing capacity decreased | 3 - 5 units below LLN; for<br>follow-up, a decrease of 3 - 5<br>units (ml/min/mm Hg) below<br>the baseline value;<br>asymptomatic and<br>intervention not indicated | 6 - 8 units below LLN; for follow-up, an asymptomatic decrease of >5 - 8 units (ml/min/mm Hg) below the baseline value; symptomatic and intervention not indicated | Asymptomatic decrease of >8 units drop; >5 units drop along with the presence of pulmonary symptoms (e.g., >Grade 2 hypoxia or >Grade 2 dyspnea); intervention indicated | | - |
| - | ng function test results that indicat | | | | |
| Navigational Note: Also conside | r Respiratory, thoracic and mediast | inal disorders: Respiratory failure o | r Dyspnea | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Investigations | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Cardiac troponin I increased | Levels above the upper limit | - | Levels consistent with | - | - |
| | of normal and below the level | | myocardial infarction as | | |
| | of myocardial infarction as | | defined by the manufacturer | | |
| | defined by the manufacturer | l | | 1 | |
| | boratory test results that indicate ir | | | | |
| | r Cardiac disorders: Heart failure or | Cardiac disorders: Myocardial infa | rction. Report Cardiac disorders: H | eart failure or Cardiac disorders: M | yocardial |
| infarction if same grade event. | | | | | |
| Cardiac troponin Tincreased | Levels above the upper limit | - | Levels consistent with | - | - |
| | of normal and below the level | | myocardial infarction as | | |
| | of myocardial infarction as | | defined by the manufacturer | | |
| | defined by the manufacturer | l | | 1 | |
| Definition: A finding based on la | boratory test results that indicate ir | ncreased levels of cardiac troponin | T in a biological specimen. | | |
| Navigational Note: Also conside | r Cardiac disorders: Heart failure or | Cardiac disorders: Myocardial infa | rction. Report Cardiac disorders: H | eart failure or Cardiac disorders: M | yocardial |
| infarction if same grade event. | | | | | |
| CD4 lymphocytes decreased | <lln -="" 0.5="" 500="" <lln="" mm3;="" td="" x<=""><td>&lt;500 - 200/mm3; &lt;0.5 - 0.2 x</td><td>&lt;200 - 50/mm3; &lt;0.2 x 0.05 -</td><td>&lt;50/mm3; &lt;0.05 x 10e9 /L</td><td>-</td></lln> | <500 - 200/mm3; <0.5 - 0.2 x | <200 - 50/mm3; <0.2 x 0.05 - | <50/mm3; <0.05 x 10e9 /L | - |
| | 10e9/L | 10e9 /L | 10e9 /L | 1 | |
| Definition: A finding based on la | boratory test results that indicate a | n decrease in levels of CD4 lympho | cytes in a blood specimen. | | |
| Navigational Note: - | | | | | |
| Cholesterol high | >ULN - 300 mg/dL; >ULN - | >300 - 400 mg/dL; >7.75 - | >400 - 500 mg/dL; >10.34 - | >500 mg/dL; >12.92 mmol/L | - |
| | 7.75 mmol/L | 10.34 mm ol/L | 12.92 mmol/L | 1 | |
| Definition: A finding based on la | boratory test results that indicate h | igher than normal levels of cholest | erol in a blood specimen. | • | • |
| Navigational Note: - | • | | | | |
| CPK increased | >ULN - 2.5 x ULN | >2.5 x ULN - 5 x ULN | >5 x ULN - 10 x ULN | >10 x ULN | - |
| Definition: A finding based on la | i<br>boratory test results that indicate a | n increase in levels of creatine pho | snhokinase in a blood snecimen | • | |
| | r Cardiac disorders: Heart failure or | | | eart failure or Cardiac disorders: M | vocardial |
| infarction if same grade event. | r car alab albor across rical citatian con | car and another across stripe and and a man | Cool in Report Caranac disorders. | | youaranan |
| Creatinine increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x baseline: >1.5 - 3.0 | >3.0 x baseline: >3.0 - 6.0 x | >6.0 x ULN | T - |
| | | × ULN | ULN ULN | | |
| Definition: A finding based on la | ।<br>boratory test results that indicate ir | • | | • | 1 |
| • | • | | pioBicai specificii. | | |
| ivavigational ivote: Also conside | r Renal and urinary disorders: Acute | e kianey injury | | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Investigations | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Ejection fraction decreased | - | Resting ejection fraction (EF)<br>50 - 40%; 10 - 19% drop from<br>baseline | Resting ejection fraction (EF)<br>39 - 20%; >=20% drop from<br>baseline | Resting ejection fraction (EF)<br><20% | - |
| contraction. | outed when the amount of blood ej | • | , , | | the |
| | r Cardiac disorders: Left ventricular | | | | |
| Electrocardiogram QT corrected interval prolonged | Average QTc 450 - 480 ms | Average QTc 481 - 500 ms | Average QTc >= 501 ms; >60<br>ms change from baseline | Torsade de pointes;<br>polymorphic ventricular<br>tachycardia; signs/symptoms<br>of serious arrhythmia | - |
| Definition: A finding of a cardiac | dysrhythmia characterized by an a | bnormally long corrected QT interv | al. | | |
| Navigational Note: - | | | | | |
| Electrocardiogram T wave abnormal | T wave flattening | Nonspecific ST segment<br>change | - | - | - |
| Definition: A disorder characteri | ized by Electrocardiogram T wave a | mplitude changes. | • | • | |
| Navigational Note: - | · · | - | | | |
| Fibrinogen decreased | <1.0 - 0.75 x LLN; if abnormal,<br><25% decrease from baseline | <0.75 - 0.5 x LLN; if abnormal,<br>25 - <50% decrease from<br>baseline | <0.5 - 0.25 x LLN; if abnormal,<br>50 - <75% decrease from<br>baseline | <0.25 x LLN; if abnormal, 75%<br>decrease from baseline;<br>absolute value <50 mg/dL | - |
| Definition: A finding based on la | boratory test results that indicate a | in decrease in levels of fibrinogen ir | n a blood specimen. | | |
| Navigational Note: - | | | | | |
| Forced expiratory volume decreased | FEV1% (percentages of<br>observed FEV1 and FVC<br>related to their respective<br>predicted values) 99 - 70%<br>predicted | FEV1 60 - 69% | 50 - 59% | <= 49% | - |
| Definition: A finding based on te | est results that indicate a relative de | ecrease in the fraction of the forced | vital capacity that is exhaled in a s | pecific number of seconds. | |
| Navigational Note: Also conside | r Respiratory, thoracic and mediast | inal disorders: Respiratory failure o | | | |
| GGT increased | >ULN - 2.5 x ULN if baseline<br>was normal; 2.0 - 2.5 x<br>baseline if baseline was<br>abnormal | >2.5 - 5.0 x ULN if baseline<br>was normal; >2.5 - 5.0 x<br>baseline if baseline was<br>abnormal | >5.0 - 20.0 x ULN if baseline<br>was normal; >5.0 - 20.0 x<br>baseline if baseline was<br>abnormal | >20.0 x ULN if baseline was<br>normal; >20.0 x baseline if<br>baseline was abnormal | - |
| | boratory test results that indicate h<br>he transfer of a gamma glutamyl gr | igher than normal levels of the enz | | | i<br>i- |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Investigations | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Growth hormone abnormal | Asymptomatic; clinical or | Symptomatic; medical | - | - | - |
| | diagnostic observations only; | intervention indicated; | | | |
| | intervention not indicated | limiting instrumental ADL | | l | |
| <b>Definition:</b> A finding based on l | aboratory test results that indicate al | bnormal levels of growth hormone | in a biological specimen. | | |
| Navigational Note: - | | | | | |
| Haptoglobin decreased | <lln< td=""><td>-</td><td>-</td><td>-</td><td>-</td></lln<> | - | - | - | - |
| Definition: A finding based on I | aboratory test results that indicate a | n decrease in levels of haptoglobin | in a blood specimen. | • | |
| Navigational Note: - | | | | | |
| Hemoglobin increased | Increase in >0 - 2 g/dL | Increase in >2 - 4g/dL | Increase in >4 g/dL | - | - |
| Definition: A finding based on la | aboratory test results that indicate in | •<br>ncreased levels of hemoglobin abov | e normal. | • | , |
| Navigational Note: - | , | 3 | | | |
| INR increased | >1.2 - 1.5; >1 - 1.5 x baseline if | >1.5 - 2.5; >1.5 - 2.5 x baseline | >2.5: >2.5 x baseline if on | l - | - |
| | on anticoagulation; | if on anticoagulation; dose | anticoagulation; bleeding | | |
| | monitoring only indicated | adjustment indicated | | | |
| Definition: A finding based on I | aboratory test results that indicate a | n increase in the ratio of the patier | nt's prothrombin time to a control s | ample in the blood. | |
| Navigational Note: - | | | | | |
| Lipase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN; >2.0 - 5.0 x | >2.0 - 5.0 x ULN with signs or | >5.0 x ULN and with signs or | - |
| | 1 | ULN and asymptomatic | symptoms; >5.0 x ULN and | symptoms | |
| | | | asymptomatic | | |
| Definition: A finding based on la | aboratory test results that indicate a | n increase in the level of lipase in a | biological specimen. | | |
| Navigational Note: - | | | | | |
| Lymphocyte count decreased | <lln -="" 0.8="" 800="" <lln="" mm3;="" td="" x<=""><td>&lt;800 - 500/mm3; &lt;0.8 - 0.5 x</td><td>&lt;500 - 200/mm3; &lt;0.5 - 0.2 x</td><td>&lt;200/mm3; &lt;0.2 x 10e9 /L</td><td>-</td></lln> | <800 - 500/mm3; <0.8 - 0.5 x | <500 - 200/mm3; <0.5 - 0.2 x | <200/mm3; <0.2 x 10e9 /L | - |
| | 10e9/L | 10e9 /L | 10e9 /L | l | |
| <b>Definition:</b> A finding based on la | 10e9/L<br>aboratory test results that indicate a | /- | | | |
| • | | decrease in number of lymphocyte | es in a blood specimen. | | |
| <b>Definition:</b> A finding based on land Navigational Note: - Lymphocyte count increased | | /- | | <br> - | - |
| Navigational Note: -<br>Lymphocyte count increased | | decrease in number of lymphocyte >4000/mm3 - 20,000/mm3 | >20,000/mm3 | - ions or bone marrow. | - |
| Navigational Note: -<br>Lymphocyte count increased | aboratory test results that indicate a | decrease in number of lymphocyte >4000/mm3 - 20,000/mm3 | >20,000/mm3 | -<br>ions or bone marrow. | <br> - |
| Navigational Note: -<br>Lymphocyte count increased<br>Definition: A finding based on I: | aboratory test results that indicate a | decrease in number of lymphocyte >4000/mm3 - 20,000/mm3 | >20,000/mm3 | -<br>ions or bone marrow.<br><500/mm3; <0.5 x 10e9 /L | <br> - |
| Navigational Note: -<br>Lymphocyte count increased<br>Definition: A finding based on l<br>Navigational Note: - | aboratory test results that indicate a - aboratory test results that indicate a | decrease in number of lymphocyte >4000/mm3 - 20,000/mm3 n abnormal increase in the number | s in a blood specimen. >20,000/mm3 of lymphocytes in the blood, effus | | <br> -<br> - |
| Navigational Note: -<br>Lymphocyte count increased<br>Definition: A finding based on I:<br>Navigational Note: -<br>Neutrophil count decreased | aboratory test results that indicate a - aboratory test results that indicate a <lln -="" 1.5="" 1500="" <lln="" mm3;="" p="" x<=""></lln> | decrease in number of lymphocyte >4000/mm3 - 20,000/mm3 n abnormal increase in the number <1500 - 1000/mm3; <1.5 - 1.0 x 10e9 /L | s in a blood specimen. >20,000/mm3 of lymphocytes in the blood, effus <1000 - 500/mm3; <1.0 - 0.5 x 10e9 /L | | - |
| Navigational Note: -<br>Lymphocyte count increased<br>Definition: A finding based on I:<br>Navigational Note: -<br>Neutrophil count decreased | aboratory test results that indicate a - aboratory test results that indicate a <pre></pre> | decrease in number of lymphocyte >4000/mm3 - 20,000/mm3 n abnormal increase in the number <1500 - 1000/mm3; <1.5 - 1.0 x 10e9 /L | s in a blood specimen. >20,000/mm3 of lymphocytes in the blood, effus <1000 - 500/mm3; <1.0 - 0.5 x 10e9 /L | | - |
| Navigational Note: -<br>Lymphocyte count increased<br>Definition: A finding based on I:<br>Navigational Note: -<br>Neutrophil count decreased<br>Definition: A finding based on I: | aboratory test results that indicate a - aboratory test results that indicate a <pre></pre> | decrease in number of lymphocyte >4000/mm3 - 20,000/mm3 n abnormal increase in the number <1500 - 1000/mm3; <1.5 - 1.0 x 10e9 /L | s in a blood specimen. >20,000/mm3 of lymphocytes in the blood, effus <1000 - 500/mm3; <1.0 - 0.5 x 10e9 /L | | - |
| Navigational Note: - Lymphocyte count increased Definition: A finding based on languagational Note: - Neutrophil count decreased Definition: A finding based on languagational Note: - | aboratory test results that indicate a - aboratory test results that indicate a <lln -1.5="" -1500="" 10e9="" <lln="" a<="" aboratory="" indicate="" l="" mm3;="" results="" td="" test="" that="" x=""><td>decrease in number of lymphocyte &gt;4000/mm3 - 20,000/mm3 n abnormal increase in the number &lt;1500 - 1000/mm3; &lt;1.5 - 1.0 x 10e9 /L decrease in number of neutrophils</td><td>&gt; sin a blood specimen. &gt;20,000/mm3 of lymphocytes in the blood, effus &lt;1000 - 500/mm3; &lt;1.0 - 0.5 x 10e9 /L in a blood specimen.</td><td></td><td> <br/> -<br/> -</td></lln> | decrease in number of lymphocyte >4000/mm3 - 20,000/mm3 n abnormal increase in the number <1500 - 1000/mm3; <1.5 - 1.0 x 10e9 /L decrease in number of neutrophils | > sin a blood specimen. >20,000/mm3 of lymphocytes in the blood, effus <1000 - 500/mm3; <1.0 - 0.5 x 10e9 /L in a blood specimen. | | <br> -<br> - |
| Navigational Note: - Lymphocyte count increased Definition: A finding based on I: Navigational Note: - Neutrophil count decreased Definition: A finding based on I: Navigational Note: - Pancreatic enzymes decreased | aboratory test results that indicate a - aboratory test results that indicate a <lln -1.5="" -1500="" 10e9="" <lln="" a<="" aboratory="" indicate="" l="" mm3;="" results="" td="" test="" that="" x=""><td>decrease in number of lymphocyte &gt;4000/mm3 - 20,000/mm3 n abnormal increase in the number &lt;1500 - 1000/mm3; &lt;1.5 - 1.0 x 10e9 /L decrease in number of neutrophils Increase in stool frequency, bulk, or odor; steatorrhea</td><td>sin a blood specimen. &gt;20,000/mm3 of lymphocytes in the blood, effus &lt;1000 - 500/mm3; &lt;1.0 - 0.5 x 10e9 /L in a blood specimen. Sequelae of absorption deficiency</td><td></td><td> <br/> -<br/> -</td></lln> | decrease in number of lymphocyte >4000/mm3 - 20,000/mm3 n abnormal increase in the number <1500 - 1000/mm3; <1.5 - 1.0 x 10e9 /L decrease in number of neutrophils Increase in stool frequency, bulk, or odor; steatorrhea | sin a blood specimen. >20,000/mm3 of lymphocytes in the blood, effus <1000 - 500/mm3; <1.0 - 0.5 x 10e9 /L in a blood specimen. Sequelae of absorption deficiency | | <br> -<br> - |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Investigations | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Platelet count decreased | <lln -="" -<="" 75,000="" <lln="" mm3;="" td=""><td>&lt;75,000 - 50,000/mm3; &lt;75.0</td><td>&lt;50,000 - 25,000/mm3; &lt;50.0</td><td>&lt;25,000/mm3; &lt;25.0 x 10e9 /L</td><td>-</td></lln> | <75,000 - 50,000/mm3; <75.0 | <50,000 - 25,000/mm3; <50.0 | <25,000/mm3; <25.0 x 10e9 /L | - |
| | 75.0 x 10e9 /L | -50.0 x 10e9 /L | - 25.0 x 10e9 /L | 1 | |
| Definition: A finding based on I | aboratory test results that indicate a | a decrease in number of platelets ir | n a blood specimen. | | |
| Navigational Note: - | | | | | |
| Serum amylase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN; >2.0 - 5.0 x | >2.0 - 5.0 x ULN with signs or | >5.0 x ULN and with signs or | - |
| | | ULN and asymptomatic | symptoms; >5.0 x ULN and | symptoms | |
| | | | asymptomatic | 1 | |
| Definition: A finding based on I | aboratory test results that indicate a | an increase in the levels of amylase | in a serum specimen. | | |
| Navigational Note: - | | | | | |
| Thyroid stimulating hormone | TSH increased and no | - | - | - | - |
| increased | intervention initiated | | | | |
| Definition: A disorder character | rized by an increase in thyroid stimu | lating hormone. | | | |
| Navigational Note: If interventi | on initiated or symptomatic, report | as Endocrine disorders: Hypothyro | idism. | | |
| Urine output decreased | - | - | Adult: Oliguria (<80 ml in 8 | Adult: Anuria (<240 ml in 24 | - |
| | | | hr); | hr); | |
| | | | Infants: < 0.5 mL/kg per hour | Pediatric: No urine output | |
| | | | for 24 hours; | over 12 hours | |
| | | | Children: < 500 mL/1.73 m2 | | |
| | 1 | 1 | body surface area per day | I | |
| • | est results that indicate urine produ | iction is less relative to previous ou | tput. | | |
| Navigational Note: - | | | | | |
| Vital capacity abnormal | 90 - 75% of predicted value | <75 - 50% of predicted value; | <50% of predicted value; | - | - |
| | 1 | limiting instrumental ADL | limiting self care ADL | 1 | |
| | oulmonary function test results that | indicate an abnormal vital capacity | । (amount of exhaled after a maximı | ım inhalation) when compared to t | he |
| predicted value. | | | | | |
| | er Investigations: Forced Expiratory | | | ailure or Dyspnea | |
| Weightgain | 5 - <10% from baseline | 10 - <20% from baseline | >=20% from baseline | - | - |
| Definition: A finding characteria | zed by an unexpected or abnormal i | ncrease in overall body weight; for | pediatrics, greater than the baselin | e growth curve. | |
| Navigational Note: Do not use l | Metabolism and nutrition disorders | : Obesity, this term is being retired. | | | |
| <b>W</b> eight loss | 5 to <10% from baseline; | 10 - <20% from baseline; | >=20% from baseline; tube | - | - |
| | intervention not indicated | nutritional support indicated | feeding or TPN indicated | 1 | |
| Definition: A finding characteri: | zed by a decrease in overall body we | eight; for pediatrics, less than the b | aseline growth curve. | | |
| Navigational Note: - | | | | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| Investigations | | | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| White blood cell decreased | <lln -="" 3.0="" 3000="" <lln="" mm3;="" x<br="">10e9 /L</lln> | <3000 - 2000/mm3; <3.0 - 2.0<br>x 10e9 /L | <2000 - 1000/mm3; <2.0 - 1.0<br>x 10e9 /L | <1000/mm3; <1.0 x 10e9 /L | - |
| Definition: A finding based on la | boratory test results that indicate a | n decrease in number of white blo | od cells in a blood specimen. | | |
| Navigational Note: - | | | | | |
| Investigations - Other, specify | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: - | | | | | |
| Navigational Note: - | | | | | |

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade ! |
|---|---|---|---|---|---|
| Acidosis | pH <normal, but="">=7.3</normal,> | - | pH <7.3 | Life-threatening consequences | Death |
| Definition: A disorder chara<br>Navigational Note: - | cterized by abnormally high acidity (high | n hydrogen-ion concentration) of ti | ne blood and other body tissues. | | |
| Alcohol intolerance | - | Present | Severe symptoms; limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder chara<br>vomiting, indigestion and he<br><b>Navigational Note:</b> - | icterized by an increase in sensitivity to t<br>eadaches. | he adverse effects of alcohol, whic | h can include nasal congestion, skin | flushes, heart dysrhythmias, nause | ea, |
| Alkalosis | pH >normal, but <=7.5 | - | pH >7.5 | Life-threatening consequences | Death |
| Definition: A disorder chara<br>Navigational Note: - | cterized by abnormally high alkalinity (lo | ow hydrogen-ion concentration) of | the blood and other body tissues. | • | • |
| Anorexia | Loss of appetite without<br>alteration in eating habits | Oral intake altered without<br>significant weight loss or<br>malnutrition; oral nutritional<br>supplements indicated | Associated with significant<br>weight loss or malnutrition<br>(e.g., inadequate oral caloric<br>and/or fluid intake); tube<br>feeding or TPN indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder chara<br><b>Navigational Note:</b> - | cterized by a loss of appetite. | <u>.</u> | , | <u>.</u> | |
| Dehydration | Increased oral fluids indicated;<br>dry mucous membranes;<br>diminished skin turgor | IV fluids indicated | Hospitalization indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder chara<br><b>Navigational Note:</b> - | acterized by excessive loss of water from | the body. It is usually caused by se | vere diarrhea, vomiting or diaphore | esis. | • |
| Glucose intolerance | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; dietary<br>modification or oral agent<br>indicated | Severe symptoms; insulin indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder chara<br>Navigational Note: - | cterized by an inability to properly meta | bolize glucose. | | | |
| H <b>y</b> percalcemia | Corrected serum calcium of<br>>ULN - 11.5 mg/dL; >ULN - 2.9<br>mmol/L; lonized calcium >ULN<br>- 1.5 mmol/L | Corrected serum calcium of<br>>11.5 - 12.5 mg/dL; >2.9 - 3.1<br>mmol/L; Ionized calcium >1.5<br>-1.6 mmol/L; symptomatic | Corrected serum calcium of<br>>12.5 - 13.5 mg/dL; >3.1 - 3.4<br>mmol/L; lonized calcium >1.6<br>- 1.8 mmol/L; hospitalization<br>indicated | Corrected serum calcium of >13.5 mg/dL; >3.4 mmol/L; lonized calcium >1.8 mmol/L; life-threatening consequences | Death |

CTCAE v5.0 – November 27, 2017 Back to TOC


| | | Metabolism and nutrition of | lisorders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Hyperglycemia | Abnormal glucose above | Change in daily management | Insulin therapy initiated; | Life-threatening | Death |
| | baseline with no medical | from baseline for a diabetic; | hospitalization indicated | consequences; urgent | |
| | intervention | oral antiglycemic agent | | intervention indicated | |
| | | initiated; workup for diabetes | | | |
| | cterized by laboratory test results that | indicate an elevation in the concen | tration of blood sugar. It is usually a | n indication of diabetes mellitus or | glucose |
| intolerance. | | | | | |
| Navigational Note: - | | | | | |
| Hyperkalemia | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L; | >6.0 - 7.0 mmol/L; | >7.0 mmol/L; life-threatening | Death |
| | | intervention initiated | hospitalization indicated | consequences | |
| Definition: A disorder chara- | cterized by laboratory test results that | indicate an elevation in the concen | tration of potassium in the blood; as | ssociated with kidney failure or som | etimes |
| with the use of diuretic drug | ξs. | | | | |
| Navigational Note: - | | | | | |
| Hyperlipidemia | Requiring diet changes | Requiring pharmaceutical | Hospitalization; pancreatitis | Life-threatening | - |
| | | intervention | | consequences | |
| Definition: A disorder chara- | cterized by laboratory test results that | indicate an elevation in the concen | tration of lipids in blood. | • | |
| Navigational Note: - | | | · | | |
| Hypermagnesemia | >ULN - 3.0 mg/dL; >ULN - 1.23 | - | >3.0 - 8.0 mg/dL; >1.23 - 3.30 | >8.0 mg/dL; >3.30 mmol/L; | Death |
| 3 | mmol/L | | mmol/L | life-threatening consequences | |
| Definition: A disorder chara- | cterized by laboratory test results that | indicate an elevation in the concen | tration of magnesium in the blood. | • | • |
| Navigational Note: - | orange and the second state of the second stat | | | | |
| Hypernatremia | >ULN - 150 mmol/L | >150 - 155 mmol/L; | >155 -160 mmol/L: | >160 mmol/L; life-threatening | Death |
| riypemaaema | 7021 130 mmoly2 | intervention initiated | hospitalization indicated | consequences | Doddi |
| Definition: A disorder chara- | cterized by laboratory test results that | • | | barracqueribes | 1 |
| Navigational Note: - | cterized by rabbilatory test results that | indicate an elevatorim the concern | dador or socialitim the blood. | | |
| Hyperphosphatemia | Laboratory finding only and | Noninvasive intervention | Severe or medically significant | Life-threatening | Death |
| Пурегрітозрітасенна | intervention not indicated | indicated | but not immediately life- | consequences; urgent | Deau |
| | intervendonnot indicated | Indicated | threatening; hospitalization or | intervention indicated (e.g., | |
| | | | prolongation of existing | dialysis) | |
| | | | hospitalization indicated | ulaiysis <i>j</i> | |
| Definition: A disaudar above | l<br>cterized by laboratory test results that | I | | ı | ı |
| | cterized by laboratory test results that | iliuluate an elevation in the concen | наноп от priospriate in a brood. | | |
| Navigational Note: - | 450 | . 200 (-) | - F00 /-ll | L +4000 /- /- +44 4 // - | D 4b |
| Hypertriglyceridemia | 150 mg/dL - 300 mg/dL; 1.71 | >300 mg/dL - 500 mg/dL; | >500 mg/dL - 1000 mg/dL; | >1000 mg/dL; >11.4 mmol/L; | Death |
| | mmol/L - 3.42 mmol/L | >3.42 mmol/L - 5.7 mmol/L | >5.7 mmol/L - 11.4 mmol/L | life-threatening consequences | I |
| | cterized by laboratory test results that | indicate an elevation in the concen | tration of triglyceride concentration | in the blood. | |
| Navigational Note: - | | | | | |

| | Metabolism and nutrition disorders | | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Hyperuricemia | >ULN without physiologic | - | >ULN with physiologic | Life-threatening | Death |
| | consequences | 1 | consequences | consequences | |
| Definition: A disorder chara | acterized by laboratory test results that i | indicate an elevation in the concen | tration of uric acid. | | |
| Navigational Note: - | | | | | |
| Hypoalbuminemia | <lln -="" 3="" 30="" <lln="" dl;="" g="" l<="" td=""><td>&lt;3 - 2g/dL; &lt;30 - 20g/L</td><td>&lt;2 g/dL; &lt;20 g/L</td><td>Life-threatening</td><td>Death</td></lln> | <3 - 2g/dL; <30 - 20g/L | <2 g/dL; <20 g/L | Life-threatening | Death |
| | | | | consequences; urgent | |
| | | 1 | 1 | intervention indicated | |
| Definition: A disorder chara | acterized by laboratory test results that i | 'ndicate a low concentration of albu | ımin in the blood. | | |
| Navigational Note: - | | | | | |
| Hypocalcemia | Corrected serum calcium of | Corrected serum calcium of | Corrected serum calcium of | Corrected serum calcium of | Death |
| | <lln -="" 2.0<="" 8.0="" <lln="" dl;="" mg="" td=""><td>&lt;8.0 - 7.0 mg/dL; &lt;2.0 - 1.75</td><td>&lt;7.0 - 6.0 mg/dL; &lt;1.75 - 1.5</td><td>&lt;6.0 mg/dL; &lt;1.5 mmol/L;</td><td></td></lln> | <8.0 - 7.0 mg/dL; <2.0 - 1.75 | <7.0 - 6.0 mg/dL; <1.75 - 1.5 | <6.0 mg/dL; <1.5 mmol/L; | |
| | mmol/L; Ionized calcium <lln< td=""><td>mmol/L; Ionized calcium &lt;1.0</td><td>mmol/L; Ionized calcium &lt;0.9</td><td>lonized calcium &lt;0.8 mmol/L;</td><td></td></lln<> | mmol/L; Ionized calcium <1.0 | mmol/L; Ionized calcium <0.9 | lonized calcium <0.8 mmol/L; | |
| | - 1.0 mmol/L | - 0.9 mmol/L; symptomatic | - 0.8 mmol/L; hospitalization | life-threatening consequences | |
| | | I | indicated | 1 | |
| Definition: A disorder chara | acterized by laboratory test results that i | 'ndicate a low concentration of calc | ium (corrected for albumin) in the l | olood. | |
| Navigational Note: - | | | | | |
| Hypoglycemia | <lln -="" 3.0<="" 55="" <lln="" dl;="" mg="" td=""><td>&lt;55 - 40 mg/dL; &lt;3.0 - 2.2</td><td>&lt;40 - 30 mg/dL; &lt;2.2 - 1.7</td><td>&lt;30 mg/dL; &lt;1.7 mmol/L; life-</td><td>Death</td></lln> | <55 - 40 mg/dL; <3.0 - 2.2 | <40 - 30 mg/dL; <2.2 - 1.7 | <30 mg/dL; <1.7 mmol/L; life- | Death |
| | mmol/L | mmol/L | mmol/L | threatening consequences; | |
| | | 1 | | seizures | |
| <b>Definition:</b> A disorder chara | <br>acterized by laboratory test results that i | <br>indicate a low concentration of glud | cose in the blood. | seizures | |
| | acterized by laboratory test results that i | hdicate a low concentration of gluc | cose in the blood. | seizures | |
| Navigational Note: - | cterized by laboratory test results that i | indicate a low concentration of gluc Symptomatic with <lln -="" 3.0<="" td=""><td>cose in the blood.</td><td>seizures &lt;2.5 mmol/L; life-threatening</td><td>Death</td></lln> | cose in the blood. | seizures <2.5 mmol/L; life-threatening | Death |
| Navigational Note: - | | | | , | Death |
| <b>Definition:</b> A disorder chara<br><b>Navigational Note:</b> -<br>Hypokalemia | | Symptomatic with <lln -="" 3.0<="" td=""><td>&lt;3.0 - 2.5 mmol/L;</td><td>&lt;2.5 mmol/L; life-threatening</td><td>Death</td></lln> | <3.0 - 2.5 mmol/L; | <2.5 mmol/L; life-threatening | Death |
| Navigational Note: -<br>Hypokalemia | | Symptomatic with <lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" td=""><td>&lt;3.0 - 2.5 mmol/L;<br/>hospitalization indicated</td><td>&lt;2.5 mmol/L; life-threatening</td><td>Death</td></lln> | <3.0 - 2.5 mmol/L;<br>hospitalization indicated | <2.5 mmol/L; life-threatening | Death |
| Navigational Note: -<br>Hypokalemia<br>Definition: A disorder chara | <lln -="" 3.0="" l<="" mmol="" td=""><td>Symptomatic with <lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" td=""><td>&lt;3.0 - 2.5 mmol/L;<br/>hospitalization indicated</td><td>&lt;2.5 mmol/L; life-threatening</td><td>Death</td></lln></td></lln> | Symptomatic with <lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" td=""><td>&lt;3.0 - 2.5 mmol/L;<br/>hospitalization indicated</td><td>&lt;2.5 mmol/L; life-threatening</td><td>Death</td></lln> | <3.0 - 2.5 mmol/L;<br>hospitalization indicated | <2.5 mmol/L; life-threatening | Death |
| Navigational Note: -<br>Hypokalemia | <lln -="" 3.0="" l<="" mmol="" td=""><td>Symptomatic with <lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" td=""><td>&lt;3.0 - 2.5 mmol/L;<br/>hospitalization indicated</td><td>&lt;2.5 mmol/L; life-threatening</td><td>Death</td></lln></td></lln> | Symptomatic with <lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" td=""><td>&lt;3.0 - 2.5 mmol/L;<br/>hospitalization indicated</td><td>&lt;2.5 mmol/L; life-threatening</td><td>Death</td></lln> | <3.0 - 2.5 mmol/L;<br>hospitalization indicated | <2.5 mmol/L; life-threatening | Death |
| Navigational Note: -<br>Hypokalemia<br>Definition: A disorder chara<br>Navigational Note: - | < | Symptomatic with <lln -="" 3.0="" a="" concentration="" indicated="" intervention="" l;="" low="" mmol="" ndicate="" of="" pot<="" td=""><td>&lt;3.0 - 2.5 mmol/L;<br/>hospitalization indicated<br/>assium in the blood.</td><td>&lt;2.5 mmol/L; life-threatening consequences</td><td> </td></lln> | <3.0 - 2.5 mmol/L;<br>hospitalization indicated<br>assium in the blood. | <2.5 mmol/L; life-threatening consequences | |
| Navigational Note: -<br>Hypokalemia<br>Definition: A disorder chara<br>Navigational Note: -<br>Hypomagnesemia | <pre>cLLN - 3.0 mmol/L scterized by laboratory test results that i </pre> | Symptomatic with <lln -="" 3.0="" <a="" a="" concentration="" href="father: 41.2 - 0.9 mg/dL; &lt;0.5 - 0.4" indicated="" intervention="" l;="" low="" mmol="" ndicate="" of="" pot="">father: 41.2 - 0.9 mg/dL; &lt;0.5 - 0.4 mmol/L</lln> | <3.0 - 2.5 mmol/L;<br>hospitalization indicated<br>assium in the blood.<br><0.9 - 0.7 mg/dL; <0.4 - 0.3<br>mmol/L | <2.5 mmol/L; life-threatening consequences | |
| Navigational Note: - Hypokalemia Definition: A disorder chara Navigational Note: - Hypomagnesemia Definition: A disorder chara | <pre>cLLN - 3.0 mmol/L scterized by laboratory test results that i</pre> | Symptomatic with <lln -="" 3.0="" <a="" a="" concentration="" href="father: 41.2 - 0.9 mg/dL; &lt;0.5 - 0.4" indicated="" intervention="" l;="" low="" mmol="" ndicate="" of="" pot="">father: 41.2 - 0.9 mg/dL; &lt;0.5 - 0.4 mmol/L</lln> | <3.0 - 2.5 mmol/L;<br>hospitalization indicated<br>assium in the blood.<br><0.9 - 0.7 mg/dL; <0.4 - 0.3<br>mmol/L | <2.5 mmol/L; life-threatening consequences | |
| Navigational Note: - Hypokalemia Definition: A disorder chara Navigational Note: - Hypomagnesemia Definition: A disorder chara Navigational Note: - | <pre>cLLN - 3.0 mmol/L scterized by laboratory test results that i</pre> | Symptomatic with <lln -="" 3.0="" <a="" a="" concentration="" href="father: 41.2 - 0.9 mg/dL; &lt;0.5 - 0.4" indicated="" intervention="" l;="" low="" mmol="" ndicate="" of="" pot="">father: 41.2 - 0.9 mg/dL; &lt;0.5 - 0.4 mmol/L</lln> | <3.0 - 2.5 mmol/L;<br>hospitalization indicated<br>assium in the blood.<br><0.9 - 0.7 mg/dL; <0.4 - 0.3<br>mmol/L | <2.5 mmol/L; life-threatening consequences <0.7 mg/dL; <0.3 mmol/L; life-threatening consequences | |
| Navigational Note: -<br>Hypokalemia Definition: A disorder chara Navigational Note: - Hypomagnesemia | <pre>cterized by laboratory test results that i</pre> | Symptomatic with <lln -="" 0.4="" 0.9="" 3.0="" <0.5="" <1.2="" a="" and="" concentratio<="" concentration="" dl;="" indicate="" indicated="" intervention="" l="" l;="" low="" magnetic="" mg="" mmol="" of="" pot="" some="" states="" td=""><td>&lt;3.0 - 2.5 mmol/L;<br/>hospitalization indicated<br/>assium in the blood.<br/>&lt;0.9 - 0.7 mg/dL; &lt;0.4 - 0.3<br/>mmol/L<br/>gnesium in the blood.</td><td>&lt;2.5 mmol/L; life-threatening consequences</td><td>Death</td></lln> | <3.0 - 2.5 mmol/L;<br>hospitalization indicated<br>assium in the blood.<br><0.9 - 0.7 mg/dL; <0.4 - 0.3<br>mmol/L<br>gnesium in the blood. | <2.5 mmol/L; life-threatening consequences | Death |
| Navigational Note: - Hypokalemia Definition: A disorder chara Navigational Note: - Hypomagnesemia Definition: A disorder chara Navigational Note: - | <pre>cterized by laboratory test results that i</pre> | Symptomatic with <lln -="" 0.4="" 0.9="" 3.0="" <0.5="" <1.2="" a="" concentration="" dl;="" indicate="" indicated="" intervention="" l="" l;="" low="" maging="" mg="" mmol="" ndicate="" of="" pot="" s<="" second="" td="" the="" to=""><td>&lt;3.0 - 2.5 mmol/L;<br/>hospitalization indicated<br/>assium in the blood.<br/>&lt;0.9 - 0.7 mg/dL; &lt;0.4 - 0.3<br/>mmol/L<br/>gnesium in the blood.</td><td>&lt;2.5 mmol/L; life-threatening consequences &lt;0.7 mg/dL; &lt;0.3 mmol/L; life-threatening consequences &lt;120 mmol/L; life-threatening</td><td>Death</td></lln> | <3.0 - 2.5 mmol/L;<br>hospitalization indicated<br>assium in the blood.<br><0.9 - 0.7 mg/dL; <0.4 - 0.3<br>mmol/L<br>gnesium in the blood. | <2.5 mmol/L; life-threatening consequences <0.7 mg/dL; <0.3 mmol/L; life-threatening consequences <120 mmol/L; life-threatening | Death |
| Navigational Note: - Hypokalemia Definition: A disorder chara Navigational Note: - Hypomagnesemia Definition: A disorder chara Navigational Note: - | <pre>cterized by laboratory test results that i</pre> | Symptomatic with <lln -="" 0.4="" 0.9="" 3.0="" <0.5="" <1.2="" a="" concentration="" dl;="" indicate="" indicated="" intervention="" l="" l;="" low="" maging="" mg="" mmol="" ndicate="" of="" pot="" s<="" second="" td="" the="" to=""><td>&lt;3.0 - 2.5 mmol/L;<br/>hospitalization indicated<br/>assium in the blood. &lt;0.9 - 0.7 mg/dL; &lt;0.4 - 0.3<br/>mmol/L<br/>gnesium in the blood. 125-129 mmol/L<br/>symptomatic; 120-124</td><td>&lt;2.5 mmol/L; life-threatening consequences &lt;0.7 mg/dL; &lt;0.3 mmol/L; life-threatening consequences &lt;120 mmol/L; life-threatening</td><td>Death</td></lln> | <3.0 - 2.5 mmol/L;<br>hospitalization indicated<br>assium in the blood. <0.9 - 0.7 mg/dL; <0.4 - 0.3<br>mmol/L<br>gnesium in the blood. 125-129 mmol/L<br>symptomatic; 120-124 | <2.5 mmol/L; life-threatening consequences <0.7 mg/dL; <0.3 mmol/L; life-threatening consequences <120 mmol/L; life-threatening | Death |
| Navigational Note: - Hypokalemia Definition: A disorder chara Navigational Note: - Hypomagnesemia Definition: A disorder chara Navigational Note: - Hyponatremia | <pre>cterized by laboratory test results that i</pre> | Symptomatic with <lln -="" 0.4="" 0.9="" 125-129="" 3.0="" <0.5="" <1.2="" a="" and="" asymptomatic<="" concentration="" dl;="" indicate="" indicated="" intervention="" l="" l;="" low="" mag="" mg="" mmol="" of="" pot="" td=""><td>&lt;3.0 - 2.5 mmol/L; hospitalization indicated assium in the blood. &lt;0.9 - 0.7 mg/dL; &lt;0.4 - 0.3 mmol/L gnesium in the blood. 125-129 mmol/L symptomatic; 120-124 mmol/L regardless of symptoms</td><td>&lt;2.5 mmol/L; life-threatening consequences &lt;0.7 mg/dL; &lt;0.3 mmol/L; life-threatening consequences &lt;120 mmol/L; life-threatening</td><td>Death</td></lln> | <3.0 - 2.5 mmol/L; hospitalization indicated assium in the blood. <0.9 - 0.7 mg/dL; <0.4 - 0.3 mmol/L gnesium in the blood. 125-129 mmol/L symptomatic; 120-124 mmol/L regardless of symptoms | <2.5 mmol/L; life-threatening consequences <0.7 mg/dL; <0.3 mmol/L; life-threatening consequences <120 mmol/L; life-threatening | Death |

| | | Metabolism and nutrition d | isorders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| H <b>y</b> pophosphatemia | Laboratory finding only and intervention not indicated | Oral replacement therapy<br>indicated | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated | Life-threatening<br>consequences | Death |
| Definition: A disorder charact | erized by laboratory test results that | indicate a low concentration of pho | sphates in the blood. | | |
| Navigational Note: - | | | | | |
| Iron overload | - | Moderate symptoms;<br>intervention not indicated | Severe symptoms;<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder charact <b>Navigational Note:</b> - | erized by accumulation of iron in the | tissues. | | • | • |
| Obesity | - | BMI 25 - 29.9 kg/m2 | BMI 30 - 39.9 kg/m2 | BMI >=40 kg/m2 | - |
| <b>Definition:</b> A disorder charact<br><b>Navigational Note:</b> Use term I<br>gain | erized by having a high amount of bo<br>nvestigations: Weight | dy fat | ' | • | ' |
| Tumor lysis syndrome | - | - | Present | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder charact | erized by metabolic abnormalities tha | it result from a spontaneous or the | rapy-related cytolysis of tumor cells | • | |
| Navigational Note: - | | | | | |
| Metabolism and nutrition disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: - | | | | | |
| Navigational Note: - | | | | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| CTCAE Term | | Musculoskeletal and connective | tissue disorders | | |
|---|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Abdominal soft tissue necros | is - | Local wound care; medical | Operative debridement or | Life-threatening | Death |
| | | intervention indicated (e.g., | other invasive intervention | consequences; urgent | |
| | | dressings or topical | indicated (e.g., tissue | intervention indicated | |
| | | medications) | reconstruction, flap, or | | |
| | | 1 | grafting) | 1 | |
| Definition: A disorder charac | terized b <b>y</b> a necrotic process occurring | ; in the soft tissues of the abdomir | nal wall. | | |
| Navigational Note: - | | | | | |
| Arthralgia | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | - | - |
| | | instrumental ADL | ADL | [ | |
| Definition: A disorder charac | terized by a sensation of marked disco | mfort in a joint. | | | |
| Navigational Note: - | | | | | |
| Arthritis | Mild pain with inflammation, | Moderate pain associated | Severe pain associated with | - | - |
| | erythema, or joint swelling | with signs of inflammation, | signs of inflammation, | | |
| | | erythema, or joint swelling; | erythema, or joint swelling; | | |
| | | limiting instrumental ADL | irreversible joint damage; | | |
| | | | limiting self care ADL | | |
| Definition: A disorder charac | terized by inflammation involving a joi | nt | | | |
| Navigational Note: - | | | | | |
| Avascular necrosis | Asymptomatic; clinical or | Symptomatic; limiting | Severe symptoms; limiting self | Life-threatening | Death |
| | diagnostic observations only; | instrumental ADL | care ADL; elective operative | consequences; urgent | |
| | intervention not indicated | | intervention indicated | intervention indicated | |
| Definition: A disorder charac | terized by necrotic changes in the bon | e tissue due to interruption of blo | od supply. Most often affecting the e | piphysis of the long bones, the nec | rotic |
| changes result in the collapse | and the destruction of the bone struc | cture. | | - | |
| Navigational Note: Use new | term: Musculoskeletal and connective | tissue disorders: Osteonecrosis | | | |
| Back pain | Mildpain | Moderate pain; limiting | Severe pain; limiting self care | - | - |
| • | · · | instrumental ADL | ADL | | |
| | tarizad by a consation of marked disco | mfort in the back region. | • | • | • |
| Definition: A disorder charac | terizeu dy a serisation or market discu | | | | |
| <b>Definition:</b> A disorder charac<br><b>Navigational Note:</b> - | terized by a serisation of marked disco | | | | |
| Navigational Note: - | | Moderate pain: limiting | Severe pain: limiting self care | | _ |
| | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care | - | - |
| Navigational Note: -<br>Bone pain | Mild pain | instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Navigational Note: -<br>Bone pain<br>Definition: A disorder charac | | instrumental ADL | | - | - |
| Navigational Note: -<br>Bone pain | Mild pain | instrumental ADL | | | - |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Musculoskeletal and connective ti | ssue disorders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Chest wall necrosis | - | Local wound care; medical<br>intervention indicated (e.g.,<br>dressings or topical<br>medications) | Operative debridement or<br>other invasive intervention<br>indicated (e.g., tissue<br>reconstruction, flap, or<br>grafting) | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder character <b>Navigational Note:</b> - | ized by a necrotic process occurring | in the soft tissues of the chest wall | including breast. | • | |
| Chest wall pain Definition: A disorder character | Mild pain ized by a sensation of marked disco | Moderate pain; limiting instrumental ADL mfort in the chest wall. | Severe pain; limiting self care<br>ADL | - | - |
| Navigational Note: - | , | | | | |
| Exostosis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; limiting instrumental ADL | Severe symptoms; limiting self<br>care ADL; elective operative<br>intervention indicated | - | - |
| Definition: A disorder character | ized by non-neoplastic overgrowth | of bone. | ' | • | |
| Navigational Note: - | · | | | | |
| Fibrosis deep connective tissue | Mild induration, able to move<br>skin parallel to plane (sliding)<br>and perpendicular to skin<br>(pinching up) | Moderate induration, able to<br>slide skin, unable to pinch<br>skin; limiting instrumental ADL | Severe induration; unable to<br>slide or pinch skin; limiting<br>joint or orifice movement<br>(e.g., mouth, anus); limiting<br>self care ADL | Generalized; associated with<br>signs or symptoms of impaired<br>breathing or feeding | Death |
| Definition: A disorder character | ized by fibrotic degeneration of the | deep connective tissues. | ' | • | |
| Navigational Note: - | | | | | |
| Flank pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| <b>Definition:</b> A disorder character <b>Navigational Note:</b> - | ized by a sensation of marked disco | mfort on the lateral side of the bod | y in the region below the ribs and a | bove the hip. | |
| Generalized muscle weakness | Symptomatic; perceived by<br>patient but not evident on<br>physical exam | Symptomatic; evident on<br>physical exam; limiting<br>instrumental ADL | Limiting self care ADL | - | - |
| Definition: A disorder character | ized by a reduction in the strength | of muscles in multiple anatomic site | s. | | |
| Navigational Note: - | | | | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Musculoskeletal and connective ti | ssue disorders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Growth suppression | Reduction in growth velocity<br>by 10 - 29% ideally measured<br>over the period of a year | Reduction ingrowth velocity<br>by 30 - 49% ideally measured<br>over the period of a year or 0 -<br>49% reduction in growth from<br>the baseline growth curve | Reduction in growth velocity<br>of >=50% ideally measured<br>over the period of a year | - | - |
| <b>Definition:</b> A disorder character Navigational Note: - | terized by stature that is smaller than | normal as expected for age. | | | |
| Head soft tissue necrosis | - | Local wound care; medical<br>intervention indicated (e.g.,<br>dressings or topical<br>medications) | Operative debridement or<br>other invasive intervention<br>indicated (e.g., tissue<br>reconstruction, flap, or<br>grafting) | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder charactional Note: - | terized by a necrotic process occurring | in the soft tissues of the head. | | | · |
| Joint effusion | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; invasive<br>intervention indicated | - | - |
| Definition: A disorder charac | terized by excessive fluid in a joint, usu | •<br>ually as a result of joint inflammatic | n. | • | |
| Navigational Note: - | | • | | | |
| Joint range of motion<br>decreased | <=25% loss of ROM (range of<br>motion); decreased ROM<br>limiting athletic activity | >25 - 50% decrease in ROM;<br>limiting instrumental ADL | >50% decrease in ROM;<br>limiting self care ADL | - | - |
| Definition: A disorder charac | terized by a decrease in joint flexibility | of any joint. | | | |
| Navigational Note: - | | | | | |
| Joint range of motion<br>decreased cervical spine | Mild restriction of rotation or<br>flexion between 60 - 70<br>degrees | Rotation <60 degrees to right<br>or left; <60 degrees of flexion | Ankylosed/fused over<br>multiple segments with no C-<br>spine rotation | - | - |
| Definition: A disorder charact | terized by a decrease in flexibility of a | cervical spine joint. | • | • | • |
| Navigational Note: - | | | | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Musculoskeletal and connective ti | ssue disorders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Joint range of motion<br>decreased lumbar spine | Stiffness; difficulty bending to<br>the floor to pick up a very light<br>object but able to do athletic<br>activity | Pain with range of motion (ROM) in lumbar spine; requires a reaching aid to pick up a very light object from the floor | <50% lumbar spine flexion;<br>associated with symptoms of<br>ankylosis or fused over<br>multiple segments with no L-<br>spine flexion (e.g., unable to<br>reach to floot up a very<br>light object) | - | - |
| <b>Definition:</b> A disorder character <b>Navigational Note:</b> - | ized by a decrease in flexibility of a l | umbar spine joint. | | | |
| Kyphosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate accentuation;<br>limiting instrumental ADL | Severe accentuation;<br>operative intervention<br>indicated; limiting self care<br>ADL | - | - |
| <b>Definition:</b> A disorder character <b>Navigational Note:</b> - | ized by an abnormal increase in the | curvature of the thoracic portion o | f the spine. | | · |
| Lordosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate accentuation;<br>limiting instrumental ADL | Severe accentuation;<br>operative intervention<br>indicated; limiting self care<br>ADL | - | - |
| | ized by an abnormal increase in the | curvature of the lumbar portion of | the spine. | | |
| Navigational Note: -<br>Muscle cramp | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| <b>Definition:</b> A disorder character <b>Navigational Note:</b> Synonym: N | ized by marked cramping sensation<br>Juscle spasm | • | 1 | • | 1 |
| Muscle weakness lower limb | Symptomatic; perceived by<br>patient but not evident on<br>physical exam | Symptomatic; evident on<br>physical exam; limiting<br>instrumental ADL | Limiting self care ADL | - | - |
| | ized by a reduction in the strength o | of the lower limb muscles. | • | • | • |
| Navigational Note: -<br>Muscle weakness trunk | Symptomatic; perceived by<br>patient but not evident on<br>physical exam | Symptomatic; evident on<br>physical exam; limiting<br>instrumental ADL | Limiting self care ADL | - | - |
| <b>Definition:</b> A disorder character <b>Navigational Note:</b> - | ized b <b>y</b> a reduction in the strength o | of the trunk muscles. | | | |

| | | Musculoskeletal and connective t | issue disorders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Muscle weakness upper limb | Symptomatic; perceived by<br>patient but not evident on<br>physical exam | Symptomatic; evident on<br>physical exam; limiting<br>instrumental ADL | Limiting self care ADL | - | - |
| | F | • | I | 1 | I |
| Navigational Note: - | rized by a reduction in the strength | of the upper limb muscles. | | | |
| Musculoskeletal deformity | Cosmetically and functionally insignificant hypoplasia | Deformity, hypoplasia, or<br>asymmetry able to be<br>remediated by prosthesis<br>(e.g., shoe insert) or covered<br>by clothing | Significant deformity,<br>hypoplasia, or asymmetry,<br>unable to be remediated by<br>prosthesis or covered by<br>clothing; limiting self care ADL | - | - |
| Definition: A disorder characte | rized b <b>y</b> a malformation of the musc | uloskeletal system. | | | |
| Navigational Note: - | | | | | |
| Myalgia | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | - | = |
| Definition: A disorder characte | rized b <b>y</b> marked discomfort sensatio | n originating from a muscle or grou | up of muscles. | • | • |
| Navigational Note: - | | | | | |
| Myositis | Mild pain | Moderate pain associated<br>with weakness; pain limiting<br>instrumental ADL | Pain associated with severe<br>weakness; limiting self care<br>ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | - |
| Definition: A disorder character | rized by inflammation involving the | skeletal muscles. | • | • | • |
| Navigational Note: - | , , | | | | |
| Neck pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characte | rized by a sensation of marked disco | mfort in the neck area. | · | • | • |
| Navigational Note: - | | | | | |
| Neck soft tissue necrosis | - | Local wound care; medical intervention indicated (e.g., dressings or topical medications) | Operative debridement or<br>other invasive intervention<br>indicated (e.g., tissue<br>reconstruction, flap, or<br>grafting) | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder character | rized b <b>y</b> a necrotic process occurring | in the soft tissues of the neck. | | | |
| Navigational Note: - | | | | | |

| | | Musculoskeletal and connective ti | ssue disorders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Osteonecrosis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; medical<br>intervention indicated (e.g.,<br>analgesics or<br>bisphosphonates); limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; elective operative<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| changes result in the collapse | terized by necrotic changes in the bone<br>and the destruction of the bone struc | | d supply. Most often affecting the e | piphysis of the long bones, the | necrotic |
| Navigational Note: - | | | | | |
| Osteonecrosis of jaw | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical<br>intervention indicated (e.g.,<br>topical agents); limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; elective operative<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | terized by a necrotic process occurring | in the bone of the mandible. | | | |
| Navigational Note: - | | | | | |
| Osteoporosis | Adult: Radiologic evidence of osteoporosis or Bone Mineral Density (BMD) t-score -1 to - 2.5 (osteopenia); Pediatric: Radiologic evidence | Adult: BMD t-score < -2.5; loss of height < 2 cm; therapy to improve BMD indicated; limiting instrumental ADL; Pediatric: Low BMD (z-score | Adult: Loss of height >=2 cm;<br>hospitalization indicated;<br>limiting self care ADL;<br>Pediatric: Limiting self care<br>ADL | - | - |
| | of low BMD with z score of <=<br>-2.0 and no history of<br>significant fractures | <= -2.0) and significant<br>fracture history (defined as a<br>long bone fracture of the<br>lower extremity, vertebral<br>compression, 2 or more long<br>bone fractures of the upper<br>extremities); therapy to<br>improve BMD indicated | | | |
| <b>Definition:</b> A disorder charact composition), resulting in incr | l<br>cerized by reduced bone mass, with a c<br>eased fracture incidence. | | <br> the number and size of the trabec | <br>ulae of cancellous bone (but no | rmal chemical |
| Navigational Note: - | | | | | |
| Pain in extremity | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder charact | erized by a sensation of marked disco | mfort in the upper or lower extrem | ities. | • | • |
| Navigational Note: - | | | | | |

| CTCAE Term Pelvic soft tissue necrosis | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Dalvic soft tissua pacrosis | | | | Olduc 4 | Grade 5 |
| reme sore assue near osis | - | Local wound care; medical<br>intervention indicated (e.g.,<br>dressings or topical<br>medications) | Operative debridement or<br>other invasive intervention<br>indicated (e.g., tissue<br>reconstruction, flap, or<br>grafting) | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder characteriz<br>Navigational Note: - | red by a necrotic process occurring | in the soft tissues of the pelvis. | | | |
| Rhabdomyolysis | Asymptomatic, intervention not indicated; laboratory findings only | Non-urgent intervention indicated | Symptomatic, urgent intervention indicated | Life-threatening<br>consequences; dial <b>y</b> sis | Death |
| Definition: A disorder characteriz<br>Navigational Note: - | ed by the breakdown of muscle tis | sue resulting in the release of mu | scle fiber contents into the bloodstre | am. | |
| Rotator cuff injury | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting<br>instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>limiting self care ADL | - | - |
| Definition: A disorder characteriz<br>Navigational Note: - | red by an injury of the rotator cuff. | | | | |
| Scoliosis | <20 degrees; dinically<br>undetectable | >20 - 45 degrees; visible by<br>forward flexion; limiting<br>instrumental ADL | >45 degrees; scapular<br>prominence in forward<br>flexion; operative intervention<br>indicated; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz Navigational Note: - | red by a malformed, lateral curvatu | re of the spine. | • | • | • |
| Soft tissue necrosis lower limb | - | Local wound care; medical<br>intervention indicated (e.g.,<br>dressings or topical<br>medications) | Operative debridement or<br>other invasive intervention<br>indicated (e.g., tissue<br>reconstruction, flap, or<br>grafiting) | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |

| | | Musculoskeletal and connective tis | ssue disorders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Soft tissue necrosis upper limb | - | Local wound care; medical<br>intervention indicated (e.g.,<br>dressings or topical<br>medications) | Operative debridement or<br>other invasive intervention<br>indicated (e.g., tissue<br>reconstruction, flap, or<br>grafting) | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | ized by a necrotic process occurring | in the soft tissues of the upper extr | emity. | • | • |
| Navigational Note: - | | | | | |
| Superficial soft tissue fibrosis | Mild induration, able to move<br>skin parallel to plane (sliding)<br>and perpendicular to skin<br>(pinching up) | Moderate induration, able to<br>slide skin, unable to pinch<br>skin; limiting instrumental ADL | Severe induration; unable to<br>slide or pinch skin; limiting<br>joint or orifice movement<br>(e.g., mouth, anus); limiting<br>self care ADL | Generalized; associated with<br>signs or symptoms of impaired<br>breathing or feeding | Death |
| Definition: A disorder character | ized by fibrotic degeneration of the | superficial soft tissues. | | • | |
| Navigational Note: - | | | | | |
| Trismus | Decreased ROM (range of motion) without impaired eating | Decreased ROM requiring<br>small bites, soft foods or<br>purees | Decreased ROM with inability<br>to adequately aliment or<br>hydrate orally | - | - |
| Definition: A disorder character<br>Navigational Note: - | ized by lack of ability to open the m | outh fully due to a decrease in the r | ange of motion of the muscles of m | nastication. | |
| Unequal limb length | Mild length discrepancy <2 cm | Moderate length discrepancy 2 - 5 cm; shoe lift indicated; limiting instrumental ADL | Severe length discrepancy >5<br>cm; limiting self care ADL;<br>operative intervention<br>indicated | - | - |
| Navigational Note: - | ized by a discrepancy between the i | enguis or the lower of upper extre | illues. | | |
| Musculoskeletal and<br>connective tissue disorder -<br>Other, specify | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: - | | | | | |
| Navigational Note: - | | | | | |

| | Neoplasm | s benign, malignant and unspecifie | ed (incl cysts and polyps) | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Leukemia secondary to | - | - | - | Present | Death |
| oncology chemotherapy | | l | | | |
| Definition: A disorder characteri | zed by leukemia arising as a result o | of the mutagenic effect of chemoth | erapy agents. | | |
| Navigational Note: - | | | | | |
| Myelodysplastic syndrome | - | - | - | Life-threatening | Death |
| | | | | consequences; urgent | |
| | | I | l | intervention indicated | J |
| | zed by insufficiently healthy hemat | apoletic cell production by the bone | e marrow. | | |
| Navigational Note: - | | Intervention initiated | 1 | | |
| Skin papilloma | Asymptomatic; intervention not indicated | Intervention initiated | - | - | - |
| Definition: A disorder characteri | zed by the presence of one or more | l | l | l | J |
| Navigational Note: - | zed by the presence of one of more | e waits. | | | |
| Treatment related secondary | I - | Ι. | Non life-threatening | Acute life-threatening | Death |
| malignancy | | | secondary malignancy | secondary malignancy; blast | Deadi |
| , | | | , | crisis in leukemia | |
| Definition: A disorder characteri | zed by development of a malignand | •<br>cy most probably as a result of treat | ment for a previously existing malig | nancy. | ' |
| Navigational Note: - | | | | | |
| Tumor hemorrhage | Mild symptoms; intervention | Moderate symptoms; | Transfusion indicated; | Life-threatening | Death |
| | not indicated | intervention indicated | invasive intervention | consequences; urgent | |
| | | l | indicated; hospitalization | intervention indicated | |
| <b>Definition:</b> A disorder characteri | zed b <b>y</b> bleeding in a tumor. | | | | |
| Navigational Note: - | T | | | | |
| Tumor pain | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | = | - |
| Definition: A discuster above stari | | instrumental ADL | ADL pressing on a nerve, blocking blood | l | <u> </u> |
| metastasis. | zed by a sensation of marked disco- | ппогстопта пеоргазит втасттау ве | e pressing or a nerve, brocking brook | d vessels, il illamed or mactured no | ''' |
| Navigational Note: - | | | | | |
| Neoplasms benign, malignant | Asymptomatic or mild | Moderate: minimal, local or | Severe or medically significant | Life-threatening | Death |
| and unspecified (incl cysts and | symptoms; clinical or | noninvasive intervention | but not immediately life- | consequences; urgent | |
| polyps) - Other, specify | diagnostic observations only; | indicated; limiting age- | threatening; hospitalization or | intervention indicated | |
| | intervention not indicated | appropriate instrumental ADL | prolongation of existing | | |
| | | | hospitalization indicated; | | |
| | | l | limiting self care ADL | | I |
| Definition: - | | | | | |
| Navigational Note: - | | | | | |

| | | Nervous system disord | ers | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Abducens nerve disorder | Asymptomatic; clinical or | Moderate symptoms; limiting | Severe symptoms; limiting self | - | - |
| | diagnostic observations only; | instrumental ADL | care ADL | | |
| | intervention not indicated | I | | 1 | |
| Definition: A disorder characte<br>Navigational Note: - | erized by dysfunction of the abducen | s nerve (sixth cranial nerve). | | | |
| Accessory nerve disorder | Asymptomatic; clinical or | Moderate symptoms; limiting | Severe symptoms; limiting self | - | - |
| • | diagnostic observations only; | instrumental ADL | care ADL | | |
| | intervention not indicated | | | | |
| Definition: A disorder characte | erized by dysfunction of the accessor | nerve (eleventh cranial nerve). | • | • | • |
| Navigational Note: - | | • | | | |
| Acoustic nerve disorder NOS | Asymptomatic; clinical or | Moderate symptoms; limiting | Severe symptoms; limiting self | - | - |
| | diagnostic observations only; | instrumental ADL | care ADL | | |
| | intervention not indicated | | | | |
| Definition: A disorder characte | erized by dysfunction of the acoustic | nerve (eighth cranial nerve). | | | • |
| Navigational Note: - | | | | | |
| Akathisia | Mild restlessness or increased | Moderate restlessness or | Severe restlessness or | - | - |
| | motor activity | increased motor activity; | increased motor activity; | | |
| | | limiting instrumental ADL | limiting self care ADL | | |
| Definition: A disorder characte | erized by an uncomfortable feeling of | inner restlessness and inability to s | stay still; this is a side effect of some | e psychotropic drugs. | |
| Navigational Note: - | | • | • | | |
| Amnesia | Mild; transient memory loss | Moderate; short term | Severe; long term memory | - | - |
| | • | memory loss; limiting | loss; limiting self care ADL | | |
| | | instrumental ADL | 1 | | |
| Definition: A disorder characte | erized by systematic and extensive lo | ss of memor <b>v</b> . | • | • | |
| Navigational Note: - | | • | | | |
| Anosmia | Present | - | _ | - | - |
| | erized by a change in the sense of sm | I<br>all | 1 | 1 | ı |
| Navigational Note: Also consid | | aı. | | | |
| Aphonia | der Orlactory Herve disorder | 1 | Voicelessness: unable to | 1 | |
| Aprionia | <sup>-</sup> | - | speak | - | 1 - |
| D-61-161 6 -1/ | | I | 1 -1 | 1 | ı |
| | erized by the inability to speak. It may | result from injuries to the vocal co | iras or may be tunctional (psychoge | nic). | |
| Navigational Note: - | 1 | | | 1 | |
| Arachnoiditis | Mild symptoms | Moderate symptoms; limiting | Severe symptoms; limiting self | Life-threatening | Death |
| | | instrumental ADL | care ADL | consequences, urgent | |
| | 1 | I | | intervention indicated | |
| Definition: A disorder characte | erized by inflammation of the arachno | oid membrane and adjacent subara | chnoid space. | | |
| Navigational Note: - | | | | | |

| | | Nervous system disord | ers | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Ataxia | Asymptomatic; clinical or | Moderate symptoms; limiting | Severe symptoms; limiting self | - | - |
| | diagnostic observations only; | instrumental ADL | care ADL; mechanical | | |
| | intervention not indicated | | assistance indicated | 1 | |
| Definition: A disorder charact | erized by lack of coordination of musc | de movements resulting in the impa | airment or inability to perform volu | ntar <b>y</b> activities. | |
| Navigational Note: - | | | | | |
| Brachial plexopathy | Asymptomatic; clinical or | Moderate symptoms; limiting | Severe symptoms; limiting self | - | - |
| | diagnostic observations only; | instrumental ADL | care ADL | | |
| | intervention not indicated | l | 1 | l | l |
| | erized by regional paresthesia of the b | orachial plexus, marked discomfort | and muscle weakness, and limited i | movement in the arm or hand. | |
| Navigational Note: - | | | 1 | | |
| Central nervous system | Asymptomatic; clinical or | Moderate symptoms; | Severe symptoms; medical | Life-threatening | Death |
| necrosis | diagnostic observations only; | corticosteroids indicated | intervention indicated | consequences; urgent | |
| | intervention not indicated | <u>.</u> | 1 | intervention indicated | 1 |
| | erized by a necrotic process occurring | in the brain and/or spinal cord. | | | |
| Navigational Note: - | Ta | I a | I a | Luci | 1 |
| Cerebrospinal fluid leakage | Post-craniotomy:<br>asymptomatic; Post-lumbar | Post-craniotomy: moderate<br>symptoms; medical | Severe symptoms; medical<br>intervention indicated | Life-threatening | Death |
| | puncture: transient headache: | intervention indicated: Post- | intervention indicated | consequences; urgent<br>intervention indicated | |
| | postural care indicated | lumbar puncture: persistent | | litter veridori indicated | |
| | posturar care mulcated | moderate symptoms; blood | | | |
| | | patch indicated | | | |
| Definition: A disorder charact | erized by loss of cerebrospinal fluid in | • ' | 1 | • | |
| Navigational Note: - | " | 3 | | | |
| Cognitive disturbance | Mild cognitive disability; not | Moderate cognitive disability: | Severe cognitive disability; | - | - |
| | interfering with | interfering with | significant impairment of | | |
| | work/school/life | work/school/life performance | work/school/life performance | | |
| | performance; specialized | but capable of independent | | | |
| | educational services/devices | living; specialized resources | | | |
| | not indicated | on part time basis indicated | | 1 | |
| | erized by a conspicuous change in cog | nitive function. | | | |
| Navigational Note: - | | | | | |
| Concentration impairment | Mild inattention or decreased | Moderate impairment in | Severe impairment in | - | - |
| | level of concentration | attention or decreased level | attention or decreased level | ĺ | |
| | | of concentration; limiting | of concentration; limiting self | ĺ | |
| | I | instrumental ADL | care ADL | I | I |
| | erized by a deterioration in the ability | to concentrate. | | | |
| Navigational Note: - | | | | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Nervous system disord | ers | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Depressed level of consciousness | Decreased level of alertness | Sedation; slow response to<br>stimuli; limiting instrumental<br>ADL | Difficult to arouse | Life-threatening<br>consequences; coma; urgent<br>intervention indicated | Death |
| Definition: A disorder chara- | cterized by a decrease in ability to perc | eive and respond. | • | • | • |
| Navigational Note: - | | | | | |
| Dizziness | Mild unsteadiness or<br>sensation of movement | Moderate unsteadiness or<br>sensation of movement;<br>limiting instrumental ADL | Severe unsteadiness or<br>sensation of movement;<br>limiting self care ADL | - | - |
| Definition: A disorder chara- | cterized by a disturbing sensation of ligi | ntheadedness, unsteadiness, giddir | ess, spinning or rocking. | • | • |
| Navigational Note: - | | | | | |
| Dysarthria | Mild slurred speech | Moderate impairment of<br>articulation or slurred speech | Severe impairment of<br>articulation or slurred speech | - | - |
| <b>Definition:</b> A disorder chara-<br><b>Navigational Note:</b> - | cterized by slow and slurred speech res | ulting from an inability to coordina | te the muscles used in speech. | | |
| Dysesthesia | Mild sensory alteration | Moderate sensory alteration;<br>limiting instrumental ADL | Severe sensory alteration;<br>limiting self care ADL | - | - |
| <b>Definition:</b> A disorder chara- | cterized by distortion of sensory percep | tion, resulting in an abnormal and | unpleasant sensation. | | |
| Navigational Note: - | | | | | |
| Dysgeusia | Altered taste but no change in diet | Altered taste with change in<br>diet (e.g., oral supplements);<br>noxious or unpleasant taste;<br>loss of taste | - | - | - |
| Definition: A disorder chara- | cterized by abnormal sensual experienc | e with the taste of foodstuffs; it can | nbe related to a decrease in the ser | nse of smell. | • |
| Navigational Note: - | | | | | |
| Dysphasia | Awareness of receptive or<br>expressive characteristics; not<br>impairing ability to<br>communicate | Moderate receptive or<br>expressive characteristics;<br>impairing ability to<br>communicate spontaneously | Severe receptive or expressive<br>characteristics; impairing<br>ability to read, write or<br>communicate intelligibly | - | - |
| Definition: A disorder chara- | cterized by impairment of verbal comm | unication skills, often resulting fror | n brain damage. | | |
| Navigational Note: - | | | | | |
| Edema cerebral | - | - | New onset; worsening from baseline | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder chara- | cterized by swelling due to an excessive | accumulation of fluid in the brain. | - | - | - |
| Navigational Note: - | | | | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Nervous system disord | lers | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Encephalopathy | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder charact | erized by a pathologic process involvi | ng the brain. | | | |
| Navigational Note: - | | | | | |
| Extrapyramidal disorder | Mild involuntary movements | Moderate involuntary<br>movements; limiting<br>instrumental ADL | Severe involuntary<br>movements or torticollis;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder charact | erized by abnormal, repetitive, involu | ntary muscle movements, frenzied | speech and extreme restlessness. | | • |
| Navigational Note: Synonym: | Restless legs | | | | |
| Facial muscle weakness | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder charact | erized by a reduction in the strength | of the facial muscles. | | | |
| Navigational Note: - | | | | | |
| Facial nerve disorder | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| | erized by dysfunction of the facial ner | ve (seventh cranial nerve). | | | |
| Navigational Note: - | | T | T | Lie | |
| Glossopharyngeal nerve<br>disorder | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder charact | erized by dysfunction of the glossoph | aryngeal nerve (ninth cranial nerve | ). | • | • |
| Navigational Note: - | | | | | |
| Guillain-Barre syndrome | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self<br>care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated;<br>intubation | Death |
| Definition: A disorder charact | erized by the body's immune system | attacking the peripheral nervous sy | stem causing ascending paralysis. | | |
| Navigational Note: - | | | | | |
| Headache | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder charact | erized b <b>y</b> a sensation of marked disco | mfort in various parts of the head, | not confined to the area of distribut | tion of any nerve. | |
| Navigational Note: - | | | | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Nervous system disord | lers | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Hydrocephalus | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms;<br>intervention not indicated | Severe symptoms or<br>neurological deficit;<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder character | ized by an abnormal increase of cer | ebrospinal fluid in the ventricles of | the brain. | • | · |
| Navigational Note: - | | | | | |
| Hypersomnia | Mild increased need for sleep | Moderate increased need for<br>sleep | Severe increased need for<br>sleep | - | - |
| Definition: A disorder character | rized by characterized by excessive s | leepiness during the daytime. | • | | · |
| Navigational Note: - | | | | | |
| Hypoglossal nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder character | ized by dysfunction of the hypoglos | sal nerve (twelfth cranial nerve). | • | • | |
| Navigational Note: - | | | | | |
| Intracranial hemorrhage | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms;<br>intervention indicated | Ventriculostomy, ICP<br>monitoring, intraventricular<br>thrombolysis, or invasive<br>intervention indicated;<br>hospitalization | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder character | ized by bleeding from the cranium. | | | • | |
| Navigational Note: - | | | | | |
| Ischemia cerebrovascular | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms | - | - | - |
| Definition: A disorder character | rized by a decrease or absence of blo | ood supply to the brain caused by c | bstruction (thrombosis or embolism | n) of an artery resulting in neuro | ological |
| damage. | | | | | |
| Navigational Note: Prior to usin | ng this term consider Nervous systen | | | | |
| Lethargy | Mild symptoms; reduced<br>alertness and awareness | Moderate symptoms; limiting<br>instrumental ADL | - | - | - |
| Definition: A disorder character | rized b <b>y</b> a decrease in consciousness | characterized by mental and physi | ical inertness. | | |
| Navigational Note: - | | | | | |

| | | Nervous system disord | ers | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Leukoencephalopathy | Asymptomatic; small focal T2/FLAIR hyperintensities; involving periventricular white matter or <1/3 of susceptible areas of cerebrum +/- mild increase in subarachnoid space (SAS) and/or mild ventriculomegaly | Moderate symptoms; focal T2/FLAIR hyperintensities, involving periventricular white matter extending into centrum semiovale or involving 1/3 to 2/3 of susceptible areas of cerebrum +/- moderate increase in SAS and/or moderate | Severe symptoms; extensive T2/FLAIR hyperintensities, involving periventricular white matter involving 2/3 or more of susceptible areas of cerebrum +/- moderate to severe increase in SAS and/or moderate to severe ventriculomegaly | Life-threatening consequences; extensive TZ/FLAIR hyperintensities, involving periventricular white matter involving most of susceptible areas of cerebrum +/- moderate to severe increase in SAS and/or moderate to severe | Death |
| | | ventriculomegaly | | ventriculomegaly | |
| | ized by diffuse reactive astrocytosis | with multiple areas of necrotic foci | without inflammation. | | |
| Navigational Note: - | T | | T | | |
| Memory impairment | Mild memory impairment | Moderate memory<br>impairment; limiting<br>instrumental ADL | Severe memory impairment;<br>limiting self care ADL | - | - |
| Definition: A disorder character | ized by a deterioration in memory f | unction. | • | | - |
| Navigational Note: - | | | | | |
| Meningismus | Mild symptoms | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder character | ized b <b>y</b> neck stiffness, headache, an | d photophobia resulting from irrita | tion of the cerebral meninges. | • | • |
| Navigational Note: - | | | | | |
| Movements involuntary | Mild symptoms | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL | - | - |
| Definition: A disorder character | ized by uncontrolled and purposele: | ss movements. | • | • | |
| Navigational Note: - | | | | | |
| Muscle weakness left-sided | Symptomatic; perceived by<br>patient but not evident on<br>physical exam | Symptomatic; evident on<br>physical exam; limiting<br>instrumental ADL | Limiting self care ADL | - | - |
| Definition: A disorder character | ized by a reduction in the strength o | of the muscles on the left side of the | e bod <b>y.</b> | • | • |
| Navigational Note: - | | | | | |
| Muscle weakness right-sided | Symptomatic; perceived by<br>patient but not evident on<br>physical exam | Symptomatic; evident on<br>physical exam; limiting<br>instrumental ADL | Limiting self care ADL | - | - |
| <b>Definition:</b> A disorder character | ized by a reduction in the strength o | of the muscles on the right side of th | ne bod <b>y.</b> | | |
| Navigational Note: - | | | | | |

| | | Nervous system disord | ers | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Myasthenia gravis | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | zed b <b>y</b> weakness and rapid fatigue o | of any of the skeletal muscles. | | | |
| Navigational Note: - | | | | | |
| Neuralgia | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| | zed b <b>y</b> intense painful sensation ald | ong a nerve or group of nerves. | | | |
| Navigational Note: - | | | | | |
| Nystagmus | - | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL | - | - |
| Definition: A disorder characteri | zed by involuntary movements of th | ne eyeballs. | - | - | |
| Navigational Note: - | | | | | |
| Oculomotor nerve disorder | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by dysfunction of the oculomot | or nerve (third cranial nerve). | | | |
| Navigational Note: - | | | | | |
| Olfactory nerve disorder | - | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL | - | - |
| Definition: A disorder characteri | zed by dysfunction of the olfactory | nerve (first cranial nerve). | • | • | • |
| Navigational Note: - | | | | | |
| Paresthesia | Mild symptoms | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL | - | - |
| Definition: A disorder characteri | zed by functional disturbances of se | • | ! | numbness, pressure, cold. and/or | warmth. |
| Navigational Note: - | | , | | .,,,, | |
| Peripheral motor neuropathy | Asymptomatic; clinical or | Moderate symptoms; limiting | Severe symptoms; limiting self | Life-threatening | Death |
| | diagnostic observations only | instrumental ADL | care ADL | consequences; urgent<br>intervention indicated | |
| Definition: A disorder characteri | zed by damage or dysfunction of th | e peripheral motor nerves. | | | |
| | Nervous system disroders: Periphe | | | | |

| OTO 4 E T | | Nervous system disord | ers | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Peripheral sensory | Asymptomatic | Moderate symptoms; limiting | Severe symptoms; limiting self | Life-threatening | - |
| neuropathy | | instrumental ADL | care ADL | consequences; urgent | |
| | | | | intervention indicated | |
| Definition: A disorder characte | erized by damage or dysfunction of th | ne peripheral sensory nerves. | | | |
| Navigational Note: - | | | | | |
| Phantom pain | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | - | - |
| | | instrumental ADL | ADL | | |
| Definition: A disorder characte | erized by a sensation of marked disco | mfort related to a limb or an organ | that is removed from or is not phys | ically part of the body. | • |
| Navigational Note: - | | | | | |
| Presyncope | - | Present (e.g., near fainting) | - | - | - |
| Definition: A disorder characte | erized by an episode of lightheadedn | ess and dizziness which may preced | e an episode of syncope. | • | • |
| Navigational Note: - | - · · | | | | |
| Pyramidal tract syndrome | Asymptomatic; clinical or | Moderate symptoms; limiting | Severe symptoms; limiting self | Life-threatening | Death |
| | diagnostic observations only: | instrumental ADL | care ADL | consequences; urgent | |
| | intervention not indicated | | | intervention indicated | |
| Definition: A disorder characte | erized by dysfunction of the corticosp | inal (pyramidal) tracts of the spinal | cord. Symptoms include an increas | e in the muscle tone in the lowe | r extremities, |
| hyperreflexia, positive Babinsk | i and a decrease in fine motor coordi | nation. | • • | | |
| Navigational Note: - | | | | | |
| Radiculitis | Mild symptoms | Moderate symptoms; medical | Severe symptoms; limiting self | Life-threatening | Death |
| | | intervention indicated; | care ADL | consequences; urgent | |
| | | limiting instrumental ADL | | intervention indicated | |
| <b>Definition:</b> A disorder characte | erized by inflammation involving a ne | | <br>ed discomfort radiating along a nen | | re on the |
| <b>Definition:</b> A disorder characte connecting nerve root. | rized by inflammation involving a ne | | <br>ed discomfort radiating along a nen | | re on the |
| connecting nerve root. | | | <br>ed discomfort radiating along a nen | | re on the |
| connecting nerve root.<br>Navigational Note: - | erized by inflammation involving a ne Asymptomatic; clinical or | | ed discomfort radiating along a nen | | re on the |
| | | rve root. Patients experience mark | | e path because of spinal pressu | |
| connecting nerve root. Navigational Note: - Recurrent laryngeal nerve | Asymptomatic; clinical or | rve root. Patients experience mark | Severe symptoms; medical | e path because of spinal pressu Life-threatening | |
| connecting nerve root. Navigational Note: - Recurrent laryngeal nerve | Asymptomatic; clinical or diagnostic observations only; | rve root. Patients experience mark | Severe symptoms; medical intervention indicated (e.g., | Life-threatening consequences; urgent | |
| connecting nerve root. Navigational Note: - Recurrent laryngeal nerve palsy | Asymptomatic; clinical or diagnostic observations only; | ve root. Patients experience mark | Severe symptoms; medical intervention indicated (e.g., thyroplasty, vocal cord | Life-threatening consequences; urgent | |
| connecting nerve root. Navigational Note: - Recurrent laryngeal nerve palsy Definition: A disorder characte | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | ve root. Patients experience mark | Severe symptoms; medical intervention indicated (e.g., thyroplasty, vocal cord | Life-threatening consequences; urgent | |
| connecting nerve root. Navigational Note: - Recurrent laryngeal nerve palsy Definition: A disorder characte Navigational Note: - | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | ve root. Patients experience mark | Severe symptoms; medical intervention indicated (e.g., thyroplasty, vocal cord | Life-threatening consequences; urgent | |
| connecting nerve root. Navigational Note: - Recurrent laryngeal nerve palsy Definition: A disorder characte Navigational Note: - Reversible posterior | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | rve root. Patients experience mark | Severe symptoms; medical intervention indicated (e.g., thyroplasty, vocal cord injection) | e path because of spinal pressu<br>Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| connecting nerve root. Navigational Note: - Recurrent laryngeal nerve palsy | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms Woderate symptoms Tyngeal nerve. Moderate symptoms; limiting | Severe symptoms; medical intervention indicated (e.g., thyroplasty, vocal cord injection) Severe symptoms; limiting self | e path because of spinal pressu Life-threatening consequences; urgent intervention indicated Life-threatening | Death |
| connecting nerve root. Navigational Note: - Recurrent laryngeal nerve palsy Definition: A disorder characte Navigational Note: - Reversible posterior leukoencephalopathy syndrome | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms ryngeal nerve. Moderate symptoms; limiting instrumental ADL | Severe symptoms; medical intervention indicated (e.g., thyroplasty, vocal cord injection) Severe symptoms; limiting self care ADL; hospitalization | e path because of spinal pressu Life-threatening consequences; urgent intervention indicated Life-threatening consequences | Death |
| connecting nerve root. Navigational Note: - Recurrent laryngeal nerve palsy Definition: A disorder characte Navigational Note: - Reversible posterior leukoencephalopathy syndrome Definition: A disorder characte | Asymptomatic; clinical or diagnostic observations only; intervention not indicated erized by paralysis of the recurrent la | Moderate symptoms Moderate symptoms Moderate symptoms; limiting instrumental ADL nanges, visual disturbances, and/or | Severe symptoms; medical intervention indicated (e.g., thyroplasty, vocal cord injection) Severe symptoms; limiting self care ADL; hospitalization selzures associated with imaging fire | e path because of spinal pressu Life-threatening consequences; urgent intervention indicated Life-threatening consequences udings of posterior leukoenceph | Death Death alopathy, It |
| connecting nerve root. Navigational Note: - Recurrent laryngeal nerve palsy Definition: A disorder characte Navigational Note: - Reversible posterior leukoencephalopathy syndrome Definition: A disorder characte has been observed in associati | Asymptomatic; clinical or diagnostic observations only; intervention not indicated erized by paralysis of the recurrent la | Moderate symptoms Moderate symptoms ryngeal nerve. Moderate symptoms; limiting instrumental ADL nanges, visual disturbances, and/or y, eclampsia, and immunosuppress | Severe symptoms; medical intervention indicated (e.g., thyroplasty, vocal cord injection) Severe symptoms; limiting self care ADL; hospitalization selzures associated with imaging fire | e path because of spinal pressu Life-threatening consequences; urgent intervention indicated Life-threatening consequences udings of posterior leukoenceph | Death Death alopathy, It |
| | Nervous system disorders | | | | | |
|---|---|---|---|---|---|--|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 | |
| Seizure | Brief partial seizure and no<br>loss of consciousness | Brief generalized seizure | New onset seizures (partial or<br>generalized); multiple seizures<br>despite medical intervention | Life-threatening<br>consequences; prolonged<br>repetitive seizures | Death | |
| Definition: A disorder characteria | zed by a sudden, involuntary skelet | al muscular contractions of cerebra | or brain stem origin. | | | |
| Navigational Note: - | | | | | | |
| Somnolence | Mild but more than usual<br>drowsiness or sleepiness | Moderate sedation; limiting<br>instrumental ADL | Obtundation or stupor | Life-threatening<br>consequences; urgent<br>intervention indicated | Death | |
| Definition: A disorder characteria | zed by characterized by excessive sl | eepiness and drowsiness. | | | | |
| Navigational Note: - | | | | | | |
| Spasticity | Mild or slight increase in muscle tone | Moderate increase in muscle<br>tone and increase in<br>resistance through range of<br>motion | Severe increase in muscle<br>tone and increase in<br>resistance through range of<br>motion | Life-threatening<br>consequences; unable to<br>move active or passive range<br>of motion | Death | |
| disturbances. | zed by increased involuntary muscl | e tone that affects the regions inter | fering with voluntary movement. It | results in gait, movement, and spec | ech | |
| Navigational Note: - | | | | | | |
| Spinal cord compression | - | - | Severe symptoms; limiting self<br>care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death | |
| Definition: A disorder characteria | zed by pressure on the spinal cord. | | | | | |
| Navigational Note: - | | | | | | |
| Stroke | Incidental radiographic findings only | Mild to moderate neurologic<br>deficit; limiting instrumental<br>ADL | Severe neurologic deficit;<br>limiting self care ADL;<br>hospitalization | Life-threatening<br>consequences; urgent<br>intervention indicated | Death | |
| Definition: A disorder characteria<br>damage.<br>Navigational Note: - | red by a decrease or absence of blo | od supply to the brain caused by ob | struction (thrombosis or embolism | ) of an artery resulting in neurologi | cal | |
| Syncope | - | - | Fainting; orthostatic collapse | - | - | |
| Definition: A disorder characteria<br>Navigational Note: - | zed b <b>y</b> spontaneous loss of conscio | usness caused by insufficient blood | supply to the brain. | | ' | |
| Tendon reflex decreased | Ankle reflex reduced | Ankle reflex absent; other<br>reflexes reduced | Absence of all reflexes | - | - | |
| Definition: A disorder characteria | zed by less than normal deep tendo | n reflexes. | | | | |
| Navigational Note: Also consider | Nervous system disorders: Periphe | eral motor neuropath <b>y</b> or Periphera | l sensor <b>y</b> neuropath <b>y</b> | | | |

| | | Nervous system disord | ers | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Transient ischemic attacks | Mild neurologic deficit with or | Moderate neurologic deficit | - | - | - |
| | without imaging confirmation | with or without imaging | | | |
| | | confirmation | | | |
| | rized by a brief attack (less than 24 h<br>s. Consider Nervous system disorders | | scular origin, with no persistent neu | rological deficit. | |
| Tremor | Mild symptoms | Moderate symptoms; limiting | Severe symptoms; limiting self | I - | - I |
| Tremor | 14ma symptoms | instrumental ADL | care ADL | | |
| Definition: A disorder characte | rized by the uncontrolled shaking mo | • | · | ' | 1 |
| Navigational Note: - | a ized by the discord offed shaking int | overner cor are writte body or mark | iduai pai is. | | |
| Trigeminal nerve disorder | Asymptomatic; clinical or | Moderate symptoms; limiting | Severe symptoms; limiting self | Ι. | Τ. |
| ringerminal rich ve disorder | diagnostic observations only: | instrumental ADL | care ADL | | |
| | intervention not indicated | Iliad difficilital ADE | Carcabe | | |
| Definition: A disarder electrosta | rized by dysfunction of the trigemina | I nonce (fifth granial name) | I . | 1 | J |
| Navigational Note: - | erized by dysiunction of the trigernina | ii nerve (iii in craniai nerve). | | | |
| Trochlear nerve disorder | Asymptomatic; clinical or | Moderate symptoms; limiting | Severe symptoms; limiting self | ı | |
| Trodilear Herve disorder | diagnostic observations only; | instrumental ADL | care ADI | l <sup>-</sup> | - |
| | intervention not indicated | instrumental ADL | Care ADL | | |
| B. C. St A. P In In | l . | <br> | I | ı | I |
| | rized by dysfunction of the trochlear | nerve (fourth cranial nerve). | | | |
| Navigational Note: - | T | Landa de la companya | T | Lugar | 1 8 3 |
| Vagus nerve disorder | Asymptomatic; clinical or | Moderate symptoms; limiting | Severe symptoms; limiting self | Life-threatening | Death |
| | diagnostic observations only; | instrumental ADL | care ADL | consequences; urgent | |
| | intervention not indicated | l | | intervention indicated | |
| | erized by dysfunction of the vagus ner | ve (tenth cranial nerve). | | | |
| Navigational Note: - | | | | | |
| Vasovagal reaction | - | - | Present | Life-threatening | Death |
| | | | | consequences; urgent | |
| | | 1 | | intervention indicated | |
| | rized b <b>y</b> a sudden drop of the blood | pressure, bradycardia, and periphe | ral vasodilation that may lead to los | s of consciousness. It results fro | om an increase |
| in the stimulation of the vagus | nerve. | | | | |
| Navigational Note: - | _ | | | | |
| Nervous system disorders - | Asymptomatic or mild | Moderate; minimal, local or | Severe or medically significant | Life-threatening | Death |
| Other, specify | symptoms; clinical or | noninvasive intervention | but not immediately life- | consequences; urgent | |
| | diagnostic observations only; | indicated; limiting age- | threatening; hospitalization or | intervention indicated | |
| | intervention not indicated | appropriate instrumental ADL | prolongation of existing | l | |
| | | | hospitalization indicated; | | |
| | | I | limiting self care ADL | l | |
| Definition: - | | | | | |
| Navigational Note: - | | | | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Pregnancy, puerperium and perina | tal conditions | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Fetal growth retardation | - | <10% percentile of weight for<br>gestational age | <5% percentile of weight for<br>gestational age | <1% percentile of weight for<br>gestational age | - |
| Definition: A disorder character | ized by inhibition of fetal growth res | sulting in the inability of the fetus to | achieve its potential weight. | | |
| Navigational Note: - | | | | | |
| Pregnancy loss | - | - | - | Fetal loss at any gestational age | - |
| Definition: Death in utero. | | - | | | |
| Navigational Note: - | | | | | |
| Premature delivery | Delivery of a liveborn infant at<br>>34 to 37 weeks gestation | Delivery of a liveborn infant at<br>>28 to 34 weeks gestation | Delivery of a liveborn infant at<br>24 to 28 weeks gestation | Delivery of a liveborn infant at<br>24 weeks of gestation or less | - |
| <b>Definition:</b> A disorder character gestation. | ized by delivery of a viable infant be | fore the normal end of gestation. T | ypically, viability is achievable betw | een the twentieth and thirty-sever | th week of |
| Navigational Note: - | | | | | |
| Pregnancy, puerperium and<br>perinatal conditions - Other,<br>specify | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: - | | - | | | |
| Navigational Note: - | | | | | |

| CTCAE Term | | | 5 | | |
|---|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade ! |
| gitation | Mild mood alteration | Moderate mood alteration | Severe agitation;<br>hospitalization not indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | - |
| Pefinition: A disorder charact<br>Javigational Note: - | erized by a state of restlessness assoc | iated with unpleasant feelings of ir | ritability and tension. | | |
| norgasmia | Inability to achieve orgasm<br>not adversely affecting<br>relationship | Inability to achieve orgasm<br>adversely affecting<br>relationship | - | - | - |
| Definition: A disorder charact<br>Navigational Note: - | erized by an inability to achieve orgas | m. | | | |
| nxiety | Mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self<br>care ADL; hospitalization<br>indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | - |
| Definition: A disorder charact<br>Javigational Note: - | erized by apprehension of danger and | l dread accompanied by restlessnes | ss, tension, tachycardia, and dyspne | a unattached to a clearly identifiabl | le stimulus |
| Confusion | Mild disorientation | Moderate disorientation;<br>limiting instrumental ADL | Severe disorientation; limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | - |
| Definition: A disonder charact<br>Navigational Note: - | erized by a lack of clear and orderly th | nought and behavior. | | • | • |
| elayed orgasm | Delay in achieving orgasm not<br>adversely affecting<br>relationship | Delay in achieving orgasm<br>adversely affecting<br>relationship | - | - | - |
| Definition: A disorder charact<br>Navigational Note: - | erized by sexual dysfunction characte | rized by a delay in dimax. | | • | • |
| elirium | Mild acute confusional state | Moderate and acute confusional state; limiting instrumental ADL | Severe and acute confusional<br>state; limiting self care ADL;<br>urgent intervention indicated;<br>new onset | Life-threatening<br>consequences, threats of<br>harm to self or others; urgent<br>intervention indicated | Death |
| Definition: A disorder charact<br>eversible condition.<br>lavigational Note: - | erized by the acute and sudden devel | opment of confusion, illusions, mov | vement changes, inattentiveness, ag | itation, and hallucinations. Usuall <b>y</b> , | itisa |
| elusions | - | Moderate delusional<br>symptoms | Severe delusional symptoms;<br>hospitalization not indicated;<br>new onset | Life-threatening<br>consequences, threats of<br>harm to self or others: | Death |

| | | Psychiatric disorder | 's | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Depression | Mild depressive symptoms | Moderate depressive | Severe depressive symptoms; | Life-threatening | Death |
| | | symptoms; limiting | limiting self care ADL; | consequences, threats of | |
| | | instrumental ADL | hospitalization not indicated | harm to self or others; | |
| | | 1 | | hospitalization indicated | |
| | terized b <b>y</b> melancholic feelings of grie | f or unhappiness. | | | |
| Navigational Note: - | | | | | _ |
| Euphoria | Mild mood elevation | Moderate mood elevation | Severe mood elevation (e.g., | = | - |
| | | I | hypomania) | I | I |
| | terized by an exaggerated feeling of w | ell-being which is disproportionate | e to events and stimuli. | | |
| Navigational Note: - | | | 1 | | |
| Hallucinations | Mild hallucinations (e.g., | Moderate hallucinations | Severe hallucinations; | Life-threatening | Death |
| | perceptual distortions) | | hospitalization not indicated | consequences, threats of | |
| | | | | harm to self or others;<br>hospitalization indicated | |
| Definite and Advanced an element | <br>terized by a false sensory perception i | <br> | 1 | nospitalization indicated | I |
| | terized by a raise sensory perception i | n the absence of an external sumul | ius. | | |
| Navigational Note: - | Battal difficulty fulling and and | N 4 | Course difficulty to follow | | 1 |
| Insomnia | Mild difficulty falling asleep,<br>staying asleep or waking up | Moderate difficulty falling<br>asleep, staying asleep or | Severe difficulty in falling<br>asleep, staying asleep or | - | |
| | early | waking up early | waking up early | | |
| Definition: A disorder charact | terized by difficulty in falling asleep an | | and the ap carry | 1 | ı |
| Navigational Note: - | terized by difficulty in failing asieep ar | фоттентантів азгеер. | | | |
| Irritability | Mild; easily consolable | Moderate; limiting | Severe abnormal or excessive | - | - |
| | ,, | instrumental ADL: increased | response; limiting self care | | |
| | | attention indicated | ADL; inconsolable; medical or | | |
| | | | psychiatric intervention | | |
| | | | indicated | | |
| Definition: A disorder charac | terized b <b>y</b> an abnormal responsivenes | s to stimuli or physiological arousal | l; may be in response to pain, fright, | a drug, an emotional situation or | a medical |
| condition. | | | | | |
| Navigational Note: - | | | | | |
| Libido decreased | Decrease in sexual interest | Decrease in sexual interest | - | - | - |
| | not adversely affecting | adversely affecting | | | 1 |
| | relationship | relationship | 1 | I | 1 |
| | terized by a decrease in sexual desire. | | | | |
| Navigational Note: - | | | | | |
| Libido increased | Present | - | <del>-</del> | - | - |
| <b>Definition:</b> A disorder charac | terized by an increase in sexual desire | | | | |
| Navigational Note: - | | | | | |

CTCAE v5.0 – November 27, 2017 Back to TOC


| | | Psychiatric disorders | s | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Mania | Mild manic symptoms (e.g.,<br>elevated mood, rapid<br>thoughts, rapid speech,<br>decreased need for sleep) | Moderate manic symptoms<br>(e.g., relationship and work<br>difficulties; poor hygiene) | Severe manic symptoms (e.g.,<br>hypomania; major sexual or<br>financial indiscretions);<br>hospitalization not indicated;<br>new onset | Life-threatening<br>consequences, threats of<br>harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder chara | acterized by excitement of psychotic pro | pportions manifested by mental and | I physical hyperactivity, disorganizat | ion of behavior and elevation of m | ood. |
| Navigational Note: - | | | | | |
| Personality change | Mild personality change | Moderate personality change | Severe personality change;<br>hospitalization not indicated | Life-threatening<br>consequences, threats of<br>harm to self or others;<br>hospitalization indicated | - |
| | acterized by a conspicuous change in a p | person's behavior and thinking. | | | |
| Navigational Note: - | | | | | |
| Psychosis | Mild psychotic symptoms | Moderate psychotic<br>symptoms (e.g., disorganized<br>speech; impaired reality<br>testing) | Severe psychotic symptoms<br>(e.g., paranolid, extreme<br>disorganization);<br>hospitalization not indicated;<br>new onset | Life-threatening<br>consequences, threats of<br>harm to self or others;<br>hospitalization indicated | Death |
| <b>Definition:</b> A disorder chara<br>tumor.<br><b>Navigational Note:</b> - | acterized by personality change, impaire | d functioning, and loss of touch wit | h reality. It may be a manifestation | of schizophrenia, bipolar disorder ( | or brain |
| Restlessness | Mild symptoms; intervention<br>not indicated | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL | - | - |
| Definition: A disorder chara | acterized by an inability to rest, relax or | be still. | • | • | • |
| Navigational Note: - | | | | | |
| Suicidal ideation | Increased thoughts of death<br>but no wish to kill oneself | Suicidal ideation with no<br>specific plan or intent | Specific plan to commit<br>suicide without serious intent<br>to die which may not require<br>hospitalization | Specific plan to commit<br>suicide with serious intent to<br>die which requires<br>hospitalization | - |
| Definition: A disorder chara | acterized by thoughts of taking one's ow | n life. | | | |
| Navigational Note: - | | | | | |
| Navigational Note, - | | | Suicide attempt or gesture | Suicide attempt with intent to | Death |
| Suicide attempt | - | | without intent to die | die which requires<br>hospitalization | |
| Suicide attempt | -<br>acterized by self-inflicted harm in an att | empt to end one's own life. | | die which requires | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| Psychiatric disorders | | | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Psychlatric disorders - Other,<br>specify | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; limiting self care<br>ADL | Life-threatening<br>consequences; hospitalization<br>or urgent intervention<br>indicated | Death |
| Definition: - | | | | | |
| Navigational Note: - | | | | | |

| Renal and urinary disorders | | | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Acute kidney injury | - | - | Hospitalization indicated | Life-threatening<br>consequences; dialysis<br>indicated | Death |
| Definition: A disorder characteri: | zed by the acute loss of renal functi | on (within 2 weeks) and is tradition | ally classified as pre-renal (low bloo | od flow into kidney), renal (kidney d | amage) |
| and post-renal causes (ureteral c | r bladder outflow obstruction). | | | | |
| Navigational Note: Also consider | Investigations: Creatinine increase | d | | | |
| Bladder perforation | - | Invasive intervention not indicated | Invasive intervention indicated | Life-threatening<br>consequences; organ failure;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characteri: | zed b <b>y</b> a rupture in the bladder wall | | | | |
| Navigational Note: - | | | | | |
| Bladder spasm | Intervention not indicated | Antispasmodics indicated | Hospitalization indicated | - | - |
| <b>Definition:</b> A disorder characteri: | zed by a sudden and involuntary co | ntraction of the bladder wall. | | | |
| Navigational Note: - | | | | | |
| Chronic kidney disease | eGFR (estimated Glomerular Filtration Rate) or CrCl (creatinine clearance) <lln -="" 1.73="" 2+="" 60="" creatinine="" m2="" min="" ml="" or="" present;="" protein="" proteinuria="" urine="">0.5 ted by gradual and usually permanezed</lln> | eGFR or CrCl 59 - 30<br>ml/min/1.73 m2 | eGFR or CrCl 29 - 15<br>ml/min/1.73 m2 | eGFR or CrCl <15 ml/min/1.73<br>m2; dialysis or renal<br>transplant indicated | Death |
| | zed by gradual and usually permane | ent loss of klaney function resulting | in renai failure. | | |
| Navigational Note: - Cystitis noninfective | Microscopic hematuria; | Moderate hematuria: | Gross hematuria; transfusion, | Life-threatening | Death |
| Cysaus Ioninective | minimal increase in<br>frequency, urgency, dysuria,<br>or nocturia; new onset of<br>incontinence | moderate increase in<br>frequency, urgency, dysuria,<br>nocturia or incontinence;<br>urinary catheter placement or<br>bladder irrigation indicated;<br>limiting instrumental ADL | IV medications, or<br>hospitalization indicated;<br>elective invasive intervention<br>indicated | consequences; urgent invasive intervention indicated | Beauti |
| Definition: A disorder characteri: | zed b <b>y</b> inflammation of the bladder | which is not caused by an infection | of the urinary tract. | | |
| Navigational Note: - | | | | | |
| Dysuria | Present | - | - | - | - |
| Definition: A disorder characteri | zed b <b>y</b> painful urination. | | | | |
| Navigational Note: If associated<br>Infections and infestations: Urina | | on. For grades higher than Grade 1, | . consider Renal and urinary disord | ers: Bladder spasm or Cystitis nonin | fective; |

| Renal and urinary disorders | | | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Glucosuria | Present | - | - | - | - |
| Definition: A disorder characteri | zed by laboratory test results that in | ndicate glucose in the urine. | | | ' |
| Navigational Note: - | | | | | |
| Hematuria | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; urinary catheter<br>or bladder irrigation indicated;<br>limiting instrumental ADL | Gross hematuria; transfusion,<br>IV medications, or<br>hospitalization indicated;<br>elective invasive intervention<br>indicated; limiting self care<br>ADL | Life-threatening<br>consequences; urgent invasive<br>intervention indicated | Death |
| Definition: A disorder characteri | zed by laboratory test results that in | ndicate blood in the urine. | | | |
| Navigational Note: - | | | | | |
| Hemoglobinuria | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | - | - | - | - |
| Definition: A disorder characteri | zed by laboratory test results that in | ndicate the presence of free hemog | lobin in the urine. | • | ' |
| Navigational Note: Report under | rlying AE if > Grade 1 | _ | | | |
| Nephrotic syndrome | - | - | Not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder characteri | zed by symptoms that include sever | re edema, proteinuria, and hypoalb | uminemia; it is indicative of renal d | ysfunction. | ' |
| Navigational Note: - | | | | | |
| Proteinuria | 1+ proteinuria; urinary protein<br>≥ULN -<1.0 g/24 hrs | Adult: 2+ and 3+ proteinuria;<br>urinary protein 1.0 - <3.5 g/24<br>hrs; | Adult: Urinary protein >= 3.5<br>g/24 hrs; 4+ proteinuria;<br>Pediatric: Urine P/C | - | - |
| | | Pediatric: Urine P/C<br>(Protein/Creatinine) ratio 0.5 -<br>1.9 | (Protein/Creatinine) ratio >1.9 | | |
| Definition: A disorder characteri | zed by laboratory test results that ir | ndicate the presence of excessive p | rotein in the urine. It is predominar | ntly albumin, but also globulin. | |
| Navigational Note: 24-hour uring | e collection takes precedence over ( | dipstick | | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| c; oral antiemetics c; oral antiemetics ound the clock tion analgesics or cotic analgesics the pelvis of the kid ain; limiting I ADL; medication mfort radiating to the | intervention (e.g., analgesics,<br>antiemetics); elective invasive<br>intervention indicated | Grade 4 Life-threatening consequences; urgent invasive intervention indicated | Grade 5 Death |
|---|---|---|---|
| ound the clock tion analgesics or cotic analgesics the pelvis of the kid ain; limiting I ADL; medication | intervention (e.g., analgesics, antiemetics); elective invasive intervention indicated intervention indicated; | consequences; urgent invasive | Death |
| ain; limiting<br>il ADL;<br>medication | Hospitalization indicated; | <u> </u> | |
| l ADL;<br>medication | | T - | |
| l ADL;<br>medication | | - | |
| nfort radiating to th | | | - |
| | he inguinal area. Often, the cause is | is the passage of crystals/kidney stone | es. |
| nd hematocrit<br>Indicated | Transfusion indicated;<br>invasive intervention<br>indicated; hospitalization | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | • | • | • |
| c, invasive<br>not indicated | Invasive intervention indicated | Life-threatening<br>consequences; urgent invasive<br>intervention indicated | Death |
| part of the urinary | system and another organ or anato | omic site. | • |
| rumental ADL;<br>nagement | - | - | - |
| s; pads indicated; | Intervention indicated (e.g., clamp, collagen injections); operative intervention indicated; limiting self care ADL | | = |
| r | rumental ADL<br>he bladder. | operative intervention indicated; limiting self care ADL | operative intervention<br>indicated; limiting self care<br>ADL |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Renal and urinary disor | ders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Urinary retention | Urinary, suprapubic or<br>intermittent catheter<br>placement not indicated; able<br>to void with some residual | Placement of urinary,<br>suprapubic or intermittent<br>catheter placement indicated;<br>medication indicated | Elective invasive intervention<br>indicated; substantial loss of<br>affected kidney function or<br>mass | Life-threatening<br>consequences; organ failure;<br>urgent operative intervention<br>indicated | Death |
| <b>Definition:</b> A disorder characte | rized by accumulation of urine within | n the bladder because of the inabili | ty to urinate. | | |
| Navigational Note: - | | | | | |
| Urinary tract obstruction | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic but no<br>hydronephrosis, sepsis, or<br>renal dysfunction; urethral<br>dilation, urinary or suprapubic<br>catheter indicated | Altered organ function (e.g.,<br>hydronephrosis or renal<br>dysfunction); invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder character<br><b>Navigational Note:</b> - | rized by blockage of the normal flow | of contents of the urinary tract. | | | |
| Urinary tract pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characte | erized by a sensation of marked disco | mfort in the urinary tract. | | | |
| Navigational Note: - | | | | | |
| Urinary urgency | Present | Limiting instrumental ADL;<br>medical management<br>indicated | - | - | - |
| Definition: A disorder characte | rized by a sudden compelling urge to | urinate. | | • | |
| Navigational Note: - | | | | | |
| Urine discoloration | Present | - | = | - | - |
| Definition: A disorder characte | erized by a change in the color of the | urine. | • | • | • |
| Navigational Note: - | | | | | |
| Renal and urinary disorders -<br>Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: - | | | | | |
| Navigational Note: - | | | | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| Reproductive system and breast disorders | | | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Amenorrhea | - | Present | - | - | - |
| Definition: A disorder characteri: | zed b <b>y</b> the abnormal absence of me | enses for at least three consecutive | menstrual cycles. | • | |
| Navigational Note: - | | | | | |
| Azoospermia | - | Absence of sperm in ejaculate | - | - | - |
| Definition: A disorder characteri: | zed by laboratory test results that i | ndicate complete absence of sperm | atozoa in the semen. | | |
| Navigational Note: - | | | | | |
| Breast atrophy | Minimal asymmetry; minimal | Moderate asymmetry; | Asymmetry >1/3 of breast | - | - |
| | atroph <b>y</b> | moderate atrophy | volume; severe atrophy | l | |
| | zed b <b>y</b> underdevelopment of the br | east. | | | |
| Navigational Note: - | | | | | |
| Breast pain | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | - | - |
| | | instrumental ADL | ADL | I | |
| | zed by a sensation of marked discor | mfort in the breast region. | | | |
| Navigational Note: - | Lager to the second | L | | ı | |
| Dysmenorrhea | Mild symptoms; intervention<br>not indicated | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL | l - | - |
| Definition: A disorder characteri | zed by abnormally painful abdomin | • | Care ADL | 1 | |
| Navigational Note: - | zed by abilionnally painful abdomin | ar cramps during menses. | | | |
| Dyspareunia | Mild discomfort or pain | Moderate discomfort or pain | Severe discomfort or pain | l - | - |
| D / 0 P G 1 C G 1 1 G | associated with vaginal | associated with vaginal | associated with vaginal | | |
| | penetration; discomfort | penetration; discomfort or | penetration; discomfort or | | |
| | relieved with use of vaginal | pain partially relieved with | pain unrelieved by vaginal | | |
| | lubricants or estrogen | use of vaginal lubricants or | lubricants or estrogen | | |
| | | estrogen | | l | |
| <b>Definition:</b> A disorder characteri: | zed b <b>y</b> painful or difficult coitus. | | | | |
| Navigational Note: - | | | | | |
| Ejaculation disorder | Diminished ejaculation | Anejaculation or retrograde | - | - | - |
| | l | ejaculation | l | ! | |
| | zed b <b>y</b> problems related to ejaculat | ion. This category includes premat. | ire, delayed, retrograde and paintu | l ejaculation. | |
| Navigational Note: - | | | | | |

| | | Reproductive system and breas | st disorders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Erectile dysfunction | Decrease in erectile function<br>(frequency or rigidity of<br>erections) but intervention<br>not indicated (e.g., medication<br>or use of mechanical device,<br>penile pump) | Decrease in erectile function<br>(frequency/rigidity of<br>erections), erectile<br>intervention indicated, (e.g.,<br>medication or mechanical<br>devices such as penile pump) | Decrease in erectile function<br>(frequency/rigidity of<br>erections) but erectile<br>intervention not helpful (e.g.,<br>medication or mechanical<br>devices such as penile pump);<br>placement of a permanent<br>penile prosthesis indicated<br>(not previously present) | - | - |
| Definition: A disorder character | rized by the persistent or recurrent i | nability to achieve or to maintain a | n erection during sexual activity. | • | · · |
| Navigational Note: - | | | | | |
| Fallopian tube obstruction | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; elective<br>intervention indicated | Severe symptoms; invasive<br>intervention indicated | - | - |
| Definition: A disorder character | ized by blockage of the normal flow | of the contents in the fallopian tub | e. | • | • |
| Navigational Note: - | | | | | |
| Feminization acquired | Mild symptoms; intervention<br>not indicated | Moderate symptoms; medical<br>intervention indicated | - | - | = |
| Definition: A disorder character | rized by the development of seconda | ary female sex characteristics in ma | les due to extrinsic factors. | | |
| Navigational Note: - | | | | | |
| Genital edema | Mild swelling or obscuration<br>of anatomic architecture on<br>close inspection | Readily apparent obscuration<br>of anatomic architecture;<br>obliteration of skin folds;<br>readily apparent deviation<br>from normal anatomic<br>contour | Lymphorrhea; gross deviation<br>from normal anatomic<br>contour; limiting self care ADL | - | - |
| <b>Definition:</b> A disorder character <b>Navigational Note:</b> - | rized by swelling due to an excessive | accumulation of fluid in the genita | is. | | |
| Gynecomastia | Asymptomatic | Symptomatic (e.g., pain or<br>psychosocial impact) | Severe symptoms; elective<br>operative intervention<br>indicated | - | - |
| Definition: A disorder characte | ized by excessive development of th | e breasts in males. | • | • | • |
| Navigational Note: - | | | | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Reproductive system and breas | st disorders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Hematosalpin <b>x</b> | Minimal bleeding identified | Moderate bleeding; medical | Transfusion indicated; | Life-threatening | Death |
| | on imaging study or | intervention indicated | invasive intervention | consequences; urgent | |
| | laparoscopy; intervention not | | indicated | operative intervention | |
| | indicated | | | indicated | |
| <b>Definition:</b> A disorder characte | rized by the presence of blood in a f | allopian tube. | | | |
| Navigational Note: - | | | | | |
| Irregular menstruation | Intermittent/irregular menses | Intermittent/irregular menses | - | - | - |
| | for no more than 3 | for more than 3 consecutive | | | |
| | consecutive menstrual cycles | menstrual cycles | | | |
| Definition: A disorder characte | rized by a change in cycle or duratio | n of menses from baseline. | • | • | • |
| | ler Reproductive system and breast o | | menorrhea. | | |
| Lactation disorder | Mild changes in lactation, not | Changes in lactation, | - | - | - |
| | significantly affecting | significantly affecting breast | | | |
| | production or expression of | production or expression of | | | |
| | breast milk | breast milk | | | |
| Definition: A disorder characte | rized by disturbances of milk secreti | on. It is not necessarily related to pr | egnancy that is observed in female | s and can be observed in males. | |
| Navigational Note: - | · | , | -3 | | |
| Menorrhagia | Mild; iron supplements | Moderate symptoms; medical | Severe; transfusion indicated; | Life-threatening | Death |
| _ | indicated | intervention indicated (e.g., | operative intervention | consequences; urgent | |
| | | hormones) | indicated (e.g., hysterectomy) | intervention indicated | |
| Definition: A disorder characte | rized by abnormally heavy vaginal bl | eeding during menses. | | • | • |
| Navigational Note: - | | 3 3 | | | |
| Nipple deformity | Asymptomatic; asymmetry | Symptomatic; asymmetry of | - | - | - |
| | with slight retraction and/or | nipple areolar complex with | | | |
| | thickening of the nipple | moderate retraction and/or | | | |
| | areolar complex | thickening of the nipple | | | |
| | | areolar complex | | | |
| Definition: A disorder characte | rized by a malformation of the nippl | e. | • | • | • |
| Navigational Note: - | , | | | | |
| Oligospermia | Sperm concentration > 0 to < | - | - | - | - |
| 3 . | 15 million/ml | | | | |
| Definition: A disorder characte | rized by a decrease in the number o | f snermatozoa in the semen | 1 | • | |
| Navigational Note: - | in zod by a dobi edec in a le namber b | op a mateza a m ano coma n | | | |
| Ovarian hemorrhage | Mild symptoms; intervention | Moderate symptoms: | Transfusion indicated: | Life-threatening | Death |
| o tarrarricano mage | not indicated | intervention indicated | invasive intervention | consequences; urgent | Dead |
| | not maicacca | intervention in lateated | indicated; hospitalization | intervention indicated | |
| Definition & discorder 1 | <br> | ı | murcateu, nospitanzauon | I intervendon murated | I |
| | rized by bleeding from the ovary. | | | | |
| Navigational Note: - | | | | | |

| | | Reproductive system and breas | t disorders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Ovarian rupture | Asymptomatic clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic and intervention<br>not indicated | Transfusion; invasive intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder character | ized by tearing or disruption of the | ovarian tissue. | | | |
| Navigational Note: - | | | | | |
| Ovulation pain | - | Present | - | - | - |
| <b>Definition:</b> A disorder character ovarian follicle. | ized by a sensation of marked disco | mfort in one side of the abdomen b | etween menstrual cycles, around t | he time of the discharge of the ov | um from the |
| Navigational Note: - | | | | | |
| Pelvic floor muscle weakness | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic, not interfering<br>with bladder, bowel, or<br>vaginal function; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL | - | - |
| Definition: A disorder character | ized by a reduction in the strength o | of the muscles of the pelvic floor. | | | |
| Navigational Note: - | | | | | |
| Pelvic pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder character | ized b <b>y</b> a sensation of marked disco | mfort in the pelvis. | | • | • |
| Navigational Note: - | | | | | |
| Penile pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder character | ized by a sensation of marked disco | mfort in the penis. | ' | • | · |
| Navigational Note: - | • | | | | |
| Perineal pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder character | ized by a sensation of marked disco | mfort in the area between the geni | tal organs and the anus. | • | • |
| Navigational Note: - | | | | | |
| Premature menopause | - | Present | - | - | - |
| | ized by premature ovarian failure. S<br>mone (LH) and follicle-stimulating h | | night sweats, mood swings, and a d | ecrease in sex drive. Laboratory f | ndings |
| Navigational Note: - | | | | | |
| Prostatic hemorrhage | Mild symptoms; intervention not indicated | Moderate symptoms;<br>intervention indicated | Transfusion indicated;<br>invasive intervention<br>indicated; hospitalization | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder character | ized by bleeding from the prostate ( | sland. | • | • | • |
| Navigational Note: - | | _ | | | |

| | | Reproductive system and bre | ast disorders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Prostatic obstruction | Asymptomatic; clinical or | Symptomatic; elective | Severe symptoms; invasive | - | - |
| | diagnostic observations only; | intervention indicated | intervention indicated | | |
| | intervention not indicated | 1 | 1 | I | |
| | | secondary to enlargement of the | prostate gland. This results in voiding | g difficulties (straining to void, sk | ow urine |
| stream, and incomplete emptyi | ng of the bladder). | | | | |
| Navigational Note: - | Lami | T | T | | |
| Prostatic pain | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | - | - |
| | 1 | instrumental ADL | ADL | I | J |
| | ized by a sensation of marked disco | omfort in the prostate gland. | | | |
| Navigational Note: - | T | | T | | |
| Scrotal pain | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | - | - |
| | 1 | instrumental ADL | ADL | I | |
| | ized b <b>y</b> a sensation of marked disco | omfort in the scrotal area. | | | |
| Navigational Note: - | T | | | | |
| Spermatic cord hemorrhage | Mild symptoms; intervention | Moderate symptoms; | Transfusion indicated; | Life-threatening | Death |
| | not indicated | intervention indicated | invasive intervention | consequences; urgent | |
| | 1 | 1 | indicated; hospitalization | intervention indicated | |
| | ized by bleeding from the spermati | c cord. | | | |
| Navigational Note: - | | | _ | | |
| Spermatic cord obstruction | Asymptomatic; clinical or | Symptomatic, elective | Severe symptoms; invasive | - | - |
| | diagnostic observations only; | intervention indicated | intervention indicated | | |
| magnetic and the second | intervention not indicated | 1 | 1 | ı | |
| | ized by blockage of the normal flow | or the contents of the spermatic | cora. | | |
| Navigational Note: - | T | | 1- | Luci | |
| Testicular disorder | Asymptomatic; clinical or | Symptomatic but not | Severe symptoms; interfering | Life-threatening | - |
| | diagnostic observations only;<br>intervention not indicated | interfering with sexual | with sexual function; limiting | consequences; urgent | |
| | Intervention not indicated | function; intervention not | self care ADL; intervention indicated | intervention indicated | |
| | | indicated; limiting<br>instrumental ADL | Indicated | | |
| Definition Advanded house | l<br>ized by abnormal function or appea | • | 1 | I | I |
| | | | AE terms in the Renal and urinary di | carders SOC or Reproductive syst | am and breast |
| disorders SOC. | inteproductive system and breast | disorders. Gerillar ederria or ourier | AL terms in the items and drinking dr | solders 300 of Reproductive syst | cerri ariu bi east |
| Testicular hemorrhage | Mild symptoms; intervention | Moderate symptoms; | Transfusion indicated: | Life-threatening | Death |
| resussiai ricinormage | not indicated | intervention indicated | invasive intervention | consequences; urgent | DCGGT |
| | The markets a | co. ro. ia o i larea coa | indicated; hospitalization | intervention indicated | |
| Definition: A disorder character | ized by bleeding from the testis. | • | 1 | | ı |
| Navigational Note: - | iza z y z iza z i o i i dio costa. | | | | |
| ivavigational ivote: - | | | | | |

CTCAE v5.0 – November 27, 2017 Back to TOC


**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Reproductive system and breas | st disorders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Testicular pain | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | - | - |
| | 1 | instrumental ADL | ADL | 1 | 1 |
| Definition: A disorder charact | erized by a sensation of marked disco | mfort in the testis. | | | |
| Navigational Note: - | | | | | |
| Uterine fistula | Asymptomatic | Symptomatic, invasive | Invasive intervention | Life-threatening | Death |
| | | intervention not indicated | indicated | consequences; urgent<br>intervention indicated | |
| Definition: A disaudar days at | I<br>terized by an abnormal communication | I | I | Intervention indicated | į |
| Navigational Note: - | enzeu by an abnormal communication | in petween the aterus and another | bigan or anatomic site. | | |
| Uterine hemorrhage | Mild symptoms; intervention | Moderate symptoms; | Transfusion indicated: | Life-threatening | Death |
| Otermenemonnage | not indicated | intervention indicated | invasive intervention | consequences; urgent | Deau |
| | not indicated | intervention indicated | indicated; hospitalization | intervention indicated | |
| Definition: A disorder charact | terized by bleeding from the uterus. | • | marcacca, mospitanzacom | I III Col Vollador I II la cacca | 1 |
| Navigational Note: - | terized by breeding from the decide. | | | | |
| Uterine obstruction | Asymptomatic: clinical or | Symptomatic: elective | Severe symptoms; invasive | - | - |
| | diagnostic observations only; | intervention indicated | intervention indicated | | |
| | intervention not indicated | | | | |
| Definition: A disorder charact | terized by blockage of the uterine out | et. | • | • | • |
| Navigational Note: - | | | | | |
| Uterine pain | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | - | - |
| | | instrumental ADL | ADL | 1 | |
| Definition: A disorder charact | terized by a sensation of marked disco | mfort in the uterus. | | | |
| Navigational Note: - | | | | | |
| Vaginal discharge | Mild vaginal discharge | Moderate to heavy vaginal | - | - | - |
| | (greater than baseline for | discharge; use of perineal pad | | | |
| | patient) | or tampon indicated | | 1 | 1 |
| Definition: A disorder charact | erized by vaginal secretions. Mucus p | roduced by the cervical glands is dis | scharged from the vagina naturally, | especially during the childbear | ing years. |
| Navigational Note: - | | | | | |
| Vaginal dryness | Mild vaginal dryness not | Moderate vaginal dryness | Severe vaginal dryness | - | - |
| | interfering with sexual | interfering with sexual | resulting in dyspareunia or | | 1 |
| | function | function or causing frequent | severe discomfort | | 1 |
| | ĺ | discomfort | 1 | | 1 |
| | terized b <b>y</b> an uncomfortable feeling of | itching and burning in the vagina. | | | |
| Navigational Note: - | | | | | |

| Reproductive system and breast disorders | | | | |
|---|---|---|---|---|
| Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Asymptomatic | Symptomatic, invasive<br>intervention not indicated | Invasive intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| cterized by an abnormal communicatio | n between the vagina and another | organ or anatomic site. | | |
| Mild symptoms; intervention not indicated | Moderate symptoms;<br>intervention indicated | Transfusion indicated;<br>invasive intervention<br>indicated; hospitalization | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| cterized by bleeding from the vagina. | • | | | |
| Mild discomfort or pain, edema, or redness | Moderate discomfort or pain,<br>edema, or redness; limiting<br>instrumental ADL | Severe discomfort or pain,<br>edema, or redness; limiting<br>self care ADL; small areas of<br>mucosal ulceration | Life-threatening<br>consequences; widespread<br>areas of mucosal ulceration;<br>urgent intervention indicated | - |
| cterized by inflammation involving the | vagina. Symptoms may include redi | ness, edema, marked discomfort ar | nd an increase in vaginal discharge. | |
| Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; elective intervention indicated | Severe symptoms; invasive intervention indicated | - | - |
| cterized by blockage of vaginal canal. | | | | |
| Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| cterized by a sensation of marked disco | mfort in the vagina. | | • | |
| - | Invasive intervention not<br>indicated | Invasive intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| cterized by a rupture in the vaginal wal | i. | • | • | |
| Asymptomatic; mild vaginal shortening or narrowing | Vaginal narrowing and/or<br>shortening not interfering<br>with physical examination | Vaginal narrowing and/or<br>shortening interfering with<br>the use of tampons, sexual<br>activity or physical | - | Death |
| | Asymptomatic Mild symptoms; intervention not indicated cerized by bleeding from the vagina. Mild discomfort or pain, edema, or redness ceterized by inflammation involving the diagnostic observations only; intervention not indicated ceterized by blockage of vaginal canal. Mild pain Mild pain ceterized by a sensation of marked discompany in the diagnostic observations only; intervention not indicated ceterized by a sensation of marked discompany in the d | Asymptomatic Symptomatic Invasive Intervention not indicated | Asymptomatic Symptomatic, invasive intervention indicated intervention pot indicated intervention pot indicated intervention indicated intervention indicated intervention pot indicated invasive intervention indicated; hospitalization indicated invasive intervention indicated indic | Asymptomatic Symptomatic, invasive intervention not indicated indicated indicated intervention not indicated intervention not indicated indicated intervention indicated; invasive intervention indicated; invasive intervention indicated intervention indicated; invasive intervention indicated interve |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | Reproductive system and breast disorders | | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Reproductive system and<br>breast disorders - Other,<br>specify | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: - | | | | | |
| Navigational Note: - | | | | | |

| | Respiratory, thoracic and mediastinal disorders | | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Adult respiratory distress | - | - | Present with radiologic | Life-threatening respiratory or | Death |
| syndrome | | | findings; intubation not | hemodynamic compromise; | |
| | | | indicated | intubation or urgent | |
| m from a least to the second | | <b> </b> | | intervention indicated | |
| | zed by progressive and life-threater | ning pulmonary distress in the abser | nce of an underlying pulmonary cor | ndition, usuall <b>y</b> following major tral | ima or |
| surgery. | | | | | |
| Navigational Note: - | L Add d | Na dente commente de discol | | | |
| Allergic rhinitis | Mild symptoms; intervention<br>not indicated | Moderate symptoms; medical<br>intervention indicated | - | - | - |
| Definition: A disorder characteri | | Intervention indicated<br> mucous membranes caused by an | IgE-madiated response to external | l<br>allergens. The inflammation may al | sa involve |
| | | nx. Symptoms include sneezing, nas | | | somione |
| Navigational Note: - | mases, eyes, madre ear, and phary | nx. symptoms meduce sheezing, nas | ar congestion, minorinea and item | 6. | |
| Apnea | | | Present: medical intervention | Life-threatening respiratory or | Death |
| Aprilea | | | indicated | hemodynamic compromise; | DCau |
| | | | Transacca | intubation or urgent | |
| | | | | intervention indicated | |
| Definition: A disorder characteri | zed by cessation of breathing. | • | | | • |
| Navigational Note: - | , | | | | |
| Aspiration | Asymptomatic; clinical or | Altered eating habits; | Dyspnea and pneumonia | Life-threatening respiratory or | Death |
| • | diagnostic observations only; | coughing or choking episodes | symptoms (e.g., aspiration | hemodynamic compromise; | |
| | intervention not indicated | after eating or swallowing; | pneumonia); hospitalization | intubation or urgent | |
| | | medical intervention indicated | indicated; unable to aliment | intervention indicated | |
| | | (e.g., suction or oxygen) | orally | | |
| Definition: A disorder characteri | zed b <b>y</b> inhalation of solids or liquids | into the lungs. | | | |
| Navigational Note: - | | | | | |
| Atelectasis | Asymptomatic; clinical or | Symptomatic (e.g., dyspnea, | Supplemental oxygen | Life-threatening respiratory or | Death |
| | diagnostic observations only; | cough); medical intervention | indicated; hospitalization or | hemodynamic compromise; | |
| | intervention not indicated | indicated (e.g., chest | elective operative | intubation or urgent | |
| | | physiotherapy, suctioning); | intervention indicated (e.g., | intervention indicated | |
| | l | bronchoscopic suctioning | stent, laser) | | |
| | zed by the collapse of part or the er | ntire lung. | | | |
| Navigational Note: - | | | | | |
| Bronchial fistula | Asymptomatic | Symptomatic, invasive | Invasive intervention | Life-threatening | Death |
| | | intervention not indicated | indicated | consequences; urgent | |
| Deficial and Advander described | l | <br> | | intervention indicated | |
| | zea by an abnormal communication | n between the bronchus and anothe | er organ or anatomic site. | | |
| Navigational Note: - | | | | | |

| | | Respiratory, thoracic and mediast | tinal disorders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Bronchial obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., mild wheezing); endoscopic evaluation indicated; radiographic evidence of atelectasis/lobar collapse; medical management indicated (e.g., steroids, bronchodilators) | Shortness of breath with stridor; endoscopic intervention indicated (e.g., laser, stent placement) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent<br>intervention indicated | Death |
| Definition: A disorder charact<br>Navigational Note: - | erized by blockage of a bronchus pass | age, most often by bronchial secre | tions and exudates. | | |
| Bronchial stricture | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., rhonchi or<br>wheezing) but without<br>respiratory distress; medical<br>intervention indicated (e.g.,<br>steroids, bronchodilators) | Shortness of breath with stridor; endoscopic intervention indicated (e.g., laser, stent placement) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent<br>intervention indicated | Death |
| | erized by a narrowing of the bronchia | l tube. | | | |
| Navigational Note: - | | T | The state of the s | Luci | 1 8 0 |
| Bronchopleural fistula | Asymptomatic | Symptomatic, invasive intervention not indicated | Hospitalization; invasive<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | erized by an abnormal communicatio | n between a bronchus and the pleu | ral cavity. | • | • |
| Navigational Note: -<br>Bronchopulmonary | Mild symptoms; intervention | Moderate symptoms; invasive | Transfusion indicated: | Life-threatening | Death |
| hemorrhage | not indicated | intervention not indicated | invasive intervention indicated; hospitalization | consequences; intubation or<br>urgent intervention indicated | Deadi |
| Definition: A disorder charact | erized by bleeding from the bronchial | wall and/or lung parenchyma. | • | | • |
| Navigational Note: - | | | | | |
| Bronchospasm | Mild symptoms; intervention<br>not indicated | Symptomatic; medical<br>intervention indicated;<br>limiting instrumental ADL | Limiting self care ADL;<br>supplemental oxygen<br>indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder charact<br><b>Navigational Note:</b> - | erized by a sudden contraction of the | smooth muscles of the bronchial w | vall. | | |

| Respiratory, thoracic and mediastinal disorders | | | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Chylothorax | Asymptomatic; clinical or | Symptomatic; medical | Severe symptoms; elective | Life-threatening respiratory or | Death |
| | diagnostic observations only; | intervention indicated (e.g., | operative intervention | hemodynamic compromise; | |
| | intervention not indicated | fat-restricted diet); | indicated | intubation or urgent | |
| | | thoracentesis or tube | | intervention indicated | |
| | | drainage indicated | | l | |
| | terized b <b>y</b> milk <b>y</b> pleural effusion (abno | rmal collection of fluid) resulting fro | om accumulation of l <b>y</b> mph fluid in t | he pleural cavity. | |
| lavigational Note: - | | | | | |
| Cough | Mild symptoms; | Moderate symptoms, medical | Severe symptoms; limiting self | - | - |
| | nonprescription intervention | intervention indicated; | care ADL | | |
| | indicated | limiting instrumental ADL | 1 | <b>!</b> | l . |
| | terized b <b>y</b> sudden, often repetitive, sp | asmodic contraction of the thoracic | cavity, resulting in violent release | of air from the lungs and usually acc | companied |
| y a distinctive sound. | | | | | |
| lavigational Note: - | Shortness of breath with | Shortness of breath with | Shortness of breath at rest: | 126- 4 | D#- |
| yspnea | moderate exertion | | Snortness of breath at rest;<br>limiting self care ADL | Life-threatening | Death |
| | moderate exertion | minimal exertion; limiting | limiting self care AUL | consequences; urgent | |
| | 1 | instrumental ADL | l | intervention indicated | l |
| | terized b <b>y</b> an uncomfortable sensatior | of difficulty breathing. | | | |
| lavigational Note: - | | | | | |
| pistaxis | Mild symptoms; intervention | Moderate symptoms; medical | Transfusion; invasive | Life-threatening | Death |
| | not indicated | intervention indicated (e.g., | intervention indicated (e.g., | consequences; urgent | |
| | | nasal packing, cauterization; | hemostasis of bleeding site) | intervention indicated | |
| | | topical vasoconstrictors) | | l | |
| | terized by bleeding from the nose. | | | | |
| lavigational Note: - | | | | | |
| liccups | Mild symptoms; intervention | Moderate symptoms; medical | Severe symptoms; interfering | - | - |
| | not indicated | intervention indicated; | with sleep; limiting self care | | |
| | | limiting instrumental ADL | ADL | 1 | |
| | terized by repeated gulp sounds that r | esult from an involuntar <b>y</b> opening a | and closing of the glottis. This is attr | ibuted to a spasm of the diaphragn | ١. |
| lavigational Note: - | | | | | |
| loarseness | Mild or intermittent voice | Moderate or persistent voice | Severe voice changes | - | - |
| | change; fully understandable; | changes; may require | including predominantly | l | |
| | self-resolves | occasional repetition but | whispered speech | l | |
| | | understandable on telephone; | | l | |
| | | medical evaluation indicated | | I | |
| efinition: A disorder charac | terized by harsh and raspy voice arisin | g from or spreading to the larynx. | | | |
| lavigational Note: - | | • | | | |

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| | Si Bate 1 | | | | |
| Hypoxia | | Decreased oxygen saturation | Decreased oxygen saturation | Life-threatening airway | Death |
| | | with exercise (e.g., pulse | at rest (e.g., pulse oximeter | compromise; urgent | |
| | | oximeter <88%); intermittent | <88% or PaO2 <=55 mm Hg) | intervention indicated (e.g., | |
| | I | supplemental oxygen | | tracheotomy or intubation) | 1 |
| <b>Definition:</b> A disorder charac | terized by a decrease in the level of ox | ygen in the body. | | | |
| Navigational Note: - | | | | | |
| Laryngeal edema | Asymptomatic; clinical or | Symptomatic; medical | Stridor; respiratory distress; | Life-threatening airway | Death |
| | diagnostic observations only; | intervention indicated (e.g., | hospitalization indicated | compromise; urgent | |
| | intervention not indicated | dexamethasone, epinephrine, | | intervention indicated (e.g., | |
| | | antihistamines) | | tracheotomy or intubation) | |
| Definition: A disorder charac | terized by swelling due to an excessive | accumulation of fluid in the larvox | | • | • |
| Navigational Note: - | , | ,,,,, | | | |
| Laryngeal fistula | Asymptomatic | Symptomatic, invasive | Invasive intervention | Life-threatening | Death |
| zar ji godi notara | , reyring contrado | intervention not indicated | indicated | consequences; urgent | |
| | | intervendonnochidicated | Indicated | intervention indicated | |
| Definition: A disarder above | I<br>terized by an abnormal communication | I<br>n h atrugan the lenguy and another s | l<br>vzan az anatazzia elta | Intervendormacated | 1 |
| | cenzed by an abnormal communication | n between the larynx and another t | ngari or anatomic site. | | |
| Navigational Note: - | L satisficación de la companya de la | I Na danata manatana | Transfusion indicated: | 125- 41 | D |
| Laryngeal hemorrhage | Mild cough or trace | Moderate symptoms; | , | Life-threatening | Death |
| | hemoptysis; laryngoscopic | intervention indicated | invasive intervention | consequences, urgent | |
| | findings | | indicated; hospitalization | intervention indicated (e.g., | |
| | 1 | I | | tracheotomy or intubation) | |
| <b>Definition:</b> A disorder charac | terized by bleeding from the larynx. | | | | |
| Navigational Note: - | | | | | |
| Laryngeal inflammation | Mild sore throat; raspy voice | Moderate sore throat; | Severe throat pain; | - | - |
| | | analgesics indicated | endoscopic intervention | | |
| | | | indicated | | |
| Definition: A disorder charac | terized by an inflammation involving th | ne larvnx. | • | • | • |
| Navigational Note: - | | | | | |
| Laryngeal mucositis | Endoscopic findings only; mild | Moderate pain, analgesics | Severe pain; severely altered | Life-threatening airway | Death |
| Early in Coal InfoCoaldia | discomfort with normal intake | indicated; altered oral intake; | eating/swallowing; medical | compromise; urgent | Dead |
| | uiscomione with normal intake | limiting instrumental ADL | intervention indicated | intervention indicated (e.g., | |
| | | imiting instrumental ADL | intervention indicated | | |
| | 1 | I . | I <sub>e</sub> | tracheotomy or intubation) | 1 |
| <b>Definition:</b> A disorder charac | terized by ulceration or inflammation i | 'nvolving the mucous membrane of | the larynx. | | |
| Navigational Note: - | | | | | |

| | | Respiratory, thoracic and mediast | inal disorders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Laryngeal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., noisy airway breathing), no respiratory distress; medical intervention indicated (e.g., steroids); limiting instrumental ADL | Limiting self care ADL; stridor;<br>endoscopic intervention<br>indicated (e.g., stent, laser) | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | terized by blockage of the laryngeal ai | rway. | | | |
| Navigational Note: - | Asymptomatic; clinical or | Symptomatic (e.g., noisy | Limiting self care ADL; stridor; | Life-threatening | Death |
| Laryngeal stenosis | Asymptomate; clinical or diagnostic observations only; intervention not indicated | airway breathing), no<br>respiratory distress; medical<br>intervention indicated (e.g.,<br>steroids); limiting<br>instrumental ADL | endoscopic intervention<br>indicated (e.g., stent, laser) | consequences; urgent intervention indicated | Death |
| Definition: A disorder charac | terized by a narrowing of the laryngea | l airway. | | • | • |
| Navigational Note: - | | | | | |
| Laryngopharyngeal<br>dysesthesia | Mild symptoms; no anxiety;<br>intervention not indicated | Moderate symptoms; mild<br>anxiety, but no dyspnea; short<br>duration of observation<br>and/or anxiolytic indicated;<br>limiting instrumental ADL | Severe symptoms; dyspnea<br>and swallowing difficulty;<br>limiting self care ADL | Life-threatening<br>consequences | Death |
| Definition: A disorder charact | terized by an uncomfortable persisten | it sensation in the area of the laryng | opharynx. | • | |
| Navigational Note: - | | | | | |
| Laryngospasm | - | Transient episode;<br>intervention not indicated | Recurrent episodes;<br>noninvasive intervention<br>indicated (e.g., breathing<br>technique, pressure point<br>massage) | Persistent or severe episodes<br>associated with syncope;<br>urgent intervention indicated<br>(e.g., fiberoptic laryngoscopy,<br>intubation, botox injection) | Death |
| | terized by paroxysmal spasmodic mus | cular contraction of the vocal cords. | • | | |
| Navigational Note: - | T | | T | | |
| Mediastinal hemorrhage | Mild symptoms; intervention<br>not indicated; radiologic<br>evidence only | Moderate symptoms;<br>intervention indicated | Transfusion indicated;<br>invasive intervention<br>indicated; hospitalization | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder charac | terized by bleeding from the mediastir | num. | | | |
| Navigational Note: - | | | | | |

| | | Respiratory, thoracic and mediast | inal disorders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Nasal congestion | Mild symptoms; intervention<br>not indicated | Moderate symptoms; medical<br>intervention indicated | Associated with bloody nasal discharge or epistaxis | - | - |
| Definition: A disorder charac | terized by obstruction of the nasal pas | ssage due to mucosal edema. | | | • |
| Navigational Note: - | | | | | |
| Orophar <b>y</b> ngeal pain | Mild pain | Moderate pain; altered oral<br>intake; non-narcotics<br>initiated; topical analgesics<br>initiated | Severe pain; severely altered<br>eating/swallowing; narcotics<br>initiated; requires parenteral<br>nutrition | - | - |
| Definition: A disorder charac | terized by a sensation of marked disco | omfort in the oropharynx. | • | • | • |
| Navigational Note: - | | | | | |
| Pharyngeal fistula | Asymptomatic | Symptomatic, invasive intervention not indicated | Invasive intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder charac | terized by an abnormal communicatio | n between the pharynx and anothe | r organ or anatomic site. | | |
| Navigational Note: - | | | | | |
| Pharyngeal hemorrhage | Mild symptoms; intervention<br>not indicated | Moderate symptoms;<br>intervention indicated | Transfusion indicated;<br>invasive intervention<br>indicated; hospitalization | Life-threatening<br>consequences; intubation or<br>urgent intervention indicated | Death |
| Definition: A disorder charac | terized by bleeding from the pharynx. | • | • | • | • |
| Navigational Note: - | | | | | |
| Pharyngeal mucositis | Endoscopic findings only;<br>minimal symptoms with<br>normal oral intake; mild pain<br>but analgesics not indicated | Moderate pain, analgesics<br>indicated; altered oral intake;<br>limiting instrumental ADL | Severe pain; unable to<br>adequately aliment or hydrate<br>orally; limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder charac | terized by ulceration or inflammation | involving the mucous membrane of | the pharynx. | • | • |
| Navigational Note: - | | | | | |
| Pharyngeal necrosis | - | - | Inability to aliment adequately<br>by GI tract; invasive<br>intervention indicated; tube<br>feeding or TPN indicated | Life-threatening<br>consequences; urgent<br>operative intervention<br>indicated | Death |
| Definition: A disorder charac | terized by a necrotic process occurring | g in the pharynx. | | | |
| Navigational Note: - | | | | | |

| | | Respiratory, thoracic and medias | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade |
| Pharyngeal stenosis | Asymptomatic; clinical or | Symptomatic (e.g., noisy | Limiting self care ADL; stridor; | Life-threatening airway | Death |
| | diagnostic observations only; | airway breathing), no | endoscopic intervention | compromise; urgent | |
| | intervention not indicated | respiratory distress; medical | indicated (e.g., stent, laser) | intervention indicated (e.g., | |
| | | intervention indicated (e.g., | | tracheotomy or intubation) | |
| | | steroids); limiting | | | |
| | | instrumental ADL | 1 | | |
| <b>Definition:</b> A disorder charac | cterized by a narrowing of the pharyng | eal airway. | | | |
| Navigational Note: - | | | | | |
| Pharyngolaryngeal pain | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | - | - |
| | | instrumental ADL | ADL | | |
| Definition: A disorder charac | cterized by a sensation of marked disco | mfort in the pharyngolaryngeal re | gion. | | • |
| Navigational Note: - | | | | | |
| Pleural effusion | Asymptomatic; clinical or | Symptomatic; intervention | Symptomatic with respiratory | Life-threatening respiratory or | Death |
| | diagnostic observations only; | indicated (e.g., diuretics or | distress and hypoxia; | hemodynamic compromise; | |
| | intervention not indicated | therapeutic thoracentesis) | operative intervention | intubation or urgent | |
| | | , | including chest tube or | intervention indicated | |
| | | | pleurodesis indicated | | |
| Definition: A disorder charac | cterized by an increase in amounts of fl | uid within the pleural cavity. Symp | 1 ' | ugh and marked chest discomfort | • |
| Navigational Note: - | , | and the first and balley to your | | | |
| Pleural hemorrhage | Asymptomatic; mild | Symptomatic or associated | >1000 ml of blood evacuated; | Life-threatening | Death |
| - | hemorrhage confirmed by | with pneumothorax; chest | persistent bleeding (150-200 | consequences; intubation or | |
| | thoracentesis | tube drainage indicated | ml/hr for 2 - 4 hr); persistent | urgent intervention indicated | |
| | | | transfusion indicated; elective | | |
| | | | operative intervention | | |
| | | | indicated; hospitalization | | |
| <b>Definition:</b> A disorder charac | cterized by bleeding from the pleural ca | evity. | | • | • |
| Navigational Note: - | storizons, stooding to the displaced at | | | | |
| Pleuritic pain | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | - | - |
| | | instrumental ADL | ADL | | |
| Definition: A disorder charac | terized by a sensation of marked disco | | 1 7.02 | ' | 1 |
| Navigational Note: - | startzea by a scrisa don or marked disco | into cirrate picara. | | | |
| Pneumonitis | Asymptomatic: clinical or | Symptomatic: medical | Severe symptoms; limiting self | Life-threatening respiratory | Death |
| | diagnostic observations only: | intervention indicated: | care ADL; oxygen indicated | compromise: urgent | DCaai |
| | intervention not indicated | 1 | care ADE, Oxygermiuicated | intervention indicated (e.g., | |
| | intervendon not indicated | limiting instrumental ADL | | tracheotomy or intubation) | |
| | 1 | 1 | 1 | a acrieowiny or intubation) | 1 |
| | cterized by inflammation focally or diffu | usely affecting the lung parenchym | ia. | | |
| Navigational Note: - | , | , | | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Respiratory, thoracic and mediast | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade |
| Pneumothorax | Asymptomatic; clinical or | Symptomatic; intervention | Sclerosis and/or operative | Life-threatening | Death |
| | diagnostic observations only; | indicated | intervention indicated; | consequences; urgent | |
| | intervention not indicated | 1 | hospitalization indicated | intervention indicated | |
| Definition: A disorder chara- | cterized b <b>y</b> abnormal presence of air in | the pleural cavity resulting in the co | ollapse of the lung. | | |
| Navigational Note: - | | | | | |
| Postnasal drip | Mild symptoms; intervention | Moderate symptoms; medical | - | - | - |
| | not indicated | intervention indicated | | | |
| Definition: A disorder chara- | cterized by excessive mucous secretion | in the back of the nasal cavity or th | roat, causing sore throat and/or co | ughing. | |
| Navigational Note: - | | | | | |
| Productive cough | Occasional/minimal | Moderate sputum production; | Persistent or copious | - | - |
| | production of sputum with | limiting instrumental ADL | production of sputum; limiting | | |
| | cough | | self care ADL | | |
| Definition: A disorder chara- | cterized by expectorated secretions up | on coughing. | | | |
| Navigational Note: - | | | | | |
| Pulmonary edema | Radiologic findings only; | Moderate dyspnea on | Severe dyspnea or dyspnea at | Life-threatening respiratory | Death |
| | minimal dyspnea on exertion | exertion; medical intervention | rest; oxygen indicated; | compromise; urgent | |
| | | indicated; limiting | limiting self care ADL | intervention or intubation | |
| | | instrumental ADL | | with ventilatory support | |
| | | | | indicated | |
| Definition: A disorder chara- | cterized b <b>y</b> accumulation of fluid in the | lung tissues that causes a disturban | ice of the gas exchange that may le | ad to respiratory failure. | |
| Navigational Note: - | | | | | |
| Pulmonary fibrosis | Radiologic pulmonary fibrosis | Evidence of pulmonary | Severe hypoxia; evidence of | Life-threatening | Death |
| | <2.5% of lung volume | hypertension; radiographic | right-sided heart failure; | consequences (e.g., | |
| | associated with hypoxia | pulmonary fibrosis 25 - 50% | radiographic pulmonary | hemodynamic/pulmonary | |
| | | associated with hypoxia | fibrosis >50 - <b>7</b> 5% | complications); intubation | |
| | | | | with ventilatory support | |
| | | | | indicated; radiographic | |
| | | | | pulmonary fibrosis >75% with | |
| | | 1 | | severe honeycombing | |
| Definition: A disorder chara- | cterized by the replacement of the lung | g tissue by connective tissue, leading | to progressive dyspnea, respirator | y failure or right heart failure. | |
| Navigational Note: - | | | | | |
| Pulmonary fistula | Asymptomatic | Symptomatic, invasive | Invasive intervention | Life-threatening | Death |
| | | intervention not indicated | indicated | consequences; urgent | 1 |
| | | | | intervention indicated | 1 |
| | and the second second | 1 4 4 4 4 4 | | | |
| <b>Definition:</b> A disorder chara- | cterized by an abnormal communicatio | n between the lung and another org | gan or anatomic site. | | |

| | | Respiratory, thoracic and mediast | inal disorders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Pulmonary hypertension | Minimal dyspnea; findings on<br>physical exam or other<br>evaluation | Moderate dyspnea, cough;<br>requiring evaluation by<br>cardiac catheterization and<br>medical intervention | Severe symptoms, associated<br>with hypoxia, right heart<br>failure; oxygen indicated | Life-threatening airway<br>consequences; urgent<br>intervention indicated (e.g.,<br>tracheotomy or intubation) | Death |
| Definition: A disorder characteri | zed by an increase in pressure with | in the pulmonary circulation due to | lung or heart disorder. | | |
| Navigational Note: - | | | | | |
| Respiratory failure | - | - | - | Life-threatening<br>consequences; urgent<br>intervention, intubation, or<br>ventilatory support indicated | Death |
| <b>Definition:</b> A disorder characterian increase in arterial levels of ca | zed by impaired gas exchange by tharbon dioxide. | ne respiratory system resulting in hy | poxia and a decrease in oxygenation | | iated with |
| Navigational Note: - | | | | | |
| Retinoic acid syndrome | Fluid retention; <3 kg of<br>weight gain; intervention with<br>fluid restriction and/or<br>diuretics indicated | Moderate signs or symptoms;<br>steroids indicated | Severe symptoms;<br>hospitalization indicated | Life-threatening<br>consequences; ventilatory<br>support indicated | Death |
| <b>Definition:</b> A disorder characteri retinoic acid. | zed by weightgain, dyspnea, pleura | al and pericardial effusions, leukocy | tosis and/or renal failure originally | described in patients treated with | all-trans |
| Navigational Note: - | | | | | |
| Rhinorrhea | Present | - | - | - | - |
| Definition: A disorder characteri | zed by excessive mucous secretions | draining from the nose. | • | • | • |
| Navigational Note: - | | | | | |
| Sinus disorder | Asymptomatic mucosal<br>crusting; blood-tinged<br>secretions | Symptomatic stenosis or<br>edema/narrowing interfering<br>with airflow; limiting<br>instrumental ADL | Stenosis with significant nasal<br>obstruction; limiting self care<br>ADL | Necrosis of soft tissue or<br>bone; urgent operative<br>intervention indicated | Death |
| Definition: A disorder characteri | zed by involvement of the paranasa | al sinuses. | | | • |
| Navigational Note: - | · · | | | | |
| Sinus pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| <b>Definition:</b> A disorder characteri<br><b>Navigational Note:</b> - | zed by a sensation of marked disco | mfort in the face, between the eye: | s, or upper teeth originating from t | ne sinuses. | - |

| | | Respiratory, thoracic and mediast | tinal disorders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Sleep apnea | Snoring and nocturnal sleep<br>arousal without apneic<br>periods | Moderate apnea and oxygen desaturation; excessive daytime sleepiness; medical evaluation indicated; limiting instrumental ADL | Oxygen desaturation;<br>associated with pulmonary<br>hypertension; medical<br>intervention indicated;<br>limiting self care ADL | Cardiovascular or<br>neuropsychiatric symptoms;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder chara-<br>Navigational Note: - | cterized by cessation of breathing for s | hort periods during sleep. | | | |
| Sneezing Definition: A disorder chara- | Mild symptoms; intervention not indicated cterized by the involuntary expulsion o | Moderate symptoms; medical intervention indicated | - | - | - |
| Navigational Note: - | started by the involuntary apparation of | | | | |
| Sore throat | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL; limiting ability to<br>swallow | - | - |
| <b>Definition:</b> A disorder chara-<br><b>Navigational Note:</b> - | cterized by marked discomfort in the t | nroat | ' | • | |
| Stridor | - | - | Respiratory distress limiting self care ADL; medical intervention indicated | Life-threatening airway<br>compromise; urgent<br>intervention indicated (e.g.,<br>tracheotomy or intubation) | Death |
| | cterized by a high pitched breathing so | und due to laryngeal or upper airwa | y obstruction. | , , | • |
| Navigational Note: - | | T | T | Luci | 1 |
| Tracheal fistula | Asymptomatic | Symptomatic, invasive<br>intervention not indicated | Invasive intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder characteristic Navigational Note: - | cterized by an abnormal communicatio | on between the trachea and another | organ or anatomic site. | | |
| Tracheal mucositis | Endoscopic findings only;<br>minimal hemoptysis, pain, or<br>respiratory symptoms | Moderate symptoms; medical<br>intervention indicated;<br>limiting instrumental ADL | Severe pain; hemorrhage or<br>respiratory symptoms;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder chara- | cterized b <b>y</b> an inflammation or ulcerati | on involving the mucous membrane | of the trachea. | - | • |
| Navigational Note: - | | | | | |

| | | Respiratory, thoracic and mediast | inal disorders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Tracheal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated lized by a narrowing of the trachea. | Symptomatic (e.g., noisy airway breathing), no respiratory distress; medical intervention indicated (e.g., steroids); limiting instrumental ADL | Stridor or respiratory distress<br>limiting self care ADL; invasive<br>intervention indicated (e.g.,<br>stent, laser) | Life-threatening airway<br>compromise; urgent<br>intervention indicated (e.g.,<br>tracheotomy or intubation) | Death |
| Navigational Note: - | ized by a harrowing of the trachea. | | | | |
| Voice alteration | Mild or intermittent change from normal voice | Moderate or persistent<br>change from normal voice;<br>still understandable | Severe voice changes including predominantly whispered speech; may require frequent repetition or face-to-face contact for understandability; may require assistive technology | - | - |
| Definition: A disorder character | ized by a change in the sound and/o | or speed of the voice. | , | • | 1 |
| Navigational Note: - | | · | | | |
| Wheezing | Detectable airway noise with minimal symptoms | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | Severe respiratory symptoms<br>limiting self care ADL; oxygen<br>therapy or hospitalization<br>indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder character | ized by a high-pitched, whistling sou | und during breathing. It results from | n the narrowing or obstruction of th | ne respiratory airways. | • |
| Navigational Note: - | | | | | |
| Respiratory, thoracic and mediastinal disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: - | | - | | - | |
| Navigational Note: - | | | | | |

| | | Skin and subcutaneous tissue | disorders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Alopecia | Hair loss of <50% of normal | Hair loss of >=50% normal for | - | - | - |
| | for that individual that is not | that individual that is readily | | | |
| | obvious from a distance but | apparent to others; a wig or | | | |
| | only on close inspection; a | hair piece is necessary if the | | | |
| | different hair style may be | patient desires to completely | | | |
| | required to cover the hair loss | camouflage the hair loss; | | | |
| | but it does not require a wig | associated with psychosocial | | | |
| | or hair piece to camouflage | impact | | | |
| Definition: A disorder chara | acterized by a decrease in density of hair | compared to normal for a given in | dividual at a given age and body loc | ation. | |
| Navigational Note: - | | | | | |
| Body odor | Mild odor; physician | Pronounced odor; | - | - | - |
| | intervention not indicated; | psychosocial impact; patient | | | |
| | self care interventions | seeks medical intervention | | | |
| Definition: A disorder chara | acterized by an abnormal body smell res | ulting from the growth of bacteria | on the body. | | - |
| Navigational Note: - | | | | | |
| Bullous dermatitis | Asymptomatic; blisters | Blisters covering 10 - 30% | Blisters covering >30% BSA; | Blisters covering >30% BSA; | Death |
| | covering <10% BSA | BSA; painful blisters; limiting | limiting self care ADL | associated with fluid or | |
| | , and the second | instrumental ADL | | electrolyte abnormalities; ICU | |
| | | | | care or burn unit indicated | |
| Definition: A disorder chara | acterized by inflammation of the skin cha | aracterized by the presence of bulla | e which are filled with fluid. | • | • |
| Navigational Note: If infect | ious, consider Infections and infestation | s: Rash pustular or other site-speci | ic Infections and infestations term. | | |
| Dry skin | Covering < 10% BSA and no | Covering 10 - 30% BSA and | Covering >30% BSA and | I - | - |
| / | associated erythema or | associated with erythema or | associated with pruritus: | | |
| | pruritus | pruritus; limiting instrumental | limiting self care ADL | | |
| | p. a | ADL | | | |
| Definition: A disorder chara | acterized by flaky and dull skin; the pores | s are generally fine, the texture is a | nanery thin texture. | • | • |
| Navigational Note: - | second and and administration per or | a a a gonoran y mio, a lo tomal o lo a | paper, am restar of | | |
| Eczema | Asymptomatic or mild | Moderate; topical or oral | Severe or medically significant | - | - |
| 2 DE OTTO | symptoms: additional medical | intervention indicated: | but not immediately life- | | |
| | intervention over baseline not | additional medical | threatening; IV intervention | | |
| | indicated | intervention over baseline | indicated | | |
| | | indicated | The sea that | l | |
| <b>Definition:</b> A disorder obers | I<br>acterized by skin which becomes itchy, re | • | I<br>d/or forme blisters | • | 1 |
| | acterized by skill writer becomes iteny, re | ou, mmameu, crusty, critck, scary, an | ayor rorms birsters. | | |
| Navigational Note: - | | | | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Skin and subcutaneous tissue | disorders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Erythema multiforme | Target lesions covering <10%<br>BSA and not associated with<br>skin tenderness | Target lesions covering 10 -<br>30% BSA and associated with<br>skin tenderness | Target lesions covering >30%<br>BSA and associated with oral<br>or genital erosions | Target lesions covering >30%<br>BSA; associated with fluid or<br>electrolyte abnormalities; ICU<br>care or burn unit indicated | Death |
| <b>Definition:</b> A disorder charac<br><b>Navigational Note:</b> - | terized by target lesions (a pink-red rin | g around a pale center). | | | |
| Erythroderma | - | Erythema covering >90% BSA<br>without associated symptoms;<br>limiting instrumental ADL | Erythema covering >90% BSA<br>with associated symptoms<br>(e.g., pruritus or tenderness);<br>limiting self care ADL | Erythema covering >90% BSA<br>with associated fluid or<br>electrolyte abnormalities; ICU<br>care or burn unit indicated | Death |
| <b>Definition:</b> A disorder charac<br><b>Navigational Note:</b> - | terized by generalized inflammatory er | ythema and exfoliation. The inflam | matory process involves > 90% of t | the body surface area. | |
| Fat atrophy | Covering <10% BSA and asymptomatic | Covering 10 - 30% BSA and<br>associated with erythema or<br>tenderness; limiting<br>instrumental ADL | Covering >30% BSA;<br>associated with erythema or<br>tenderness; limiting self-care<br>ADL | - | - |
| <b>Definition:</b> A disorder charac<br><b>Navigational Note:</b> - | terized by shrinking of adipose tissue. | | • | • | |
| Hair color changes | Present | l - | - | T - | Ι- |
| • | terized by change in hair color or loss o | f normal nigmentation | ı | • | ı |
| Navigational Note: - | and the state of t | or normal pignionadora | | | |
| Hair texture abnormal | Present | - | - | - | - |
| <b>Definition:</b> A disorder charac<br><b>Navigational Note:</b> - | terized by a change in the way the hair | feels. | ' | • | |
| Hirsutism | In women, increase in length, thickness or density of hair in a male distribution that the patient is able to camouflage by periodic shaving, bleaching, or removal of hair | In women, increase in length, thickness or density of hair in a male distribution that requires daily shaving or consistent destructive means of hair removal to camouflage; associated with psychosocial impact | - | - | - |
| <b>Definition:</b> A disorder charac<br>androgen control (beard, mo<br><b>Navigational Note:</b> - | terized by the presence of excess hair<br>ustache, chest, abdomen). | growth in women in anatomic sites | where growth is considered to be | a secondary male characteristic and | l under |

| Hyperhidrosis Limited to one site (palms, soles, or axillae); self care interventions Definition: A disorder characterized by excessive sweating. Navigational Note: Synonym: Night sweats, diaphoresis Hyperkratosis Present Pefinition: A disorder characterized by a thickening of the outer layer of the skin. Navigational Note: Hypertrichosis Increase in length, thickness or density of hair that the patient is either able to camouflage by periodic shaving or removal of hairs or is not concerned enough about the overgrowth to use any form of hair removal Definition: A disorder characterized by hair density or length beyond the accepted limits of normal in a particular body region, for a particular age. | Grade 4 | Grade |
|---|---|---|
| soles, or axillae); self care intervention; associated with psychosocial impact Definition: A disorder characterized by excessive sweating. Navigational Note: Synonym: Night sweats, diaphoresis Hyperkeratosis Present - Limiting self-care ADLs - Definition: A disorder characterized by a thickening of the outer layer of the skin. Navigational Note: - Hypertrichosis Increase in length, thickness or density of hair that the patient is either able to camouflage by periodic shaving or removal of hairs or is not concerned enough about the overgrowth to use any form of hair removal Increase in length, thickness or density of hair at least on the usual exposed areas of the body [face (not limited to beard/moustache area) plus/minus arms] that requires frequent shaving or use of destructive means of hair removal to camouflage; associated with psychosocial impact | | |
| Interventions associated with psychosocial impact Definition: A disorder characterized by excessive sweating. Navigational Note: Synonym: Night sweats, diaphoresis Hyperkeratosis Present - Limiting self-care ADLs - Definition: A disorder characterized by a twickening of the outer layer of the skin. Navigational Note: Hypertrichosis Increase in length, thickness or density of hair that the patient is either able to camouflage by periodic shaving or removal of hairs or is not concerned enough about the overgrowth to use any form of hair removal to camouflage; associated with psychosocial impact impact impact impact impact impact impact Increase in length, thickness or density of hair at least on the usual exposed areas of the body [face (not limited to beard/moustache area) plus/minus arms] that requires frequent shaving or use of destructive means of hair removal to camouflage; associated with psychosocial impact | | <br> |
| Definition: A disorder characterized by excessive sweating. Navigational Note: Synonym: Night sweats, diaphoresis Hyperkeratosis Present - Limiting self-care ADLs - Definition: A disorder characterized by a thickening of the outer layer of the skin. Navigational Note: Hypertrichosis Increase in length, thickness or density of hair that the patient is either able to camouflage by periodic shaving or removal of hairs or is not concerned enough about the overgrowth to use any form of hair removal any form of hair removal impact Limiting self-care ADLs - characterized by a thickening of the outer layer of the skin. Increase in length, thickness or density of hair at least on the usual exposed areas of the body [face (not limited to beard/moustache area) plus/minus arms] that requires frequent shaving or use of destructive means of hair removal to camouflage; associated with psychosocial impact | | - |
| Definition: A disorder characterized by excessive sweating. Navigational Note: Synonym: Night sweats, diaphoresis Hyperkeratosis Present - Limiting self-care ADLs - Definition: A disorder characterized by a thickening of the outer layer of the skin. Navigational Note: - Hypertrichosis Increase in length, thickness or density of hair that the patient is either able to camouflage by periodic shaving or removal of hairs or is not concerned enough about the overgrowth to use any form of hair removal any form of hair removal The service of the skin. Increase in length, thickness or density of hair at least on the usual exposed areas of the body [face (not limited to beard/moustache area) plus/minus arms] that requires frequent shaving or use of destructive means of hair removal to camouflage; associated with psychosocial impact | | - |
| Navigational Note: Synonym: Night sweats, diaphoresis Present - Limiting self-care ADLs - Definition: A disorder characterized by a thickening of the outer layer of the skin. Navigational Note: Hypertrichosis Increase in length, thickness or density of hair that the patient is either able to camouflage by periodic shaving or removal of hairs or is not concerned enough about the overgrowth to use any form of hair removal Increase in length, thickness or density of hair at least on the usual exposed areas of the body [face (not limited to beard/moustache area) plus/minus arms] that requires frequent shaving or use of destructive means of hair removal to camouflage; associated with psychosocial impact | | - |
| diaphoresis Hyperkeratosis Present - Limiting self-care ADLs - Definition: A disorder characterized by a thickening of the outer layer of the skin. Navigational Note: - Hypertrichosis Increase in length, thickness or density of hair that the patient is either able to camouflage by periodic shaving or removal of hairs or is not concerned enough about the overgrowth to use any form of hair removal Increase in length, thickness or density of hair at least on the usual exposed areas of the body (face (not limited to beard/moustache area) plus/minus arms] that requires frequent shaving or use of destructive means of hair removal to camouflage; associated with psychosocial impact | | - |
| Hyperkeratosis Present - Limiting self-care ADLs - Definition: A disorder characterized by a thickening of the outer layer of the skin. Navigational Note: - Hypertrichosis Increase in length, thickness or density of hair that the patient is either able to camouflage by periodic shaving or removal of hairs or is not concerned enough about the overgrowth to use any form of hair removal end of the skin. Increase in length, thickness or density of hair at least on the usual exposed areas of the body (face (not limited to beard/moustache area) plus/minus arms] that requires frequent shaving or use of destructive means of hair removal to camouflage; associated with psychosocial impact | | |
| Definition: A disorder characterized by a thickening of the outer layer of the skin. Navigational Note: - Hypertrichosis Increase in length, thickness or density of hair that the patient is either able to camouflage by periodic shaving or removal of hairs or is not concerned enough about the overgrowth to use any form of hair removal of hair removal to camouflage; associated with psychosocial impact. | | - |
| Navigational Note: - Hypertrichosis Increase in length, thickness or density of hair that the patient is either able to camouflage by periodic shaving or removal of hairs or is not concerned enough about the overgrowth to use any form of hair removal Increase in length, thickness or density of hair at least on the usual exposed areas of the body [face (not limited to beard/moustache area) plus/minus arms] that requires frequent shaving or use of destructive means of hair removal to camouflage; associated with psychosocial impact | | - |
| Navigational Note: - Hypertrichosis Increase in length, thickness or density of hair that the patient is either able to camcuflage by periodic shaving or removal of hairs or is not concerned enough about the overgrowth to use any form of hair removal any form of hair removal Increase in length, thickness or density of hair at least on the usual exposed areas of the body [face (not limited to beard/moustache area) plus/minus arms] that requires frequent shaving or use of destructive means of hair removal to camouflage; associated with psychosocial impact | | - |
| Hypertrichosis Increase in length, thickness or density of hair that the patient is either able to camouflage by periodic shaving or removal of hairs or is not concerned enough about the overgrowth to use any form of hair removal Increase in length, thickness or density of hair at least on the usual exposed areas of the body [face (not limited to beard/moustache area) plus/minus arms] that requires frequent shaving or use of destructive means of hair removal to camouflage; associated with psychosocial impact | | - |
| or density of hair that the patient is either able to camouflage by periodic shaving or removal of hairs or is not concerned enough about the overgrowth to use any form of hair removal or hair removal or density of hair at least on the usual exposed areas of the body [face (not limited to beard/moustache area) plus/minus arms] that requires frequent shaving or use of destructive means of hair removal to camouflage; associated with psychosocial impact | | |
| patient is either able to camouflage by periodic shaving or removal of hairs or is not concerned enough about the overgrowth to use any form of hair removal use of destructive means of hair removal to camouflage; associated with psychosocial impact | | |
| camouflage by periodic shaving or removal of hairs or is not concerned enough about the overgrowth to use any form of hair removal about the overgrowth to use any form of hair removal about the overgrowth to use any form of hair removal body [face (not limited to beard/moustache area) plus/minus arms] that requires frequent shaving or use of destructive means of hair removal to camouflage; associated with psychosocial impact | | |
| shaving or removal of hairs or is not concerned enough about the overgrowth to use any form of hair removal any form of hair removal the owners of the provided of the provided in the provide | | |
| is not concerned enough about the overgrowth to use any form of hair removal use of destructive means of hair removal to camouflage; associated with psychosocial impact | | |
| about the overgrowth to use any form of hair removal use of destructive means of hair removal to camouflage; associated with psychosocial impact | | |
| any form of hair removal use of destructive means of hair removal to camouflage; associated with psychosocial impact | | |
| hair removal to camouflage; associated with psychosocial impact | | |
| associated with psychosocial impact | | |
| Impact | | |
| | | l |
| | ge or race. | |
| Navigational Note: - | | |
| -/ | at stroke | Death |
| instrumental ADL limiting self care ADL | | l |
| Definition: A disorder characterized by reduced sweating. | | |
| Navigational Note: - | | |
| Lipohypertrophy Asymptomatic and covering Covering 10 - 30% BSA and Covering > 30% BSA and - | | - |
| <10% BSA associated tenderness; associated tenderness and | | |
| limiting instrumental ADL narcotics or NSAIDs indicated; | | |
| lipohypertrophy; limiting self | | |
| care ADL | | |
| Definition: A disorder characterized by hypertrophy of the subcutaneous adipose tissue at the site of multiple subcutaneous injections of insulin. | ١. | • |
| Navigational Note: - | | |
| Nail changes Present - - - | | - |
| Definition: A disorder characterized by a change in the nails. | | • |
| Navigational Note: - | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Skin and subcutaneous tissue | disorders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Nail discoloration | Asymptomatic; clinical or<br>diagnostic observations only | - | - | - | - |
| Definition: A disorder characteri | ized by a change in the color of the i | nail plate. | • | | • |
| Navigational Note: - | | | | | |
| Nail loss | Asymptomatic separation of<br>the nail bed from the nail<br>plate or nail loss | Symptomatic separation of<br>the nail bed from the nail<br>plate or nail loss; limiting<br>instrumental ADL | - | - | - |
| Definition: A disorder characteri | ized by loss of all or a portion of the | nail. | | | |
| Navigational Note: - | | | | | |
| Nail ridging | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | - | - | - | - |
| Definition: A disorder characteri | ized by vertical or horizontal ridges | on the nails. | | | |
| Navigational Note: - | | | | | |
| Pain of skin | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteri | ized by a sensation of marked discor | mfort in the skin. | • | • | • |
| Navigational Note: - | | | | | |
| Palmar-plantar<br>erythrodysesthesia syndrome | Minimal skin changes or<br>dermatitis (e.g., erythema,<br>edema, or hyperkeratosis)<br>without pain | Skin changes (e.g., peeling,<br>blisters, bleeding, fissures,<br>edema, or hyperkeratosis)<br>with pain; limiting<br>instrumental ADL | Severe skin changes (e.g.,<br>peeling, blisters, bleeding,<br>fissures, edema, or<br>hyperkeratosis) with pain;<br>limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by redness, marked discomfort, | , swelling, and tingling in the palms | of the hands or the soles of the fee | t. Also known as Hand-Foot Synd | drome. |
| Navigational Note: - | | | | | |
| Photosensitivity | Painless erythema and<br>erythema covering <10% BSA | Tender erythema covering 10<br>-30% BSA | Erythema covering >30% BSA<br>and erythema with blistering;<br>photosensitivity; oral<br>corticosteroid therapy<br>indicated; pain control<br>indicated (e.g., narcotics or<br>NSAIDs) | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder characteri<br><b>Navigational Note:</b> - | zed by an increase in sensitivity of t | he skin to light. | | | |

| | | Skin and subcutaneous tissue | disorders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade |
| Pruritus | Mild or localized; topical | Widespread and intermittent; | Widespread and constant; | - | - |
| | intervention indicated | skin changes from scratching | limiting self care ADL or sleep; | | |
| | | (e.g., edema, papulation, | systemic corticosteroid or | | |
| | | excoriations, lichenification, | immunosuppressive therapy | | |
| | | oozing/crusts); oral | indicated | | |
| | | intervention indicated;<br>limiting instrumental ADL | | | |
| | | , - | I | I | l |
| Definition: A disorder characti<br>Navigational Note: - | erized by an intense itching sensation. | • | | | |
| Purpura | Combined area of lesions | Combined area of lesions | Combined area of lesions | | - |
| ai pai a | covering <10% BSA | covering 10 - 30% BSA: | covering >30% BSA; | | |
| | | bleeding with trauma | spontaneous bleeding | | |
| Definition: A disorder characte | erized by hemorrhagic areas of the ski | | | er lesions are usually a darker purple | e color an |
| eventually become a brownish | | | outrio appour roughornir seren era | a resignical o dedain, a dancer parpr | 0 00101 a.i. |
| Navigational Note: - | • | | | | |
| Rash acneiform | Papules and/or pustules | Papules and/or pustules | Papules and/or pustules | Life-threatening | Death |
| | covering <10% BSA, which | covering 10 - 30% BSA, which | covering >30% BSA with | consequences; papules and/or | |
| | may or may not be associated | may or may not be associated | moderate or severe | pustules covering any % BSA, | |
| | with symptoms of pruritus or | with symptoms of pruritus or | symptoms; limiting self-care | which may or may not be | |
| | tenderness | tenderness; associated with | ADL; associated with local | associated with symptoms of | |
| | | psychosocial impact; limiting | superinfection with oral | pruritus or tenderness and are | |
| | | instrumental ADL; papules | antibiotics indicated | associated with extensive | |
| | | and/or pustules covering > | | superinfection with IV | |
| | | 30% BSA with or without mild | | antibiotics indicated | |
| | 1 | symptoms | <b>I</b> | l | l |
| | erized by an eruption of papules and p | oustules, typically appearing in face | , scalp, upper chest and back. | | |
| Navigational Note: -<br>Rash maculo-papular | Macules/papules covering | Macules/papules covering 10 - | Macules/papules covering | T | |
| rasn maculo-papular | <10% BSA with or without | 30% BSA with or without | >30% BSA with moderate or | l <sup>-</sup> | - |
| | symptoms (e.g., pruritus, | symptoms (e.g., pruritus, | severe symptoms; limiting self | | |
| | burning, tightness) | burning, tightness); limiting | care ADL | l | |
| | buttillig, agridless) | instrumental ADL: rash | Cale ADL | l | |
| | | covering > 30% BSA with or | | l | |
| | | without mild symptoms | | l | |
| Dafinition: A disarder aborest | <br>erized by the presence of macules (fla | | l<br>un as marbillfarm rash, it is and af | I<br>the most common sutaneous advan | l<br>se events |
| | trunk, spreading centripetally and as | | wir as morbimonii rasii, it is one or | are most common tartaneous adver | se events |
| Vavigational Note: - | unit, spreading certained and as | aociacca wia i prartus. | | | |
| iavigational Note: - | | | | | |

| | Skin and subcutaneous tissue | disorders | | |
|---|---|---|---|---|
| Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| terized by a sensation of marked disco | mfort in the skin covering the top a | nd the back of the head. | | |
| Covering <10% BSA;<br>associated with<br>telangiectasias or changes in<br>skin color | Covering 10 - 30% BSA;<br>associated with striae or<br>adnexal structure loss | Covering >30% BSA;<br>associated with ulceration | - | - |
| cterized by the degeneration and thinni | ng of the epidermis and dermis. | • | | • |
| Hyperpigmentation covering<br><10% BSA; no psychosocial<br>impact | Hyperpigmentation covering<br>>10% BSA; associated<br>psychosocial impact | - | - | - |
| cterized by darkening of the skin due to | excessive melanin deposition. | • | • | • |
| Hypopigmentation or<br>depigmentation covering<br><10% BSA; no psychosocial<br>impact | Hypopigmentation or<br>depigmentation covering<br>>10% BSA; associated<br>psychosocial impact | - | - | = |
| cterized by loss of skin pigment (e.g., vi | tiligo). | • | • | • |
| Mild induration, able to move<br>skin parallel to plane (sliding)<br>and perpendicular to skin<br>(pinching up) | Moderate induration, able to<br>slide skin, unable to pinch<br>skin; limiting instrumental ADL | Severe induration; unable to<br>slide or pinch skin; limiting<br>joint or orifice movement<br>{e.g., mouth, anus}; limiting<br>self care ADL | Generalized; associated with<br>signs or symptoms of impaired<br>breathing or feeding | Death |
| cterized by an area of hardness in the s | kin. | • | - | • |
| Combined area of ulcers <1<br>cm; nonblanchable erythema<br>of intact skin with associated<br>warmth or edema | Combined area of ulcers 1 - 2<br>cm; partial thickness skin loss<br>involving skin or<br>subcutaneous fat | Combined area of ulcers >2<br>cm; full-thickness skin loss<br>involving damage to or<br>necrosis of subcutaneous<br>tissue that may ex tend down<br>to fascia | Any size ulcer with extensive destruction, tissue necrosis, or damage to muscle, bone, or supporting structures with or without full thickness skin loss | Death |
| | Mild pain cterized by a sensation of marked disco Covering <10% BSA; associated with telangiectasias or changes in skin color cterized by the degeneration and thinni Hyperpigmentation covering <10% BSA; no psychosocial impact terized by darkening of the skin due to Hypopigmentation or depigmentation covering <10% BSA; no psychosocial impact terized by loss of skin pigment (e.g., vi Mild induration, able to move skin parallel to plane (sliding) and perpendicular to skin (pinching up) terized by an area of hardness in the si Combined area of ulcers <1 cm; nonblanchable erythema of intact skin with associated | Grade 1 Grade 2 Mild pain Moderate pain; limiting instrumental ADL Sterized by a sensation of marked discomfort in the skin covering the top at | Mild pain Moderate pain; limiting Severe pain; limiting Instrumental ADL Severe pain; limiting Severe pain; limiting | Mild pain Moderate pain; limiting Severe pain; limiting self care ADL |

| | | Skin and subcutaneous tissue | disorders | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| | -<br>rized by less than 10% total body ski | -<br>n area separation of dermis. The sy | Skin sloughing covering <10%<br>BSA with associated signs<br>(e.g., erythema, purpura,<br>epidermal detachment, and<br>mucous membrane<br>detachment)<br>androme is thought to be a hyperser | Skin sloughing covering 10 -<br>30% BSA with associated signs<br>(e.g., erythema, purpura,<br>epidermal detachment and<br>mucous membrane<br>detachment)<br>nsitivity complex affecting the skin a | Death<br>Ind the |
| mucous membranes. | | | | | |
| Navigational Note: - | | | | | |
| Subcutaneous emphysema | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>limiting self care ADL | - | - |
| Definition: A disorder character | rized by air in the subcutaneous tissa | | | • | • |
| Navigational Note: - | nzed by an in the subcutanced susse | | | | |
| Telangiectasia | Telangiectasias covering < 10% | Telangiectasias covering | | 1 | 1 |
| Terangrectasia | BSA BSA | >=10% BSA; associated with psychosocial impact | - | | = |
| Definition: A disorder character | rized by local dilatation of small vess | | the skin or mucous membranes. | • | • |
| Navigational Note: - | , | | | | |
| Toxic epidermal necrolysis | - | - | - | Skin sloughing covering >=30%<br>BSA with associated<br>symptoms (e.g., erythema,<br>purpura, or epidermal<br>detachment) | Death |
| Definition: A disorder character | rized by greater than 30% total body | skin area separation of dermis. Th | e syndrome is thought to be a hype | rsensitivity complex affecting the sk | in and the |
| mucous membranes. | , 3 | | | ,, | |
| Navigational Note: - | | | | | |
| Urticaria | Urticarial lesions covering<br><10% BSA; topical<br>intervention indicated | Urticarial lesions covering 10 -<br>30% BSA; oral intervention<br>indicated | Urticarial lesions covering<br>>30% BSA; IV intervention<br>indicated | - | - |
| Definition: A disorder character | rized by an itchy skin eruption chara | -<br>cterized by wheals with pale interio | ors and well-defined red margins. | • | • |
| Navigational Note: - | | | | | |
| Maniferioriei More: - | | | | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| Skin and subcutaneous tissue disorders | | | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Skin and subcutaneous tissue<br>disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: - | | | | | |
| Navigational Note: - | | | | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| Social circumstances | | | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Social circumstances - Other,<br>specify | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: - | | | | | |
| Navigational Note: - | | | | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| Surgical and medical procedures | | | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Surgical and medical<br>procedures - Other, specify | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: - | | | | | |
| Navigational Note: - | | | | | |

| | | Vascular disorders | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Arterial thromboembolism | - | - | Urgent intervention indicated | Life-threatening<br>consequences; hemodynamic<br>or neurologic instability; organ<br>damage; loss of extremity(ies) | Death |
| Definition: A disorder character | ized by occlusion of an arterial vess | el b <b>y</b> a blood clot that develops in a | n arter <b>y.</b> | | |
| Navigational Note: Consider Ne | rvous system disorders: TIA or Stro | ke for CNS-related events or Cardia | disorders: Myocardial infarction | | |
| Capillary leak syndrome | Asymptomatic | Symptomatic; medical intervention indicated | Severe symptoms;<br>intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| | | | | who demonstrate a state of general<br>eneralized edema and multiple orga | |
| Flushing | Asymptomatic; clinical or diagnostic observations only | Moderate symptoms; limiting instrumental ADL | Symptomatic, associated with<br>hypotension and/or<br>tachycardia; limiting self care<br>ADL | - | - |
| Definition: A disorder character | ized by episodic reddening of the sl | kin, especially face, neck, or chest. | | | • |
| Navigational Note: - | | | | | |
| Hematoma | Mild symptoms; intervention<br>not indicated | Minimally invasive evacuation<br>or aspiration indicated | Transfusion; invasive intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| <b>Definition:</b> A disorder character <b>Navigational Note:</b> - | ized by a localized collection of bloo | od, usually dotted, in an organ, spa | te, or tissue, due to a break in the w | vall of a blood vessel. | |
| Hot flashes | Mild symptoms; intervention<br>not indicated | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL | - | - |
| Definition: A disorder character | ized by an uncomfortable and temp | porary sensation of intense body wa | rmth, flushing, sometimes accompa | anied by sweating upon cooling. | • |
| Navigational Note: - | | | | | |

| | | Vascular disorders | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Hypertension | Adult: Systolic BP 120 - 139<br>mm Hg or diastolic BP 80 - 89<br>mm Hg;<br>Pediatric: Systolic/diastolic BP<br>>90th percentile but< 95th<br>percentile; | Adult: Systolic BP 140 - 159<br>mm Hg or diastolic BP 90 - 99<br>mm Hg if previously WNL;<br>change in baseline medical<br>intervention indicated;<br>recurrent or persistent (>=24<br>hrs); symptomatic increase by<br>>20 mm Hg (diastolic) or to | Adult: Systolic BP >=160 mm<br>Hg or diastolic BP >=100 mm<br>Hg; medical intervention<br>indicated; more than one drug<br>or more intensive therapy<br>than previously used<br>indicated; | Adult and Pediatric: Life-<br>threatening consequences<br>(e.g., malignant hypertension,<br>transient or permanent<br>neurologic deficit,<br>hypertensive crisis); urgent<br>intervention indicated | Death |
| | Adolescent: BP ≥120/80 even if < 95th percentile | >140/90 mm Hg;<br>monotherapy indicated<br>initiated; | Pediatric and adolescent: Systolic and/or diastolic > 5 mmHg above the 99th percentile | | |
| | | Pediatric and adolescent: Recurrent or persistent (>=24 hrs) BP >ULN; monotherapy indicated; systolic and /or diastolic BP between the 95th percentile and 5 mmHg above the 99th percentile; Adolescent: Systolic between 130-139 or diastolic between 80-89 even if < 95th percentile | | | |
| Definition: A disorder charact<br>Navigational Note: - | erized b <b>y</b> a pathological increase in bl | ood pressure. | | | |
| Hypotension | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Medical intervention<br>indicated; hospitalization<br>indicated | Life-threatening<br>consequences and urgent<br>intervention indicated | Death |
| Definition: A disorder charact<br>Navigational Note: - | erized by a blood pressure that is belo | ow the normal expected for an indiv | idual in a given environment. | • | • |
| Lymph leakage | - | Symptomatic; medical intervention indicated | Severe symptoms; invasive intervention indicated | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder charact | erized by the loss of lymph fluid into t | he surrounding tissue or body cavit | у. | • | • |
| Navigational Note: - | | | | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Vascular disorders | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Lymphedema | Trace thickening or faint discoloration | Marked discoloration;<br>leathery skin texture; papillary<br>formation; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL | - | - |
| Definition: A disorder character | rized by excessive fluid collection in | tissues that causes swelling. | • | • | • |
| Navigational Note: - | | | | | |
| Lymphocele | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; invasive intervention indicated | - | - |
| Definition: A disorder character | rized by a cystic lesion containing ly | mph. | • | • | • |
| Navigational Note: - | | | | | |
| Peripheral ischemia | - | Brief (<24 hrs) episode of<br>ischemia managed medically<br>and without permanent<br>deficit | Prolonged (>=24 hrs) or<br>recurring symptoms and/or<br>invasive intervention<br>indicated | Life-threatening<br>consequences; evidence of<br>end organ damage; urgent<br>operative intervention<br>indicated | Death |
| <b>Definition:</b> A disorder character <b>Navigational Note:</b> - | rized by impaired circulation to an e | extremity. | | | |
| Phlebitis | - | Present | - | - | - |
| Definition: A disorder character | rized by inflammation of the wall of | a vein. | • | • | • |
| Navigational Note: - | • | | | | |
| Superficial thrombophlebitis | = | Present | = | = | - |
| Definition: A disorder character | rized by a blood clot and inflammat | ion involving a superficial vein of the | e extremities. | • | • |
| Navigational Note: - | | | | | |
| Superior vena cava syndrome | Asymptomatic; incidental finding of SVC thrombosis | Symptomatic; medical intervention indicated (e.g., anticoagulation, radiation or chemotherapy) | Severe symptoms; multi-<br>modality intervention<br>indicated (e.g.,<br>anticoagulation,<br>chemotherapy, radiation,<br>stenting) | Life-threatening<br>consequences; urgent multi-<br>modality intervention<br>indicated (e.g., lysis,<br>thrombectomy, surgery) | Death |
| | | w in the superior vena cava. Signs a | and symptoms include swelling and | cyanosis of the face, neck, and upp | er arms, |
| cough, orthopnea and headach<br>Navigational Note: - | e. | | | | |
| Navigational Note: - | | | | | |

**Title**: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients undergoing Complex Cardiac Surgery Procedures (the ReCePI study)

| | | Vascular disorders | | | |
|---|---|---|---|---|---|
| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Thromboembolic event | Medical intervention not indicated (e.g., superficial thrombosis) | Medical intervention indicated | Urgent medical intervention<br>indicated (e.g., pulmonary<br>embolism or intracardiac<br>thrombus) | Life-threatening<br>consequences with<br>hemodynamic or neurologic<br>instability | Death |
| Definition: A disorder character | ized by occlusion of a vessel by a th | -<br>rombus that has migrated from a di | stal site via the blood stream. | | |
| Navigational Note: Consider Ne | rvous system disorders: TIA or Strok | e for CNS-related events. Use Vasc | ular disorders: Arterial thromboem | bolism for arterial thrombi. | |
| Vasculitis | Asymptomatic, intervention not indicated | Moderate symptoms, medical intervention indicated | Severe symptoms, medical intervention indicated (e.g., steroids) | Life-threatening<br>consequences; evidence of<br>peripheral or visceral<br>ischemia; urgent intervention<br>indicated | Death |
| <b>Definition:</b> A disorder character | ized by inflammation involving the v | wall of a vessel. | | | |
| Navigational Note: - | | | | | |
| Vascular disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: - | • | - | • | • | • |
| Navigational Note: - | | | | | |